# The GlaxoSmithKline group of companies

| Division | : | Worldwide Development |
|------------------|---|-----------------------------------|
| Information Type | : | Reporting and Analysis Plan (RAP) |

| Title | : | Reporting and Analysis Plan for A 6-month, open label, randomised, efficacy study to evaluate fluticasone furoate (FF, GW685698)/vilanterol (VI, GW642444) Inhalation Powder delivered once daily via the Dry Powder Inhaler Ellipta compared with usual ICS/LABA maintenance therapy delivered by Dry Powder Inhaler in subjects with Persistent Asthma |
|---|---|---|
| <b>Compound Number</b> | : | GW685698+GW642444 |
| Effective Date | : | 21-AUG-2017 |

# **Description:**

The purpose of this document is to describe the final planned analyses and output to be included in the Clinical Study Report for Protocol HZA116492.

This RAP is intended to describe the planned efficacy and safety analyses required for the study.

This RAP will be provided to the study team members to convey the content of the final Statistical Analysis Complete (SAC) deliverable.

#### **Author's Name and Functional Area:**

| PPD | 05-DEC-2016 |
|----------------------------------------------|-------------|
| Principal Statistician (Clinical Statistics) | 03-DEC-2010 |
| PPD | 16-AUG-2017 |
| Statistics Leader (Clinical Statistics) | 10-AUG-201/ |

# Approved by:

| PPD | 18-AUG-2017 |
|---|---|
| Director, Statistics & Programming (Clinical Statistics) | 16-AUG-2017 |
| PPD | 21-AUG-2017 |
| Programming Manager (Clinical Programming) | 21 <b>-</b> AUG-201/ |

Copyright 2017 the GlaxoSmithKline group of companies. All rights reserved. Unauthorised copying or use of this information is prohibited.

# **TABLE OF CONTENTS**

| | | | | PAGE |
|---|---|---|---|---|
| 1. | REPO | RTING & | ANALYSIS PLAN SYNPOSIS | 5 |
| 2. | RAP A | MENDME | ENTS | 8 |
| _ | | | .,_,, | |
| 3. | | | KEY PROTOCOL INFORMATION | |
| | 3.1. | | s to the Protocol Defined Statistical Analysis Plan | |
| | 3.2. | | bjectives and Endpoints | |
| | 3.3. | Sample | al Hypotheses | 10 |
| | 3.4. | Sample | Size Assumptions | 10 |
| 4. | PLANI | NED ANA | LYSES | 17 |
| | 4.1. | | Analyses | |
| | 4.2. | | ok | |
| | 4.3. | | alyses | |
| 5. | | | PULATIONS | |
| | 5.1. | Protocol | Deviations | 19 |
| 6. | | | ONS FOR DATA ANALYSES AND DATA HANDLING | 20 |
| 7. | | | ATION ANALYSES | |
| | 7.1. | Overviev | v of Planned Analyses | 21 |
| 8. | PRIMA | ARY STAT | TISTICAL ANALYSES | 22 |
| 0. | 8.1. | | Analyses | |
| | 0.1. | 8.1.1. | Overview of Planned Efficacy Analyses | |
| | | 8.1.2. | | |
| | | | • | |
| 9. | SECO | NDARY S | STATISTICAL ANALYSES | 26 |
| | 9.1. | Efficacy | Analyses | |
| | | 9.1.1. | | |
| | | 9.1.2. | Planned Efficacy Statistical Analyses | |
| | 9.2. | | nalyses | 29 |
| | | 9.2.1. | Overview of Planned Analyses | |
| | | 9.2.2. | Benefit:Risk analyses | 30 |
| 10 | OTHE | R STATIS | STICAL ANALYSES | 32 |
| 10. | 10.1. | | nalyses | |
| | 10.1. | | Overview of Planned Other Analyses | |
| | | | Planned Other Statistical Analyses | |
| | | | , | |
| 11. | REFE | RENCES. | | 37 |
| 12 | APPEI | VDICES | | 32 |
| 14. | 12.1. | | x 1: Protocol Deviation Management and Definitions for PP | |
| | | | on | 39 |
| | | | Protocol Deviations | |
| | | | Exclusions from PP Population | |

| 12.2. | | x 2: Time & Events | |
|---|---|---|---|
| 40.0 | | Protocol Defined Time & Events | |
| 12.3. | | x 3: Assessment Windows | |
| 12.4. | | x 4: Treatment States and Phases | |
| | | Treatment Phases | |
| | 12.4.2. | Treatment States | |
| | | 12.4.2.1. Treatment States for Concomitant Medications | |
| | | 12.4.2.2. Treatment States for Efficacy Measurements | |
| | | 12.4.2.3. Treatment States for Exacerbation Data | |
| 40.5 | ۸ا!. | 12.4.2.4. Treatment States for AE Data | |
| 12.5. | | x 5: Data Display Standards & Handling Conventions | |
| | 12.5.1. | 3 - 1 - 1 - 1 - 1 | |
| | 12.5.2. | Baseline Definition & Derivations | |
| | | 12.5.2.1. Baseline Definitions | 40 |
| | | 12.5.2.2. Derivations and Handling of Missing Baseline | 40 |
| | 40.50 | Data | |
| 10.6 | 12.5.3. | Reporting Process & Standards | |
| 12.6. | 12.6.1. | x 6: Derived and Transformed DataGeneral | |
| | _ | | |
| | 12.6.2. | Study Population | |
| | 12.6.3.<br>12.6.4. | Efficacy | |
| 12.7. | | Safetyx 7: Premature Withdrawals & Handling of Missing Data | |
| 12.7. | 12.7.1. | | |
| | 12.7.1. | Handling of Missing Data | |
| | 12.7.2. | 12.7.2.1. Handling of Missing or Partial Dates | |
| | | 12.7.2.1. Handling of Missing Data for Statistical | 57 |
| | | Analysis | 58 |
| 12.8. | Annendiy | x 8: Values of Potential Clinical Importance | |
| 12.0. | | Vital Signs | |
| 12.9. | | x 9: Multicenter Studies | |
| 12.0. | | Methods for Handling Centres | |
| 12 10 | | x 10: Examination of Covariates, Subgroups & Other Strata | |
| 12.10. | | Examination of Strata and Covariates | |
| | | Examination of subgroups | |
| | | Examination of seasonal effect | |
| 12.11. | | x 11: Multiple Comparisons & Multiplicity | |
| | | Handling of Multiple Comparisons & Multiplicity | |
| 12.12. | | x 12: Model Checking and Diagnostics for Statistical | |
| | | S | 64 |
| | 12.12.1. | Statistical Analysis Assumptions | 64 |
| 12.13. | | x 13: Blinding Strategy | |
| 12.14. | Appendix | x 14: Abbreviations & Trade Marks | 67 |
| | | Abbreviations | |
| | 12.14.2. | Trademarks | 68 |
| 12.15. | Appendix | x 15: List of Data Displays | 69 |
| | | Data Display Numbering | |
| | | Mock Example Shell Referencing | |
| | | Deliverable [Priority] | |
| | | Study Population Tables | |
| | | Study Population Figures | |
| | | Efficacy Tables | |

# 2017N339371\_00 HZA116492


| | 12.15.7. | Efficacy Figures | 93 |
|--------|----------|---------------------------------------------|-----|
| | 12.15.8. | Safety Tables | 97 |
| | 12.15.9. | Safety Figures | 100 |
| | | .ICH Listings | |
| | | .Non-ICH Listings | |
| 12.16. | | c 16: Example Mock Shells for Data Displays | |
| | | Study Population Table Shells | |
| | | Study Population Figure Shells | |
| | | Efficacy Table Shells | |
| | | Efficacy Figure Shells | |
| | | Safety Table Shells | |
| | | Safety Figure Shells | |
| | | Non-ICH Listing Shells | |

# 1. REPORTING & ANALYSIS PLAN SYNPOSIS

| Overview | Key Elements of the RAP |
|---|---|
| Purpose | This RAP details all planned analyses and output required for the final Clinical Study Report of study HZA116492. |
| Protocol | This RAP is based on the protocol amendment 02 (Dated: 28-APR-2016) of study HZA116492 (GSK Document No.: 2014N190259_02). |
| Primary<br>Objective | To compare the efficacy of fluticasone furoate (FF)/vilanterol(VI) 92 mcg/22 mcg or FF 184 mcg/22 mcg with usual fixed combinations inhaled corticosteroid / long-acting beta agonist (ICS/LABA) for asthma maintenance therapy at Week 12 (Visit 4). |
| Primary<br>Endpoint | Change from baseline in the Asthma Control Test (ACT) total score at Week 12 (Visit 4). |
| Study<br>Design | This is a Phase IIIb multi-center randomised open label, parallel group study performed in subjects in primary and in respiratory specialist care / research sites who have a diagnosis of asthma and a regular treatment for asthma. Subjects with unsatisfactorily controlled asthma (defined as an ACT < 20) and intended to be treated by usual ICS/LABA maintenance therapy to seek a better control of their asthma will be randomised to receive either FF/VI (FF/VI 92 mcg/22 mcg or FF/VI 184 mcg/22 mcg) once daily or another usual ICS/LABA combination therapy in inhalation powder twice daily (fluticasone propionate[FP]/salmeterol [S] or budesonide[BUD]/formoterol [F]) decided by the physician. |
| | Physicians will be allowed during the treatment period to adapt prescription to different doses if necessary as well as to adapt doses of any comparative treatment according to products label. |
| Planned | No interim analysis is planned for this study. |
| Analyses | All decisions regarding final analysis for the reporting effort, as defined in this RAP document, will be made prior to Database Freeze (DBF) (unblinding) of the study data. |
| | All planned analyses will be carried out once DBF has taken place. Once this has been achieved, unblinding will occur and the analyses will be performed. |
| | The open-label study design and the method of recording study medication data in the datasets means that extra steps must be taken to ensure that Statistics and Programming (S&P) remain blinded to study investigator prescribing of study medication until the formal unblinding takes place at DBF. See Section 12.13 for more details. |

| Overview | Key Elements of the RAP |
|---|---|
| Analysis<br>Populations | All Subjects Enrolled (ASE) population: All subjects screened (provided consent) and for whom a record exists on the study database. Note, this population is not identified in the protocol, but is needed for displays that include subjects screened but not in the intent-to-treat (ITT) population (e.g. tabulation of reasons for withdrawal before randomisation). |
| | Intent-to-treat (ITT) population: All randomized subjects having received at least one dose of the prescription of study medication (either FF/VI or usual ICS/LABA asthma maintenance therapy). The ITT population will be used to analyze the primary efficacy endpoint analysis, the secondary efficacy endpoint and other efficacy endpoints. Subjects will be assigned to the treatment group as randomized for the ITT population. |
| | Per protocol (PP) population: all ITT subjects without any protocol deviations specifically defined in this RAP. Protocol deviations will be reviewed and will be classified as important or not important during data review meetings that will be held before DBF. Deviations classified as important will be further defined according to whether they require the patient to be excluded from the PP population. Deviations that exclude a patient from the PP population are defined in this RAP (see Section 12.1.2). Subjects will be assigned to the treatment group as treated for the PP population. |
| | <u>Safety population:</u> All enrolled subjects having received at least one dose of the prescription of study medication (either FF/VI or usual ICS/LABA asthma maintenance therapy) and considered as-treated. The Safety population will be the basis for safety analyses. Subjects will be assigned to the treatment group as treated for the Safety population. |
| Hypothesis | The primary analysis is designed to determine whether the fixed combination FF/VI is non-inferior to any other ICS/LABA combinations in inhalation powder assuming a non-inferiority margin of 1.5. Non-inferiority will be claimed if the 95% two-sided confidence interval (CI) on the difference in mean primary efficacy endpoints (FF/VI versus ICS/LABA comparator) precludes the non-inferiority margin of -1.5. |
| | If (and only if) non-inferiority is significantly achieved at Week 12 (Visit 4) with regard to the primary endpoint, then non-inferiority of the fixed combination FF/VI to any other ICS/LABA combinations will be tested at Week 24 (Visit 6) considering the same non-inferiority margin of 1.5. Non-inferiority will be claimed if the 95% two-sided CI on the difference in mean primary efficacy endpoints (FF/VI versus ICS/LABA comparator) at Week 24 (Visit 6) precludes the non-inferiority margin of -1.5. This step-down testing procedure strongly controls the overall type I error of the non-inferiority endpoints at the 0.05 two-sided level. |
| Primary<br>Analyses | The primary endpoint will be analysed using a mixed model repeated measures (MMRM) approach. The model will include factors and covariates as follows: randomised treatment, scheduled visit time point (Week 6 and Week 12), baseline ACT total score, randomised treatment-by-visit interaction, baseline ACT total score-by-visit interaction, gender, age, country and patient will be fitted as a random factor. The Restricted Maximum Likelihood (REML) estimation approach will be used, and the default covariance structure will be unstructured. Consistent with MMRM model fitting, no explicit imputation of missing assessments for a given time point will be performed. The adjusted means for each treatment and the estimated treatment differences for the treatment comparisons will be presented together with the 95% CIs for the differences (FF/VI versus ICS/LABA comparator) and p-values at Week 12 (Visit 4). |
| | If non-inferiority is statistically achieved at Week 12 (Visit 4), then superiority of FF/VI to any other comparator will be tested at the usual 0.05 two-sided nominal level of significance. |

| Overview | Key Elements of the RAP |
|---|---|
| | The same models and analyses mentioned above will be used to assess the superiority hypothesis. |
| Secondary<br>Analyses | Key secondary analysis |
| Allalyses | The key secondary endpoint assessed at Week 24 (Visit 6) will also be analyzed using a MMRM approach where data up to and including Week 24 (Visit 6) will be used in the model. The model will include factors and covariates as follows: randomised treatment, scheduled visit time point (Week 6, Week 12, Week 18 and Week 24), baseline ACT total score, randomised treatment-by-visit interaction, baseline ACT total score-by-visit interaction, gender, age, country and patient will be fitted as a random factor. The REML estimation approach will be used, and the default covariance structure will be unstructured. Consistent with MMRM model fitting, no explicit imputation of missing assessments for a given time point will be performed. The adjusted means for each treatment and the estimated treatment difference for the treatment comparison will be presented together with the 95% CI for the difference (FF/VI versus ICS/LABA comparator) and p-value at Week 24 (Visit 6). If non-inferiority is statistically achieved at Week 24 (Visit 6), then superiority of FF/VI versus any other comparator will be tested at the usual 0.05 two-sided nominal level of significance. The same models and analyses mentioned above will be used to assess the superiority |
| | hypothesis. Other secondary analyses |
| | The other key secondary endpoint will be the correct use of the inhaler device assessed at randomisation (Visit 2), at Week 12 (Visit 4) and at Week 24 (Visit 6). The device will be considered as correctly used if the patient didn't make any critical or non-critical errors at the corresponding visits (randomisation [Visit 2], Week 12 [Visit 4] and Week 24 [Visit 6]). Percentages of subjects correctly using the device will be calculated within each group. A corresponding 95% CI of the difference in percentages will also be provided. |
| | An exploratory analysis of the categorised data will be performed using logistic regression models with covariates as follows: randomised treatment, correct use of inhaler device at baseline, randomised treatment-by-visit interaction, gender, age and country. The estimated treatment differences will be displayed as odds ratios together with 95% CIs and p-values. |

# 2. RAP AMENDMENTS

A summary of the amendments made to the RAP are listed here.

## **Amendment Details**

# RAP-HZA116492 [05-DEC-2016]

# GSK2285997-116492 Statistical Analysis Plan Reporting and Analysis Plan (Amendment 1) Version 001 [21-AUG-2017]

Subjects with a missed or out of window Visit 4 will no longer lead to exclusion from the PP population.

Treatment compliance calculation now covers changes in dose.

Clarified age range to be used, multiple sections

Updated standard shell references in Section 12.15

Added time since last dose derivation.

Resolved discrepancies between main body and example shells for terms included in subgroup analyses

Clarified labelling: "Day 0" to be labelled as "Randomisation (Day 0)"

Clarified labelling for MARS-A subgroups

Other label ordering clarifications

Removed references to PCI values for Vital Signs and updated tables accordingly

# 3. SUMMARY OF KEY PROTOCOL INFORMATION

# 3.1. Changes to the Protocol Defined Statistical Analysis Plan

Any changes from the originally planned statistical analysis specified in the protocol are outlined in Table 1.

Table 1 Changes to Protocol Defined Analysis Plan

| Protocol | Reporting & Analysis Plan | |
|---|---|---|
| Statistical Analysis Plan | Statistical Analysis Plan | Rationale for Changes |
| • N/A | The open-label study design and the method of recording study medication data in the datasets means that extra steps must be taken to ensure that S&P remain blinded to study investigator prescribing of study medication until the formal unblinding takes place at DBF. See Section 12.13 for more details. | To preserve the integrity of<br>the analyses, S&P will<br>remain blinded prior to<br>formal unblinding at DBF.<br>All planned analyses will be<br>carried out after this point. |
| • N/A | All Subjects Enrolled (ASE) Population: All subjects screened (provided consent) and for whom a record exists on the study database. Note, this population is not identified in the protocol, but is needed for displays that include subjects screened but not in the ITT Population (e.g. tabulation of reasons for withdrawal before randomisation). | Population needed for displays that include subjects screened but not in the ITT population. |
| <ul> <li>Continuous variables will be summarized using descriptive statistics (number of observed and missing data, mean, standard deviation (SD), median, Q1, Q3, minimum, and maximum).</li> <li>Categorical variables will be summarized as numbers of observed and missing data, counts and percentage for each category (reported to the number of non-missing values). For binary variables, 95% confidence</li> </ul> | See Appendix 16: Example Mock Shells for Data Displays for example mock shells for data displays | Continuous and categorical<br>variables will be<br>summarized in line with<br>GSK Integrated Data<br>Standards Library (IDSL)<br>data standards |

| Protocol | Reporting & Analysis Plan | |
|---|---|---|
| Statistical Analysis Plan | Statistical Analysis Plan | Rationale for Changes |
| intervals for proportions will be estimated based on the Clopper-Pearson method. | | |
| If treatment is withdrawn, then the missing ACT score at the nearest visit after treatment withdrawal will be replaced by the ACT score assessed at withdrawal time. If no ACT score is assessed at withdrawal time, then the ACT missing score at the nearest visit after treatment withdrawal will not be replaced. | Consistent with MMRM model fitting, no explicit imputation of missing assessments for a given time point will be performed. | The protocol inconsistently describes whether or not missing scores will be imputed. Consistent with MMRM models and the MAR assumption they are based upon, no missing data will be imputed for the primary efficacy analysis. Sensitivity analyses for the primary endpoint are proposed in Section 8.1.2 and will consider imputation of missing data. |
| The primary endpoint will be analysed using a mixed model repeated measures (MMRM) approach. The model will include factors and covariates as follows: treatment, scheduled visit time point (Week 6 and Week 12), baseline ACT, treatment by visit interaction, baseline ACT by visit interaction, gender, age and patient will be fitted as a random factor. | The primary endpoint will be analysed using a MMRM approach. The model will include factors and covariates as follows: randomised treatment, scheduled visit time point (Week 6 and Week 12), baseline ACT total score, randomised treatment-by-visit interaction, baseline ACT total score-by-visit interaction, gender, age, country and patient will be fitted as a random factor. | Clarified that randomised treatment and baseline ACT total score will be included. Additionally country will be included in the model due to the addition of Germany, and separate randomisation schedules for France and Germany achieving stratification by country Same changes for secondary and other analyses |
| Sensitivity analyses (for the primary endpoint) | Text changed and clarified | The text from the protocol regarding sensitivity analyses has been updated and clarified where necessary. Description of the multiple imputation (MI) process has been brought in line with GSK standard text. |
| Usual ICS/LABA maintenance<br>therapy | Usual ICS/LABA | The comparator arm is described as "Usual ICS/LABA" for consistency with reporting of the HZA115150 study (GSK Document No.: 2011N129785_02). |

| Protocol | Reporting & Analysis Plan | |
|---|---|---|
| Statistical Analysis Plan | Statistical Analysis Plan | Rationale for Changes |
| | Statistical Analysis Plan EQ-5D-5L This endpoint will be analysed using a logistic regression model adjusting for randomised treatment, gender, country, baseline ACT total score, baseline ACT total score squared and age | <ul> <li>Clarity as to which version of the EuroQol questionnaire is being used</li> <li>Clarified that randomised treatment will be included.</li> <li>Country will be included in the model due to the addition of Germany, and separate randomisation schedules for France and Germany achieving stratification by country</li> <li>Due to this being a composite endpoint, a quadratic relationship is expected between baseline score and probability of response. Baseline ACT total score and baseline ACT total score squared will be included (instead of "baseline ACT score categorised into two classes") to account for this</li> <li>All patients are on the same</li> </ul> |
| | | baseline asthma therapy class (ICS), therefore this will not be included as a covariate • Season at randomisation will not be included; this is only considered as sensitivity analysis for the primary efficacy endpoint |
| • N/A | <ul> <li>≥ 3 point increase from baseline in ACT total score at Week 12 (Visit 4) and Week 24 (Visit 6)</li> <li>Time to first severe asthma exacerbation</li> </ul> | These endpoints have been added for consistency with the HZA115150 study (GSK Document No.: 2011N129785_02). |

# 3.2. Study Objectives and Endpoints

| Objectives | | Endpoints |
|---|---|---|
| Pri | mary Objective | Primary Endpoint |
| • | To compare the efficacy of FF/VI 92 mcg/ 22 mcg or FF 184 mcg/22 mcg with usual fixed combinations ICS/LABA for asthma maintenance therapy at Week 12 (Visit 4). | <ul> <li>Change from baseline in the ACT total score at<br/>Week 12 (Visit 4).</li> </ul> |
| Sec | condary Objectives | Secondary Endpoints |
| • | To assess effect of FF/VI on asthma control compared with usual ICS/LABA fixed combination at Week 24 (Visit 6). | Change from baseline in ACT score at Week 24 (Visit 6). |
| • | To assess Ellipta™ inhaler correct use compared with other dry powder inhaler (DPI) (Diskus and Turbuhaler) at Week 12 (Visit 4) and at Week 24 (Visit 6) independently of the use at Week 12 (Visit 4). | <ul> <li>Percentage of subjects with correct use of device<br/>(defined as not making any critical error or non-<br/>critical error) at Week 12 (Visit 4) and at Week 24<br/>(Visit 6) independently of the use at Week 12 (Visit<br/>4).</li> </ul> |
| Oth | ner Objectives | Other Endpoints |
| • | To assess effect of FF/VI on trough (predose) forced expiratory volume in 1 second (FEV1) compared with usual ICS/LABA fixed combination at Week 12 (Visit 4) | Change from baseline in trough (pre-dose) FEV1 at Week 12 (Visit 4). |
| • | To assess the effect of FF/VI on response to treatment at Week 12 (Visit 4) and Week 24 (Visit 6) | <ul> <li>ACT score ≥ 20 or ≥ 3 point increase from baseline in ACT at Week 12 (Visit 4) and Week 24 (Visit 6). Note: A 3 point increase in ACT total score was suggested as the Minimal Clinically Important Difference (MCID) in the literature (Schatz, 2009).</li> <li>ACT score ≥ 20 at Week 12 (Visit 4) and Week 24 (Visit 6).</li> <li>≥ 3 Point Increase from Baseline in ACT Total Score at Week 12 (Visit 4) and Week 24 (Visit 6).</li> <li>Change from baseline in individual question scores for ACT at Weeks 12, 24</li> </ul> |
| • | To assess the compliance with study medication and self-reported adherence to study medication at Week 12 (Visit 4) and Week 24 (Visit 6) | <ul> <li>Compliance with study medication from Randomisation (Day 0) to Week 12 (Visit 4), from Week 12 (Visit 4) to Week 24 (Visit 6) and from randomisation (Day 0) to Week 24 (Visit 6).</li> <li>Score of the Medication Adherence Report Scale for Asthma (MARS-A) questionnaire at Randomisation (Day 0), Week 12 (Visit 4) and Week 24 (Visit 6).</li> </ul> |
| • | To assess the effect of FF/VI on severe asthma exacerbation over the study period | Number of subject with at least 1 severe asthma<br>exacerbation*, number of severe asthma<br>exacerbation and annual severe exacerbation rate<br>over the study period. |

| Objectives | Endpoints |
|---|---|
| | Time to first severe asthma exacerbation |
| To assess the effect of FF/VI on Health<br>Related Quality of Life at Week 24 (Visit 6) | <ul> <li>Change from baseline in total score and domain scores of standardised Asthma Quality of Life Questionnaire (AQLQ[S]) at Week 24 (Visit 6).</li> <li>An increase from baseline of ≥ 0.5 in AQLQ(s) total score at Week 24 (Visit 6).</li> <li>An increase from baseline of ≥ 0.5 in AQLQ(s) environmental stimuli domain score at Week 24 (Visit 6).</li> <li>Percentage of subjects who have an increase from baseline of ≥ 0.5 in AQLQ(S) individual domain scores at Week 24 (Visit 6).</li> <li>Change from baseline in total score and domain scores of AQLQ(S) at Week 24 (Visit 6).</li> <li>Health status using the EuroQol Questionnaire (EQ-5D-5L) at Week 24 (Visit 6).</li> </ul> |
| To assess Patient Satisfaction and<br>Preference assessment with different<br>inhalers at Week 12 (Visit 4) | Score of Patient Satisfaction and Preference<br>Questionnaire (PASAP-Q) at Week 12 (Visit 4). |
| To evaluate the Safety of FF/VI compared with usual ICS/LABA (FP/S and BUD/F). | <ul> <li>Serious Adverse Events (SAE) and non-serious Adverse Drug Reactions (ADR):</li> <li>Frequency and type of SAEs,</li> <li>Frequency and type of non-serious ADRs related to treatment.</li> </ul> |

<sup>\*</sup> A severe asthma exacerbation will be defined as deterioration of asthma requiring the use of systemic corticosteroids<sup>2</sup> (tablets, suspension, or injection) for at least 3 days or an inpatient hospitalisation, or emergency department visit due to asthma that required systemic corticosteroids <sup>1,2,3</sup>.

## Notes defining endpoints:

- 1. Contacts with a doctor or hospitalisation are defined as exacerbation-related contacts if these contacts were a direct result of an acute worsening of asthma symptoms.
- 2. A prescription of systemic corticosteroid is defined as exacerbation-related if the reason the drug was given, in whole or in part, was to treat an acute worsening of asthma symptoms.
- 3. Exacerbation-related hospitalisation includes hospitalisation that is prolonged as a result of an asthma exacerbation.



- A phone call is provided at Week 6 and Week 18 in order to check whether the subject has experienced any AEs and then the Investigator calling the patient must determine whether the event is related to study medication (either arm) and whether the event is serious. At these telephone calls subjects will also be asked to complete the ACT questionnaire and to send it back to the Investigator.
- Week 12 (Visit 4) should be scheduled at the same time of day as the randomisation visit (Visit 2).

# Design Features

- This is a Phase IIIb multi-center randomised open label, parallel group study performed in subjects in primary and respiratory specialist care / research sites who have a diagnosis of asthma and a regular treatment for asthma.
- Subjects with unsatisfactorily controlled asthma (defined as ACT total score < 20) and
  intended to be treated by usual ICS/LABA maintenance therapy to seek a better
  control of their asthma will be randomised to receive either FF/VI once daily or another
  usual ICS/LABA combination therapy in inhalation powder twice daily (FP/S or BUD/F)
  decided by the physician.</li>

## **Overview of Study Design and Key Features**

# Treatment Assignment

Subjects will be assigned to study treatment in accordance with the randomisation schedule.

Subjects will be randomised in a 1:1 ratio to one of the 2 following treatment groups:

FF/VI (as per dose guidance below)

Initiate on usual inhaled dry powder ICS/LABA fixed combination for asthma maintenance therapy (i.e. Seretide Diskus or Symbicort Turbuhaler) according to usual physician's prescription.

#### **Dose Guidance:**

For subjects randomised to FF/VI, Investigator can make dosing decision based on the guidance below:

- FF/VI 92 mcg/22mcg dose once a day is approximately equivalent to FP/S medium dose (250 mcg/50mcg) and BUD/F medium dose (200 mcg/6 mcg) twice a day. See Table 2 for further guidance for doses conversion for other corticosteroids.
- FF/VI 184 mcg/22 mcg dose once a day is approximately equivalent to FP/S high dose (500 mcg/50 mcg) and to BUD/F high dose (400 mcg/12 mcg) twice a day. See Table 2 for guidance for dose conversion for other corticosteroids.
- Starting doses are: 92 mcg/22 mcg once daily for FF/VI; 250 mcg/50 mcg twice daily for FP/S and 200 mcg/6 mcg twice daily for BUD/F.

Table 2 ICS/LABA Daily Dose (SmPC Seretide Diskus; Symbicort Turbuhaler)

| Formulation | Inhaler Devices | Doses Available (mcg)<br>ICS/LABA and<br>Inhalations/day |
|---|---|---|
| Fluticasone propionate/salmeterol | DPI (Diskus) | 1 inhalation x 2 Medium-dose 250/50 |
| | | High-dose 500/50 |
| Budesonide/formoterol | DPI (Turbuhaler) | 1-2 inhalations x 2 Medium-dose 200/6 High-dose 400/12 |

Information extracted from Global Initiative for Asthma (GINA, 2012).

For patients with moderate to severe hepatic impairment, the 92/22 micrograms dose of FF/VI should be used and patients should be monitored for systemic corticosteroid-related adverse reactions.

| Overview of St | udy Design and Key Features |
|---|---|
| | Planned Dose Adjustments Subjects for whom it is considered appropriate/necessary to adjust treatment can have their dose increased from the starting dose as would be normal clinical practice at the Investigator's discretion. This will not require the subject to be withdrawn from the study. |
| | It is not permitted for patients to be switched to a different treatment i.e. patients randomised to the usual ICS/LABA arm cannot change to a different ICS/LABA or receive FF/VI. Patients randomised to the FF/VI arm cannot receive usual ICS/LABA. If a switch between products is required, the patient should be withdrawn from the study. |
| Interim<br>Analysis | No interim analysis is planned for this study. |

From this point onwards in the RAP, usual ICS/LABA maintenance therapy will be referred to as usual ICS/LABA.

# 3.3. Statistical Hypotheses

The primary endpoint is defined as the change from baseline in the ACT total score assessed at Week 12 (Visit 4). The primary analysis will assess the non-inferiority of fixed combination FF/VI to usual ICS/LABA in inhalation powder assuming a non-inferiority margin of 1.5. Non-inferiority will be claimed if the 95% two-sided confidence interval on the difference in mean primary efficacy endpoints (FF/VI versus usual ICS/LABA) precludes the non-inferiority margin of -1.5.

If (and only if) non-inferiority is significantly achieved at Week 12 (Visit 4) with regard to the primary endpoint, then non-inferiority of the fixed combination FF/VI to usual ICS/LABA will be tested at Week 24 (Visit 6) considering the same non-inferiority margin of 1.5. Non-inferiority will be claimed if the 95% two-sided confidence interval on the difference in mean primary efficacy endpoints (FF/VI versus usual ICS/LABA) at Week 24 (Visit 6) precludes the non-inferiority margin of -1.5.

Of note, as the two tests for non-inferiority are sequentially performed, the closure principle holds and there is no need to adjust the two-sided nominal level of significance (i.e. 0.05) for each test.

# 3.4. Sample Size Assumptions

Results based on the HZA106829 study have shown that the estimated SD of the change in ACT score was 3.7. Unpublished data have shown that the standard deviation of change of ACT ranged from 3.8 to 4.8. Therefore, a somewhat conservative choice of SD of 4.5 point is retained.

Based on the literature (Schatz, 2009), the Minimally Important Difference (MID) of the ACT could be considered as 3 points. Half this MID (i.e. 1.5) could therefore be used to define the non-inferiority margin.

Assuming a 4.5 point standard deviation for the change in ACT total score at Week 12 (Visit 4), a 1.5 point non-inferiority margin, and a two-sided nominal significance level of 0.05, the sample size needed per group to achieve at least a 90% power is 191 (i.e. a total of 382 subjects).

Assuming a 10% dropout rate, around 422 subjects must be randomized either to FF/VI or to usual ICS/LABA in 1:1 ratio to achieve at least a 90% power.

## 4. PLANNED ANALYSES

# 4.1. Interim Analyses

Not applicable.

## 4.2. Data Look

At a date agreed by the study team and the contract research organisation (CRO) (selected to execute the statistical analyses specified in this RAP), a data look will be performed using blinded treatment codes on a subset of the data. The aim of the data look is solely to ensure that all of the required tables, figures and listings are being produced and formatted correctly, such that the output produced on unblinded data at the end of the study is correct and complete. This data look will be performed when sufficient data are available, but early enough to leave time for changes to be made to the planned outputs and methods prior to database release (DBR). Any changes will be documented before DBR.

# 4.3. Final Analyses

All planned analyses will be performed after the completion of the following sequential steps:

- 1. All subjects have completed the study as defined in the protocol
- 2. All required database cleaning activities have been completed and final DBR has been declared by Data Management.
- 3. All protocol deviations (PDs) have been confirmed
- 4. All criteria for unblinding the randomisation codes have been met.
- 5. Randomisation codes have been distributed according to RandAll NG procedures.
- 6. DBF has been declared by Data Management.

# 5. ANALYSIS POPULATIONS

| Population | Definition / Criteria | Analyses Evaluated |
|---|---|---|
| All Subjects<br>Enrolled (ASE) | Comprise of all subjects screened (provided consent) and for whom a record exists on the study database. | Subject disposition tables |
| | Note, this population is not identified in the protocol, but is needed for displays that include subjects screened but not in the ITT Population (e.g. tabulation of reasons for withdrawal before randomisation) | |
| Intent-to-Treat (ITT) | Comprise of all randomized subjects having<br>received at least one dose of the prescription of<br>study medication (either FF/VI or usual ICS/LABA) | Study Population Efficacy |
| | Subjects will be assigned to the treatment group as randomized for the ITT population | |
| Per Protocol (PP) | Comprise of all randomized subjects who receive<br>at least one dose of study treatment and who<br>comply with the protocol. | This population will be<br>used for summaries<br>and re-analyses of the |
| | <ul> <li>Protocol deviations that would exclude subjects<br/>from the PP population are defined in Section 5.1<br/>(Protocol Deviations) and Appendix 1 (Protocol<br/>Deviation Management and Definition for Per-<br/>Protocol Population).</li> </ul> | primary efficacy<br>secondary efficacy<br>endpoints. |
| Safety | <ul> <li>Comprise of all enrolled subjects having received at least one dose of study medication (either FF/VI or usual ICS/LABA) and considered as-treated.</li> <li>Subjects will be assigned to the treatment group as treated for the Safety population</li> </ul> | Safety |

# NOTES:

• Please refer to Appendix 15: List of Data Displays which details the population to be used for each displays being generated.

# 5.1. Protocol Deviations

All PDs (any deviation from the protocol) are tracked and monitored during the study. Important PDs are those deviations that may compromise subject rights, safety, or well-being, and/or data integrity, and/or study end-points, and are defined in the protocol deviation management plan (PDMP). Apart from any incorrect treatment deviations, all protocol deviations will be agreed upon prior the unblinding and the freezing of the database. All deviations from the inclusion/exclusion criteria, and important PDs will be summarised. A listing of treatment misallocations will be produced.

# 6. CONSIDERATIONS FOR DATA ANALYSES AND DATA HANDLING CONVENTIONS

Table 3 provides an overview of appendices within the RAP for outlining general considerations for data analyses and data handling conventions.

Table 3 Overview of Appendices

| Section | Component |
|---|---|
| 12.1 | Appendix 1: Protocol Deviation Management and Definitions for PP Population |
| 12.2 | Appendix 2: Time & Events |
| 12.3 | Appendix 3: Assessment Windows |
| 12.4 | Appendix 4: Treatment States and Phases |
| 12.5 | Appendix 5: Data Display Standards & Handling Conventions |
| 12.6 | Appendix 6: Derived and Transformed Data |
| 12.7 | Appendix 7: Premature Withdrawals & Handling of Missing Data |
| 12.8 | Appendix 8: Values of Potential Clinical Importance |
| 12.9 | Appendix 9: Multicenter Studies |
| 12.10 | Appendix 10: Examination of Covariates, Subgroups & Other Strata |
| 12.11 | Appendix 11: Multiple Comparisons & Multiplicity |
| 12.12 | Appendix 12: Model Checking and Diagnostics for Statistical Analyses |
| 12.13 | Appendix 13: Blinding Strategy |
| 12.14 | Appendix 14: Abbreviations & Trade Marks |
| 12.15 | Appendix 15: List of Data Displays |
| 12.16 | Appendix 16: Example Mock Shells for Data Displays |

# 7. STUDY POPULATION ANALYSES

# 7.1. Overview of Planned Analyses

The study population analyses will be based on the ITT population, unless otherwise specified.

Table 4 provides an overview of the planned study population analyses, with full details of data displays being presented in Appendix 15: List of Data Displays.

Table 4 Overview of Planned Study Population Analyses

| Display Type | Data | rated | |
|---|---|---|---|
| | Table | Figure | Listing |
| Subject Disposition | | <u> </u> | |
| Subject Populations | <b>Y</b> [1] | | Υ |
| Inclusion/exclusion Criteria Failures for Subjects Not | <b>Y</b> [1] | | |
| Starting Treatment | • | | |
| End of Study Record | <b>Y</b> [2] | | Υ |
| Attendance at Each Clinic Visit and Phone Call Visit | Υ | | |
| Number of Subjects by Country and Centre | <b>Y</b> [2,3] | | |
| Randomised and Actual Treatments | | | Υ |
| Protocol Deviations | | | |
| Deviations from the Inclusion/Exclusion Criteria | Υ | | Υ |
| Important Protocol Deviations | Υ | | Υ |
| Important Protocol Deviations Resulting in Exclusion from | Υ | | Υ |
| the PP Population | ī | | T |
| Treatment Misallocations | | | Υ |
| Demographic and Baseline Characteristics | | | |
| Demographic Characteristics | <b>Y</b> [2,4] | | Υ |
| Race and Racial Combinations | Υ | | Υ |
| Race and Racial Combinations Details | Υ | | |
| Current and Past Medical Conditions | Υ | | |
| Asthma Duration at Baseline | <b>Y</b> [2] | | Υ |
| Asthma Exacerbation History at Baseline | <b>Y</b> [2] | | Y |
| Lung Function at Baseline | Υ | | |
| Smoking History at Baseline | <b>Y</b> [2] | | Y |
| Concomitant Medications | | | |
| Pre-Treatment Concomitant Medications | Υ | | Υ |
| On-Treatment Concomitant Medications | Υ | | Υ |
| On-Treatment Asthma Concomitant Medications | Υ | | |
| Relationship between Ingredient and Verbatim Text | | | Y |
| Exposure and Medication Modifications | | | |
| Study Medication Dosage Modification | Υ | | |
| Extent of Exposure to Study Medication (Regardless of | V | Υ | Υ |
| Modification to Study Medication Dosage) | Υ | Y | Y |
| Extent of Exposure to Study Medication (up to First | V | | |
| Modification of Study Medication Dosage) | Υ | | |
| Extent of Exposure to Study Medication by Medication and | Υ | | |
| Dosage | Y | | |
| Number of Subjects by Subgroup | Υ | | |

#### NOTES:

- Y = Yes display generated.
- [1] Display will be based on ASE population
- [2] Display will be repeated for the PP population
- [3] Display will be repeated for the ASE population
- [4] Display will be repeated for the Safety population

# 8. PRIMARY STATISTICAL ANALYSES

# 8.1. Efficacy Analyses

## 8.1.1. Overview of Planned Efficacy Analyses

The primary efficacy analyses will be based on the ITT population and repeated for the PP population, unless otherwise specified.

Table 5 provides an overview of the planned efficacy analyses, with full details of data displays being presented in: List of Data Displays.

Table 5 Overview of Planned Efficacy Analyses

| Endpoint | Data displays generated | | | | | | |
|---|---|---|---|---|---|---|---|
| | St | Stats Analysis Summary Individual | | | | | |
| | T | F | L | T | F | F | L |
| ACT Total Score | | | | | | | |
| Change from Baseline | Y[1,2,3,4,5,6, | | | <b>Y</b> [1,2,3,4,5,7] | <b>Y</b> [1] | | Y[8] |
| in the ACT Total Score | 7] | | | | | | |
| at Week 12 (Visit 4) | | | | | | | |

#### NOTES:

- T = Table, F = Figure, L = Listing, Y = Yes display generated.
- Stats Analysis = Represents TFL related to any formal statistical analyses (i.e. modelling) conducted.
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.
- Display will be repeated for the following subgroups (ITT only) (see Section 12.10 for more details):
  - [1]: Country
  - [2]: Number of severe asthma exacerbations in the previous year prior to randomisation
  - [3]: Smoking status at baseline
  - [4]: Age group
  - [5]: Gender
- [6] Sensitivity analyses will be produced for the following approaches:
  - Last observation carried forward (LOCF) (ITT only)
  - MI analyses utilizing covariates (ITT only)
  - Semi-parametric Hodges-Lehmann (HL) approach (ITT only)
  - Worst observation carried forward (WOCF) for treatment withdrawals (ITT only)
  - Adjusting for seasonal effect
- [7] Display will be repeated for:
  - FF/VI versus the subset of Usual ICS/LABA subjects prescribed FP/S at randomisation (only if ≥25% of Usual ICS/LABA patients are prescribed FP/S at randomisation)
  - FF/VI versus the subset of Usual ICS/LABA subjects prescribed BUD/F at randomisation (only if ≥25% of Usual ICS/LABA patients are prescribed BUD/F at randomisation)
- [8] Display will be produced for the ITT population only.

# 8.1.2. Planned Efficacy Statistical Analyses

## **Primary Statistical Analyses**

## Endpoint(s)

Change from Baseline in the ACT Total Score at Week 12 (Visit 4)

#### **Model Specification**

- The primary endpoint will be performed on both the ITT and the PP populations, and analysed using an MMRM model utilizing the REML estimation approach and a default covariance structure of unstructured
- Terms fitted in the model will include:

Response : Change from Baseline in ACT Total Score

Fixed Categorical : Randomised treatment, visit (Week 6 and Week 12), gender, country

Fixed Continuous : Baseline ACT total score, age

Interaction terms : Randomised treatment-by-visit, baseline ACT total score-by-visit

Random effect : Subject

# SAS Code to Perform Analysis

```
proc mixed data=input_data;
```

class trtcd gender country visit subjid;

model ACT = trtcd gender country age baseline

visit visit\*baseline visit\*trtcd / ddfm=kr;

repeated visit / subject=subjid type=un;

random intercept / subject=subjid;

Ismeans visit\*trtcd / cl diff e om=OMdset at (baseline age)=(&blm. &agem.);

run ;

where OMdset is a dataset with a row for every visit-subject combination that contains all of the covariates and blm and agem are macro variables containing the means for baseline and age for the subjects used in the analysis. These are used to derive the adjusted means using coefficients which are based on the subjects used in the analysis.

#### **Model Checking & Diagnostics**

• Refer to Appendix 12: Model Checking and Diagnostics for Statistical Analyses.

### **Model Results Presentation**

- For Week 12 (Visit 4), the adjusted (least squares [LS]) mean change from baseline for each treatment and the estimated treatment difference for FF/VI versus Usual ICS/LABA (i.e. the difference in LS mean change from baseline) will be presented together with the associated 95% CI and p-value.
- Summary statistics will be produced for absolute value of and change from baseline in ACT total score at each post-baseline visit (Week 6 [Visit 3], Week 12 [Visit 4], Week 18 [Visit 5] and Week 24 [Visit 6]).
- A listing of ACT total and change from baseline scores will be provided.
- Mean ACT total score ± SD will be plotted by visit.

#### **Subgroup Analyses**

- For the analyses by country (France, Germany) and gender (male, female), the model will additionally
  include the randomised treatment-by-subgroup and randomised treatment-by-subgroup-by-visit
  interactions as a covariate.
  - For the analyses by number of severe asthma exacerbations in the previous year prior to randomisation (0, >1) and smoking status at baseline (Current smoker, Former smoker and Never smoked), the model will additionally include the subgroup, randomised treatment-by-subgroup interaction and randomised treatment-by-subgroup-by-visit interaction as covariates.
- For the analysis by age group (≤50 years, >50 years), the continuous covariate age will be replaced by age group, randomised treatment-by-age group interaction and randomised treatment-by-age group-by-visit interaction.

## **Sensitivity and Supportive Statistical Analyses**

## **Justification for Sensitivity Analyses Handling Missing Data**

• While subjects missing Week 12 (Visit 4) data but having earlier data will be included in the MMRM primary analysis, the interpretability of the results from the primary model will depend on the missing data satisfying the Missing at Random (MAR) assumption. To support the validity of the conclusions drawn from this analysis, several sensitivity analyses will be performed to explore the dropout pattern and its possible impact on treatment comparisons. These sensitivity analyses will be performed on the ITT population only.

#### **Last Observation Carried Forward**

• Missing values at Week 12 (Visit 4) will be replaced by the last available post-randomization value (either the Week 6 (Visit 2) ACT score or the ACT score at treatment withdrawal time, if applicable), i.e. based on the LOCF method. The change from baseline in ACT at Week 12 (Visit 4) will be analyzed using an analysis of covariance (ANCOVA) model adjusting for randomised treatment, baseline ACT score, gender, country and age. For Week 12 (Visit 4), the LS mean change from baseline for each treatment and estimated LS mean change from baseline difference for FF/VI versus Usual ICS/LABA will be presented together with the associated 95% CI and p-value.

# **Multiple Imputation**

- Sensitivity analyses will be performed using MI methods based on pattern mixture models. First, a
  repeated measures Normal model will be fitted to the data using a Bayesian approach, with noninformative priors for the mean and variance-covariance matrix to provide a joint posterior for the
  parameters in this model. The repeated measures Normal model will include separate mean profiles for
  each treatment group and the same covariates as those in the primary efficacy analysis.
- Independent samples will then be drawn from the posterior distributions for the mean and variance-covariance matrix to provide inputs into an imputation model. For each subject with missing data, these sampled values of the parameters for mean vectors and the variance-covariance matrices specify a joint distribution for their observed and unobserved outcome data.
- The post-withdrawal part of each pattern-specific distribution will be modelled using the approach discussed below. This imputation model will have the same covariates as those in the primary efficacy analysis.
- Based on this imputation model, a single set of data will be sampled for the missing data based on the
  distribution for the subject's missing data conditional upon their observed data. Each imputed data set
  will then be analysed using simple ANCOVA at Week 12 (Visit 4) and the resulting treatment
  differences and their standard errors combined using Rubin's rules.
- The post-withdrawal part of each pattern-specific distribution will be modelled using these two approaches:
  - MAR Approach. The means and variance-covariances following withdrawal are chosen to reflect the subject's own treatment group. This approach will provide similar results to using a mixed effects model where the unstructured covariance matrix is estimated separately for each arm, and all covariates are crossed with treatment. As such it is not truly a sensitivity analysis as we expect to get very similar results. Like the MMRM this answers an on-treatment question.
  - Copy Differences from Reference Approach. This approach addresses a potential pattern of informative missingness, in which subjects withdrawn from the test groups would have followed the same trend over time (difference in mean value between time-points) as those in the reference group, had they continued in the study. Therefore, this approach may be considered conservative because it will assume that following withdrawal from a test treatment arm, imputation for their missingness will be derived from observed reference data. The intention is to represent an ITT-like approach.
- For each method, the LS mean change from baseline at Week 12 (Visit 4) for each treatment and
  estimated LS mean change from baseline difference for FF/VI versus Usual ICS/LABA will be
  presented together with the associated 95% CI and p-value.

## **Sensitivity and Supportive Statistical Analyses**

#### **Hodges-Lehmann Approach**

 A sensitivity analysis based on the semi parametric HL approach will be proposed to assess the robustness of the MMRM Model-based non-inferiority results. The HL difference between groups at Week 12 (Visit 4) and corresponding 95% CI will be provided.

#### **Worst Observation Carried Forward**

• When treatment withdrawal occurs, an alternative method for imputing the missing value at the nearest visit after withdrawal time will be proposed: the primary endpoint missing value will be estimated by the worst ACT score observed between baseline visit and withdrawal time, inclusive – i.e. using the WOCF method. An ANCOVA model adjusting for randomised treatment, baseline ACT score, gender, country and age will be used to analyse this imputed data, with the LS mean change from baseline for each treatment presented at Week 12 (Visit 4) together with the estimated LS mean change from baseline difference and associated 95% CI

# **Summary of Sensitivity Statistical Analyses**

 A plot will be produced displaying the treatment differences and 95% CIs for the primary analysis and each of the sensitivity analyses described above.

#### Seasonal effect

A sensitivity analysis adjusting for seasonal effect will be performed by repeating the primary efficacy analysis with the addition of season at randomisation, season-by-visit, randomised treatment-by-season at randomisation interaction and randomised treatment-by-season at randomisation-by-visit interaction. See Section 12.10.3 for the definition of season at randomisation. The LS mean change from baseline at Week 12 (Visit 4) for each treatment and estimated LS mean change from baseline difference will be displayed for each season at randomisation together with the associated 95% CI and p-value, and the interaction p-value.

# 9. SECONDARY STATISTICAL ANALYSES

# 9.1. Efficacy Analyses

# 9.1.1. Overview of Planned Efficacy Analyses

The secondary efficacy analyses will be based on the ITT population, unless specified otherwise.

Table 6 provides an overview of the planned efficacy analyses, with further details of data displays being presented in Appendix 15: List of Data Displays.

Table 6 Overview of Planned Efficacy Analyses

| Endpoint | Data displays generated | | | | | | |
|---|---|---|---|---|---|---|---|
| • | St | Stats Analysis Summary | | Indiv | ridual | | |
| | T | F | L | T | F | F | L |
| ACT Total Score | | | | | | | |
| Change from Baseline | Y[1,2,3,4] | Υ | | Y[1,2,4,5,6,7, | <b>Y</b> [1,2] | | |
| in the ACT Total Score | | | | 8] | | | |
| at Week 24 (Visit 4) | | | | | | | |
| Correct Use of Device | | | | | | | |
| Percentage of Subjects | <b>Y</b> [1] | | | Y[1] | | | Υ |
| with Correct Use of | | | | | | | |
| Inhaler Device at Week | | | | | | | |
| 12 (Visit 4) and at | | | | | | | |
| Week 24 (Visit 6) | | | | | | | |
| Independently of the | | | | | | | |
| Use at Week 12 (Visit | | | | | | | |
| 4) | | | | | | | |

#### NOTES:

- T = Table, F = Figure, L = Listing, Y = Yes display generated.
- Stats Analysis = Represents TFL related to any formal statistical analyses (i.e. modelling) conducted.
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.
- [1] Display will be repeated for the PP population
- [2] Display will be repeated by Country (ITT only)
- [3] Sensitivity analyses will be produced for the following approaches:
  - LOCF (ITT only)
  - MI analyses utilizing covariates (ITT only)
  - Semi-parametric HL approach (ITT only)
  - WOCF for treatment withdrawals (ITT only)
  - Adjusting for seasonal effect
- [4] Display will be repeated for:
  - FF/VI versus the subset of Usual ICS/LABA subjects prescribed FP/S at randomisation (only if ≥25% of Usual ICS/LABA patients are prescribed FP/S at randomisation)
  - FF/VI versus the subset of Usual ICS/LABA subjects prescribed BUD/F at randomisation (only if ≥25% of Usual ICS/LABA patients are prescribed BUD/F at randomisation)
- Display will be repeated for the following subgroups (ITT only) (see Section 12.10 for more details):
  - [5]: Number of severe asthma exacerbations in the previous year prior to randomisation
  - [6]: Smoking status at baseline
  - [7]: Age group
  - [8]: Gender

# 9.1.2. Planned Efficacy Statistical Analyses

#### **Secondary Statistical Analyses**

## Endpoint(s)

Change from Baseline in the ACT Total Score at Week 24 (Visit 6)

#### **Model Specification**

 This endpoint will be performed on both the ITT and the PP populations, and analysed using an MMRM model utilizing the REML estimation approach and a default variance-covariance structure of unstructured

• Terms fitted in the model will include:

Response : Change from Baseline in ACT Total Score

Fixed Categorical: Randomised treatment, visit (Week 6, Week 12, Week 18 and Week 24),

gender, country

Fixed Continuous : Baseline ACT total score, age

Interaction terms : Randomised treatment-by-visit, baseline ACT total score-by-visit

Random effect : Subject

## **Model Checking & Diagnostics**

Refer to Appendix 12: Model Checking and Diagnostics for Statistical Analyses.

#### **Model Results Presentation**

- For Week 24 (Visit 6), the LS mean change from baseline for each treatment and the estimated difference in LS mean change from baseline for FF/VI versus Usual ICS/LABA will be presented together with the associated 95% CI and p-value.
- Summary statistics, a listing and plots of mean ACT total score  $\pm$  SD will be produced as part of the primary efficacy endpoint analysis (see Section 8.1.2).

## **Subgroup Analysis**

• For the analysis by country (France, Germany), the model will additionally include the randomised treatment-by-country, country-by-visit and randomised treatment-by-country-by-visit interactions as a covariate.

#### **Sensitivity and Supportive Statistical Analyses**

• The same sensitivity analyses as those described for the primary endpoint will be performed for the key secondary endpoint of change from baseline in the ACT total score at Week 24 (Visit 6).

#### **Secondary Statistical Analyses**

## Endpoint(s)

Percentage of subjects with correct use of inhaler device at Week 12 (Visit 4) and at Week 24 (Visit 6) independently of the use at Week 12 (Visit 4)

# **Model Specification**

- These endpoints will be analysed for both the ITT and the PP populations using logistic regression models
- Terms fitted in the model will include:
   Response : Endpoint

Fixed Categorical : Randomised treatment, correct use of inhaler device at baseline, gender,

country

Fixed Continuous : Age

# SAS Code to Perform Analysis

proc logistic data=input\_data plots=(all);

class trtcd country baseline gender / ref=first param=ref:

model corr\_use (event="Y") = trtcd baseline age gender country;

contrast "Trt\_effect" trtcd 1 / estimate=exp:

run;

# **Secondary Statistical Analyses**

# **Model Checking & Diagnostics**

Refer to Appendix 12: Model Checking and Diagnostics for Statistical Analyses.

# **Model Results Presentation**

- The number and percentage of subjects with correct use within each randomised treatment group will be presented by visit, together with the adjusted odds ratio comparing FF/VI with Usual ICS/LABA, associated p-value and 95% CI.
- A summary and listing of correct use / errors of inhaler use will be produced.

# 9.2. Safety Analyses

# 9.2.1. Overview of Planned Analyses

The safety analyses will be based on the Safety population.

Table 7 provides an overview of the planned analyses, with further details of data displays being presented in Appendix 15: List of Data Displays.

 Table 7
 Overview of Planned Safety Analyses

| Endpoint | Data displays generated | | | | | |
|---|---|---|---|---|---|---|
| · | Stats / | Analysis | | mary | | ridual |
| | Т | F | Т | F | F | L |
| Adverse Events | | | | | | |
| SAEs and ADRs Overview | | | Υ | | | |
| Non-Serious ADRs | | | Υ | | | Υ |
| Serious ADRs | | | Υ | | | |
| All ADRs | | | Υ | | | |
| SAEs | | | Υ | | | Υ |
| SAEs and ADRs Leading to Permanent | | | Υ | | | Υ |
| Discontinuation of Study Medication or | | | | | | |
| Withdrawal from Study | | | | | | |
| SAEs Leading to Permanent | | | Υ | | | |
| Discontinuation of Study Medication or | | | | | | |
| Withdrawal from Study | | | | | | |
| ADRs Leading to Permanent | | | Υ | | | |
| Discontinuation of Study Medication or | | | | | | |
| Withdrawal from Study | | | | | | |
| Non-Serious ADRs Leading to | | | | | | Y |
| Permanent Discontinuation of Study | | | | | | |
| Medication or Withdrawal from Study | | | | | | |
| Most Frequent Non-Serious ADRs, | | | Υ | | | |
| Reported by ≥1% or More of Subjects in | | | | | | |
| Any Treatment Group | | | | | | |
| Non-Serious ADRs of Special Interest | | | Y | | | |
| Serious ADRs of Special Interest | | | Y | | | |
| All ADRs of Special Interest | | | Y | | | |
| SAEs of Special Interest | | | Y | | | \ <u>'</u> |
| Fatal SAEs | | | Y | | | Y |
| Fatal Serious ADRs | | | Y | | | |
| Fatal SAEs of Special Interest | | | Y | | | |
| Non-Fatal SAEs | | | Y | | | Y |
| Non-Fatal SAEs of Special Interest | | | Υ | | | \ |
| AE terms of Special Interest | | | | | | Υ |
| Top Ten Most Commonly Reported On- | | | Υ | | | |
| treatment ADRs per Treatment Group | | | | | | <u> </u> |
| Vital Signs | | | \/ | | | |
| Vital Signs | | | Υ | | | Y |

| Endpoint | Data displays generated | | | | | |
|---|---|---|---|---|---|---|
| | Stats Analysis | | Summary | | Indiv | idual |
| | T | F | T | F | F | L |
| Inhaler Device Malfunctions | Inhaler Device Malfunctions | | | | | |
| Inhaler Device Malfunctions | | | | | | Y |
| Liver chemistry | | | | | | |
| Liver event | | | | | | Υ |
| Liver biopsy | | | | | | Υ |
| Liver imaging | | | | | | Υ |
| Other | | | | | | |
| Pregnancy | | | | | | Υ |

#### NOTES:

- T = Table, F = Figure, L = Listing, Y = Yes display generated.
- Stats Analysis = Represents TFL related to any formal statistical analyses (i.e. modelling) conducted.
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.

# 9.2.2. Benefit:Risk analyses

Benefit:Risk analyses will be based on the ITT population for Benefit, and Safety population for Risk.

Table 8 provides an overview of the planned analyses, with further details of data displays being presented in Appendix 15: List of Data Displays.

Table 8 Overview of Planned Benefit:Risk Analyses

| Endpoint | Data displays generated | | | | |
|---|---|---|---|---|---|
| | Stats Analysis | | Summary | | Individual |
| | T | F | T | F | L |
| Summary of Benefit:Risk | | Y | | | |

#### NOTES:

- T = Table, F = Figure, L = Listing, Y = Yes display generated.
- Stats Analysis = Represents TFL related to any formal statistical analyses (i.e. modelling) conducted.
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.

# **Benefit Risk Statistical Safety Analyses**

#### Endpoint(s)

 Summary of Benefit:Risk: various endpoints analyses in the context of safety and effectiveness analyses

## **Model Specification**

- Estimates and their 95% CIs obtained from selected safety and effectiveness analyses will be
  presented for the ITT population on a multiple panel forest plot which will display effectiveness and
  safety data.
- For certain endpoints, the x-axis may be reversed to ensure benefit/risk to either FF/VI or Usual ICS/LABA is shown accurately.
- Due to endpoints being presented using different scales, the forest plot will be split into additional panels to allow better visibility of the results.

## **Benefit Risk Statistical Safety Analyses**

#### **Model Checking & Diagnostics**

Model checking and diagnostics are described in each endpoint analysis section.

## **Model Results Presentation**

- The top panel ("Benefits") of the forest plot will display:
  - difference in LS mean change from baseline from the MMRM analysis of the primary efficacy endpoint, defined as the change from baseline in ACT total score at Week 12 (Visit 4), as described in Section 8.1.2
  - o difference in LS mean change from baseline from the MMRM analysis of the change from baseline in ACT total score at Week 24 (Visit 6), as described in Section 9.1.2
  - adjusted odds ratio from the logistic regression analysis of percentage of subjects with correct use of inhaler device at Week 12 (Visit 4), as described in Section 9.1.2
  - adjusted odds ratio from the logistic regression analysis of percentage of subjects with correct use of inhaler device at Week 24 (Visit 6) independently of the use at Week 12 (Visit 4), as described in Section 9.1.2
- The bottom panel ("Risks") of the forest plot will display the risk difference for FF/VI vs. usual ICS/LABA
  of the incidence of the following SAEs of special interest:
  - Asthma/bronchospasm, cardiovascular effects, decreased bone mineral density and associated fractures, hypersensitivity, local steroid effects, lower respiratory tract infection (LRTI) excluding pneumonia, pneumonia, adrenal suppression, ocular effects, effects on glucose, effects on potassium, tremor

# 10. OTHER STATISTICAL ANALYSES

# 10.1. Other Analyses

# 10.1.1. Overview of Planned Other Analyses

The other statistical analyses will be based on the ITT population, unless otherwise specified.

Table 9 provides an overview of the planned other analyses, with full details of data displays being presented in Appendix 15: List of Data Displays.

Table 9 Overview of Planned Other Analyses

| Endpoint | Absolute | | | | | | |
|---|---|---|---|---|---|---|---|
| | Stats Analysis | | | Sum | mary | Individual | |
| | Т | F | L | T | F | F | L |
| Trough (Pre-dose) FEV | | | | | | | |
| Change from Baseline | Y | | | Υ | | | Υ |
| in Trough (Pre-dose) | | | | | | | |
| FEV1 at Week 12 | | | | | | | |
| (Visit 4) | | | | | | | |
| ACT | | T | | | | | T |
| ACT Total Score ≥ 20 | Υ | | | Υ | Υ | | |
| or ≥ 3 Point Increase | | | | | | | |
| from Baseline in ACT | | | | | | | |
| Total Score at Week | | | | | | | |
| 12 (Visit 4) and Week | | | | | | | |
| 24 (Visit 6) | | | | | | | |
| ACT Total Score ≥ 20 | | | | Υ | Υ | | |
| at Week 12 (Visit 4) | | | | | | | |
| and Week 24 (Visit 6) | | | | | | | |
| ≥ 3 Point Increase | | | | Υ | Υ | | |
| from Baseline in ACT | | | | | | | |
| Total Score at Week | | | | | | | |
| 12 (Visit 4) and Week | | | | | | | |
| 24 (Visit 6) | | | | | | | |
| Change from Baseline | | | | Y | | | |
| in Individual ACT | | | | | | | |
| Questions at Week 12 | | | | | | | |
| (Visit 4) and Week 24 | | | | | | | |
| (Visit 6) | | | | | | | |
| Compliance with Study | Medication | | ı | T | 1 | 1 | T |
| Compliance with Study | | | | <b>Y</b> [1] | Υ | | Y |
| Medication from | | | | | | | |
| Randomisation (Day 0) | | | | | | | |
| to Week 12 (Visit 4), | | | | | | | |
| from Week 12 (Visit 4) | | | | | | | |
| to Week 24 (Visit 6) | | | | | | | |
| and from | | | | | | | |
| Randomisation (Day 0) | | | | | | | |
| to Week 24 (Visit 6) | | | | | | | |

| Endpoint | Absolute | | | | | | |
|---|---|---|---|---|---|---|---|
| • | Stats Analysis | | | Summary Individual | | | |
| | T | F | L | Т | F | F | L |
| MARS-A Score at | | | | <b>Y</b> [2] | <b>Y</b> [2] | | Υ |
| Randomisation (Day | | | | | | | |
| 0), Week 12 (Visit 4) | | | | | | | |
| and Week 24 (Visit 6). | | | | | | | |
| Severe asthma exacerb | ations | • | | • | | | |
| Number of Subjects | | | | <b>Y</b> [3] | | | Υ |
| With at Least 1 Severe | | | | | | | |
| Asthma Exacerbation | | | | | | | |
| and Number of Severe | | | | | | | |
| Asthma Exacerbations | | | | | | | |
| Annual Severe Asthma | Υ | Υ | | | | | |
| Exacerbation Rate | | | | | | | |
| over the Study Period | | | | | | | |
| Time to First Severe | Υ | Υ | | | | | |
| Asthma Exacerbation | | | | | | | |
| <b>Asthma Quality of Life</b> | Questionna | aire (AQLQIS | S1) | | | | |
| Change from Baseline | | | | Υ | | | Υ |
| in Total Score and | | | | - | | | • |
| Domain Scores of | | | | | | | |
| AQLQ(S) at Week 24 | | | | | | | |
| (Visit 6) | | | | | | | |
| An Increase from | Υ | | | Υ | | | |
| Baseline of ≥ 0.5 in | • | | | | | | |
| AQLQ(s) Total Score | | | | | | | |
| at Week 24 (Visit 6) | | | | | | | |
| An Increase from | Υ | | | Υ | | | |
| Baseline of ≥ 0.5 in | • | | | | | | |
| AQLQ(s) | | | | | | | |
| Environmental Stimuli | | | | | | | |
| Domain Score at Week | | | | | | | |
| 24 (Visit 6) | | | | | | | |
| An Increase from | | | | Y | | | |
| Baseline of ≥ 0.5 in | | | | | | | |
| AQLQ(S) Individual | | | | | | | |
| Domain Scores | | | | | | | |
| (Symptoms, Activity | | | | | | | |
| limitations and | | | | | | | |
| Emotional Function) at | | | | | | | |
| Week 24 (Visit 6) | | | | | | | |
| EQ-5D-5L | | 1 | l . | | | | |
| EQ-5D-5L Descriptive | Y | | | Υ | | | Υ |
| System Dimensions at | • | | | | | | • |
| Week 24 (Visit 6) | | | | | | | |
| EQ-5D-5L Utility Score | Υ | | | Υ | | | Υ |
| at Week 24 (Visit 6) | | | | | | | |
| EQ-5D-5L Visual | Υ | | | Υ | | | Υ |
| Analogue Scale (VAS) | ' | | | ' | | | ' |
| Score at Week 24 | | | | | | | |
| (Visit 6) | | | | | | | |
| (*1010) | | 1 | 1 | 1 | <u> </u> | | |

| Endpoint | Absolute | | | | | | |
|-------------------|----------------|---|---|---------|---|------------|---|
| | Stats Analysis | | | Summary | | Individual | |
| | T | F | L | T | F | F | L |
| PASAP-Q | | | | | | | |
| PASAP-Q Scores at | | | | Υ | | | Υ |
| Week 12 (Visit 4) | | | | | | | |

#### NOTES:

- T = Table, F = Figure, L = Listing, Y = Yes display generated.
- Stats Analysis = Represents TFL related to any formal statistical analyses (i.e. modelling) conducted.
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.
- [1] Display will be repeated for the PP population
- [2] A reminder was sent to centres in France instructing that the MARS-A questionnaire refers to the patient's preventer inhaler (i.e. their maintenance therapy prior to entering the study, and study medication while on-study). See Section 12.6.3 for further details. Display will be repeated split by:
  - Patients in France, all MARS-A assessments completed pre-reminder
  - Patients in France, some MARS-A assessments completed pre-reminder, some post-reminder
  - Patients in France, all MARS-A assessments completed post-reminder
  - Patients in Germany
- [3] Display will be repeated by season.

# 10.1.2. Planned Other Statistical Analyses

#### **Other Statistical Analyses**

#### Endpoint(s)

- Change from baseline in trough (pre-dose) FEV1 at Week 12 (Visit 4)
- Change from baseline in EQ-5D-5L Utility Score at Week 24 (Visit 6)
- Change from baseline in EQ-5D-5L VAS Score at Week 24 (Visit 6)

## **Model Specification**

- These endpoints will be analysed for the ITT population using ANCOVA models
- Terms fitted in the model will include:

Response : Endpoint

Fixed Categorical : Randomised treatment, gender, country

Fixed Continuous FEV1 endpoint: Baseline trough (pre-dose) FEV1 and age

EQ-5D-5L Utility Score endpoint: Baseline EQ-5D-5L Utility Score

and age

EQ-5D-5L VAS Score endpoint: Baseline EQ-5D-5L VAS Score

and age

#### **Model Checking & Diagnostics**

• Refer to Appendix 12: Model Checking and Diagnostics for Statistical Analyses.

# SAS Code to Perform Analysis

proc mixed data=input\_data;

class trtcd gender country;

model FEV1 = trtcd gender country age baseline / ddfm=kr;

Ismeans trtcd / cl diff e;

run ;

#### **Model Results Presentation**

- The LS mean change from baseline for each treatment and the difference in estimated LS mean change from baseline for FF/VI versus Usual ICS/LABA will be presented together with the associated 95% CI and p-value.
- Summary statistics.
- Listings will be provided.

## **Other Statistical Analyses**

#### Endpoint(s)

- Percentage of subjects who had either an ACT total score ≥ 20 or ≥ 3 point increase from baseline in ACT total score at Week 12 (Visit 4) and Week 24 (Visit 6)
- Percentage of subjects who have an increase from baseline of ≥ 0.5 in AQLQ(S) total score at Week 24 (Visit 6)
- Percentage of subjects who have an increase from baseline of ≥ 0.5 in AQLQ(S) environmental stimuli domain score at Week 24 (Visit 6)
- Percentage of subjects with 'no problems' in each dimension of the EQ-5D-5L questionnaire at Week 24 (Visit 6)

# **Model Specification**

- These endpoints will be analysed for the ITT population using logistic regression models
- Terms fitted in the model will include:

Response : Endpoint

Fixed Categorical : Randomised treatment, gender, country

Fixed Continuous ACT endpoints: Baseline ACT total score, baseline ACT total

score squared and age

AQLQ(S) endpoints: Baseline AQLQ(S) score and age

EQ-5D-5L endpoints: Baseline EQ-5D-5L dimension score and

age

## **Model Checking & Diagnostics**

Refer to Appendix 12: Model Checking and Diagnostics for Statistical Analyses.

#### **Model Results Presentation**

- The number and percentage of subjects with a response within each randomised treatment group will be presented by visit, together with the adjusted odds ratio comparing FF/VI with Usual ICS/LABA, associated 95% CIs and p-values.
- The number and percentage of subjects with ACT total score ≥20 or ≥3 point increase from baseline in ACT total score will be summarized by visit to include the tabulations of frequencies together and separately.
- The number and percentage of subjects with an increase from baseline of ≥ 0.5 in AQLQ(S) total and
  individual domain scores at Week 24 (Visit 6) will be summarized.
- The responses to each EQ-5D-5L dimension will be descriptively summarised

#### **Other Statistical Analyses**

#### Endpoint(s)

• Annual severe asthma exacerbation rate over the study period

#### **Model Specification**

- This endpoint will be analysed for the ITT population using a generalised linear model (GLM), assuming the Negative Binomial distribution
- Terms fitted in the model will include:

Response : Annual severe asthma exacerbation rate over the study period

Fixed Categorical : Randomised treatment, gender, country, number of severe

asthma exacerbations in the previous year prior to randomisation

(0, ≥1)

Fixed Continuous : Age

Offset variable : Logarithm of time on treatment

## **Model Checking & Diagnostics**

Refer to Appendix 12: Model Checking and Diagnostics for Statistical Analyses.

### **Other Statistical Analyses**

#### **SAS Code to Perform Analysis**

proc genmod data=input\_data;

class trtcd gender country;

model no\_exac = trtcd exacbl gender country age / dist=negbin link=log offset=log\_tm type3; lsmeans trtcd /cl diff=control("0") om exp;

run:

## **Model Results Presentation**

- The LS mean number / annual rate, adjusted treatment ratio and associated 95% CI and p-value will be presented.
- Percentage reduction in mean number / annual rate and associated 95% CI will also be presented.
- The severe asthma exacerbation data will be summarized to include the tabulations of exacerbation frequencies, exacerbation duration (days) and the outcome, the prescription of oral corticosteroids and/or antibiotics to treat exacerbations, hospitalisations and emergency department visits due to an exacerbation, intubations due to an exacerbation and withdrawal of IP or withdrawal from the study as a result of an exacerbation.
- A listing of severe exacerbations will be provided.
- Box plots will be provided for the severe annual exacerbation rates.

### **Other Statistical Analyses**

## Endpoint(s)

Time to first severe asthma exacerbation

## **Model Specification**

- The cumulative distribution of this endpoint will be illustrated for the ITT population using Kaplan-Meier estimates and evaluated using the Wald Chi-Square test based on a Cox proportional hazards model.
- The analyses and summaries will include on-treatment exacerbations, from start date of exposure to min(stop date of exposure + 1 day, date of study discontinuation).
- The exact method for handling ties in times will be used.
- Terms fitted in the model will include:

Response : Time to first severe asthma exacerbation Fixed Categorical : Randomised treatment, gender, country

Fixed Continuous : Age

## **Model Checking & Diagnostics**

• Refer to Appendix 12: Model Checking and Diagnostics for Statistical Analyses.

#### **Model Results Presentation**

- The hazard ratio for FF/VI versus Usual ICS/LABA with associated 95% CI and p-value will be presented.
- Cumulative incidence curves of time to first severe asthma exacerbation will be presented.
- Summary statistics will also be presented.
#### 11. REFERENCES

Devlin N., Shah K., Feng Y., Mulhern B., Van Hou, B. Valuing Health-Related Quality of Life: An EQ-5D-5L Value Set for England. Office of Health Economics. January 2016.

Efron, B. The Efficiency of Cox's Likelihood Function for Censored Data. J Am Stat Assoc. 1977;72:557–565.

EuroQol. EQ-5D-3L User Guide. EuroQol, Europe: 2013. Version 5.

Firth D. Bias Reduction of Maximum Likelihood Estimates. Biometrika. 1993;80:27–38.

GINA 2012, http://www.ginasthma.org/local/uploads/files/GINA Report March13.pdf

GlaxoSmithKline Document Number 2011N129785\_02 Study ID HZA115150. A 12-month, open label, randomised, effectiveness study to evaluate fluticasone furoate (FF, GW685698)/vilanterol (VI, GW642444) Inhalation Powder delivered once daily via a Novel Dry Powder Inhaler compared with usual maintenance therapy in subjects with Asthma. Report Date 11-Mar-2014.

GlaxoSmithKline Document number 2014N190259\_02 Study HZA116492: A 6-month, open label, randomised, efficacy study to evaluate fluticasone furoate (FF, GW685698)/vilanterol (VI, GW642444) Inhalation Powder delivered once daily via the Dry Powder Inhaler Ellipta<sup>TM</sup> compared with usual ICS/LABA maintenance therapy delivered by Dry Powder Inhaler in subjects with Persistent Asthma. Report Date 28-APR-2016

Juniper E.F., Guyatt G.H, Ferrie P.J., Griffith L.E. Measuring quality of life in asthma. Am Rev Respir Dis. 1993;147:832–838.

Kozma C.M., Slaton T.L., Monz B.U., Hodder R., Reese P.R. Development and Validation of a Patient Satisfaction and Preference Questionnaire for Inhalation Devices (PASAPQ). Treat Respir Med. 2005; 4 (1): 41-52.

Schatz M., Kosinski M., Yarlas A.S., Hanlon J., Watson M.E., Jhingran P. The minimally important difference of the Asthma Control Test. J Allergy Clin Immunol. 2009;124(4):719–23.

# 12. APPENDICES

| Section | Appendix |
|---|---|
| RAP Section 5: | RAP Section 5 : Analysis Populations |
| Section 12.1 | Appendix 1: Protocol Deviation Management and Definitions for PP Population |
| RAP Section 6: | RAP Section 6 : General Considerations for Data Analyses & Data Handling Conventions |
| Section 12.2 | Appendix 2: Time & Events |
| Section 12.3 | Appendix 3: Assessment Windows |
| Section 12.4 | Appendix 4: Treatment States and Phases |
| Section 12.5 | Appendix 5: Data Display Standards & Handling Conventions |
| Section 12.6 | Appendix 6: Derived and Transformed Data |
| Section 12.7 | Appendix 7: Premature Withdrawals & Handling of Missing Data |
| Section 12.8 | Appendix 8: Values of Potential Clinical Importance |
| Section 12.9 | Appendix 9: Multicenter Studies |
| Section 12.10 | Appendix 10: Examination of Covariates, Subgroups & Other Strata |
| Section 12.11 | Appendix 11: Multiple Comparisons & Multiplicity |
| Section 12.12 | Appendix 12: Model Checking and Diagnostics for Statistical Analyses |
| Other RAP Appe | ndices |
| Section 12.13 | Appendix 13: Blinding Strategy |
| Section 12.14 | Appendix 14: Abbreviations & Trade Marks |
| Section 12.15 | Appendix 15: List of Data Displays |
| Section 12.16 | Appendix 16: Example Mock Shells for Data Displays |

# 12.1. Appendix 1: Protocol Deviation Management and Definitions for PP Population

#### 12.1.1. Protocol Deviations

All PDs (any deviation from the protocol) are tracked and monitored during the study. Important PDs are those deviations that may compromise subject rights, safety, or well-being, and/or data integrity, and/or study end-points, and are defined in the PDMP. Apart from any incorrect treatment deviations, all protocol deviations will be agreed upon prior the unblinding and the freezing of the database. All deviations from the inclusion/exclusion criteria, and important PDs will be summarised. A listing of treatment misallocations will be produced.

#### 12.1.2. Exclusions from PP Population

**Important** PDs that will result in exclusion from the PP population are specified in Table 10, and will be summarised in a data display.

Table 10 PDs resulting in exclusion from the PP population

| <b>Deviation Category</b> | <b>Deviation Subcategory</b> |
|---|---|
| Informed consent | <ul> <li>Signed informed consent/assent not available on site<sup>[1]</sup></li> <li>Wrong informed consent/assent version signed<sup>[1]</sup></li> </ul> |
| | <ul> <li>Informed consent/assent not signed and/or dated by<br/>subject (parent/Legally Acceptable representative, if<br/>applicable)</li> </ul> |
| | • Informed consent/assent not signed and/or dated by appropriate site staff. [1] |
| | • Informed consent/assent not signed prior to any study procedure <sup>[1]</sup> |
| | Other informed consent/assent deviations <sup>[1]</sup> |
| Eligibility criteria not met – | Informed consent |
| inclusion criteria | • Gender and Age <sup>[2]</sup> |
| | Type of subject |
| | Current Asthma Therapy |
| | <ul> <li>Inability of subject to complete questionnaires</li> </ul> |
| Eligibility criteria not met – | History of Life-threatening asthma |
| exclusion criteria | Subjects having a severe and unstable asthma |
| | COPD Respiratory Disease |
| | • Other diseases/abnormalities <sup>[1]</sup> |
| | • Subjects with a history of adverse reaction to any |
| | intranasal, inhaled, or systemic corticosteroid and LABA |
| | therapy and to components of the inhalation powder <sup>[1]</sup> |
| | • Investigational Medications used within 30 days or five half-lives of prior study <sup>[1]</sup> |
| | Chronic user of systemic corticosteroids |
| | • Subjects treated by the monoclonal antibody omalizumab (Xolair) or mepolizumab (Nucala <sup>TM</sup> ) |
| | • Subjects involved in other clinical trials <sup>[1]</sup> |

| <b>Deviation Category</b> | Deviation Subcategory |
|---|---|
| Not withdrawn after developing | Not withdrawn from study <sup>[1]</sup> |
| withdrawal criteria | Not discontinued from study treatment <sup>[1]</sup> |
| | • Other deviation of not being withdrawn after developing withdrawal criteria <sup>[1]</sup> |
| Excluded medication, vaccine | • Medication, excluded by the protocol, was administered <sup>[3]</sup> |
| or device | • Other excluded medication, vaccine or device deviation <sup>[3]</sup> |
| Wrong study treatment / | Study treatment not administered per protocol <sup>[1]</sup> |
| administration / dose | Wrong study treatment or assignment administered |
| | Expired study treatment administered <sup>[1]</sup> |
| | Use of study treatment impacted by a temperature |
| | excursion which was not reported or approved or which was disapproved for further use. [1] |
| | • Study treatment not available at site for administration <sup>[1]</sup> |
| | Other deviations related to wrong study |
| | treatment/administration/dose <sup>[1]</sup> |
| Study procedures | Non study treatment supply procedures <sup>[1]</sup> |
| | Equipment procedures <sup>[1]</sup> |
| | Other deviations from study procedures <sup>[1]</sup> |

- [1] To be reviewed on a case-by-case basis[2] Patients < 18 years will be excluded from PP population, others will be reviewed on a case-</li> by-case basis
  [3] To be judged by the medical monitor

# 12.2. Appendix 2: Time & Events

# 12.2.1. Protocol Defined Time & Events

| Study Visits | Visit 1*<br>Screening | Visit 2*<br>Randomisation | Visit 3<br>Phone<br>call 1 | Visit<br>4** | Visit 5<br>Phone<br>call 2 | Visit 6 | Early<br>Withdrawal |
|---|---|---|---|---|---|---|---|
| Study Week (± | Day -7 to - | Day 0 | Week | Week | Week | Week | Early |
| specified no. of | 1 | - | 6 (±3 | 12 | 18 (±3 | 24 | Withdrawal |
| days) | | | days) | (±7 | days) | (±14 | |
| | | | | days) | | days) | |
| Visit | X | X | | X | | X | X |
| Phone interview | | | X | | Х | | |
| Assessments | | | | | | | |
| Informed Consent | х | | | | | | |
| Eligibility criteria | х | х | | | | | |
| Demography | х | | | | | | |
| Smoking status | х | | | | | | |
| Medical/Family history | Х | | | | | | |
| of consented subjects | | | | | | | |
| including CV Risk | | | | | | | |
| factors and | | | | | | | |
| exacerbation history | | | | | | | |
| PGx (saliva sample)*** | | X | | | | | |
| Physical examination | x | X | | X | | X | X |
| Safety Assessments | | | | | | | |
| Urine Pregnancy<br>Test¥ | | X | | X | | X | X |
| Exacerbation | | Х | х | х | х | х | х |
| Assessment | | | | | | | |
| Vital signs | х | Х | | Х | | X | X |
| Serious Adverse Event | | X | Х | Х | Х | Х | X |
| and Adverse Drug | | | | | | | |
| Reaction Assessment <sup>1</sup> | | | | | | | |
| Efficacy | | | | | | | |
| Assessments | | | | | | | |
| Spirometry Testing | | x | | X | | | x **** |
| (Pre-dose trough | | | | | | | |
| FEV1) | | | | | | | |
| Subject | | | | | | | |
| Questionnaires | | | | | | | |
| Asthma Control Test | X | X | X | X | X | X | Х |
| EQ-5D | | X | | | | X | Х |
| Asthma Quality of | | X | | | | X | х |
| Life Questionnaire | | | | | | | |
| MARS-A questionnaire | | X | | X | | X | X |
| Patient Satisfaction | | | | X | | | х |
| and Preference | | | | | | | |

| Study Visits | Visit 1*<br>Screening | Visit 2*<br>Randomisation | Visit 3<br>Phone<br>call 1 | Visit<br>4** | Visit 5<br>Phone<br>call 2 | Visit 6 | Early<br>Withdrawal |
|---|---|---|---|---|---|---|---|
| Study Week (± specified no. of days) | Day -7 to -<br>1 | Day 0 | Week<br>6 (±3<br>days) | Week<br>12<br>(±7<br>days) | Week<br>18 (±3<br>days) | Week<br>24<br>(±14<br>days) | Early<br>Withdrawal |
| Visit | X | X | | X | | X | X |
| Phone interview | | | X | | X | | |
| (PASAP-Q) | | | | | | | |
| Inhaler correct use | | | | | | | |
| assessment | | | | | | | |
| Type A/overall errors record | | X | | X | | X | |
| Medication | | | | | | | |
| Assessments | | | | | | | |
| Concomitant<br>Medication<br>Assessment | х | X | | X | | X | X |
| Dispense Study<br>Medication <sup>2</sup> | | x | | X | | | |
| Collect Study<br>Medication <sup>2</sup> | | | | X | | X | X |
| RAMOS/eCRF | | | | | | | |
| RAMOS NG | | X | | X | | | |
| eCRF | X | X | X | X | X | X | X |

<sup>1.</sup> SAE and ADR monitoring will occur from Day 1. SAE related to study participation should begin from signing of informed consent form (ICF). An additional safety and ACT check is provided by phone at Week 6 and 18.

<sup>2.</sup> Throughout the study the study medication will be dispensed and collected by the investigator site.

<sup>\*</sup> Visit 1 and Visit 2 can be combined if the subject did not take his usual asthma medication before coming on site. Then this visit will be Randomisation (Day 0) and all baseline characteristics will be collected at this visit. Written Informed Consent must be obtained prior to initiation of study procedures or initiating changes in medications.

<sup>\*\*</sup> Visit 4 (Week 12) should be scheduled at the same time of day as Visit 2 (Randomisation visit).

<sup>\*\*\*</sup>PGx saliva sample collected at Visit 2 (Randomisation) or any scheduled clinic visit thereafter.

<sup>\*\*\*\*</sup> Only if early withdrawal occurs before Week 12.

<sup>¥</sup> Only for childbearing women.

# 12.3. Appendix 3: Assessment Windows

Clinic visits/phone calls are scheduled to take place as specified in the protocol. For the ACT and MARS-A questionnaires, measurements that are not within  $\pm 7$  days of the visit target day for Week 6 (Visit 3) and Week 18 (Visit 5), or  $\pm 14$  days for Week 12 (Visit 4) and Week 24 (Visit 6) will be excluded from the analyses. For EQ-5D-5L and AQLQ(S), measurements that are not within  $\pm 14$  days of the visit target day of Week 24 (Visit 6) will be excluded from the summaries. For PASAP-Q, measurements that are not within  $\pm 14$  days of the visit target day of Week 12 (Visit 4) will be excluded from the summaries.

Table 11 Visit slotting rules for ACT and MARS-A

| Days relative to randomisation * | Target Study Day | Visit Slot |
|--------------------------------------|------------------|-------------------|
| 35 – 49 | 42 | Week 6 (Visit 3) |
| 70 – 98 | 84 | Week 12 (Visit 4) |
| 119 – 133 | 126 | Week 18 (Visit 5) |
| 154 – 182 | 168 | Week 24 (Visit 6) |
| * Date of assessment – Randomisation | date + 1 | |

Table 12 Visit slotting rules for EQ-5D-5L and AQLQ(S)

| Days relative to randomisation * | Target Study Day | Visit Slot |
|---|---|---|
| 154 – 182 | 168 | Week 24 (Visit 6) |
| * Date of assessment – Randomisation date + 1 | | |

Table 13 Visit slotting rules for PASAP-Q

| Days relative to randomisation * | Target Study Day | Visit Slot |
|---|---|---|
| 70 – 98 | 84 | Week 12 (Visit 4) |
| * Date of assessment – Randomisation date + 1 | | |

For all other endpoints, individual measurements collected outside of the assessment window for scheduled visits will be included in the ITT and PP analyses without adjustment.

All available data will be assigned to an assessment window where possible, including Early Withdrawal visits. If multiple measurements are collected within the same assessment window, the last valid value prior to randomisation will be used as the baseline value and the value closest to the target day for that window will be used for all post-randomisation visits. If values are the same distance from the target, then the earlier value will be taken.

# 12.4. Appendix 4: Treatment States and Phases

#### 12.4.1. Treatment Phases

In general, assessments and events will be classified according to the time of occurrence relative to study treatment, unless otherwise specified. Endpoint/measurement specific definitions are defined in Section 12.4.2.

| Treatment Phase | Definition |
|---|---|
| Pre-Treatment | Date < Study Treatment Start Date |
| On-Treatment | Study Treatment Start Date ≤ Date ≤ Study Treatment Stop Date + 1 |
| Post-Treatment | Date > Study Treatment Stop Date + 1 |

#### NOTES:

• If it is not possible to determine the treatment phase of an assessment or event, it will be considered as On-Treatment.

#### 12.4.2. Treatment States

Assessments and events will be classified according to time of occurrence relative to the start and/or stop date of the study treatment. The earliest and latest exposure treatment start and stop dates will be used to determine whether an assessment or event was pre-treatment, on-treatment or post-treatment. If it is not possible to tell whether an assessment or event was on-treatment or not, it will be considered as on-treatment.

#### 12.4.2.1. Treatment States for Concomitant Medications

| Treatment State | Definition |
|---|---|
| Pre-Treatment | (Start Date of Medication < Study Treatment Start Date) and (End Date of Medication < Study Treatment Start Date) |
| On-Treatment | [(Start Date of Medication < Study Treatment Start Date) and (End Date of Medication ≥ Study Treatment Start Date)] or (Study Treatment Start Date ≤ Start Date of Medication ≤ Study Treatment Stop Date + 1) |
| Post-Treatment | Start Date of Medication > Study Treatment Stop Date +1 |

# 12.4.2.2. Treatment States for Efficacy Measurements

| Treatment State | Definition |
|---|---|
| Pre-Treatment | Date of Measurement ≤ Study Treatment Start Date |
| On-Treatment | Study Treatment Start Date < Date of Measurement ≤ Study Treatment Stop Date + 1 |
| Post-Treatment | Date of Measurement > Study Treatment Stop Date +1 |

#### 12.4.2.3. Treatment States for Exacerbation Data

| Treatment State | Definition |
|---|---|
| Pre-Treatment | Exacerbation Onset Date < Study Treatment Start Date |
| On-Treatment | Study Treatment Start Date ≤ Exacerbation Onset Date ≤ Study Treatment Stop Date + 1 |
| Post-Treatment | Exacerbation Onset Date > Study Treatment Stop Date + 1 |

#### NOTES:

- If the study treatment stop date is missing, then the exacerbation will be considered to be On-Treatment
- See Section 12.6.3 for details on missing onset and/or resolution dates.

#### 12.4.2.4. Treatment States for AE Data

Treatment states for adverse events are described below. Severe asthma exacerbations will be treated in the same way, with the exacerbation start date used in place of the AE start date.

| Treatment State | Definition |
|---|---|
| Pre-Treatment | AE Onset Date < Study Treatment Start Date |
| On-Treatment | Study Treatment Start Date ≤ AE Onset Date ≤ Study Treatment Stop Date + 1 |
| Post-Treatment | AE Onset Date > Study Treatment Stop Date + 1 |
| Onset Time<br>Since 1st Dose<br>(Days) | If Study Treatment Start Date > AE Onset Date = AE Onset Date - Study Treatment Start Date If Study Treatment Start Date ≤ AE Onset Date = AE Onset Date - Study Treatment Start Date +1 Missing otherwise. |
| Duration (Days) | AE Resolution Date – AE Onset Date + 1 |
| Drug-related | If relationship is marked 'YES' or is missing on the AE case report form (CRF) page. |

#### NOTES:

• If the study treatment stop date is missing, then the AE will be considered to be On-Treatment.

# 12.5. Appendix 5: Data Display Standards & Handling Conventions

#### 12.5.1. Study Treatment & Sub-group Display Descriptors

| Treatment Group Descriptions | | | |
|---|---|---|---|
| RandAll NG Data Displays for Reporting | | | g |
| Code Description | | Description | Order [1] |
| А | Fluticasone furoate /vilanterol inhalation<br>Powder delivered once daily | FF/VI | 2 |
| В | Usual ICS/LABA maintenance therapy delivered by Dry Powder Inhaler | Usual ICS/LABA | 1 |

#### NOTES:

#### 12.5.2. Baseline Definition & Derivations

#### 12.5.2.1. Baseline Definitions

For all endpoints the baseline value will be the last assessment prior to randomisation.

#### 12.5.2.2. Derivations and Handling of Missing Baseline Data

| Definition | Reporting Details |
|---|---|
| Change from Baseline | = Post-Dose Visit Value – Baseline |
| % Change from Baseline | = 100 x [(Post-Dose Visit Value – Baseline) / Baseline] |
| Maximum Change from Baseline | = Calculate the change from baseline at each given timepoint and determine the maximum change |

#### NOTES:

- Unless otherwise specified, the baseline definitions specified in Section 12.5.2.1 will be used for derivations for endpoints / parameters and indicated on summaries and listings.
- Unless otherwise stated, if baseline data is missing no derivation will be performed and will be set to missing.
- The baseline definition will be footnoted on all change from baseline displays.

#### 12.5.3. Reporting Process & Standards

| Reporting Process | |
|---|---|
| Software | |
| The currently supported versions of SAS software will be used. | |
| Reporting Area | |
| HARP Server | : uk1salx00175 |
| HARP Area | : /arenv/arprod/gw685698_gw642444/hza116492/final |
| QC Spreadsheet : /arenv/arwork/gw685698_gw642444/hza116492/final/qc | |
| Analysis Datasets | |
| Analysis datasets will be created according to CDISC standards. | |

<sup>1.</sup> Order represents treatments being presented in data displays, as appropriate.

#### **Reporting Process**

 For creation of ADaM datasets (e.g. ADCM, ADAE) the same version of dictionary datasets will be implemented for conversion from SI to SDTM.

#### **Generation of RTF Files**

RTF files will be generated for all tables in the final reporting effort.

#### **Reporting Standards**

#### General

- The current GSK IDSL will be applied for reporting, unless otherwise stated:
  - 4.03 to 4.23: General Principles
  - 5.01 to 5.08: Principles Related to Data Listings
  - o 6.01 to 6.11: Principles Related to Summary Tables
  - 7.01 to 7.13: Principles Related to Graphics

#### **Formats**

- All data will be reported according to the treatment the subject was randomised to unless otherwise stated.
- GSK IDSL Statistical Principles (5.03 & 6.06.3) for decimal places (DPs) will be adopted for reporting of data based on the raw data collected.
- Numeric data will be reported at the precision collected on the electronic case report form (eCRF) or recorded in the raw dataset if from non eCRF sources.
- The reported precision from non eCRF sources will follow the IDSL statistical principles but may be adjusted to a clinically interpretable number of DP's.

#### **Planned and Actual Times**

- Reporting for tables, figures and formal statistical analyses:
  - Planned time relative to dosing will be used in figures, summaries, statistical analyses and calculation of any derived parameters, unless otherwise stated.
  - The impact of any major deviation from the planned assessment times and/or scheduled visit days
    on the analyses and interpretation of the results will be assessed as appropriate.
- Reporting for Data Listings:
  - Planned and actual time relative to study drug dosing will be shown in listings (Refer to IDSL Statistical Principle 5.05.1).
  - Unscheduled or unplanned readings will be presented within the subject's listings.
  - For visits outside the time-windows, please see Section 12.3.

#### **Unscheduled Visits**

- Unscheduled visits will not be included in summary tables or figures.
- All unscheduled visits will be included in listings.

#### **Descriptive Summary Statistics**

| Continuous Data Refer to IDSL Statistical Principle 6.06.1 | |
|---|---|
| Categorical Data | N, n, frequency, % |
| 0 11 101 1 | |

#### **Graphical Displays**

Refer to IDSL Statistical Principals 7.01 to 7.13.

# 12.6. Appendix 6: Derived and Transformed Data

#### 12.6.1. General

#### **Multiple Measurements at One Time Point**

- If there are multiples values within a time window the last valid value prior to randomisation will be used as the baseline value and the value closest to the target day for that window will be used for all post-randomisation visits. If values are the same distance from the target, then for efficacy outputs where visit slotting is used the earlier record will be used. For all other cases of multiple valid measurements the mean will be taken.
- Subjects having both High and Low values for Normal Ranges at any post-baseline visits for safety
  parameters will be counted in both the High and Low categories of "Any visit post-baseline" row of
  related summary tables. This will also be applicable to relevant Potential Clinical Importance summary
  tables.

## **Study Day**

- Calculated as the number of days from randomisation date:
  - Ref Date = Missing → Study Day = Missing
  - Ref Date < Randomisation Date → Study Day = Ref Date Randomisation Date
  - Ref Data ≥ Randomisation Date → Study Day = Ref Date (Randomisation Date) + 1

#### **Time Since First Dose**

- Calculated as the number of days from the date of first dose:
  - Ref Date = Missing → Time Since First Dose = Missing
  - Ref Date < First Dose Date → Time Since First Dose = Ref Date First Dose Date
  - Ref Date ≥ First Dose Date → Time Since First Dose = Ref Date (First Dose Date) + 1

#### Time Since Last Dose

- Calculated as the number of days from the date of last dose:
  - Ref Date = Missing → Time Since Last Dose = Missing
  - Ref Date < Last Dose Date → Time Since Last Dose = Ref Date Last Dose Date</li>
  - Ref Date ≥ Last Dose Date → Time Since Last Dose = Ref Date Last Dose Date) + 1

#### **Study Treatment Discontinuation**

• In this study, subjects who are intentionally and permanently withdrawn from study medication may not continue in the study attending the remaining visits (excluding the Follow-up contact) and completing the scheduled assessments.

#### 12.6.2. Study Population

#### **Demographics**

#### Age

- GSK standard IDSL algorithms will be used for calculating age where birth date will be imputed as follows:
  - Any subject with a missing day will have this imputed as day '15'.
  - Any subject with a missing date and month will have this imputed as '30th June'.
- Birth date will be presented in listings as 'YYYY'.
- Completely missing dates of birth will remain as missing, with no imputation applied. Consequently, the

#### **Demographics**

age of the subject will not be calculated and will remain missing.

• Age, in whole years, will be calculated with respect to the date of screening (Visit 1).

#### **Body Mass Index**

• Calculated as Weight (kg) / [Height (m)]<sup>2</sup>

#### Race

 In the demographic summary table race will be summarised as follows; White is defined as those subjects who chose only the White (Arabic/North African Heritage) and/or White (White/Caucasian/European Heritage) categories on the CRF, Black is defined as those subjects who chose only the African American/African Heritage category on the CRF, and Other is defined as those subjects who chose any of the other races on the CRF.

#### **Extent of Exposure**

Subjects for whom it is considered appropriate/necessary to adjust treatment can have their dose increased from the starting dose, and will be recorded in the eCRF. Treatment sequence identifier will be incremented by 1 each time the study medication is modified, and recorded on eCRF.

Extent of exposure will be presented in three different ways:

 The extent of exposure to study medication, regardless of study medication dosage modifications during the study, will be defined as the number of days on study medication and will be calculated for each subject as follows:

Exposure = (study medication stop date – study medication start date) + 1

If medication start date is missing, then the randomisation date (i.e. date of Visit 2) of the subject will be used for medication start date. If the medication stop date is missing, the Visit 6 date or early withdrawal visit date will be used instead. If all these dates are missing, then the extent of exposure will be set to missing.

- The extent of exposure to study medication, up to first study medication dosage modification
- The extent of exposure to each dose of study medication, presented separately for FF/VI 92 mcg/22 mcg, FF/VI 184 mcg/22mcg, FP/S 250 mcg/50 mcg, FP/S 500 mcg/50 mcg, BUD/F 200 mcg/6 mcg, BUD/F 400 mcg/12 mcg

Note: do not split by dose frequency

#### 12.6.3. **Efficacy**

#### **Primary Endpoint**

#### **ACT**

The ACT is a validated self-administered questionnaire utilising 5 questions to assess asthma control during the past 4 Weeks on a 5-point categorical scale (1 to 5).

By answering all 5 questions, a subject with asthma can obtain a score that may range between 5 and 25, with higher scores indicating better control. An ACT score of 5 to 19 suggests that the subject's asthma is unlikely to be well controlled. A score of 20 to 25 suggests that the subject's asthma is likely to be well controlled. The MID for ACT is 3 (Schatz, 2009).

#### **Primary Endpoint**

The total score is calculated as the sum of the scores from all 5 questions, provided all scores are non-missing; if any individual scores are missing then the overall score will be set to missing.

#### **Secondary Endpoint**

#### **Correct Use of Device**

Inhaler use will be assessed at Randomisation (Visit 2), Week 12 (Visit 4) and Week 24 (Visit 6). Correct use of device is defined as making no critical or non-critical errors.

#### **Critical and Non-Critical Errors for Ellipta**

#### Critical errors:

- Failed to open cover
- Shook the device upside down after dose preparation
- Exhaled directly into mouthpiece
- No seal by the lips around the mouthpiece during the inhalation

#### Non-critical errors:

- No exhalation before an inhalation
- Inhalation manoeuvre was not:
  - long
  - steady
  - deep
- Blocked air inlet during inhalation manoeuvre
- Did not hold breath
- Did not close the device (Note: this is an error but one which does not affect the medication that is inhaled)

#### Critical and Non-Critical Errors for Diskus

#### Critical errors:

- Failed to open cover
- Lever is not pushed back
- Shook the device after dose preparation
- Exhaled directly into mouthpiece
- No seal by the lips round the mouthpiece during the inhalation

#### Non-critical errors:

- No exhalation before an inhalation.
- Inhalation manoeuvre was not:
  - steady
  - deep
- Did not hold breath
- Did not close the device (Note: this is an error but one which does not affect the medication that is inhaled)

#### **Critical and Non-Critical Errors for Turbuhaler**

#### Critical errors:

- Failed to remove cap
- Did not hold device upright (±45° OK) during dose preparation
- Base not twisted fully backwards and forwards, no click heard

#### **Primary Endpoint**

- Shook the device after dose preparation
- Exhaled directly into mouthpiece
- No seal by the lips round the mouthpiece during the inhalation

#### Non-critical errors:

- Device tipped downwards after dose preparation
- No exhalation before an inhalation
- Inhalation manoeuvre was not:
  - forceful
  - deep
- Blocked air inlet during inhalation manoeuvre
- Did not hold breath
- Did not close the device (Note: this is an error but one which does not affect the medication that is inhaled)

#### Other Endpoints

#### FEV1

FEV1 will be measured to assess lung function at Randomisation (Visit 2) and Week 12 (Visit 4). Visit 4 should be scheduled at the same time of day as Visit 2, FEV1 measurements should be taken pre-dose and subjects should be instructed not to take their asthma medication/study drug prior to coming into the clinic at these visits. Subjects should also withhold from using their rescue medication for at least 4 hours prior to Visit 2 and Visit 4.

All sites will use standardised spirometry equipment provided by GSK. For each observation, at least 3 (with no more than 8) efforts will be obtained. At least two of the spirometry efforts should be acceptable and repeatable. The best FEV1 value will be recorded in the eCRF.

#### MARS-A

The MARS-A questionnaire is a 10-item questionnaire. The response to all ten questions will be presented and included in the calculation of the MARS-A 10-score.

The responses to the MARS-A questions will be scored as follows: Always=1, Often=2, Sometimes=3, Rarely=4, Never=5. The MARS-A 10-Score will be calculated for each subject as the sum of scores for each of the ten questions divided by the number of non-missing responses to the ten questions.

If some responses are missing the MARS-A 10-score is calculated as follows for each subject:

- If eight or more of the questions have been answered, the missing responses for that subject will be imputed to the average score
- If less than eight of the questions have been answered, the overall MARS-A 10-score for that subject will be set to missing

The French translation of the MARS-A questionnaire did not go through cognitive debriefing; therefore, while the study was ongoing it was determined that there is no word for "preventer" in French. "Preventer inhaler" was translated as "dispositif d'inhalation" (i.e., "inhalation device"). A reminder was sent to centres in France instructing that the MARS-A questionnaire refers to the patient's preventer inhaler (i.e. their maintenance therapy prior to entering the study, and study medication while on-study) as opposed to their reliever inhaler. The German translation went through cognitive debriefing and was correctly translated. The MARS-A data

#### **Other Endpoints**

displays will therefore be repeated split by:

- Patients in France, all MARS-A assessments completed pre-reminder
- Patients in France, some MARS-A assessments completed pre-reminder, some post-reminder
- Patients in France, all MARS-A assessments completed post-reminder
- Patients in Germany

The reminder was sent on 17OCT2016, and it was assumed that the centres started implementing the instructions two days after this, i.e. on 19OCT2016. If a visit occurs on the 19OCT2016 then it will be categorised as having happened before the reminder.

#### Severe Asthma Exacerbations

Missing onset or resolution dates will be handled as follows:

- Single event with missing onset and/or resolution dates:
  - (a) Missing onset date: set onset date = study treatment start date
  - (b) Missing resolution date: set resolution date = study treatment stop date
  - (c) Both missing: imputed per both (a) and (b)
- Multiple events, one event with some missing onset/resolution dates; on the assumption any partial date information does not occur during the other events:
  - (a) Missing onset date: set onset date = max[(resolution date of the nearest previous event) + 1 day, study treatment start date]
  - (b) Missing resolution date: set resolution date = min[(onset date of the nearest subsequent event) 1 day, study treatment stop date]
  - (c) Both missing: determine the largest gap between study treatment start date and first event onset date, between first event resolution date and next event(s) onset dates (if any), between last event resolution date and study treatment stop date. If there is more than one gap which is the largest, then take the first occurrence. Then impute as follows:

onset date = (onset date of largest gap) + 1 day resolution date = (resolution date of largest gap) + 1 day

#### **Time to First Severe Asthma Exacerbation**

The date of a severe asthma exacerbation is defined as the exacerbation onset date. Subjects who complete the study without a severe asthma exacerbation will be censored. Time to first severe asthma exacerbation is measured from the date of randomisation (i.e., study treatment start date) to the onset date of first severe asthma exacerbation, as recorded on eCRF, or study treatment stop date (Visit 6 or early withdrawal visit) for subject who complete the study without any severe asthma exacerbations (censored). Analyses of time to first severe asthma exacerbation will be censored at Day 168.

#### AQLQ(S) Domain and Total Scores

The AQLQ(S) contains 32 items in four domains: activity limitation (11 items), symptoms (12 items), emotional function (5 items) and environmental stimuli (4 items). The following items are included in each of the 4 domains:

Symptoms: 6, 8, 10, 12, 14, 16, 18, 20, 22, 24, 29, 30
Activity Limitation: 1, 2, 3, 4, 5, 11, 19, 25, 28, 31, 32

Emotional Function: 7, 13, 15, 21, 27Environmental Stimuli: 9, 17, 23, 26

The response format consists of a seven-point scale where a value of 1 indicates "total impairment" and a value of 7 indicates "no impairment". The total AQLQ(S) score is the mean of all 32 items in the questionnaire and each individual domain score is calculated as the mean of the items within that domain. Hence, the total and domain scores are also each defined on a range from 1 to 7 with higher scores

#### **Other Endpoints**

indicating a higher quality of life. The MID for AQLQ(S) is 0.5 (Juniper, 1993).

For the total AQLQ(S) score, the score for a subject at any time point will only be calculated if at least 90% of the questions were answered (calculated as the mean of those non-missing questions). If fewer than 90% of the questions were answered, then the mean score for that subject at that time point will be considered missing.

For each individual domain of the AQLQ(S) score, the score for a subject at any time point will only be calculated if at least 90% of the questions for that domain were answered (calculated as the mean of those non-missing questions). If fewer than 90% of the questions were answered for that domain, then the mean score for that subject and domain at that time point will be considered missing.

#### **EQ-5D-5L Utility and VAS Scores**

The EQ-5D-5L is administered at randomisation (Visit 2), Week 24 (Visit 6) and Early Withdrawal. The EQ-5D-5L consists of 2 parts: the EQ-5D-5L descriptive system and the EQ VAS.

The EQ-5D-5L descriptive system comprises the following 5 dimensions: Mobility, Self-Care, Usual Activities, Pain/Discomfort and Anxiety/Depression. Each dimension has 5 levels, where Level 1 (coded as '1') = 'No problems', Level 2 (coded as '2') = 'Slight problems', Level 3 (coded as '3') = 'Moderate problems', Level 4 (coded as '4') = 'Severe problems' and Level 5 (coded as '5') = 'Extreme problems'. Subjects indicate their health state for each dimension by ticking (or placing a cross) in the box of the most appropriate level for that dimension. Ambiguous values (e.g. 2 boxes are ticked for a single dimension) will be considered missing. Missing values will be coded as '9'. The responses (1, 2, 3, 4 or 5) to the five questions will be converted into a single utility score using the developer's instructions (EuroQol, 2013): the responses (1, 2, 3, 4 or 5) to the five questions in the descriptive system can be represented as one of 5'=3125 possible health states (11111, 11112, ..., 55555). These will be converted into a single summary index (y) that attaches value to each of the levels in each dimension by applying the formula below, which is based on the EQ-5D-5L value set for England (Devlin, 2016).

```
y = 1 - 0.9675 \times (0.051M_2 + 0.063M_3 + 0.212M_4 + 0.275M_5 + 0.057S_2 + 0.076S_3 + 0.181S_4 + 0.217S_5 + 0.051U_2 + 0.067U_3 + 0.174U_4 + 0.190U_5 + 0.060P_2 + 0.075P_3 + 0.276P_4 + 0.341P_5 + 0.079A_2 + 0.104A_3 + 0.296A_4 + 0.301A_5)
```

where variables with subscript n are indicator variables equal to 1 when the corresponding level for the dimension is 'n' and equal to 0 otherwise,  $M_m$  variables represent responses for the mobility domain,  $S_n$  variables represent responses for the self-care domain,  $U_n$  variables represent responses for the usual activities domain,  $P_n$  variables represent responses for the pain / discomfort domain, and  $A_n$  variables represent responses for the anxiety / depression domain.

For example, health state where domains MSUPA = 11223 would be equal to:

$$1 - 0.9675 \times (0.051 + 0.060 + 0.104) \approx 0.7920$$

The EQ VAS records the subject's self-rated health state on a vertical, VAS where 0='worst imaginable health state' and 100='best imaginable health state'. Subjects indicate their own health state by drawing a line from the box on the left of the scale to whichever point on the scale indicates how good or bad their own health state is that day. Ambiguous values (e.g. the line crosses the VAS twice) will be considered missing. Missing values will be coded as '999'.

Only validated EuroQoLs completed in the same language as that completed at Baseline (Visit 2) will be

#### **Other Endpoints**

summarised.

#### **PASAP-Q Domain and Total Scores**

The PASAP-Q is a self-administered 16-item questionnaire measuring satisfaction and preference with inhaler devices (Kozma, 2005). Two domains (performance and convenience) are calculated from 13 satisfaction items, measured on a Likert-type scale where a value of 1 indicates "very dissatisfied" and 7 indicates "very satisfied". The performance and convenience domains together form the total score. The other items include an overall satisfaction question (again measured from 1 to 7), a preference question (not applicable and so not asked for this study) and a question on willingness to continue using the device in the future, measured on a scale of 0 (not willing) to 100 (definitely willing).

The performance and convenience domains include the following items:

Performance: 1, 2, 3, 4, 5, 10, 11Convenience: 6, 7, 8, 9, 12, 13

If the patient completes at least half of the items in a domain, values for missing items are imputed using the mean of the completed items in that domain. The domain score is then transformed to a scale from 0 (least) to 100 (most) as follows:

Domain Score = [Mean(responses for items in domain) - 1] 
$$\times \frac{100}{6}$$

If the patient completes less than half of the items in a domain, then the missing items are not imputed and the domain score is set to missing. The total score can be calculated only when both domain scores are computable and substitution for missing items at the domain level has taken place, and is calculated on the same scale as:

Total Score = 
$$[Mean(responses for all 13 items) - 1] \times \frac{100}{6}$$

The overall satisfaction and willingness questions are summarised on their original scales of 1 to 7 and 0 to 100 respectively.

#### **Other Endpoints**

#### **Treatment Compliance**

Overall percentage treatment compliance for every subject will be calculated for each type of inhaler (Diskus, Turbuhaler and Ellipta) separately.

Compliance for Diskus, Turbuhaler and Ellipta will be based on the total number of inhalations taken from each type of inhaler and the expected number of inhalations to be taken. The expected number of inhalations will be derived as the sum over the number of days on study drug (based on the subject's treatment start and stop date for that type of inhaler) of the expected number of inhalations per day (from each inhaler). The total number of inhalations taken will be based on the dose counter for each type of inhaler, all of which are re-supplied during the study. If there is no dose counter information at all then the compliance will be missing; however, as long as the information from one dose counter is present, the compliance will be calculated assuming that all doses were taken for the missing inhalers. If a dose counter start count is missing, then it will be assumed to be 30 for Ellipta and 60 for both Diskus and Turbuhaler. In each calculation, all inhalers dispensed will be used, provided the dose counter stop counts are non-missing. The following formula will be used:

$$\frac{Total\_number\_of\_inhalations\_taken}{\sum_{i=1}^{n} Expected\_inhaltions\_for\_day_i} \times 100$$

#### Where:

- n = Stop\_date Start\_date + 1. Start\_date and Stop\_date are the earliest treatment start
  date and latest treatment stop date respectively recorded for all inhalers used during the time
  period.
- *Total\_number\_of\_inhalations\_taken* is the sum of (dose counter start count dose counter stop count) for all inhalers used during the time period
- Expected\_inhalations\_for\_day; is equal to 1 for Ellipta and 2 for Diskus and 2 or 4 for Turbuhaler for any given day, depending on the dose

#### 12.6.4. Safety

#### **SAEs of Special Interest**

SAE groups of special interest have been defined as SAEs which are included in specified areas of interest for one or more of the treatment groups (FF/VI, FF and/or VI). They are identified by groupings of preferred terms based on the Medical Dictionary for Regulatory Activities (MedDRA) dictionary version used in each reporting effort. Groupings or subgroups may be defined, based on relevant combination of preferred terms, or on Standardised MedDRA queries (SMQs).

SAEs of special interest will be confirmed prior to final data, based on the MedDRA version in use at the time.

| Special Interest SAE Group |
|---------------------------------------------------------|
| Asthma/bronchospasm |
| Cardiovascular effects |
| Decreased bone mineral density and associated fractures |
| Hypersensitivity |
| Local steroid effects |
| LRTI excluding pneumonia |
| Pneumonia |
| Adrenal suppression |
| Ocular effects |
| Effects on glucose |
| Effects on potassium |
| Tremor |

#### **Laboratory Parameters**

- If a laboratory value which is expected to have a numeric value for summary purposes, has a non-detectable level reported in the database, where the numeric value is missing, but typically a character value starting with '<x' or '>x' (or indicated as less than x or greater than x in the comment field) is present, the number of significant digits in the observed values will be used to determine how much to add or subtract in order to impute the corresponding numeric value.
  - Example 1: 2 Significant Digits = '< x ' becomes x 0.01</li>
  - Example 2: 1 Significant Digit = '> x' becomes x + 0.1
  - $\circ$  Example 3: 0 Significant Digits = '< x' becomes x 1

# 12.7. Appendix 7: Premature Withdrawals & Handling of Missing Data

#### 12.7.1. Premature Withdrawals

| Element | Reporting Detail |
|---|---|
| General | <ul> <li>Subject study completion was defined in the protocol as a subject who has completed all study visits. The end of the study is defined as the last subject's last visit.</li> <li>The definition of subject early withdrawal from the study will be any subject who is randomised and, for any reason, does not complete all study visits.</li> <li>Withdrawn subjects will not be replaced in the study.</li> <li>All available data from subjects who were withdrawn from the study will be listed and all available planned data will be included in summary tables and figures, unless otherwise specified.</li> </ul> |

# 12.7.2. Handling of Missing Data

| Element | Reporting Detail |
|---|---|
| General | Missing data occurs when any requested data is not provided, leading to blank fields on the collection instrument: |
| | <ul> <li>These data will be indicated by the use of a "blank" in subject listing displays (if applicable). Unless all data for a specific visit are missing in which case the data is excluded from the table.</li> <li>Answers such as "Not applicable" and "Not evaluable" are not considered to be missing data and should be displayed as such.</li> </ul> |
| Outliers | <ul> <li>Any subjects excluded from the summaries and/or statistical<br/>analyses will be documented along with the reason for exclusion in the clinical study<br/>report.</li> </ul> |
| Exposure start and stop date | If a subject's treatment start date is missing, then their Visit 2 date will be assumed to be the exposure start date. If a subject's treatment stop date is missing, this will be taken to be the date of Week 24 (Visit 6) (if the subject completes Visit 6) or the early withdrawal visit date. |

# 12.7.2.1. Handling of Missing or Partial Dates

| Element | Reporting Detail |
|---|---|
| General | Partial dates will be displayed as captured in subject listing displays. |
| SAEs and<br>ADRs | The eCRF does not allow the possibility of partial dates (i.e., only month and year) to be recorded for SAE and ADR start and end dates; |
| | <ul> <li>Completely missing start or end dates will remain missing, with no imputation applied.</li> <li>Consequently, time to onset and duration of such events will be missing.</li> </ul> |
| Concomitant<br>Medications | <ul> <li>Partial dates for any concomitant medications recorded in the CRF will be imputed using the following convention:</li> <li>If the partial date is a start date, a '01' will be used for the day and 'Jan' will be used for the month</li> </ul> |
| | <ul> <li>If the partial date is a stop date, a '28/29/30/31' will be used for the day<br/>(dependent on the month and year) and 'Dec' will be used for the month.</li> </ul> |

| Element | Reporting Detail |
|---------|----------------------------------------------------------|
| | The recorded partial date will be displayed in listings. |

# 12.7.2.2. Handling of Missing Data for Statistical Analysis

In general, missing data will not be imputed except for the sensitivity analyses defined in Section 8.1.2.

# 12.8. Appendix 8: Values of Potential Clinical Importance

# 12.8.1. Vital Signs

Not applicable

# 12.9. Appendix 9: Multicenter Studies

# 12.9.1. Methods for Handling Centres

In this multicentre study conducted in France and Germany, enrolment will be presented by investigative site.

# 12.10. Appendix 10: Examination of Covariates, Subgroups & Other Strata

#### 12.10.1. Examination of Strata and Covariates

The following is a list of covariates that may be used in descriptive summaries and statistical analyses, some of which may also be used for subgroup analyses.

Additional covariates of clinical interest may also be considered.

| Category | Covariates and / or Subgroups |
|---|---|
| Strata | Separate randomisation schedules were utilised for France and Germany respectively thereby stratifying the randomisation by country. Country will be included in all analyses as a covariate. A sensitivity analysis will examine the randomized treatment-by-country interaction for the primary and key secondary endpoints. |
| Covariates | For the primary efficacy analysis, the following baseline variables will be adjusted for: Randomised treatment (FF/VI, Usual ICS/LABA) Baseline ACT total score Age Gender Country Similar covariates will be considered for all other analyses; in each case the relevant baseline score (e.g. baseline AQLQ[S] score for the AQLQ[S] endpoints) will be included instead of baseline ACT total score. |

### 12.10.2. Examination of subgroups

- If the percentage of subjects is small within a particular subgroup, then the subgroup categories may be refined prior to unblinding the trial.
- If the category cannot be refined further, then descriptive rather than statistical comparisons may be performed for the particular subgroup.
- For statistical analyses by subgroup, models will include subgroup and treatment by subgroup interaction as covariates.

| Category | Subgroups |
|------------------------------------|----------------|
| Country | France |
| | Germany |
| Number of severe asthma | • 0 |
| exacerbations in the previous year | • ≥1 |
| prior to randomisation | |
| Smoking Status at Baseline | Current smoker |
| | Former smoker |

| Category | Subgroups |
|-----------|------------------|
| | Never smoked |
| Age Group | • ≤ 50 years old |
| | > 50 years old |
| Gender | Male |
| | Female |

#### 12.10.3. Examination of seasonal effect

A sensitivity analysis for the primary efficacy endpoint examining seasonal effect is defined in Section 8.1.2, specifying a season at randomisation covariate defined as follows:

| Season at Randomisation | Calendar Month of Randomisation |
|-------------------------|---------------------------------|
| Spring | March |
| | April |
| | May |
| Summer | June |
| | • July |
| | August |
| Autumn | September |
| | October |
| | November |
| Winter | December |
| | January |
| | February |

Furthermore, the summary of severe asthma exacerbations will be repeated by season using the same definition (according to calendar month) as specified above.

# 12.11. Appendix 11: Multiple Comparisons & Multiplicity

## 12.11.1. Handling of Multiple Comparisons & Multiplicity

Non inferiority of FF/VI to ICS/LABA will be first tested at the 0.05 two-sided nominal level of significance. If non-inferiority is statistically achieved, then superiority of FF/VI to ICS/LABA will be tested at the 0.05 two-sided nominal level of significance.

If and only if non-inferiority is achieved for the primary endpoint at Week 12 (Visit 4), then the key secondary endpoint, i.e. the change from baseline in the total ACT score assessed at Week 24 (Visit 6) will be tested. At Week 24 (Visit 6), non-inferiority of FF/VI to ICS/LABA will be first tested at the 0.05 two-sided nominal level of significance. If non-inferiority is achieved, then superiority of FF/VI to ICS/LABA will be tested at the 0.05 two-sided nominal level of significance.

Of note, this step-down testing procedure still strongly controls the overall type I error at the 0.05 two-sided level for the non-inferiority endpoints. The overall type I error is not controlled for the superiority tests at Week 12 (Visit 4) and Week 24 (Visit 6).

# 12.12. Appendix 12: Model Checking and Diagnostics for Statistical Analyses

#### 12.12.1. Statistical Analysis Assumptions

| Endpoint(s) | <ul> <li>Change from Baseline in the ACT Total Score at Week 12 (Visit 4)</li> <li>Change from Baseline in the ACT Total Score at Week 24 (Visit 6)</li> </ul> |
|---|---|
| Analysis | Analysis • MMRM (ANCOVA for LOCF and WOCF sensitivity analyses) |

- Should computational issues be encountered when running the model with an unstructured variancecovariance matrix, other structures including autoregressive 1 and compound symmetry will be considered.
- Distributional assumptions underlying the model will be checked with graphical methods (including quantile-quantile (Q-Q) plots of studentized residuals, plots of studentized residuals versus fitted values, etc.). To investigate the relationship between baseline ACT total score and the change from baseline in ACT total score, baseline ACT total will be categorized according to the distribution quartiles and the model will be fitted using this categorized variable in place of continuous baseline ACT total score.
- If the distributional assumption of normality fails then the LS means, estimated LS mean treatment difference and associated 95% CI from the model will be presented, with the p-value for the difference between treatment groups from a model on the rank-transformed values. Should the distributional assumption of normality also fail for the ranked model, other methods of analysis will be investigated.

| Endpoint(s) | <ul> <li>Percentage of subjects with correct use of inhaler device at Week 12 (Visit 4) and at Week 24 (Visit 6) independently of the use at Week 12 (Visit 4)</li> <li>ACT total score of ≥ 20 or ≥ 3 point increase from baseline in ACT total score at Week 12 (Visit 4) and Week 24 (Visit 6)</li> <li>Increase from baseline of ≥ 0.5 in AQLQ(S) total score at Week 24 (Visit 6)</li> <li>Increase from baseline of ≥ 0.5 in AQLQ(S) environmental stimuli domain score at Week 24 (Visit 6)</li> <li>Proportion of subjects with 'no problems' at Endpoint in the EQ-5D-5L questionnaire</li> </ul> |
|---|---|
| Analysis | Logistic regression model |
| 7 min j 010 | Logicus regression medel |

- If the likelihood maximisation algorithm fails to converge due to complete or quasi-complete separation
  of the data then Firth's penalized likelihood (Firth, 1993) will be implemented by use of the FIRTH
  option on the MODEL statement in PROC LOGISTIC.
- The fit of the logistic regression model will be assessed by examining the ROC curve and other diagnostic plots.

| Endpoint(s) | Change from baseline in trough (pre-dose) FEV1 at Week 12 (Visit 4) |
|---|---|
| | Change from baseline in EQ-5D Utility Score |
| | Change from baseline in EQ-5D VAS Score |
| Analysis | ANCOVA model |

- Distributional assumptions underlying the model will be checked with graphical methods (including quantile-quantile (Q-Q) plots of studentized residuals, plots of studentized residuals versus fitted values, etc.).
- If the distributional assumption of normality fails then the LS means, estimated LS mean treatment difference and associated 95% CI from the ANCOVA model will be presented, with the p-value for the

difference between treatment groups from an ANCOVA model on the rank-transformed values. Should the distributional assumption of normality also fail for the ranked ANCOVA, an exact p-value from a two-sample Wilcoxon Rank Sum test will be presented for the difference between treatment groups.

| Endpoint(s) | | Annual severe asthma exacerbation rate over the study period |
|---|---|---|
| Analysis | • | GLM assuming the Negative Binomial distribution |

If a GLM assuming the Negative Binomial distribution cannot be fitted due to the lack of repeat events
within a subject, a GLM assuming the Poisson distribution will be used. The underlying assumption for
the Poisson distribution that the mean and variance of the response variable are equal will be
examined. If the variance of the fitted model exceeds the mean (over-dispersion), the dispersion
parameter will be estimated as a ratio of the Pearson Chi-Square to its associated degrees of freedom
(using the PSCALE option in PROC GENMOD).

| Endpoint(s) | Time to first severe asthma exacerbation |
|-------------|------------------------------------------|
| Analysis | Cox proportional hazards model |

- Proportional hazards assumptions will be checked by plotting the log of the negative log of the
  estimated survivor functions against log time, for each treatment group. If hazards are proportional, the
  lines should be approximately parallel.
- If the assumption of proportionality is not met, the use of other models such as models including timedependent covariates will be considered.
- If there are computational issues in implementing the exact method for handling ties, then the Efron method (Efron, 1977) will be used instead.

# 12.13. Appendix 13: Blinding Strategy

The Blinding Strategy is maintained separately in a document entitled HZA116492 - Blinding Strategy.

# 12.14. Appendix 14: Abbreviations & Trade Marks

# 12.14.1. Abbreviations

| Abbreviation | Description |
|--------------|---------------------------------------------------|
| ACT | Asthma Control Test |
| ADR | Adverse Drug Reaction |
| AE | Adverse Event |
| AESI | Adverse Event of Special Interest |
| ANCOVA | Analysis of Covariance |
| AQLQ(S) | Standardised Asthma Quality of Life Questionnaire |
| ASE | All Subjects Enrolled |
| BMI | Body Mass Index |
| BUD | Budesonide |
| CI | Confidence Interval |
| CIL | Clinical Investigational Lead |
| CRF | Case Report Form |
| CRO | Contract Research Organisation |
| DBF | Database Freeze |
| DBP | Diastolic Blood Pressure |
| DBR | Database Release |
| DM | Data Management |
| DP | Decimal Place |
| DPI | Dry Powder Inhaler |
| DQL | Data Quality Lead |
| eCRF | Electronic Case Report Form |
| EQ-5D-5L | EuroQol Questionnaire |
| F | Formoterol |
| FEV1 | Forced Expiratory Volume in 1 Second |
| FF | Fluticasone Furoate |
| FP | Fluticasone Propionate |
| GINA | Global Initiative for Asthma |
| GLM | Generalised Linear Model |
| GSK | GlaxoSmithKline |
| HL | Hodges-Lehmann |
| HR | Heart Rate |
| ICF | Informed Consent Form |
| ICS | Inhaled Corticosteroid |
| IDSL | Integrated Data Standards Library |
| IP | Investigational Product |
| ITT | Intent-to-Treat |
| LABA | Long-acting Beta Agonist |
| LOCF | Last Observation Carried Forward |
| LRTI | Lower Respiratory Tract Infection |
| LS | Least Squares |
| MAR | Missing at Random |
| MARS-A | Medication Adherence Report Scale for Asthma |
| MCID | Minimal Clinically Important Difference |
| MedDRA | Medical Dictionary for Regulatory Activities |

| Abbreviation | Description |
|--------------|---------------------------------------------------|
| MI | Multiple Imputation |
| MID | Minimally Important Difference |
| MMRM | Mixed Model Repeated Measures |
| PASAP-Q | Patient Satisfaction and Preference Questionnaire |
| PD | Protocol Deviation |
| PDMP | Protocol Deviation Management Plan |
| PP | Per Protocol |
| Q-Q | Quantile-Quantile |
| RAP | Reporting and Analysis Plan |
| REML | Restricted Maximum Likelihood |
| S | Salmeterol |
| S&P | Statistics and Programming |
| SAC | Statistical Analysis Complete |
| SAE | Serious Adverse Event |
| SBP | Systolic Blood Pressure |
| SD | Standard Deviation |
| SMQ | Standardised MedDRA Query |
| VAS | Visual Analogue Scale |
| VI | Vilanterol |
| WOCF | Worst Observation Carried Forward |

# 12.14.2. Trademarks

| Trademarks of the GlaxoSmithKline Group of Companies |
|------------------------------------------------------|
| DISKUS |
| ELLIPTA |
| GSK |
| NUCALA |
| SERETIDE |

| Trademarks not owned by the GlaxoSmithKline Group of Companies |
|----------------------------------------------------------------|
| ACT |
| Asthma Quality of Life Questionnaire - |
| AQLQ(S) |
| EQ-5D |
| MARS-A Questionnaire |
| PASAP Questionnaire |
| Symbicort Turbuhaler |
| TURBUHALER |
| XOLAIR |

# 12.15. Appendix 15: List of Data Displays

#### 12.15.1. Data Display Numbering

The following numbering will be applied for RAP generated displays:

| Section | Tables Figures | |
|------------------|-----------------------|------------|
| Study Population | 1.1 to 1.n 1.1 to 1.n | |
| Efficacy | 2.1 to 2.n 2.1 to 2.n | |
| Safety | 3.1 to 3.n | 3.1 to 3.n |
| Section | Listings | |
| ICH Listings | 1 to x | |
| Other Listings | y to z | |

## 12.15.2. Mock Example Shell Referencing

Non IDSL specifications will be referenced as indicated and if required an example mock-up displays provided in Appendix 11: Example Mock Shells for Data Displays

.

| Section | Figure | Table | Listing |
|------------------|---------|---------|---------|
| Study Population | POP_Fn | POP_Tn | POP_Ln |
| Efficacy | EFF_Fn | EFF_Tn | EFF_Ln |
| Safety | SAFE_Fn | SAFE_Tn | SAFE_Ln |

#### NOTES:

• Non-Standard displays are indicated in the 'IDSL / TST ID / Example Shell' or 'Programming Notes' column as '[Non-Standard] + Reference.'

### 12.15.3. Deliverable [Priority]

| Delivery [Priority] [1] | Description |
|-------------------------|-------------------------------------|
| Data Look [1] | Data Look Outputs (blinded review) |
| SAC [2] | Final Statistical Analysis Complete |

#### NOTES:

1. Indicates priority (i.e. order) in which displays will be generated for the reporting effort.

# 12.15.4. Study Population Tables

| Study F | Study Population: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Subject Disposition | | | | | |
| 1.1. | All Enrolled<br>Subjects | Non-Standard<br>POP_T1 | Summary of Subject Populations | Randomised population line will provide the denominators for the ITT, PP and Safety percentages. | Data Look [1]<br>SAC [2] |
| 1.2. | All Enrolled<br>Subjects | IE2 | Summary of Inclusion/Exclusion Criteria Failures for Subjects Not Starting Treatment | | Data Look [1]<br>SAC [2] |
| 1.3. | ITT | ES1 | Summary of End of Study Record | | Data Look [1]<br>SAC [2] |
| 1.4. | PP | ES1 | Summary of End of Study Record Per Protocol Population | | Data Look [1]<br>SAC [2] |
| 1.5. | ITT | Non-Standard<br>POP_T2 | Summary of Attendance at Each Clinic Visit and Phone Call Visit | | Data Look [1]<br>SAC [2] |
| 1.6. | All Enrolled<br>Subjects | NS1 | Summary of Number of Subjects by Country and Centre | | SAC [2] |
| 1.7. | ITT | NS1 | Summary of Number of Subjects by Country and Centre | | Data Look [1]<br>SAC [2] |
| 1.8. | PP | NS1 | Summary of Number of Subjects by Country and Centre Per Protocol Population | | SAC [2] |
| Protoco | Protocol Deviations | | | | |
| 1.9. | ITT | IE2 | Summary of Deviations from the Inclusion/Exclusion Criteria | | Data Look [1]<br>SAC [2] |
| 1.10. | ITT | Non-Standard<br>POP_T3 | Summary of Important Protocol Deviations | | Data Look [1]<br>SAC [2] |

| Study F | Study Population: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 1.11. | ITT | Non-Standard<br>POP_T3 | Summary of Important Protocol Deviations Resulting in Exclusion from the PP Population | | Data Look [1]<br>SAC [2] |
| Demog | raphic and Bas | eline Characteris | tics | | |
| 1.12. | ITT | DM1 | Summary of Demographic Characteristics | | Data Look [1]<br>SAC [2] |
| 1.13. | PP | DM1 | Summary of Demographic Characteristics Per Protocol Population | | SAC [2] |
| 1.14. | Safety | DM1 | Summary of Demographic Characteristics Safety Population | | SAC [2] |
| 1.15. | All Enrolled<br>Subjects | DM11 | Summary of Age Ranges | | Data Look [1]<br>SAC [2] |
| 1.16. | ITT | DM5 | Summary of Race and Racial Combinations | | Data Look [1]<br>SAC [2] |
| 1.17. | ITT | DM6 | Summary of Race and Racial Combinations Details | | Data Look [1]<br>SAC [2] |
| 1.18. | ITT | MH4 | Summary of Current Medical Conditions | | Data Look [1]<br>SAC [2] |
| 1.19. | ITT | MH4 | Summary of Past Medical Conditions | | SAC [2] |
| 1.20. | ITT | Non-Standard<br>POP_T4 | Summary of Asthma Duration at Baseline | | Data Look [1]<br>SAC [2] |
| 1.21. | PP | Non-Standard<br>POP_T4 | Summary of Asthma Duration at Baseline<br>Per Protocol Population | | Data Look [1]<br>SAC [2] |
| 1.22. | ITT | Non-Standard<br>POP_T5 | Summary of Asthma Exacerbation History at Baseline | | Data Look [1]<br>SAC [2] |

| Study I | Study Population: Tables | | | | | | |
|---|---|---|---|---|---|--|--|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] | | |
| 1.23. | PP | Non-Standard<br>POP_T5 | Summary of Asthma Exacerbation History at Baseline Per Protocol Population | | Data Look [1]<br>SAC [2] | | |
| 1.24. | ITT | Non-Standard<br>POP_T6 | Summary of Smoking History at Baseline | | Data Look [1]<br>SAC [2] | | |
| 1.25. | PP | Non-Standard<br>POP_T6 | Summary of Smoking History at Baseline Per Protocol Population | | SAC [2] | | |
| Conco | Concomitant Medications | | | | | | |
| 1.26. | ITT | CM8 | Summary of Pre-Treatment Concomitant Medications | | SAC [2] | | |
| 1.27. | ITT | CM8 | Summary of On-Treatment Concomitant Medications | | SAC [2] | | |
| 1.28. | ITT | CM8 | Summary of On-Treatment Asthma Concomitant Medications | | Data Look [1]<br>SAC [2] | | |
| Exposi | Exposure | | | | | | |
| 1.29. | ITT | Non-Standard<br>POP_T7 | Summary of Study Medication Dosage Modification | | Data Look [1]<br>SAC [2] | | |
| 1.30. | ITT | Non-Standard<br>POP_T8 | Summary of Extent of Exposure to Study Medication (Regardless of Modification to Study Medication Dosage) | | Data Look [1]<br>SAC [2] | | |
| 1.31. | ITT | Non-Standard<br>POP_T8 | Summary of Extent of Exposure to Study Medication (up to First Modification to Study Medication Dosage) | | SAC [2] | | |
| Study F | Study Population: Tables | | | | | | | |
|---|---|---|---|---|---|--|--|--|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] | | | |
| 1.32. | ITT | Non-Standard<br>POP_T9 | Summary of Extent of Exposure to Study Medication by Medication and Dosage | Repeat on subsequent pages for Medication/Dosage = FF/VI 184 mcg/22 mcg OD, FP/S 250 mcg/50 mcg BID, FP/S 500 mcg/50 mcg BID, BUD/F 200 mcg/6 mcg BID (1 inhalation per dose), BUD/F 200 mcg/6 mcg BID (2 inhalations per dose), BUD/F 400 mcg/12 mcg BID (1 inhalation per dose), BUD/F 400 mcg/12 mcg BID (2 inhalations per dose). | Data Look [1]<br>SAC [2] | | | |
| Numbe | Number of Subjects by Subgroup | | | | | | | |
| 1.33. | ITT | Non-Standard<br>POP_T10 | Summary of Number of Subjects by Subgroup | | SAC [2] | | | |

# 12.15.5. Study Population Figures

| Study Pop | Study Population: Figures | | | | |
|---|---|---|---|---|---|
| No. | No. Population IDSL / TST ID / Example Shell Title Programming Notes | | | | |
| Exposure | | | | | |
| 1.1. | ITT | Non-Standard<br>POP_F1 | Plot of Exposure to Study Medication (Regardless of Modification to Study Medication Dosage) | Display increments of 6 weeks on the x-axis, up to the maximum exposure (e.g. 0, 6, 12, 18, 24, 30). | Data Look [1]<br>SAC [2] |

# 12.15.6. Efficacy Tables

| Efficacy | Efficacy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Change | from Baseline | in ACT Total Sco | re at Week 12 (Visit 4) | | |
| 2.1. | ITT | Non-Standard<br>EFF_T1 | Summary of Change from Baseline in ACT Total Score | | Data Look [1]<br>SAC [2] |
| 2.2. | PP | Non-Standard<br>EFF_T1 | Summary of Change from Baseline in ACT Total Score Per Protocol Population | | SAC [2] |
| 2.3. | ITT | Non-Standard<br>EFF_T2 | Summary of the Statistical Analysis of Change from Baseline in ACT Total Score at Week 12 (Visit 4) | | Data Look [1]<br>SAC [2] |
| 2.4. | PP | Non-Standard<br>EFF_T2 | Summary of the Statistical Analysis of Change from Baseline in ACT Total Score at Week 12 (Visit 4) Per Protocol Population | | SAC [2] |
| 2.5. | ITT | Non-Standard<br>EFF_T2 | Summary of the Statistical Analysis of Change from Baseline in ACT Total Score at Week 12 (Visit 4) (ANCOVA with LOCF) | Footnotes as follows: "Note: The analysis method was an ANCOVA model adjusted for randomised treatment, baseline ACT total score, gender, age and country. Note: Missing values at Week 12 (Visit 4) were replaced by last available post-randomization value based on the last observation carried forward (LOCF) method." | Data Look [1]<br>SAC [2] |

| Efficacy | r: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.6. | ITT | Non-Standard<br>EFF_T2 | Summary of the Statistical Analysis of Change from Baseline in ACT Total Score at Week 12 (Visit 4) (Multiple Imputation – Missing at Random Approach) | Footnotes as follows: "Note: Missing values post- randomisation were imputed using multiple imputation methods based on pattern mixture models. Note: Each imputed data set was analysed using an ANCOVA model at Week 12 (Visit 4) adjusted for randomised treatment, baseline ACT total score, gender, age and country and the resulting treatment differences and their standard errors combined using Rubin's rules." | Data Look [1]<br>SAC [2] |
| 2.7. | ITT | Non-Standard<br>EFF_T2 | Summary of the Statistical Analysis of Change from Baseline in ACT Total Score at Week 12 (Visit 4) (Multiple Imputation – Copy Differences from Reference Approach) | Footnotes as follows: "Note: Missing values post- randomisation were imputed using multiple imputation methods based on pattern mixture models. Note: Each imputed data set was analysed using an ANCOVA model at Week 12 (Visit 4) adjusted for randomised treatment, baseline ACT total score, gender, age and country and the resulting treatment differences and their standard errors combined using Rubin's rules." | Data Look [1]<br>SAC [2] |

| Efficacy | /: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.8. | ITT | Non-Standard<br>EFF_T2 | Summary of the Statistical Analysis of Change from Baseline in ACT Total Score at Week 12 (Visit 4) (Hodges-Lehmann Approach) | Present the "Difference" and "95% CI" lines of "FF/VI vs. Usual ICS/LABA" section only. Footnotes as follows: "Note: The difference between treatment groups at Week 12 (Visit 4) was calculated using the Hodges-Lehmann approach." | Data Look [1]<br>SAC [2] |
| 2.9. | ITT | Non-Standard<br>EFF_T2 | Summary of the Statistical Analysis of Change from Baseline in ACT Total Score at Week 12 (Visit 4) (ANCOVA with WOCF) | Footnotes as follows: "Note: The analysis method was an ANCOVA model adjusted for randomised treatment, baseline ACT total score, gender, age and country. Note: Missing values at Week 12 (Visit 4) due to treatment withdrawal prior to this time point were replaced by worst post-randomisation value based on the worst observation carried forward (WOCF) method." | Data Look [1]<br>SAC [2] |
| 2.10. | ITT | Non-Standard<br>EFF_T3 | Summary of the Statistical Analysis of Change from Baseline in ACT Total Score at Week 12 (Visit 4), Adjusting for Seasonal Effect | Repeat on subsequent pages for Season at randomisation = Summer, Autumn, Winter. | Data Look [1]<br>SAC [2] |
| 2.11. | PP | Non-Standard<br>EFF_T3 | Summary of the Statistical Analysis of Change from Baseline in ACT Total Score at Week 12 (Visit 4), Adjusting for Seasonal Effect Per Protocol Population | Repeat on subsequent pages for Season at randomisation = Summer, Autumn, Winter. | SAC [2] |
| 2.12. | ITT | Non-Standard<br>EFF_T1 | Summary of Change from Baseline in ACT Total Score, FF/VI Versus the Subset of Usual ICS/LABA Subjects Prescribed FP/S at Randomisation | | Data Look [1]<br>SAC [2] |

| Efficacy | Efficacy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.13. | ITT | Non-Standard<br>EFF_T2 | Summary of the Statistical Analysis of Change from Baseline in ACT Total Score at Week 12 (Visit 4), FF/VI Versus the Subset of Usual ICS/LABA Subjects Prescribed FP/S at Randomisation | Output only to be produced if ≥25% of Usual ICS/LABA patients are prescribed FP/S at randomisation. | Data Look [1]<br>SAC [2] |
| 2.14. | ITT | Non-Standard<br>EFF_T1 | Summary of Change from Baseline in ACT Total Score, FF/VI Versus the Subset of Usual ICS/LABA Subjects Prescribed BUD/F at Randomisation | | SAC [2] |
| 2.15. | ITT | Non-Standard<br>EFF_T2 | Summary of the Statistical Analysis of Change from Baseline in ACT Total Score at Week 12 (Visit 4), FF/VI Versus the Subset of Usual ICS/LABA Subjects Prescribed BUD/F at Randomisation | Output only to be produced if ≥25% of Usual ICS/LABA patients are prescribed BUD/F at randomisation. | SAC [2] |
| 2.16. | ITT | Non-Standard<br>EFF_T1S | Summary of Change from Baseline in ACT Total Score by Country | | Data Look [1]<br>SAC [2] |
| 2.17. | ITT | Non-Standard<br>EFF_T2S | Summary of the Statistical Analysis of Change from Baseline in ACT Total Score at Week 12 (Visit 4) by Country | | Data Look [1]<br>SAC [2] |
| 2.18. | ITT | Non-Standard<br>EFF_T1S | Summary of Change from Baseline in ACT Total Score by Number of Severe Asthma Exacerbations in the Previous Year Prior to Randomisation | | SAC [2] |

| Efficacy | Efficacy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.19. | ITT | Non-Standard<br>EFF_T2S | Summary of the Statistical Analysis of Change from Baseline in ACT Total Score at Week 12 (Visit 4) by Number of Severe Asthma Exacerbations in the Previous Year Prior to Randomisation | First footnote as follows: "Note: The analysis method was an MMRM adjusted for randomised treatment, visit (Week 6 and Week 12), baseline ACT total score, baseline ACT total score-by-visit interaction, gender, age, country, number of severe asthma exacerbations in the previous year prior to randomisation, two- and three- way interactions between randomised treatment, visit and number of severe asthma exacerbations in the previous year prior to randomisation, and patient fitted as a random factor." | SAC [2] |
| 2.20. | ITT | Non-Standard<br>EFF_T1S | Summary of Change from Baseline in ACT Total Score by Smoking Status at Baseline | | SAC [2] |
| 2.21. | ITT | Non-Standard<br>EFF_T2S | Summary of the Statistical Analysis of Change from Baseline in ACT Total Score at Week 12 (Visit 4) by Smoking Status at Baseline | First footnote as follows: "Note: The analysis method was an MMRM adjusted for randomised treatment, visit (Week 6 and Week 12), baseline ACT total score, baseline ACT total score-by-visit interaction, gender, age, country, smoking status at baseline, two- and three- way interactions between randomised treatment, visit and smoking status at baseline, and patient fitted as a random factor." | SAC [2] |
| 2.22. | ITT | Non-Standard<br>EFF_T1S | Summary of Change from Baseline in ACT Total Score by Age Group | | SAC [2] |

| Efficacy | Efficacy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.23. | ITT | Non-Standard<br>EFF_T2S | Summary of the Statistical Analysis of Change from Baseline in ACT Total Score at Week 12 (Visit 4) by Age Group | First footnote as follows: "Note: The analysis method was an MMRM adjusted for randomised treatment, visit (Week 6 and Week 12), baseline ACT total score, baseline ACT total score-by-visit interaction, gender, country, age group, two- and three- way interactions between randomised treatment, visit and age group, and patient fitted as a random factor." | SAC [2] |
| 2.24. | ITT | Non-Standard<br>EFF_T1S | Summary of Change from Baseline in ACT Total Score by Gender | | SAC [2] |
| 2.25. | ITT | Non-Standard<br>EFF_T2S | Summary of the Statistical Analysis of Change from Baseline in ACT Total Score at Week 12 (Visit 4) by Gender | First footnote as follows: "Note: The analysis method was an MMRM adjusted for randomised treatment, visit (Week 6 and Week 12), baseline ACT total score, baseline ACT total score-by-visit interaction, gender, age, country, two- and three- way interactions between randomised treatment, visit and gender, and patient fitted as a random factor." | SAC [2] |

| Efficacy | Efficacy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Change | Change from Baseline in ACT Total Score at Week 24 (Visit 6) | | | | |
| 2.26. | ITT | Non-Standard<br>EFF_T2 | Summary of the Statistical Analysis of Change from Baseline in ACT Total Score at Week 24 (Visit 6) | First footnote as follows: "Note: The analysis method was an MMRM adjusted for randomised treatment, visit (Week 6, Week 12, Week 18 and Week 24), baseline ACT total score, randomised treatment-by-visit interaction, baseline ACT total score-by-visit interaction, gender, age, country and patient fitted as a random factor." | Data Look [1]<br>SAC [2] |
| 2.27. | PP | Non-Standard<br>EFF_T2 | Summary of the Statistical Analysis of Change from Baseline in ACT Total Score at Week 24 (Visit 6) Per Protocol Population | First footnote as follows: "Note: The analysis method was an MMRM adjusted for randomised treatment, visit (Week 6, Week 12, Week 18 and Week 24), baseline ACT total score, randomised treatment-by-visit interaction, baseline ACT total score-by-visit interaction, gender, age, country and patient fitted as a random factor." | SAC [2] |
| 2.28. | ITT | Non-Standard<br>EFF_T2 | Summary of the Statistical Analysis of Change from Baseline in ACT Total Score at Week 24 (Visit 6) (ANCOVA with LOCF) | Footnotes as follows: "Note: The analysis method was an ANCOVA model adjusted for randomised treatment, baseline ACT total score, gender, age and country. Note: Missing values at Week 24 (Visit 6) were replaced by last available post-randomization value based on the last observation carried forward (LOCF) method." | SAC [2] |

| Efficacy | /: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.29. | ITT | Non-Standard<br>EFF_T2 | Summary of the Statistical Analysis of Change from Baseline in ACT Total Score at Week 24 (Visit 6) (Multiple Imputation – Missing at Random Approach) | Footnotes as follows: "Note: Missing values post- randomisation were imputed using multiple imputation methods based on pattern mixture models. Note: Each imputed data set was analysed using an ANCOVA model at Week 24 (Visit 6) adjusted for randomised treatment, baseline ACT total score, gender, age and country and the resulting treatment differences and their standard errors combined using Rubin's rules." | SAC [2] |
| 2.30. | ITT | Non-Standard<br>EFF_T2 | Summary of the Statistical Analysis of Change from Baseline in ACT Total Score at Week 24 (Visit 6) (Multiple Imputation – Copy Differences from Reference Approach) | Footnotes as follows: "Note: Missing values post- randomisation were imputed using multiple imputation methods based on pattern mixture models. Note: Each imputed data set was analysed using an ANCOVA model at Week 24 (Visit 6) adjusted for randomised treatment, baseline ACT total score, gender, age and country and the resulting treatment differences and their standard errors combined using Rubin's rules." | SAC [2] |

| Efficacy | /: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.31. | ITT | Non-Standard<br>EFF_T2 | Summary of the Statistical Analysis of Change from Baseline in ACT Total Score at Week 24 (Visit 6) (Hodges-Lehmann Approach) | Present the "Difference" and "95% CI" lines of "FF/VI vs. Usual ICS/LABA" section only. Footnotes as follows: "Note: The difference between treatment groups at Week 24 (Visit 6) was calculated using the Hodges-Lehmann approach." | SAC [2] |
| 2.32. | ITT | Non-Standard<br>EFF_T2 | Summary of the Statistical Analysis of Change from Baseline in ACT Total Score at Week 24 (Visit 6) (ANCOVA with WOCF) | Footnotes as follows: "Note: The analysis method was an ANCOVA model adjusted for randomised treatment, baseline ACT total score, gender, age and country. Note: Missing values at Week 24 (Visit 6) due to treatment withdrawal prior to this time point were replaced by worst post-randomisation value based on the worst observation carried forward (WOCF) method." | SAC [2] |
| 2.33. | ITT | Non-Standard<br>EFF_T3 | Summary of the Statistical Analysis of Change from Baseline in ACT Total Score at Week 24 (Visit 6), Adjusting for Seasonal Effect | First footnote as follows: "Note: The analysis method was an MMRM adjusted for randomised treatment, visit (Week 6, Week 12, Week 18 and Week 24), baseline ACT total score, baseline ACT total score, by-visit interaction, gender, age, country, season at randomisation, two-and three- way interactions between randomised treatment, visit and season at randomisation, and patient fitted as a random factor." | SAC [2] |

| Efficacy | Efficacy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.34. | PP | Non-Standard<br>EFF_T3 | Summary of the Statistical Analysis of Change from Baseline in ACT Total Score at Week 24 (Visit 6), Adjusting for Seasonal Effect Per Protocol Population | First footnote as follows: "Note: The analysis method was an MMRM adjusted for randomised treatment, visit (Week 6, Week 12, Week 18 and Week 24), baseline ACT total score, baseline ACT total score-by-visit interaction, gender, age, country, season at randomisation, two-and three- way interactions between randomised treatment, visit and season at randomisation, and patient fitted as a random factor." | SAC [2] |
| 2.35. | ITT | Non-Standard<br>EFF_T2 | Summary of the Statistical Analysis of Change from Baseline in ACT Total Score at Week 24 (Visit 6), FF/VI Versus the Subset of Usual ICS/LABA Subjects Prescribed FP/S at Randomisation | Output only to be produced if ≥25% of Usual ICS/LABA patients are prescribed FP/S at randomisation. First footnote as follows: "Note: The analysis method was an MMRM adjusted for randomised treatment, visit (Week 6, Week 12, Week 18 and Week 24), baseline ACT total score, randomised treatment-by-visit interaction, baseline ACT total score-by-visit interaction, gender, age, country and patient fitted as a random factor." | SAC [2] |

| Efficac | y: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.36. | ITT | Non-Standard<br>EFF_T2 | Summary of the Statistical Analysis of Change from Baseline in ACT Total Score at Week 12 (Visit 4), FF/VI Versus the Subset of Usual ICS/LABA Subjects Prescribed BUD/F at Randomisation | Output only to be produced if ≥25% of Usual ICS/LABA patients are prescribed BUD/F at randomisation. First footnote as follows: "Note: The analysis method was an MMRM adjusted for randomised treatment, visit (Week 6, Week 12, Week 18 and Week 24), baseline ACT total score, randomised treatment-by-visit interaction, baseline ACT total score-by-visit interaction, gender, age, country and patient fitted as a random factor." | SAC [2] |
| 2.37. | ITT | Non-Standard<br>EFF_T2S | Summary of the Statistical Analysis of Change from Baseline in ACT Total Score at Week 24 (Visit 6) by Country | First footnote as follows: "Note: The analysis method was an MMRM adjusted for randomised treatment, visit (Week 6, Week 12, Week 18 and Week 24), baseline ACT total score, baseline ACT total score-by-visit interaction, gender, age, country, two- and three- way interactions between randomised treatment, visit and country, and patient fitted as a random factor." | SAC [2] |
| Correct | Use of Inhaler | Device | | | |
| 2.38. | ITT | Non-Standard<br>EFF_T4 | Summary of Inhaler Device Use Errors | Repeat on subsequent pages for Visit = Week 12 and Week 24. "Number of patients using" line will provide the denominators for each section's percentages. | Data Look [1]<br>SAC [2] |

| Efficac | y: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.39. | PP | Non-Standard<br>EFF_T4 | Summary of Inhaler Device Use Errors Per Protocol Population | Repeat on subsequent pages for Visit = Week 12 and Week 24. "Number of patients using" line will provide the denominators for each section's percentages. | SAC [2] |
| 2.40. | ITT | Non-Standard<br>EFF_T5 | Summary of Correct Use of Inhaler Device | | Data Look [1]<br>SAC [2] |
| 2.41. | PP | Non-Standard<br>EFF_T5 | Summary of Correct Use of Inhaler Device Per Protocol Population | | SAC [2] |
| 2.42. | ITT | Non-Standard<br>EFF_T6 | Summary of the Statistical Analysis of Correct Use of Inhaler<br>Device at Week 12 (Visit 4) and at Week 24 (Visit 6)<br>Independently of the Use at Week 12 (Visit 4) | | Data Look [1]<br>SAC [2] |
| 2.43. | PP | Non-Standard<br>EFF_T6 | Summary of the Statistical Analysis of Correct Use of Inhaler<br>Device at Week 12 (Visit 4) and at Week 24 (Visit 6)<br>Independently of the Use at Week 12 (Visit 4)<br>Per Protocol Population | | SAC [2] |
| Lung F | unction Tests | | | | |
| 2.44. | ITT | Non-Standard<br>EFF_T1 | Summary of Change from Baseline in Lung Function Tests | Present an additional column to the left of "Visit", labelled "Test" with values "Trough (Pre-dose) FEV1 (L)" and "Trough (Pre-dose) Percent Predicted FEV1 (%)" to allow presentation of results by Test. Present the following visits: Randomisation (Day 0), Week 12, Change from Baseline at Week 12, Early Withdrawal and Change from Baseline at Early Withdrawal. | Data Look [1]<br>SAC [2] |

| Efficacy | y: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.45. | ITT | Non-Standard<br>EFF_T2 | Summary of the Statistical Analysis of Change from Baseline in Trough (Pre-dose) FEV1 at Week 12 (Visit 4) | Footnote as follows: "Note: The analysis method was an ANCOVA model adjusted for randomised treatment, baseline trough (pre-dose) FEV1, gender, age and country." | Data Look [1]<br>SAC [2] |
| Subject | ts Who Have Ei | ther an ACT Total | Score >= 20 or >= 3 Point Increase from Baseline in ACT Total | Score | |
| 2.46. | ITT | Non-Standard<br>EFF_T7 | Summary of Percentage of Subjects Who Have Either an ACT Total Score >= 20 or >= 3 Point Increase from Baseline in ACT Total Score | Repeat for Visit = Week 18, Week 24, Early Withdrawal. | Data Look [1]<br>SAC [2] |
| 2.47. | ITT | Non-Standard<br>EFF_T6 | Summary of the Statistical Analysis of Percentage of Subjects Who Have Either an ACT Total Score >= 20 or >= 3 Point Increase from Baseline in ACT Total Score at Week 12 (Visit 4) and Week 24 (Visit 6) | Replace "With correct use [1]" with "Responder [1]" and "Without correct use" with "Non-Responder". Footnotes as follows: "[1] Responder is defined as an ACT total score >= 20 or >= 3 point increase from baseline in ACT total score at that visit. Note: The analysis method was logistic regression adjusted for randomised treatment, baseline ACT total score, baseline ACT total score squared, gender, age and country." | SAC [2] |

| Efficac | Efficacy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Individ | ual ACT Questi | on Scores | | | |
| 2.48. | ITT | Non-Standard<br>EFF_T8 | Summary of Individual ACT Question Scores | Repeat on subsequent pages for Question = 2. Shortness of breath, 3. Asthma symptoms woken up at night or earlier than usual, 4. Used rescue inhaler or nebuliser medication, 5. Asthma control. | Data Look [1]<br>SAC [2] |
| Compli | ance with Stud | y Medication | | | |
| 2.49. | ITT | Non-Standard<br>EFF_T9 | Summary of Compliance with Study Medication | | Data Look [1]<br>SAC [2] |
| 2.50. | PP | Non-Standard<br>EFF_T9 | Summary of Compliance with Study Medication Per Protocol Population | | SAC [2] |
| MARS- | A | | | | |
| 2.51. | ITT | Non-Standard<br>EFF_T10 | Summary of Use of Medication Adherence Report Scale for Asthma (MARS-A) During the Study | Repeat on subsequent pages for Visit = Week 12, Week 24 and Early Withdrawal. | Data Look [1]<br>SAC [2] |
| 2.52. | ITT | Non-Standard<br>EFF_T10S | Summary of Use of Medication Adherence Report Scale for Asthma (MARS-A) During the Study by Status of Patient in Relation to the Reminder Sent to French Centres | Repeat on subsequent pages for Visit = Week 12, Week 24 and Early Withdrawal, and for Status = Patients in France, all MARS-A assessments completed pre-reminder, Patients in France, some MARS-A assessments completed pre-reminder, some post-reminder, Patients in France, all MARS-A assessments completed post-reminder, Patients in Germany | Data Look [1]<br>SAC [2] |

| Efficac | Efficacy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Severe | On-Treatment | Asthma Exacerba | tions | , | |
| 2.53. | ITT | Non-Standard<br>EFF_T11 | Summary of Severe On-Treatment Asthma Exacerbations | | Data Look [1]<br>SAC [2] |
| 2.54. | ITT | Non-Standard<br>EFF_T11S | Summary of Severe On-Treatment Asthma Exacerbations by Season | Repeat on subsequent pages for Season = Summer, Autumn, Winter. | Data Look [1]<br>SAC [2] |
| 2.55. | ITT | Non-Standard<br>EFF_T12 | Summary of the Statistical Analysis of Severe On-Treatment Asthma Exacerbations | | Data Look [1]<br>SAC [2] |
| 2.56. | ITT | Non-Standard<br>EFF_T13 | Summary of the Statistical Analysis of Time to First Severe On-<br>Treatment Asthma Exacerbation | | Data Look [1]<br>SAC [2] |
| AQLQ( | S) | | | | |
| 2.57. | ITT | Non-Standard<br>EFF_T1 | Summary of Change from Baseline in AQLQ(S) Total Score and Domain Scores | Present an additional column to the left of "Visit", labelled "Domain" with values "Total Score", "Environmental Stimuli", "Symptoms", "Activity Limitations" and "Emotional Function" to allow presentation of results by Domain. Present the following visits: Randomisation (Day 0), Week 24, Change from Baseline at Week 24, Early Withdrawal and Change from Baseline at Early Withdrawal. | SAC [2] |
| 2.58. | ITT | Non-Standard<br>EFF_T14 | Summary of Percentage of Subjects Who Have an Increase from Baseline of >=0.5 in AQLQ(S) Total Score and Domain Scores | Repeat on subsequent pages for Domain = Environmental Stimuli, Symptoms, Activity Limitations and Emotional Function. | Data Look [1]<br>SAC [2] |

| Efficacy | Efficacy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.59. | ITT | Non-Standard<br>EFF_T6 | Summary of the Statistical Analysis of Percentage of Subjects<br>Who Have an Increase from Baseline of >=0.5 in AQLQ(S) Total<br>Score and Environmental Stimuli Domain Score at Week 24<br>(Visit 6) | Replace "With correct use [1]" with "Responder [1]" and "Without correct use" with "Non-Responder". Do not display the "Visit" column. Footnotes as follows: "[1] Responder is defined as an increase from baseline of >= 0.5. Note: The analysis method was logistic regression adjusted for randomised treatment, baseline score, gender, age and country." | SAC [2] |
| EQ-5D- | 5L | | | | |
| 2.60. | ITT | Non-Standard<br>EFF_T15 | Summary of EQ-5D-5L Descriptive System Dimensions | Repeat on subsequent pages for Visit = Early Withdrawal and for Dimension = Self-Care, Usual Activities, Pain/Discomfort, and Anxiety/Depression. | Data Look [1]<br>SAC [2] |
| 2.61. | ITT | Non-Standard<br>EFF_T6 | Summary of the Statistical Analysis of Proportion of Responders<br>According to EQ-5D-5L Descriptive System Dimensions at Week<br>24 (Visit 6) | Replace "With correct use [1]" with "Responder [1]" and "Without correct use" with "Non-Responder". Do not display the "Visit" column. Footnotes as follows: "[1] Responder is defined as a score of 1 ('no problems'). Note: The analysis method was logistic regression adjusted for randomised treatment, baseline EQ-5D-5L domain score, gender, age and country." | SAC [2] |

| Efficacy | Efficacy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.62. | ITT | Non-Standard<br>EFF_T1 | Summary of EQ-5D-5L Utility Score | Present the following visits: Randomisation (Day 0), Week 24, Change from Baseline at Week 24, Early Withdrawal and Change from Baseline at Early Withdrawal. | Data Look [1]<br>SAC [2] |
| 2.63. | ITT | Non-Standard<br>EFF_T2 | Summary of the Statistical Analysis of Change from Baseline in EQ-5D-5L Utility Score at Week 24 (Visit 6) | Footnote as follows: "Note: The analysis method was an ANCOVA model adjusted for randomised treatment, baseline EQ-5D-5L utility score, gender, age and country." | SAC [2] |
| 2.64. | ITT | Non-Standard<br>EFF_T1 | Summary of EQ-5D-5L Visual Analogue Scale (VAS) Score | Present the following visits: Randomisation (Day 0), Week 24, Change from Baseline at Week 24, Early Withdrawal and Change from Baseline at Early Withdrawal. | SAC [2] |
| 2.65. | ITT | Non-Standard<br>EFF_T2 | Summary of the Statistical Analysis of Change from Baseline in EQ-5D-5L Visual Analogue Scale (VAS) Score at Week 24 (Visit 6) | Footnote as follows: "Note: The analysis method was an ANCOVA model adjusted for randomised treatment, baseline EQ-5D-5L VAS score, gender, age and country." | SAC [2] |

| Efficac | Efficacy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| PASAP | -Q | | | | |
| 2.66. | ITT | Non-Standard<br>EFF_T1 | Summary of PASAP-Q Scores | Present an additional column to the left of "Visit", labelled "Score" with values "Performance", "Convenience", "Overall Satisfaction", "Total Score" and "Willingness to Continue Using Inhaler" to allow presentation of results by Domain. Present the following visits: Week 12 and Early Withdrawal. Add the following footnotes: "Note: Performance, Convenience, Total Score, and Willingness to Continue Using Inhaler are expressed on a scale of 0 to 100. Note: Overall Satisfaction is expressed on a scale of 1 to 7." | SAC [2] |

# 12.15.7. Efficacy Figures

| Efficacy | Efficacy: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Change | from Baseline | in ACT Total Sco | re at Week 12 (Visit 4) | | |
| 2.1. | ITT | Non-Standard<br>EFF_F1 | Summary of Change from Baseline in ACT Total Score | Present "ACT Total Score" on y-axis and "Visit" on x-axis (Randomisation (Day 0), Week 6, Week 12, Week 18, Week 24). Present mean ACT Total Score ± SD separately for treatment group (FF/VI, Usual ICS/LABA) at each visit, connecting the means with a solid | Data Look [1]<br>SAC [2] |
| | | | | line. Distinguish the treatment groups by different line types. | |
| 2.2. | PP | Non-Standard<br>EFF_F1 | Summary of Change from Baseline in ACT Total Score<br>Per Protocol Population | Present "ACT Total Score" on y-axis and "Visit" on x-axis (Randomisation (Day 0), Week 6, Week 12, Week 18, Week 24). Present mean ACT Total Score ± SD separately for treatment group (FF/VI, Usual ICS/LABA) at each visit, connecting the means with a solid line. Distinguish the treatment groups by different line types. | SAC [2] |
| 2.3. | ITT | Non-Standard<br>EFF_F1 | Summary of Change from Baseline in ACT Total Score by Country | Present "ACT Total Score" on y-axis and "Visit" on x-axis (Randomisation (Day 0), Week 6, Week 12, Week 18, Week 24). Present mean ACT Total Score ± SD separately for treatment group (FF/VI, Usual ICS/LABA) at each visit, connecting the means with a solid line. Distinguish the treatment groups by different line types. | SAC [2] |

| Efficacy | /: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.4. | ITT/PP | Non-Standard<br>EFF_F2 | Summary of Primary and Sensitivity Analyses for Change from Baseline in ACT Total Score at Week 12 (Visit 4) | Present "Treatment difference" on the x-axis, and reverse axis so treatment difference increases from left to right. Replace "Ratio (95% CI)" with "Treatment Difference (95% CI)". Present lines for the following: Primary analysis (ITT), Primary analysis (PP), ANCOVA with LOCF (ITT), Multiple Imputation (Missing at Random) (ITT), Multiple Imputation (Copy Differences from Reference) (ITT), Hodges-Lehmann (ITT), ANCOVA with WOCF (ITT). | Data Look [1]<br>SAC [2] |
| 2.5. | ITT | Non-Standard<br>EFF_F3 | Summary of Interaction Tests for Change from Baseline in ACT Total Score at Week 12 (Visit 4) | Present "LS Mean Change" on the x-axis, and reverse axis so it increases from left to right. Replace "Ratio (95% CI)" with "LS Mean Change (95% CI)". Present the following subgroups: Country (France, Germany); Number of Severe Asthma Exacerbations in the Previous Year Prior to Randomisation (0, >= 1); Smoking Status at Baseline (Current smoker, Former smoker, Never smoked); Age Group (≤ 50 Years Old, > 50 Years Old); Gender (Male, Female). | Data Look [1]<br>SAC [2] |

| Efficacy | /: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Change | from Baseline | in ACT Total Sco | re at Week 24 (Visit 6) | | |
| 2.6. | ITT/PP | Non-Standard<br>EFF_F2 | Summary of Key Secondary and Sensitivity Analyses for Change from Baseline in ACT Total Score at Week 24 (Visit 6) | Present "Treatment difference" on the x-axis, and reverse axis so treatment difference increases from left to right. Replace "Ratio (95% CI)" with "Treatment Difference (95% CI)". Present lines for the following: Primary analysis (ITT), Primary analysis (PP), ANCOVA with LOCF (ITT), Multiple Imputation (Missing at Random) (ITT), Multiple Imputation (Copy Differences from Reference) (ITT), Hodges-Lehmann (ITT), ANCOVA with WOCF (ITT). | SAC [2] |
| Subject | s Who Have Ei | ither an ACT Total | Score >= 20 or >= 3 Point Increase from Baseline in ACT Total | Score | |
| 2.7. | ITT | Non-Standard<br>EFF_F4 | Summary of Percentage of Subjects Who Have Either an ACT Total Score >= 20 or >= 3 Point Increase from Baseline in ACT Total Score | Present "Percent of Subjects (%)" on y-axis and "Visit" on x-axis (Week 6, Week 12, Week 18, Week 24, Early Withdrawal). For each visit, present 3 vertical bars distinguished by fill pattern (similar to non-standard EFF_F6). Each bar represents: "ACT Total Score >= 20 or >= 3 Point Increase from Baseline in ACT Total Score", "ACT Total Score >= 20" and ">= 3 Point Increase from Baseline in ACT Total Score" respectively and should be labelled as such on the legend. | Data Look [1]<br>SAC [2] |

| Efficacy | Efficacy: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Complia | ance with Stud | y Medication | | | |
| 2.8. | ITT | Non-Standard<br>EFF_F5 | Box Plot of Compliance with Study Medication | Label y-axis title as "Compliance (%)", maximum of y-axis may be > 100%. | Data Look [1]<br>SAC [2] |
| MARS-A | A | | | | |
| 2.9. | ITT | Non-Standard<br>EFF_F6 | Histogram of the Questions and Answers of the MARS-A Questionnaire | Repeat on subsequent pages for Visit = Week 24, Week 52 and Early Withdrawal; and for Randomised Treatment = FF/VI. | Data Look [1]<br>SAC [2] |
| 2.10. | ITT | Non-Standard<br>EFF_F6 | Histogram of the Questions and Answers of the MARS-A Questionnaire by Status of Patient in Relation to the Reminder Sent to French Centres | Present bylines and footnotes per<br>"Repeat for" programming note on<br>shell. | SAC [2] |
| 2.11. | ITT | Non-Standard<br>EFF_F7 | Histogram of the Distribution of MARS-A Scores During the Study | Repeat on subsequent pages for Visit = Week 52 and Early Withdrawal. | Data Look [1]<br>SAC [2] |
| 2.12. | ITT | Non-Standard<br>EFF_F7 | Histogram of the Distribution of MARS-A Scores During the Study by Status of Patient in Relation to the Reminder Sent to French Centres | Present bylines and footnotes per<br>"Repeat for" programming note on<br>shell. | SAC [2] |
| Severe | On-Treatment | Asthma Exacerba | tions | | |
| 2.13. | ITT | Non-Standard<br>EFF_F8 | Box Plot of Severe On-Treatment Asthma Exacerbation Rates Adjusted for Exposure to Treatment | | Data Look [1]<br>SAC [2] |
| 2.14. | ITT | Non-Standard<br>EFF_F9 | Kaplan-Meier Plot of Time to First Severe On-Treatment Asthma Exacerbation | Display increments of 6 weeks on the x-axis, up to the maximum exposure (e.g. 0, 6, 12, 18, 24, 30). | Data Look [1]<br>SAC [2] |

# 12.15.8. Safety Tables

| Safety | : Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| SAEs a | nd ADRs | | | | |
| 3.1. | Safety | Non-Standard<br>SAFE_T1 | On-Treatment Serious Adverse Events and Adverse Drug Reactions Overview | Based on IDSL standard template AE13. | Data Look [1]<br>SAC [2] |
| 3.2. | Safety | AE1 | Summary of On-Treatment Non-Serious Adverse Drug Reactions | | SAC [2] |
| 3.3. | Safety | AE1 | Summary of On-Treatment Serious Adverse Drug Reactions | | SAC [2] |
| 3.4. | Safety | AE1 | Summary of On-Treatment Adverse Drug Reactions | | Data Look [1]<br>SAC [2] |
| 3.5. | Safety | AE1 | Summary of On-Treatment Serious Adverse Events | | Data Look [1]<br>SAC [2] |
| 3.6. | Safety | AE1 | Summary of On-Treatment or Post-Treatment Serious Adverse<br>Events and Adverse Drug Reactions Leading to Permanent<br>Discontinuation of Study Drug or Withdrawal from the Study | | SAC [2] |
| 3.7. | Safety | AE1 | Summary of On-Treatment or Post-Treatment Serious Adverse<br>Events Leading to Permanent Discontinuation of Study Drug or<br>Withdrawal from the Study | | SAC [2] |
| 3.8. | Safety | AE1 | Summary of On-Treatment or Post-Treatment Adverse Drug<br>Reactions Leading to Permanent Discontinuation of Study Drug<br>or Withdrawal from the Study | | SAC [2] |
| 3.9. | Safety | AE1 | Summary of Most Frequent On-Treatment Non-Serious Adverse Drug Reactions, Reported by 1% or More of Subjects in Any Treatment Group | | SAC [2] |

| Safety : Tables | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| SAEs a | nd ADRs of Sp | ecial Interest | | | |
| 3.10. | Safety | Non-Standard<br>SAFE_T2 | Summary of On-Treatment Non-Serious Adverse Drug Reactions of Special Interest | Based on IDSL standard template AE1. | Data Look [1]<br>SAC [2] |
| 3.11. | Safety | Non-Standard<br>SAFE_T2 | Summary of On-Treatment Serious Adverse Drug Reactions of Special Interest | Based on IDSL standard template AE1. | SAC [2] |
| 3.12. | Safety | Non-Standard<br>SAFE_T2 | Summary of On-Treatment Adverse Drug Reactions of Special Interest | Based on IDSL standard template AE1. | SAC [2] |
| 3.13. | Safety | Non-Standard<br>SAFE_T2 | Summary of On-Treatment Serious Adverse Events of Special Interest | Based on IDSL standard template AE1. | SAC [2] |
| Fatal S | AEs and ADRs | | | | |
| 3.14. | Safety | AE1 | Summary of On-Treatment Fatal Serious Adverse Events | | SAC [2] |
| 3.15. | Safety | AE1 | Summary of On-Treatment Fatal Serious Adverse Drug Reactions | | SAC [2] |
| 3.16. | Safety | Non-Standard<br>SAFE_T2 | Summary of On-Treatment Fatal Serious Adverse Events of Special Interest | Based on IDSL standard template AE1. | SAC [2] |
| Non-Fa | tal SAEs and A | DRs | | | |
| 3.17. | Safety | AE1 | Summary of On-Treatment Non-Fatal Serious Adverse Events | | SAC [2] |
| 3.18. | Safety | Non-Standard<br>SAFE_T2 | Summary of On-Treatment Non-Fatal Serious Adverse Events of Special Interest | Based on IDSL standard template AE1. | SAC [2] |
| Top Te | n Most Commo | nly Reported ADF | Rs | | |
| 3.19. | Safety | Non-Standard<br>SAFE_T3 | Top Ten Most Commonly Reported On-Treatment Adverse Drug Reactions Per Treatment Group | Present the ten most frequent preferred terms in Usual ICS/LABA, and the ten most frequent in FF/VI (do not use percentages to determine "most frequent") | Data Look [1]<br>SAC [2] |

| Safety : Tables | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Vital Si | Vital Signs | | | | |
| 3.20. | Safety | VS1 | Summary of Vital Signs | | SAC [2] |
| 3.21. | Safety | VS1 | Summary of Change from Baseline in Vital Signs | | SAC [2] |
| 3.22. | Safety | AE15 | Summary of Common (>=3%) Non-serious Adverse Events by System Organ Class and Preferred Term (Number of Subjects and Occurrences) | | SAC [2] |
| 3.23. | Safety | AE16 | Summary of Serious Adverse Events by System Organ Class and Preferred Term (Number of Subjects and Occurrences) | | SAC [2] |

# 12.15.9. Safety Figures

| Safety : Figures | | | | |
|---|---|---|---|---|
| No. | No. Population IDSL / TST ID / Example Shell Title Programming Notes Deliverable [Priority] | | | |
| Benefit | Benefit:Risk | | | |
| 3.1. | ITT/Safety | Non-Standard<br>SAFE_F1 | Summary of Benefit:Risk for FF/VI vs. Usual ICS/LABA | Data Look [1]<br>SAC [2] |

# 12.15.10. ICH Listings

| ICH : Listings | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Study F | opulation | | | | |
| 1. | ITT | ES2 | Reasons for Study Withdrawal | | SAC [2] |
| 2. | ITT | TA1 | Randomised and Actual Treatments | | SAC [2] |
| 3. | ITT | IE3 | Subjects with Inclusion, Exclusion or Randomisation Criteria Deviations | | SAC [2] |
| 4. | ITT | DM2 | Demographic Characteristics | | SAC [2] |
| 5. | ITT | DM9 | Race | | SAC [2] |
| Advers | e Events | | | | |
| 6. | Safety | AE7 | Subject Numbers for Individual Serious Adverse Events and Non-Serious Adverse Drug Reactions | | SAC [2] |
| 7. | Safety | AE8 | All Serious Adverse Events and Non-Serious Adverse Drug Reactions | | SAC [2] |
| 8. | Safety | AE8 | Fatal Serious Adverse Events | | SAC [2] |
| 9. | Safety | AE8 | Serious Adverse Events Leading to Permanent Discontinuation of Study Drug or Withdrawal from the Study | | SAC [2] |
| 10. | Safety | AE8 | Non-Serious Adverse Drug Reactions Leading to Permanent Discontinuation of Study Drug or Withdrawal from the Study | | SAC [2] |

# 12.15.11. Non-ICH Listings

| Non-ICH : Listings | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Study F | opulation | | | | |
| 11. | ASE | Non-Standard POP_L1 | Subjects Screened but Not in the Intent-to-Treat Population | | SAC [2] |
| 12. | ITT | Non-Standard<br>POP_L2 | Reasons for Important Protocol Deviations | | SAC [2] |
| 13. | ITT | MH2 | Medical Conditions | | SAC [2] |
| 14. | ITT | Non-Standard POP_L3 | Asthma History | | SAC [2] |
| 15. | ITT | Non-Standard<br>POP_L4 | Smoking History | | SAC [2] |
| 16. | ITT | CM3 | Concomitant Medications | Only include medications included in pre-treatment and on-treatment summary tables. | SAC [2] |
| 17. | ITT | CM6 | Relationship between Ingredient and Verbatim Text | | SAC [2] |
| 18. | ITT | Non-Standard<br>POP_L5 | Exposure to Study Medication | Repeat on subsequent pages for<br>Treatment = FF/VI, and use GSK drug<br>synonym as drug name. | SAC [2] |
| Efficac | y | | | | |
| 19. | ITT | Non-Standard<br>EFF_L1 | ACT Scores | Repeat on subsequent pages for Treatment = FF/VI. | SAC [2] |
| 20. | ITT | Non-Standard<br>EFF_L2 | Inhaler Device Use | Repeat on subsequent pages for Treatment = FF/VI. | SAC [2] |
| 21. | ITT | Non-Standard<br>EFF_L3 | Lung Function Tests | Repeat on subsequent pages for Treatment = FF/VI. | SAC [2] |

| Non-ICH: Listings | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 22. | ITT | Non-Standard<br>EFF_L4 | Medication Adherence Report Scale for Asthma (MARS-A)<br>Scores | Repeat on subsequent pages for Treatment = FF/VI. | SAC [2] |
| 23. | ITT | Non-Standard<br>EFF_L5 | Severe Asthma Exacerbations | Repeat on subsequent pages for Treatment = FF/VI. | SAC [2] |
| 24. | ITT | Non-Standard<br>EFF_L6 | AQLQ(S) Scores | Repeat on subsequent pages for Treatment = FF/VI. | SAC [2] |
| 25. | ITT | Non-Standard<br>EFF_L7 | EQ-5D-5L Descriptive System Dimension Scores | Repeat on subsequent pages for Treatment = FF/VI. | SAC [2] |
| 26. | ITT | Non-Standard<br>EFF_L8 | PASAP-Q Scores | Repeat on subsequent pages for Treatment = FF/VI. | SAC [2] |
| Safety | | | | | |
| 27. | Safety | Non-Standard<br>SAFE_L1 | AE Terms of Special Interest | The AE special interest dataset and the AE SMQ dataset will be set together in order to report this table and all the subgroups that come from the AE SMQ dataset will be flagged with a [1]. | SAC [2] |
| 28. | Safety | VS4 | Vital Signs | | SAC [2] |
| 29. | Safety | Non-Standard<br>SAFE_L2 | Inhaler Device Malfunctions | | SAC [2] |
| Liver C | hemistry | | | | |
| 30. | Safety | LIVER5 | Liver Event Results and Time of Event Relative to Treatment | | SAC [2] |
| 31. | Safety | LIVER6 | Liver Event Information for RUCAM Score | | SAC [2] |
| 32. | Safety | LIVER7 | Liver Biopsy Details | | SAC [2] |
| 33. | Safety | LIVER8 | Liver Imaging Details | | SAC [2] |

# 12.16. Appendix 16: Example Mock Shells for Data Displays

### 12.16.1. Study Population Table Shells

Example : POP\_T1
Protocol : HZA116492

Population : All Subjects Enrolled


Table 1.xx Summary of Subject Populations

| Population | Usual ICS/LABA | FF/VI | Total |
|-----------------------------|----------------|-----------|-----------|
| All Subjects Enrolled (ASE) | | | XXX |
| Randomised | XXX | XXX | XXX |
| Intent-to-Treat (ITT) | xxx (xx%) | xxx (xx%) | xxx (xx%) |
| Per Protocol (PP) | xxx (xx%) | xxx (xx%) | xxx (xx%) |
| Safety | xxx (xx%) | xxx (xx%) | xxx (xx%) |

ASE: All subjects screened and for whom a record exists on the study database.

ITT: All randomised subjects having received at least one dose of the prescription of study medication (FF/VI or Usual ICS/LABA).

PP: All ITT subjects who without any protocol deviations excluding them from this population.

Safety: All randomised subjects having received at least one dose of the prescription of study medication (FF/VI or Usual ICS/LABA).

Note: The randomised summary is not a defined population and consists of all subjects who were randomised and given a randomisation number.

Programming Note: randomised population line will provide the denominators for the ITT, PP and Safety percentages.

2017N339371\_00 HZA116492

Example : POP\_T2
Protocol : HZA116492
Population : Intent-to-Treat


Table 1.xx Summary of Attendance at Each Clinic Visit

| | Usual ICS/LABA<br>(N=xxx) | FF/VI<br>(N=xxx) | Total<br>(N=xxx) |
|---|---|---|---|
| Screening | xxx (xx%) | xxx (xx%) | xxx (xx%) |
| Randomisation (Day 0) | xxx (xx%) | xxx (xx%) | xxx (xx%) |
| Week 6 | xxx (xx%) | xxx (xx%) | xxx (xx%) |
| Week 12 | xxx (xx%) | xxx (xx%) | xxx (xx%) |
| Week 18 | xxx (xx%) | xxx (xx%) | xxx (xx%) |
| Week 24 | xxx (xx%) | xxx (xx%) | xxx (xx%) |
| Early Withdrawal | xxx (xx%) | xxx (xx%) | xxx (xx%) |

Note: Weeks 6 and 18 are telephone contacts.

Example : POP\_T3
Protocol : HZA116492
Population : Intent-to-Treat


Table 1.xx Summary of Important Protocol Deviations

| | Usual ICS/LABA<br>(N=xxx) | FF/VI<br>(N=xxx) | Total<br>(N=xxx) |
|---|---|---|---|
| Any Important Protocol Deviation | xxx (xx%) | xxx (xx%) | xxx (xx%) |
| Reason 1 | xxx (xx%) | xxx (xx%) | xxx (xx%) |
| Reason 2 | xxx (xx%) | xxx (xx%) | xxx (xx%) |
| Reason 3 | xxx (xx%) | xxx (xx%) | xxx (xx%) |
| | xxx (xx%) | xxx (xx%) | xxx (xx%) |

Note: A subject may have more than one protocol deviation. Note: Includes any important deviation from the protocol.

# Repeat for:

Summary of Important Protocol Deviations Resulting in Exclusion from the PP Population (ITT Population)

Example : POP\_T4

Protocol : HZA116492 Population : Intent-to-Treat 

Table 1.xx Summary of Asthma Duration at Baseline

| | Usual ICS/LABA | FF/VI | Total |
|-----------------------------|----------------|-----------|-----------|
| | (N=xxx) | (N=xxx) | (N=xxx) |
| Duration of Asthma | | | |
| < 6 months | xxx (xx%) | xxx (xx%) | xxx (xx%) |
| >= 6 months to < 1 year | xxx (xx%) | xxx (xx%) | xxx (xx%) |
| >= 1 year to < 5 years | xxx (xx%) | xxx (xx%) | xxx (xx%) |
| >= 5 years to < 10 years | xxx (xx%) | xxx (xx%) | xxx (xx%) |
| >= 10 years | xxx (xx%) | xxx (xx%) | xxx (xx%) |
| Duration of Asthma (years): | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | X.XX | X.XX | X.XX |
| Median | XX.X | XX.X | XX.X |
| Min. | XX | XX | XX |
| Max. | XX | XX | Xx |

# Repeat for:

Summary of Asthma Duration at Baseline (PP Population)

Example : POP\_T5
Protocol : HZA116492
Population : Intent-to-Treat


Table 1.xx Summary of Asthma Exacerbation History at Baseline

| | Usual ICS/LABA<br>(N=xxx) | FF/VI<br>(N=xxx) | Total<br>(N=xxx) |
|---|---|---|---|
| Did not require and/ovetonic continuatorside (not involving | | | |
| Did not require oral/systemic corticosteroids (not involving hospitalisation) | | | |
| n | XX | XX | XX |
| 0 | xx (xx%) | xx (xx%) | xx (xx%) |
| 1 | xx (xx%) | xx (xx%) | xx (xx%) |
| > 1 | xx (xx%) | xx (xx%) | xx (xx%) |
| Required oral/systemic corticosteroids (not involving hospitalisation) | | | |
| n | XX | XX | XX |
| 0 | xx (xx%) | xx (xx%) | xx (xx%) |
| 1 | xx (xx%) | xx (xx%) | xx (xx%) |
| > 1 | xx (xx%) | xx (xx%) | xx (xx%) |
| Required hospitalisation | | | |
| n | XX | XX | XX |
| 0 | xx (xx%) | xx (xx%) | xx (xx%) |
| 1 | xx (xx%) | xx (xx%) | xx (xx%) |
| >1 | xx (xx%) | xx (xx%) | xx (xx%) |

Note: Number of severe asthma exacerbations reported in the 12 months prior to Randomisation (Day 0).
Example : POP\_T5
Protocol : HZA116492
Population : Intent-to-Treat


Table 1.xx Summary of Asthma Exacerbation History at Baseline

| | Usual ICS/LABA | FF/VI | Total |
|---|---|---|---|
| | (N=xxx) | (N=xxx) | (N=xxx) |
| Total number of exacerbations during the 12 m randomisation | onths prior to | | |
| n | XX | XX | XX |
| 0 | xx (xx%) | xx (xx%) | xx (xx%) |
| 1 | xx (xx%) | xx (xx%) | xx (xx%) |
| >1 | xx (xx%) | xx (xx%) | xx (xx%) |
| Number of exacerbations during the 12 months | s prior to randomisation | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | X.XX | X.XX | X.XX |
| Median | XX.X | XX.X | XX.X |
| Min. | XX | XX | XX |
| Max. | XX | XX | XX |

Note: Number of severe asthma exacerbations reported in the 12 months prior to Randomisation (Day 0).

### Repeat for:

Summary of Asthma Exacerbation History at Baseline (PP Population)

Example : POP\_T6
Protocol : HZA116492
Population : Intent-to-Treat


Table 1.xx Summary of Smoking History at Baseline

| | | Usual ICS/LABA<br>(N=xxx) | FF/VI<br>(N=xxx) | Total<br>(N=xxx) |
|---|---|---|---|---|
| 11:1 | 0 1 | ( 0() | ( 0() | ( 0() |
| History of Smoking Use | Current smoker | xxx (xx%) | xxx (xx%) | xxx (xx%) |
| | Former smoker | xxx (xx%) | xxx (xx%) | xxx (xx%) |
| | Never smoked | xxx (xx%) | xxx (xx%) | xxx (xx%) |
| For Current and Former Smokers: | | | | |
| Years Smoked | n | XX | XX | XX |
| | Mean | XX.X | XX.X | XX.X |
| | SD | X.XX | X.XX | X.XX |
| | Median | XX.X | XX.X | XX.X |
| | Min. | XX | XX | XX |
| | Max. | XX | XX | XX |
| Cigarettes/Day | n | XX | xx | XX |
| ğ , | Mean | XX.X | XX.X | XX.X |
| | SD | X.XX | X.XX | X.XX |
| | Median | XX.X | XX.X | XX.X |
| | Min. | XX | XX | XX |
| | Max. | XX | XX | XX |

<sup>[1]</sup> Smoking Pack Years = (Number of cigarettes smoked per day/20) x number of years smoked.

Example : POP\_T6
Protocol : HZA116492
Population : Intent-to-Treat


Table 1.xx Summary of Smoking History at Baseline

| | Usual ICS/LABA<br>(N=xxx) | FF/VI<br>(N=xxx) | Total<br>(N=xxx) |
|---|---|---|---|
| n | VV | vv | XX |
| | | | XX.X |
| | | | X.XX |
| | | | XX.X |
| | | | XX |
| | | | XX |
| IVIAA. | ^^ | ** | ** |
| n | ΧΧ | XX | XX |
| | | | XX.X |
| | | | X.XX |
| | | | XX.X |
| | | | XX |
| | | | XX |
| Wax. | AA. | XX | XX |
| n | XX | XX | XX |
| | | | XX.X |
| | | | X.XX |
| | | | XX.X |
| | | | XX |
| | | | XX |
| | n<br>Mean<br>SD<br>Median<br>Min.<br>Max.<br>n<br>Mean<br>SD<br>Median<br>Min.<br>Max.<br>n<br>Mean<br>SD<br>Median<br>Min. | n XX Mean XX.X SD X.XX Median XX.X Min. XX Max. XX Mean XX.X Median XX.X Min. XX Mean XX.X Mean XX.X Median XX.X Median XX.X Median XX.X Median XX.X Median XX.X Min. XX | N XX XX Mean XX.X XX.X SD X.XX X.XX Median XX.X XX.X Min. XX XX Max. XX XX Mean XX.X XXX Median XX.X XX Min. XX XX Mean XX.X XX SD X.XX XXX Median XX.X XXX Median XX.X XXX Median XX.X XXX Median XX.X XX.X Min. XX XX.X |

<sup>[1]</sup> Smoking Pack Years = (Number of cigarettes smoked per day/20) x number of years smoked. **Repeat for:** Summary of Smoking History at Baseline (PP Population)

Example : POP\_T7
Protocol : HZA116492
Population : Intent-to-Treat


Table 1.xx Summary of Study Medication Dosage Modification

| Dosage Modification / Prescription | Usual ICS/LABA | FF/VI | Total |
|---|---|---|---|
| Treatment Path | (N=xxx) | (N=xxx) | (N=xxx) |
| Did Not Modify Dose During the Study | xxx (xx%) | xxx (xx%) | xxx (xx%) |
| Modified Dose at Least Once During the Study | xxx (xx%) | xxx (xx%) | xxx (xx%) |
| Randomised to FF/VI | | XXX | xxx |
| FF/VI 92 mcg/22 mcg OD | | xxx (xx%) | xxx (xx%) |
| FF/VI 92 mcg/22 mcg OD -> FF/VI 184 mcg/22 mcg OD | | xxx (xx%) | xxx (xx%) |
| Randomised to Usual ICS/LABA and Prescribed FP/S | XXX | | XXX |
| FP/S 250 mcg/50 mcg BID | xxx (xx%) | | xxx (xx%) |
| FP/S 250 mcg/50 mcg BID -> FP/S 500 mcg/50 mcg BID | xxx (xx%) | | xxx (xx%) |
| Randomised to Usual ICS/LABA and Prescribed BUD/F | XXX | | XXX |
| BUD/F 200 mcg/6 mcg BID (1 inh) | xxx (xx%) | xxx (xx%) | xxx (xx%) |
| BUD/F 200 mcg/6 mcg BID (1 inh) -> BUD/F 200 mcg/6 mcg BID (2 inh) | xxx (xx%) | xxx (xx%) | xxx (xx%) |
| BUD/F 200 mcg/6 mcg BID (1 inh) -> BUD/F 400 mcg/12 mcg BID (1 inh) | xxx (xx%) | xxx (xx%) | xxx (xx%) |
| BUD/F 200 mcg/6 mcg BID (2 inh) | xxx (xx%) | xxx (xx%) | xxx (xx%) |
| BUD/F 200 mcg/6 mcg BID (2 inh) -> BUD/F 400 mcg/12 mcg BID (1 inh) | xxx (xx%) | xxx (xx%) | xxx (xx%) |
| BUD/F 200 mcg/6 mcg BID (2 inh) -> BUD/F 400 mcg/12 mcg BID (2 inh) | xxx (xx%) | xxx (xx%) | xxx (xx%) |

Note: 1 inh = 1 inhalation per dose, 2 inh = 2 inhalations per dose.

Note: Subjects randomised to FF/VI initiated treatment on 92 mcg/22 mcg OD and could increase to 184 mcg/22 mcg OD.

Note: Subjects randomised to Usual ICS/LABA and prescribed FP/S initiated treatment on 250 mcg/50 mcg BID and could increase to 500 mcg/50 mcg BID.

### 2017N339371\_00 HZA116492


Note: Subjects randomised to Usual ICS/LABA and prescribed BUD/F could: initiate treatment on 200 mcg/6 mcg BID (1 inh) and increase to 200 mcg/6 mcg BID (2 inh) or 400 mcg/12 mcg BID (1 inh); or initiate on 200 mcg/6 mcg BID (2 inh) and modify to 400 mcg/12 mcg BID (1 inh) or increase to 400 mcg/12 mcg BID (2 inh).

Example : POP\_T8
Protocol : HZA116492
Population : Intent-to-Treat


Table 1.xx
Summary of Extent of Exposure to Study Medication (Regardless of Modification to Study Medication Dosage)

| Overall | | Usual ICS/LABA<br>(N=xxx) | FF/VI<br>(N=xxx) |
|---|---|---|---|
| Exposure (days) [1] | n<br>Mean<br>SD<br>Median<br>Min.<br>Max. | XX<br>XX.X<br>X.XX<br>XX.X<br>XX | XX<br>XX.X<br>X.XX<br>XX.X<br>XX |
| Total Years Exposed (yrs) | | xx | xx |
| Range of Exposure (days) | <= 6 weeks <= 12 weeks <= 18 weeks <= 24 weeks > 24 weeks | xxx (xx%)<br>xxx (xx%)<br>xxx (xx%)<br>xxx (xx%)<br>xxx (xx%) | xxx (xx%)<br>xxx (xx%)<br>xxx (xx%)<br>xxx (xx%)<br>xxx (xx%) |
| Subjects Exposed for six months (24 weeks ± 2 weeks) | | xxx (xx%) | xxx (xx%) |

<sup>[1]</sup> Exposure to study medication = treatment stop date – treatment start date + 1, regardless of dosage modification.

### Repeat for:

Summary of Summary of Extent of Exposure to Study Medication (up to First Modification to Study Medication Dosage) (ITT Population)
Footnote: "[1] Exposure to study medication = treatment stop date - treatment start date + 1."

Example : POP\_T9
Protocol : HZA116492
Population : Intent-to-Treat


Table 1.xx
Summary of Extent of Exposure to Study Medication by Medication and Dosage

| Medication/Dosage | Overall | | Usual ICS/LABA<br>(N=xxx) | FF/VI<br>(N=xxx) |
|---|---|---|---|---|
| FF/VI 92 mcg/22 mcg OD | Exposure (days) [1] | n<br>Mean<br>SD<br>Median<br>Min.<br>Max. | XX<br>XX.X<br>X.XX<br>XX.X<br>XX | XX<br>XX.X<br>X.XX<br>XX.X<br>XX |
| | Total Years Exposed (yrs) | | xx | xx |
| | Range of Exposure (days) | <= 6 weeks <= 12 weeks <= 18 weeks <= 24 weeks > 24 weeks | xxx (xx%)<br>xxx (xx%)<br>xxx (xx%)<br>xxx (xx%)<br>xxx (xx%) | xxx (xx%)<br>xxx (xx%)<br>xxx (xx%)<br>xxx (xx%)<br>xxx (xx%) |
| | Subjects Exposed for six months (24 weeks ± 2 weeks) | | xxx (xx%) | xxx (xx%) |

<sup>[1]</sup> Exposure to study medication = treatment stop date – treatment start date + 1.

Programming note: repeat on subsequent pages for Medication/Dosage = FF/VI 184 mcg/22 mcg OD, FP/S 250 mcg/50 mcg BID, FP/S 500 mcg/50 mcg BID, BUD/F 200 mcg/6 mcg BID (1 inhalation per dose), BUD/F 400 mcg/12 mcg BID (1 inhalation per dose), BUD/F 400 mcg/12 mcg BID (2 inhalations per dose).

Example : POP\_T10
Protocol : HZA116492
Population : Intent-to-Treat


Table 1.xx Summary of Number of Subjects by Subgroup

| | Usual ICS/LABA<br>(N=xxx) | FF/VI<br>(N=xxx) | Total<br>(N=xxx) |
|---|---|---|---|
| Country | | | |
| n | XXX | XXX | XXX |
| France | xxx (xx%) | xxx (xx%) | xxx (xx%) |
| Germany | xxx (xx%) | xxx (xx%) | xxx (xx%) |
| Number of Severe Asthma Exacerbations in the Previous Year Prior to Randomisation | | | |
| n | XXX | XXX | XXX |
| 0 | xxx (xx%) | xxx (xx%) | xxx (xx%) |
| >= 1 | xxx (xx%) | xxx (xx%) | xxx (xx%) |
| Smoking Status at Baseline | | | |
| n | XXX | XXX | XXX |
| Current smoker | xxx (xx%) | xxx (xx%) | xxx (xx%) |
| Former smoker | xxx (xx%) | xxx (xx%) | xxx (xx%) |
| Never smoked | xxx (xx%) | xxx (xx%) | xxx (xx%) |
| Age Group | | | |
| n | XXX | XXX | XXX |
| ≤ 50 years old | xxx (xx%) | xxx (xx%) | xxx (xx%) |
| > 50 years old | xxx (xx%) | xxx (xx%) | xxx (xx%) |
| , | ( ' ' ' ) | ( , , , ) | ( = 1, 1) |

Note: Spring = March, April and May; Summer = June, July and August; Autumn = September, October and November; Winter = December, January and February.

Example : POP\_T10
Protocol : HZA116492
Population : Intent-to-Treat


Table 1.xx
Summary of Number of Subjects by Subgroup

| | Usual ICS/LABA<br>(N=xxx) | FF/VI<br>(N=xxx) | Total<br>(N=xxx) |
|---|---|---|---|
| Gender | | | |
| n | XXX | XXX | XXX |
| Male | xxx (xx%) | xxx (xx%) | xxx (xx%) |
| Female | xxx (xx%) | xxx (xx%) | xxx (xx%) |
| Season at randomisation | | | |
| n | XXX | XXX | XXX |
| Spring | xxx (xx%) | xxx (xx%) | xxx (xx%) |
| Summer | xxx (xx%) | xxx (xx%) | xxx (xx%) |
| Autumn | xxx (xx%) | xxx (xx%) | xxx (xx%) |
| Winter | xxx (xx%) | xxx (xx%) | xxx (xx%) |

Note: Spring = March, April and May; Summer = June, July and August; Autumn = September, October and November; Winter = December, January and February.

### 12.16.2. Study Population Figure Shells

Example : POP\_F1
Protocol : HZA116492
Population : Intent-to-Treat


Figure 1.xx
Plot of Exposure to Study Medication (Regardless of Modification to Study Medication Dosage)



Programming note: display increments of 6 weeks on the x-axis, up to the maximum exposure (e.g. 0, 6, 12, 18, 24, 30).

### 12.16.3. Efficacy Table Shells

Example : EFF\_T1
Protocol : HZA116492
Population : Intent-to-Treat


Table 2.xx Summary of Change from Baseline in ACT Total Score

| Visit | | Usual ICS/LABA<br>(N=xxx) | FF/VI<br>(N=xxx) |
|---|---|---|---|
| Randomisation (Day 0) | n | xx | XX |
| , , | Mean | XX.X | XX.X |
| | SD | X.XX | X.XX |
| | Median | XX.X | XX.X |
| | Min. | XX | XX |
| | Max. | XX | XX |
| Week 6 | n | XX | XX |
| | Mean | XX.X | XX.X |
| | SD | X.XX | X.XX |
| | Median | XX.X | XX.X |
| | Min. | XX | XX |
| | Max. | XX | XX |
| Change from Baseline at Week 6 | n | XX | XX |
| <b>G</b> | Mean | XX.X | XX.X |
| | SD | X.XX | X.XX |
| | Median | XX.X | XX.X |

Min. xx xx xx Max. xx xx

Programming note: repeat for Week 12, Change from Baseline at Week 12, Week 18, Change from Baseline at Week 24, Change from Baseline at Week 24, Early Withdrawal, Change from Baseline at Early Withdrawal

### Repeat for:

Summary of Change from Baseline in ACT Total Score Per Protocol Population (PP Population)

Summary of Change from Baseline in Lung Function Tests (ITT Population)

Programming note: Present an additional column to the left of "Visit", labelled "Test" with values "Trough (Pre-dose) FEV1 (L)" and "Trough (Pre-dose) Percent Predicted FEV1 (%)" to allow presentation of results by Test. Present the following visits: Randomisation (Day 0), Week 12, Change from Baseline at Week 12, Early Withdrawal and Change from Baseline at Early Withdrawal.

Summary of Change from Baseline in AQLQ(S) Total Score and Domain Scores (ITT Population)

Programming note: Present an additional column to the left of "Visit", labelled "Domain" with values "Total Score", "Environmental Stimuli", "Symptoms", "Activity Limitations", "Emotional Function" to allow presentation of results by Domain. Present the following visits: Randomisation (Day 0), Week 24, Change from Baseline at Week 24, Early Withdrawal and Change from Baseline at Early Withdrawal.

Summary of PASAP-Q Scores (ITT Population)

Programming note: Present an additional column to the left of "Visit", labelled "Score" with values "Performance", "Convenience", "Total Score", "Overall Satisfaction", and "Willingness to Continue Using Inhaler" to allow presentation of results by Domain. Present the following visits: Week 12 and Early Withdrawal.

Add the following footnotes:

"Note: Performance, Convenience, Total Score, and Willingness to Continue Using Inhaler are expressed on a scale of 0 to 100. Note: Overall Satisfaction is expressed on a scale of 1 to 7."

Summary of EQ-5D-5L Utility Score (ITT Population)

Summary of EQ-5D-5L Visual Analogue Scale (VAS) Score (ITT Population)

Programming note: Present the following visits: Randomisation (Day 0), Week 24, Change from Baseline at Week 24, Early Withdrawal, Change from Baseline at Early Withdrawal.

Example : EFF\_T1S
Protocol : HZA116492
Population : Intent-to-Treat


## Table 2.xx

Summary of Change from Baseline in ACT Total Score by Country

Country: France

| Visit | | Usual ICS/LABA<br>(N=xxx) | FF/VI<br>(N=xxx) |
|---|---|---|---|
| Randomisation (Day 0) | n | XX | XX |
| | Mean | XX.X | XX.X |
| | SD | X.XX | X.XX |
| | Median | XX.X | XX.X |
| | Min. | XX | XX |
| | Max. | XX | XX |
| Week 6 | n | XX | XX |
| | Mean | XX.X | XX.X |
| | SD | X.XX | X.XX |
| | Median | XX.X | XX.X |
| | Min. | XX | XX |
| | Max. | XX | XX |
| Change from Baseline at Week 6 | n | XX | vv |
| Change nom baseline at week o | | | XX |
| | Mean | XX.X | XX.X |
| | SD | X.XX | X.XX |
| | Median | XX.X | XX.X |
| | Min. | XX | XX |
| | Max. | XX | XX |

Example : EFF\_T1S
Protocol : HZA116492
Population : Intent-to-Treat


# Table 2.xx Summary of Change from Baseline in ACT Total Score by Country

Country: Germany

| Visit | | Usual ICS/LABA<br>(N=xxx) | FF/VI<br>(N=xxx) |
|---|---|---|---|
| Randomisation (Day 0) | n | XX | XX |
| , , | Mean | XX.X | XX.X |
| | SD | X.XX | X.XX |
| | Median | XX.X | XX.X |
| | Min. | XX | XX |
| | Max. | XX | XX |
| Week 6 | n | XX | XX |
| | Mean | XX.X | XX.X |
| | SD | X.XX | X.XX |
| | Median | XX.X | XX.X |
| | Min. | XX | XX |
| | Max. | XX | XX |
| Change from Baseline at Week 6 | n | XX | XX |
| | Mean | XX.X | XX.X |
| | SD | X.XX | X.XX |
| | Median | XX.X | XX.X |
| | Min. | XX | XX |
| | Max. | XX | XX |

### Repeat for:

Summary of Change from Baseline in ACT Total Score by Number of Severe Asthma Exacerbations in the Previous Year Prior to Randomisation (ITT Population)

Number of Severe Asthma Exacerbations in the Previous Year Prior to Randomisation: 0

Number of Severe Asthma Exacerbations in the Previous Year Prior to Randomisation: >= 1

Summary of Change from Baseline in ACT Total Score by Smoking Status at Baseline (ITT Population)

Smoking Status at Baseline: Current smoker Smoking Status at Baseline: Former smoker Smoking Status at Baseline: Never smoked

Summary of Change from Baseline in ACT Total Score by Age Group (ITT Population)

Age Group: ≤ 50 Years Old Age Group: > 50 Years Old

Summary of Change from Baseline in ACT Total Score by Gender (ITT Population)

Gender: Male Gender: Female Example : EFF\_T2 Protocol : HZA116492

: Intent-to-Treat

Population


Table 2.xx

Summary of the Statistical Analysis of Change from Baseline in ACT Total Score at Week 12 (Visit 4)

| | Usual ICS/LABA<br>(N=xxx) | FF/VI<br>(N=xxx) |
|---|---|---|
| n<br>LS Mean Change (SE) | xx<br>xx.xx (x.xxx) | xx<br>xx.xx (x.xxx) |
| FF/VI vs. Usual ICS/LABA<br>Difference | | XX.X |
| 95% CI<br>p-value | | (xx.x, xx.x)<br>x.xxx |

Note: The analysis method was an MMRM adjusted for randomised treatment, visit (Week 6 and Week 12), baseline ACT total score, randomised treatment-by-visit interaction, baseline ACT total score-by-visit interaction, gender, age, country and patient fitted as a random factor.

Note: The Restricted Maximum Likelihood (REML) estimation approach was used with a default covariance structure of unstructured.

Programming note: Should computational issues be encountered when using an unstructured covariance structure, other structures including AR1 and CS should be considered and the second footnote updated as appropriate. Should the distributional assumption of normality fail then the p-value from a model on the rank-transformed values should be presented and the following footnote added: "Note: the p-value presented was obtained from an MMRM on the rank-transformed values of change from baseline in ACT total score at Week 12 (Visit 4) with the same specification as the untransformed model."

### Repeat for:

Summary of the Statistical Analysis of Change from Baseline in ACT Total Score at Week 12 (Visit 4) Per Protocol Population (PP Population)

Summary of the Statistical Analysis of Change from Baseline in ACT Total Score at Week 12 (Visit 4) (ANCOVA with LOCF) (ITT Population)

Programming note: Should the distributional assumption of normality fail then the p-value from a model on the rank-transformed values should be presented and the following footnote added: "Note: the p-value presented was obtained from an ANCOVA on the rank-transformed values of change from baseline in ACT total score at Week 12 (Visit 4) with the same specification as the untransformed model."

Footnotes as follows:

"Note: The analysis method was an ANCOVA model adjusted for randomised treatment, baseline ACT total score, gender, age and country.

Note: Missing values at Week 12 (Visit 4) were replaced by last available post-randomisation value based on the last observation carried forward (LOCF) method."

Summary of the Statistical Analysis of Change from Baseline in ACT Total Score at Week 12 (Visit 4) (Multiple Imputation – Missing at Random Approach) (ITT Population)

Summary of the Statistical Analysis of Change from Baseline in ACT Total Score at Week 12 (Visit 4) (Multiple Imputation – Copy Differences from Reference Approach) (ITT Population)

Programming note: Present the "FF/VI vs. Usual ICS/LABA" section only. Footnotes as follows:

"Note: Missing values post-randomisation were imputed using multiple imputation methods based on pattern mixture models.

Note: Each imputed data set was analysed using an ANCOVA model at Week 12 (Visit 4) adjusted for randomised treatment, baseline ACT total score, gender, age and country and the resulting treatment differences and their standard errors combined using Rubin's rules."

Summary of the Statistical Analysis of Change from Baseline in ACT Total Score at Week 12 (Visit 4) (Hodges-Lehmann Approach) (ITT Population)

Programming note: Present the "Difference" and "95% CI" lines of "FF/VI vs. Usual ICS/LABA" section only. Footnotes as follows:

"Note: The difference between treatment groups at Week 12 (Visit 4) was calculated using the Hodges-Lehmann approach."

Summary of the Statistical Analysis of Change from Baseline in ACT Total Score at Week 12 (Visit 4) (ANCOVA with WOCF) (ITT Population)

Programming note: Should the distributional assumption of normality fail then the p-value from a model on the rank-transformed values should be presented and the following footnote added: "Note: the p-value presented was obtained from an ANCOVA on the rank-transformed values of change from baseline in ACT total score at Week 12 (Visit 4) with the same specification as the untransformed model."

Footnotes as follows:

"Note: The analysis method was an ANCOVA model adjusted for randomised treatment, baseline ACT total score, gender, age and country.

Note: Missing values at Week 12 (Visit 4) due to treatment withdrawal prior to this time point were replaced by worst post-randomisation value based on the worst observation carried forward (WOCF) method."

Summary of the Statistical Analysis of Change from Baseline in ACT Total Score at Week 12 (Visit 4), FF/VI Versus the Subset of Usual ICS/LABA Subjects Prescribed FP/S at Randomisation (ITT Population)

Summary of the Statistical Analysis of Change from Baseline in ACT Total Score at Week 12 (Visit 4), FF/VI Versus the Subset of Usual ICS/LABA Subjects Prescribed BUD/F at Randomisation (ITT Population)

Summary of the Statistical Analysis of Change from Baseline in ACT Total Score at Week 24 (Visit 6) (ITT Population)

Summary of the Statistical Analysis of Change from Baseline in ACT Total Score at Week 24 (Visit 6) Per Protocol Population (PP Population)

Programming note: first footnote as follows:

"Note: The analysis method was an MMRM adjusted for randomised treatment, visit (Week 6, Week 12, Week 18 and Week 24), baseline ACT total score, randomised treatment-by-visit interaction, baseline ACT total score-by-visit interaction, gender, age, country and patient fitted as a random factor."

Summary of the Statistical Analysis of Change from Baseline in ACT Total Score at Week 24 (Visit 6) (ANCOVA with LOCF) (ITT Population)

Programming note: Should the distributional assumption of normality fail then the p-value from a model on the rank-transformed values should be presented and the following footnote added: "Note: the p-value presented was obtained from an ANCOVA on the rank-transformed values of change from baseline in ACT total score at Week 24 (Visit 6) with the same specification as the untransformed model."

Footnotes as follows:

"Note: The analysis method was an ANCOVA model adjusted for randomised treatment, baseline ACT total score, gender, age and country.

Note: Missing values at Week 24 (Visit 6) were replaced by last available post-randomisation value based on the last observation carried forward (LOCF) method."

Summary of the Statistical Analysis of Change from Baseline in ACT Total Score at Week 24 (Visit 6) (Multiple Imputation – Missing at Random Approach) (ITT Population)

Summary of the Statistical Analysis of Change from Baseline in ACT Total Score at Week 24 (Visit 6) (Multiple Imputation – Copy Differences from Reference Approach) (ITT Population)

Programming note: Present the "FF/VI vs. Usual ICS/LABA" section only. Footnotes as follows:

"Note: Missing values post-randomisation were imputed using multiple imputation methods based on pattern mixture models.

Note: Each imputed data set was analysed using an ANCOVA model at Week 24 (Visit 6) adjusted for randomised treatment, baseline ACT total score, gender, age and country and the resulting treatment differences and their standard errors combined using Rubin's rules."

Summary of the Statistical Analysis of Change from Baseline in ACT Total Score at Week 24 (Visit 6) (Hodges-Lehmann Approach) (ITT Population)

Present the "Difference" and "95% CI" lines of "FF/VI vs. Usual ICS/LABA" section only. Footnotes as follows:

"Note: The difference between treatment groups at Week 24 (Visit 6) was calculated using the Hodges-Lehmann approach."

Summary of the Statistical Analysis of Change from Baseline in ACT Total Score at Week 24 (Visit 6) (ANCOVA with WOCF) (ITT Population)

Programming note: Should the distributional assumption of normality fail then the p-value from a model on the rank-transformed values should be presented and the following footnote added: "Note: the p-value presented was obtained from an ANCOVA on the rank-transformed values of change from baseline in ACT total score at Week 24 (Visit 6) with the same specification as the untransformed model."

Footnotes as follows:

"Note: The analysis method was an ANCOVA model adjusted for randomised treatment, baseline ACT total score, gender, age and country.

Note: Missing values at Week 24 (Visit 6) due to treatment withdrawal prior to this time point were replaced by worst post-randomisation value based on the worst observation carried forward (WOCF) method."

Summary of the Statistical Analysis of Change from Baseline in ACT Total Score at Week 24 (Visit 6), FF/VI Versus the Subset of Usual ICS/LABA Subjects Prescribed FP/S at Randomisation (ITT Population)

Programming note: Output only to be produced if ≥25% of Usual ICS/LABA patients are prescribed FP/S at randomisation. First footnote as follows: "Note: The analysis method was an MMRM adjusted for randomised treatment, visit (Week 6, Week 12, Week 18 and Week 24), baseline ACT total score, randomised treatment-by-visit interaction, baseline ACT total score-by-visit interaction, gender, age, country and patient fitted as a random factor."

Summary of the Statistical Analysis of Change from Baseline in ACT Total Score at Week 24 (Visit 6), FF/VI Versus the Subset of Usual ICS/LABA Subjects Prescribed BUD/F at Randomisation (ITT Population)

Programming note: Output only to be produced if ≥25% of Usual ICS/LABA patients are prescribed BUD/F at randomisation. First footnote as follows:

"Note: The analysis method was an MMRM adjusted for randomised treatment, visit (Week 6, Week 12, Week 18 and Week 24), baseline ACT total score, randomised treatment-by-visit interaction, baseline ACT total score-by-visit interaction, gender, age, country and patient fitted as a random factor."

Summary of the Statistical Analysis of Change from Baseline in Trough (Pre-dose) FEV1 at Week 12 (Visit 4) (ITT Population)

Programming note: Should the distributional assumption of normality fail then the p-value from a model on the rank-transformed values should be presented and the following footnote added: "Note: the p-value presented was obtained from an ANCOVA on the rank-transformed values of change from baseline in trough (pre-dose) FEV1 at Week 12 (Visit 4) with the same specification as the untransformed model."

Footnote as follows:

"Note: The analysis method was an ANCOVA model adjusted for randomised treatment, baseline trough (pre-dose) FEV1, gender, age and country."

Summary of the Statistical Analysis of Change from Baseline in EQ-5D-5L Utility Score at Week 24 (Visit 6) (ITT Population)

Programming note: Should the distributional assumption of normality fail then the p-value from a model on the rank-transformed values should be presented and the following footnote added: "Note: the p-value presented was obtained from an ANCOVA on the rank-transformed values of change from baseline in EQ-5D-5L utility score at Week 24 (Visit 6) with the same specification as the untransformed model."

Footnote as follows:

"Note: The analysis method was an ANCOVA model adjusted for randomised treatment, baseline EQ-5D-5L utility score, gender, age and country."

Summary of the Statistical Analysis of Change from Baseline in EQ-5D-5L Visual Analogue Scale (VAS) Score at Week 24 (Visit 6) (ITT Population)

Programming note: Should the distributional assumption of normality fail then the p-value from a model on the rank-transformed values should be presented and the following footnote added: "Note: the p-value presented was obtained from an ANCOVA on the rank-transformed values of change from baseline in EQ-5D-5L VAS score at Week 24 (Visit 6) with the same specification as the untransformed model."

Footnote as follows:

"Note: The analysis method was an ANCOVA model adjusted for randomised treatment, baseline EQ-5D-5L VAS score, gender, age and country."

2017N339371\_00 HZA116492


Example : EFF\_T2S Protocol : HZA116492

Population : Intent-to-Treat

Table 2.xx

Summary of the Statistical Analysis of Change from Baseline in ACT Total Score at Week 12 (Visit 4) by Country

### Country: France

| | Usual ICS/LABA<br>(N=xxx) | FF/VI<br>(N=xxx) |
|---|---|---|
| n<br>LS Mean Change (SE) | xx<br>xx.xx (x.xxx) | xx<br>xx.xx (x.xxx) |
| FF/VI vs. Usual ICS/LABA<br>Difference<br>95% CI | | xx.x<br>(xx.x, xx.x) |

Note: The analysis method was an MMRM adjusted for randomised treatment, visit (Week 6 and Week 12), baseline ACT total score, baseline ACT total score-by-visit interaction, gender, age, country, two- and three- way interactions between randomised treatment, visit and country, and patient fitted as a random factor.

Note: The Restricted Maximum Likelihood (REML) estimation approach was used with a default covariance structure of unstructured.

2017N339371\_00 HZA116492


Example : EFF\_T2S Protocol : HZA116492

Population : Intent-to-Treat

Table 2.xx

Summary of the Statistical Analysis of Change from Baseline in ACT Total Score at Week 12 (Visit 4) by Country

### Country: Germany

| | Usual ICS/LABA<br>(N=xxx) | FF/VI<br>(N=xxx) |
|---|---|---|
| n<br>LS Mean Change (SE) | xx<br>xx.xx (x.xxx) | xx<br>xx.xx (x.xxx) |
| FF/VI vs. Usual ICS/LABA<br>Difference<br>95% CI | | xx.x<br>(xx.x, xx.x) |

Note: The analysis method was an MMRM adjusted for randomised treatment, visit (Week 6 and Week 12), baseline ACT total score, randomised treatment-by-visit interaction, baseline ACT total score-by-visit interaction, gender, age, country, randomised treatment-by-country interaction and patient fitted as a random factor. Note: The Restricted Maximum Likelihood (REML) estimation approach was used with a default covariance structure of unstructured.

Programming note: Should computational issues be encountered when using an unstructured covariance structure, other structures including AR1 and CS should be considered and the second footnote updated as appropriate.

#### Repeat for:

Summary of the Statistical Analysis of Change from Baseline in ACT Total Score at Week 12 (Visit 4) by Number of Severe Asthma Exacerbations in the Previous Year Prior to Randomisation (ITT Population)

Number of Severe Asthma Exacerbations in the Previous Year Prior to Randomisation: 0

Number of Severe Asthma Exacerbations in the Previous Year Prior to Randomisation: >= 1

Programming note: first footnote as follows:

"Note: The analysis method was an MMRM adjusted for randomised treatment, visit (Week 6 and Week 12), baseline ACT total score, baseline ACT total score-by-visit interaction, gender, age, country, number of severe asthma exacerbations in the previous year prior to randomisation, two- and three- way interactions between randomised treatment, visit and number of severe asthma exacerbations in the previous year prior to randomisation, and patient fitted as a random factor."

Summary of the Statistical Analysis of Change from Baseline in ACT Total Score at Week 12 (Visit 4) by Smoking Status at Baseline (ITT Population) Programming note: first footnote as follows:

"Note: The analysis method was an MMRM adjusted for randomised treatment, visit (Week 6 and Week 12), baseline ACT total score, baseline ACT total score-by-visit interaction, gender, age, country, smoking status at baseline, two- and three- way interactions between randomised treatment, visit and smoking status at baseline, and patient fitted as a random factor."

Summary of the Statistical Analysis of Change from Baseline in ACT Total Score at Week 12 (Visit 4) by Age Group (ITT Population) Programming note: first footnote as follows:

"Note: The analysis method was an MMRM adjusted for randomised treatment, visit (Week 6 and Week 12), baseline ACT total score, baseline ACT total score-by-visit interaction, gender, country, age group, two- and three- way interactions between randomised treatment, visit and age group, and patient fitted as a random factor."

Summary of the Statistical Analysis of Change from Baseline in ACT Total Score at Week 12 (Visit 4) by Gender (ITT Population) Programming note: first footnote as follows:

"Note: The analysis method was an MMRM adjusted for randomised treatment, visit (Week 6 and Week 12), baseline ACT total score, baseline ACT total score-by-visit interaction, gender, age, country, two- and three- way interactions between randomised treatment, visit and gender, and patient fitted as a random factor."

Summary of the Statistical Analysis of Change from Baseline in ACT Total Score at Week 24 (Visit 6) by Country (ITT Population) Programming note: first footnote as follows:

"Note: The analysis method was an MMRM adjusted for randomised treatment, visit (Week 6, Week 12, Week 18 and Week 24), baseline ACT total score, baseline ACT total score-by-visit interaction, gender, age, country, two- and three- way interactions between randomised treatment, visit and country, and patient fitted as a random factor."

2017N339371\_00 HZA116492

Example : EFF\_T3
Protocol : HZA116492

Population


: Intent-to-Treat

Table 2.xx

Summary of the Statistical Analysis of Change from Baseline in ACT Total Score at Week 12 (Visit 4), Adjusting for Seasonal Effect

| | Usual ICS/LABA<br>(N=xxx) | FF/VI<br>(N=xxx) |
|---|---|---|
| Randomised treatment-by-season at randomisation interaction p-value | | X.XXX |
| Season at randomisation: Spring<br>n<br>LS Mean Change (SE) | xx<br>xx.xx (x.xxx) | xx<br>xx.xx (x.xxx) |
| FF/VI vs. Usual ICS/LABA<br>Difference<br>95% CI | | xx.x<br>(xx.x, xx.x) |

Note: The analysis method was an MMRM adjusted for randomised treatment, visit (Week 6 and Week 12), baseline ACT total score, baseline ACT total score-by-visit interaction, gender, age, country, season at randomisation, two- and three- way interactions between randomised treatment, visit and season at randomisation, and patient fitted as a random factor.

Note: The Restricted Maximum Likelihood (REML) estimation approach was used with a default covariance structure of unstructured.

Note: Spring = March, April and May; Summer = June, July and August; Autumn = September, October and November; Winter = December, January and February.

Programming note: repeat on subsequent pages for Season at randomisation = Summer, Autumn, Winter. Should computational issues be encountered when using an unstructured covariance structure, other structures including AR1 and CS should be considered and the second footnote updated as appropriate.

### Repeat for:

Summary of the Statistical Analysis of Change from Baseline in ACT Total Score at Week 12 (Visit 4), Adjusting for Seasonal Effect Per Protocol Population (PP Population)

Summary of the Statistical Analysis of Change from Baseline in ACT Total Score at Week 24 (Visit 6), Adjusting for Seasonal Effect (ITT Population)
Summary of the Statistical Analysis of Change from Baseline in ACT Total Score at Week 24 (Visit 6), Adjusting for Seasonal Effect Per Protocol Population (PP Population)

First footnote as follows:

"Note: The analysis method was an MMRM adjusted for randomised treatment, visit (Week 6, Week 12, Week 18 and Week 24), baseline ACT total score, baseline ACT total score-by-visit interaction, gender, age, country, season at randomisation, two- and three- way interactions between randomised treatment, visit and season at randomisation, and patient fitted as a random factor."

Example : EFF\_T4
Protocol : HZA116492
Population : Intent-to-Treat


### Table 2.xx Summary of Inhaler Device Use Errors

| Visit | | Usual ICS/LABA<br>(N=xxx) | FF/VI<br>(N=xxx) |
|---|---|---|---|
| Randomisation (Day 0) | Number of patients using Ellipta | | xxx |
| | Number of patients with correct use [1] | | xxx (xx%) |
| | Number of patients without correct use | | xxx (xx%) |
| | Number of patients with at least one critical error Type of critical error: | | xxx (xx%) |
| | Failed to open cover | | xxx (xx%) |
| | Shook the device upside down after dose preparation Exhaled directly into mouthpiece | | xxx (xx%)<br>xxx (xx%) |
| | No seal by the lips around the mouthpiece during the inhalation | | xxx (xx%) |
| | Number of patients with at least one non-critical error Type of non-critical error: | | xxx (xx%) |
| | No exhalation before an inhalation | | xxx (xx%) |
| | Inhalation manoeuvre was not: long, steady and deep | | xxx (xx%) |
| | Blocked air inlet during inhalation manoeuvre | | xxx (xx%) |
| | Did not hold breath | | XXX (XX%) |
| | Did not close the device | | xxx (xx%) |

<sup>[1]</sup> Correct use is defined as not making any critical or non-critical errors at that visit.

Example : EFF\_T4
Protocol : HZA116492
Population : Intent-to-Treat


### Table 2.xx Summary of Inhaler Device Use Errors

| Visit | | Usual ICS/LABA<br>(N=xxx) | FF/VI<br>(N=xxx) |
|---|---|---|---|
| Randomisation (Day 0) | Number of patients using Diskus | xxx | |
| | Number of patients with correct use [1] | xxx (xx%) | |
| | Number of patients without correct use | xxx (xx%) | |
| | Number of patients with at least one critical error Type of critical error: | xxx (xx%) | |
| | Failed to open cover | xxx (xx%) | |
| | Lever is not pushed back | xxx (xx%) | |
| | Shook the device after dose preparation | xxx (xx%) | |
| | Exhaled directly into mouthpiece | xxx (xx%) | |
| | No seal by the lips around the mouthpiece during the inhalation | xxx (xx%) | |
| | Number of patients with at least one non-critical error Type of non-critical error: | xxx (xx%) | |
| | No exhalation before an inhalation | xxx (xx%) | |
| | Inhalation manoeuvre was not: steady and deep | xxx (xx%) | |
| | Did not hold breath | xxx (xx%) | |
| | Did not close the device | xxx (xx%) | |

<sup>[1]</sup> Correct use is defined as not making any critical or non-critical errors at that visit.

Example : EFF\_T4
Protocol : HZA116492
Population : Intent-to-Treat


### Table 2.xx Summary of Inhaler Device Use Errors

| Visit | | Usual ICS/LABA<br>(N=xxx) | FF/VI<br>(N=xxx) |
|---|---|---|---|
| Randomisation (Day 0) | Number of patients using Turbuhaler | xxx | |
| | Number of patients with correct use [1] | xxx (xx%) | |
| | Number of patients without correct use | xxx (xx%) | |
| | Number of patients with at least one critical error Type of critical error: | xxx (xx%) | |
| | Failed to remove cap | xxx (xx%) | |
| | Did not hold device upright during dose preparation | xxx (xx%) | |
| | Base not twisted fully backwards and forwards, no click heard | xxx (xx%) | |
| | Shook the device after dose preparation | xxx (xx%) | |
| | Exhaled directly into mouthpiece | xxx (xx%) | |
| | No seal by the lips around the mouthpiece during the inhalation | xxx (xx%) | |
| | Number of patients with at least one non-critical error<br>Type of non-critical error: | xxx (xx%) | |
| | Device tipped downwards after dose preparation | xxx (xx%) | |
| | No exhalation before an inhalation | xxx (xx%) | |
| | Inhalation manoeuvre was not: forceful and deep | xxx (xx%) | |
| | Blocked air inlet during inhalation manoeuvre | xxx (xx%) | |
| | Did not hold breath | xxx (xx%) | |
| | Did not close the device | xxx (xx%) | |

[1] Correct use is defined as not making any critical or non-critical errors at that visit.

Programming note: repeat on subsequent pages for Visit = Week 12 and Week 24. "Number of patients using..." line will provide the denominators for each section's percentages.

### Repeat for:

Summary of Inhaler Device Use Errors Per Protocol Population (PP Population)

Example : EFF\_T5
Protocol : HZA116492
Population : Intent-to-Treat


Table 2.xx Summary of Correct Use of Inhaler Device

| Visit | | Usual ICS/LABA<br>(N=xxx) | FF/VI<br>(N=xxx) |
|---|---|---|---|
| Randomisation (Day 0) | n | xxx | xxx |
| , , | Number of patients with correct use [1] | xxx (xx%) | xxx (xx%) |
| | Number of patients without correct use | xxx (xx%) | xxx (xx%) |
| | Number of patients with at least one critical error | xxx (xx%) | xxx (xx%) |
| | Number of patients with at least one non-critical error | xxx (xx%) | xxx (xx%) |
| Week 12 | n | XXX | XXX |
| | Number of patients with correct use [1] | xxx (xx%) | xxx (xx%) |
| | Number of patients without correct use | xxx (xx%) | xxx (xx%) |
| | Number of patients with at least one critical error | xxx (xx%) | xxx (xx%) |
| | Number of patients with at least one non-critical error | xxx (xx%) | xxx (xx%) |
| Week 24 | n | XXX | XXX |
| | Number of patients with correct use [1] | xxx (xx%) | xxx (xx%) |
| | Number of patients without correct use | xxx (xx%) | xxx (xx%) |
| | Number of patients with at least one critical error | xxx (xx%) | xxx (xx%) |
| | Number of patients with at least one non-critical error | xxx (xx%) | xxx (xx%) |

<sup>[1]</sup> Correct use is defined as not making any critical or non-critical errors at that visit.

### Repeat for:

Summary of Correct Use of Inhaler Device Per Protocol Population (PP Population)

Example : EFF\_T6
Protocol : HZA116492
Population : Intent-to-Treat


Table 2.xx

Summary of the Statistical Analysis of Correct Use of Inhaler Device at Week 12 (Visit 4) and at Week 24 (Visit 6) Independently of the Use at Week 12 (Visit 4)

| Visit | | Usual ICS/LABA<br>(N=xxx) | FF/VI<br>(N=xxx) |
|---|---|---|---|
| Week 12 | n<br>With correct use [1] | xxx<br>xxx (xx%) | xxx<br>xxx (xx%) |
| | Without correct use | xxx (xx%) | xxx (xx%) |
| | FF/VI vs. Usual ICS/LABA | | |
| | Adjusted Odds Ratio | | X.XX |
| | 95% <sub>.</sub> CI | | (x.xx, x.xx) |
| | p-value | | X.XXX |
| Week 24 | n | XXX | XXX |
| | With correct use [1] | xxx (xx%) | xxx (xx%) |
| | Without correct use | xxx (xx%) | xxx (xx%) |
| | FF/VI vs. Usual ICS/LABA | | |
| | Adjusted Odds Ratio | | X.XX |
| | 95% CI | | (x.xx, x.xx) |
| | p-value | | X.XXX |

<sup>[1]</sup> Correct use is defined as not making any critical or non-critical errors at that visit.

Note: The analysis method was logistic regression adjusted for randomised treatment, correct use of inhaler device at baseline, gender, age and country.

Programming note: If the likelihood maximisation algorithm fails to converge due to complete or quasi-complete separation of the data then implement Firth's penalized likelihood and add the following footnote: "Note: Firth's penalized likelihood was implemented due to [complete / quasi-complete] separation of data.", deleting "complete" or "quasi-complete" as appropriate.

### Repeat for:

Summary of the Statistical Analysis of Correct Use of Inhaler Device at Week 12 (Visit 4) and at Week 24 (Visit 6) Independently of the Use at Week 12 (Visit 4) Per Protocol Population (PP Population)

Summary of the Statistical Analysis of Percentage of Subjects Who Have Either an ACT Total Score >= 20 or >= 3 Point Increase from Baseline in ACT Total Score at Week 12 (Visit 4) and Week 24 (Visit 6) (ITT Population)

Programming note: Replace "With correct use [1]" with "Responder [1]" and "Without correct use" with "Non-Responder".

Footnotes as follows:

"[1] Responder is defined as an ACT total score >= 20 or >= 3 point increase from baseline in ACT total score at that visit.

Note: The analysis method was logistic regression adjusted for randomised treatment, baseline ACT total score, baseline ACT total score squared, gender, age and country."

Summary of the Statistical Analysis of Percentage of Subjects Who Have an Increase from Baseline of >= 0.5 in AQLQ(S) Total Score and Environmental Stimuli Domain Score at Week 24 (Visit 6) (ITT Population)

Domain: Total Score

Domain: Environmental Stimuli

Programming note: Replace "With correct use [1]" with "Responder [1]" and "Without correct use" with "Non-Responder". Do not display the "Visit" column. Footnotes as follows:

"[1] Responder is defined as an increase from baseline of >= 0.5.

Note: The analysis method was logistic regression adjusted for randomised treatment, baseline score, gender, age and country."

Summary of the Statistical Analysis of Proportion of Responders According to EQ-5D-5L Descriptive System Dimensions at Week 24 (Visit 6) (ITT Population)

Dimension: Mobility
Dimension: Self-care
Dimension: Usual activities
Dimension: Pain/Discomfort

Dimension: Anxiety/Depression

Programming note: Replace "With correct use [1]" with "Responder [1]" and "Without correct use" with "Non-Responder". Do not display the "Visit" column. Footnotes as follows:

"[1] Responder is defined as a score of 1 ('no problems').

Note: The analysis method was logistic regression adjusted for randomised treatment, baseline EQ-5D-5L domain score, gender, age and country."

Example : EFF\_T7
Protocol : HZA116492
Population : Intent-to-Treat


Table 2.xx

Summary of Percentage of Subjects Who Have Either an ACT Total Score of >= 20 or >= 3 Point Increase from Baseline in ACT Total Score

| Visit | | Usual ICS/LABA<br>(N=xxx) | FF/VI<br>(N=xxx) |
|---|---|---|---|
| VIOIL | | (14 ////) | (14-7/7/) |
| Week 6 | n ACT Total Score >= 20 or >= 3 Point Increase from Baseline ACT Total Score >= 20 >= 3 Point Increase from Baseline | xxx<br>xxx (xx%)<br>xxx (xx%)<br>xxx (xx%) | xxx<br>xxx (xx%)<br>xxx (xx%)<br>xxx (xx%) |
| Week 12 | n ACT Total Score >= 20 or >= 3 Point Increase from Baseline ACT Total Score >= 20 >= 3 Point Increase from Baseline | xxx<br>xxx (xx%)<br>xxx (xx%)<br>xxx (xx%) | xxx<br>xxx (xx%)<br>xxx (xx%)<br>xxx (xx%) |

...

Programming note: repeat for Visit = Week 18, Week 24, Early Withdrawal.

Example : EFF\_T8
Protocol : HZA116492
Population : Intent-to-Treat


Table 2.xx Summary of Individual ACT Question Scores

Question: 1. Getting as much done at work, school or home

| Visit | Response | Usual ICS/LABA<br>(N=xxx) | FF/VI<br>(N=xxx) |
|---|---|---|---|
| Randomisation (Day 0) | n<br>1. All of the time | xxx<br>xxx (xx%) | xxx<br>xxx (xx%) |
| | 2. Most of the time | xxx (xx%) | xxx (xx%) |
| | <ul><li>3. Some of the time</li><li>4. A little of the time</li></ul> | xxx (xx%)<br>xxx (xx%) | xxx (xx%)<br>xxx (xx%) |
| | 5. None of the time. | xxx (xx%) | xxx (xx%) |
| Week 6 | n<br> | XXX | XXX |
| | <ol> <li>All of the time</li> <li>Most of the time</li> </ol> | xxx (xx%)<br>xxx (xx%) | xxx (xx%)<br>xxx (xx%) |
| | 3. Some of the time | xxx (xx%) | xxx (xx%) |
| | <ul><li>4. A little of the time</li><li>5. None of the time.</li></ul> | xxx (xx%)<br>xxx (xx%) | xxx (xx%)<br>xxx (xx%) |
| Week 12 | n | XXX | XXX |
| | 1. All of the time | xxx (xx%) | xxx (xx%) |
| | Most of the time Some of the time | xxx (xx%)<br>xxx (xx%) | xxx (xx%)<br>xxx (xx%) |
| | 4. A little of the time | xxx (xx%) | xxx (xx%) |
| | 5. None of the time. | xxx (xx%) | xxx (xx%) |

Example : EFF\_T8
Protocol : HZA116492
Population : Intent-to-Treat


Table 2.xx Summary of Individual ACT Question Scores

Question: 1. Getting as much done at work, school or home

| Response | Usual ICS/LABA<br>(N=xxx) | FF/VI<br>(N=xxx) | |
|---|---|---|---|
| _ | NOV. | 2004 | |
| | , , | ` ' | |
| | , , | ` ' | |
| | , , | ` , | |
| 4. A little of the time | xxx (xx%) | xxx (xx%) | |
| 5. None of the time. | xxx (xx%) | xxx (xx%) | |
| n | XXX | XXX | |
| 1. All of the time | xxx (xx%) | xxx (xx%) | |
| 2. Most of the time | , , | ` ' | |
| 3. Some of the time | , , | , , | |
| 4. A little of the time | , , | ` ' | |
| 5. None of the time. | xxx (xx%) | xxx (xx%) | |
| n | XXX | XXX | |
| 1. All of the time | xxx (xx%) | xxx (xx%) | |
| 2. Most of the time | , , | , , | |
| 3. Some of the time | , , | ` ' | |
| | , , | | |
| | , , | | |
| | n 1. All of the time 2. Most of the time 3. Some of the time 4. A little of the time 5. None of the time 1. All of the time 2. Most of the time 3. Some of the time 4. A little of the time 5. None of the time 7. None of the time 8. All of the time 9. None of the time 9. None of the time 1. All of the time | Response (N=xxx) n xxx 1. All of the time xxx (xx%) 2. Most of the time xxx (xx%) 3. Some of the time xxx (xx%) 4. A little of the time. xxx (xx%) 5. None of the time xxx (xx%) 2. Most of the time xxx (xx%) 4. A little of the time xxx (xx%) 5. None of the time xxx (xx%) 1. All of the time xxx (xx%) 2. Most of the time xxx (xx%) 3. Some of the time xxx (xx%) 3. Some of the time xxx (xx%) 4. A little of the time xxx (xx%) | Response (N=xxx) (N=xxx) n xxx xxx xxx (xx%) 2. Most of the time xxx (xx%) xxx (xx%) xxx (xx%) 3. Some of the time xxx (xx%) xxx (xx%) xxx (xx%) 4. A little of the time xxx (xx%) xxx (xx%) xxx (xx%) 5. None of the time xxx (xx%) xxx (xx%) xxx (xx%) 2. Most of the time xxx (xx%) xxx (xx%) xxx (xx%) 3. Some of the time xxx (xx%) xxx (xx%) xxx (xx%) 5. None of the time xxx (xx%) xxx (xx%) xxx (xx%) 1. All of the time xxx (xx%) xxx (xx%) xxx (xx%) 2. Most of the time xxx (xx%) xxx (xx%) xxx (xx%) 3. Some of the time xxx (xx%) xxx (xx%) xxx (xx%) 3. Some of the time xxx (xx%) xxx (xx%) xxx (xx%) 4. A little of the time xxx (xx%) xxx (xx%) xxx (xx%) |
# 2017N339371\_00 HZA116492


Programming note: repeat on subsequent pages for Question = 2. Shortness of breath, 3. Asthma symptoms woken up at night or earlier than usual, 4. Used rescue inhaler or nubuliser medication, 5. Asthma control.

Example : EFF\_T9
Protocol : HZA116492
Population : Intent-to-Treat


Table 2.xx Summary of Compliance with Study Medication

| Time period | Compliance (%) | Usual ICS/LABA<br>(N=xxx) | FF/VI<br>(N=xxx) |
|---|---|---|---|
| Randomisation (Day 0) to<br>Week 24 | n | XXX | xxx |
| | < 80% | xxx (xx%) | xxx (xx%) |
| | 80% to 120% inclusive | xxx (xx%) | xxx (xx%) |
| | > 120% | xxx (xx%) | xxx (xx%) |
| | n | XX | XX |
| | Mean | XX.X | XX.X |
| | SD | X.XX | X.XX |
| | Median | XX.X | XX.X |
| | Min. | XX | XX |
| | Max. | XX | XX |

#### Note:

Compliance = {[Total no. of inhalations taken]/[Dose frequency x (Stop date – Start date)]} x 100.

Note: Total number of inhalations taken is the sum of (dose counter start count – dose counter stop count) for all inhalers used during the time period, Dose frequency is equal to 1 for Ellipta, 2 for Diskus and 2 or 4 for Turbuhaler, and Start date and Stop date are the earliest treatment start date and latest treatment stop date respectively recorded for all inhalers used during the time period.

Programming note: repeat on subsequent pages for Time period = Randomisation (Day 0) to Week 12, Week 12 to Week 24.

## Repeat for:

Summary of Compliance with Study Medication Per Protocol Population (PP Population)

Example : EFF\_T10
Protocol : HZA116492
Population : Intent-to-Treat


Table 2.xx Summary of Use of Medication Adherence Report Scale for Asthma (MARS-A) During the Study

Visit: Randomisation (Day 0)

| <br>m (Edy 0) | | Usual ICS/LABA | FF/VI |
|---|---|---|---|
| MARS-A Questions | | (N=xxx) | (N=xxx) |
| I only use it when I need it | n | XXX | XXX |
| | Always | xxx (xx%) | xxx (xx%) |
| | Often | xxx (xx%) | xxx (xx%) |
| | Sometimes | xxx (xx%) | xxx (xx%) |
| | Rarely | xxx (xx%) | xxx (xx%) |
| | Never | xxx (xx%) | xxx (xx%) |
| Only use it when I feel breathless | n | XXX | XXX |
| • | Always | xxx (xx%) | xxx (xx%) |
| | Often | xxx (xx%) | xxx (xx%) |
| | Sometimes | xxx (xx%) | xxx (xx%) |
| | Rarely | xxx (xx%) | xxx (xx%) |
| | Never | xxx (xx%) | xxx (xx%) |
| I decide to miss out a dose | n | XXX | XXX |
| | Always | xxx (xx%) | xxx (xx%) |
| | Often | xxx (xx%) | xxx (xx%) |
| | Sometimes | xxx (xx%) | xxx (xx%) |
| | Rarely | xxx (xx%) | xxx (xx%) |
| | Never | xxx (xx%) | xxx (xx%) |
| | 140401 | MM (MM/0) | AAA (AA 70) |

Note: MARS-A: Medication Adherence Report Scale for Asthma.

<sup>[1]</sup> MARS-A 10-Score is based on the mean score across all ten questions.

Example : EFF\_T10
Protocol : HZA116492
Population : Intent-to-Treat


Table 2.xx

Summary of Use of Medication Adherence Report Scale for Asthma (MARS-A) During the Study

Lloud ICC/LADA

Visit: Randomisation (Day 0)

| MARS-A Questions | | Usual ICS/LABA<br>(N=xxx) | (N=xxx) |
|---|---|---|---|
| I try to avoid using it | n | XXX | XXX |
| | Always | xxx (xx%) | xxx (xx%) |
| | Often | xxx (xx%) | xxx (xx%) |
| | Sometimes | xxx (xx%) | xxx (xx%) |
| | Rarely | xxx (xx%) | xxx (xx%) |
| | Never | xxx (xx%) | xxx (xx%) |
| I forget to take it | n | XXX | XXX |
| - | Always | xxx (xx%) | xxx (xx%) |
| | Often | xxx (xx%) | xxx (xx%) |
| | Sometimes | xxx (xx%) | xxx (xx%) |
| | Rarely | xxx (xx%) | xxx (xx%) |
| | Never | xxx (xx%) | xxx (xx%) |
| I alter the dose | n | XXX | XXX |
| | Always | xxx (xx%) | xxx (xx%) |
| | Often | xxx (xx%) | xxx (xx%) |
| | Sometimes | xxx (xx%) | xxx (xx%) |
| | Rarely | xxx (xx%) | xxx (xx%) |
| | Never | xxx (xx%) | xxx (xx%) |

Note: MARS-A: Medication Adherence Report Scale for Asthma.

[1] MARS-A 10-Score is based on the mean score across all ten questions.

Example : EFF\_T10
Protocol : HZA116492
Population : Intent-to-Treat


Table 2.xx

Summary of Use of Medication Adherence Report Scale for Asthma (MARS-A) During the Study

Visit: Randomisation (Day 0)

| MARS-A Questions | | Usual ICS/LABA<br>(N=xxx) | FF/VI<br>(N=xxx) |
|---|---|---|---|
| I stop taking it for a while | n | XXX | XXX |
| | Always | xxx (xx%) | xxx (xx%) |
| | Often<br>Sometimes | XXX (XX%) | XXX (XX%) |
| | Rarely | xxx (xx%)<br>xxx (xx%) | xxx (xx%)<br>xxx (xx%) |
| | Never | xxx (xx%) | xxx (xx%) |
| D "' | | , , | , , |
| Reserve if treatment doesn't work | n | XXX | XXX |
| | Always | xxx (xx%) | xxx (xx%) |
| | Often | xxx (xx%) | xxx (xx%) |
| | Sometimes | xxx (xx%) | xxx (xx%) |
| | Rarely | xxx (xx%) | xxx (xx%) |
| | Never | xxx (xx%) | xxx (xx%) |
| Before doing something | n | XXX | XXX |
| 3 3 | Always | xxx (xx%) | xxx (xx%) |
| | Often | xxx (xx%) | xxx (xx%) |
| | Sometimes | xxx (xx%) | xxx (xx%) |
| | Rarely | xxx (xx%) | xxx (xx%) |
| | Never | xxx (xx%) | xxx (xx%) |
| | INGVE | ^^^ (^^ /0) | ^^^ (^^ /0) |

Note: MARS-A: Medication Adherence Report Scale for Asthma.

[1] MARS-A 10-Score is based on the mean score across all ten questions.

Example : EFF\_T10
Protocol : HZA116492
Population : Intent-to-Treat


Table 2.xx

Summary of Use of Medication Adherence Report Scale for Asthma (MARS-A) During the Study

Visit: Randomisation (Day 0)

| MADS A Questions | | Usual ICS/LABA | FF/VI |
|-----------------------------|-----------|----------------|-----------|
| MARS-A Questions | | (N=xxx) | (N=xxx) |
| I take less than instructed | n | XXX | XXX |
| | Always | xxx (xx%) | xxx (xx%) |
| | Often | xxx (xx%) | xxx (xx%) |
| | Sometimes | xxx (xx%) | xxx (xx%) |
| | Rarely | xxx (xx%) | xxx (xx%) |
| | Never | xxx (xx%) | xxx (xx%) |
| MARS-A 10-Score [1] | n | XX | XX |
| • • | Mean | XX.X | XX.X |
| | SD | X.XX | X.XX |
| | Median | XX.X | XX.X |
| | Min. | XX | XX |
| | Max. | XX | XX |

Note: MARS-A: Medication Adherence Report Scale for Asthma.

[1] MARS-A 10-Score is based on the mean score across all ten questions.

Programming note: Repeat on subsequent pages for Visit = Week 12, Week 24 and Early Withdrawal.

Example : EFF\_T10S
Protocol : HZA116492
Population : Intent-to-Treat


Table 2.xx

Summary of Use of Medication Adherence Report Scale for Asthma (MARS-A) During the Study by Status of Patient in Relation to the Reminder Sent to French Centres

Status: Patients in France who had completed all MARS-A assessments prior to the reminder being implemented Visit: Randomisation (Day 0)

| | | Usual ICS/LABA | FF/VI |
|---|---|---|---|
| MARS-A Questions | | (N=xxx) | (N=xxx) |
| I only use it when I need it | n | XXX | XXX |
| • | Always | xxx (xx%) | xxx (xx%) |
| | Often | xxx (xx%) | xxx (xx%) |
| | Sometimes | xxx (xx%) | xxx (xx%) |
| | Rarely | xxx (xx%) | xxx (xx%) |
| | Never | xxx (xx%) | xxx (xx%) |
| Only use it when I feel breathless | n | XXX | XXX |
| | Always | xxx (xx%) | xxx (xx%) |
| | Often | xxx (xx%) | xxx (xx%) |
| | Sometimes | xxx (xx%) | xxx (xx%) |
| | Rarely | xxx (xx%) | xxx (xx%) |
| | Never | xxx (xx%) | xxx (xx%) |
| I decide to miss out a dose | n | XXX | XXX |
| | Always | xxx (xx%) | xxx (xx%) |
| | Often | xxx (xx%) | xxx (xx%) |
| | Sometimes | xxx (xx%) | xxx (xx%) |
| | Rarely | xxx (xx%) | xxx (xx%) |
| | Never | xxx (xx%) | xxx (xx%) |

Note: MARS-A: Medication Adherence Report Scale for Asthma.

2017N339371\_00 HZA116492


Note: Due to an issue identified with the French translation of the MARS-A, a reminder was sent to centres in France instructing that the questionnaire refers to the patient's preventer inhaler (i.e. their maintenance therapy prior to entering the study, and study medication while on-study).
[1] MARS-A 10-Score is based on the mean score across all ten questions.

Example : EFF\_T10S
Protocol : HZA116492
Population : Intent-to-Treat


Table 2.xx

Summary of Use of Medication Adherence Report Scale for Asthma (MARS-A) During the Study by Status of Patient in Relation to the Reminder Sent to French Centres

Usual ICS/LABA

FF/VI

Status: Patients in France who had completed all MARS-A assessments prior to the reminder being implemented Visit: Randomisation (Day 0)

| MARS-A Questions | | (N=xxx) | (N=xxx) | |
|-------------------------|-----------|-----------|-----------|---|
| With the At Questions | | (14-7///) | (14-7/7/) | - |
| I try to avoid using it | n | XXX | XXX | |
| | Always | xxx (xx%) | xxx (xx%) | |
| | Often | xxx (xx%) | xxx (xx%) | |
| | Sometimes | xxx (xx%) | xxx (xx%) | |
| | Rarely | xxx (xx%) | xxx (xx%) | |
| | Never | xxx (xx%) | xxx (xx%) | |
| I forget to take it | n | XXX | XXX | |
| | Always | xxx (xx%) | xxx (xx%) | |
| | Often | xxx (xx%) | xxx (xx%) | |
| | Sometimes | xxx (xx%) | xxx (xx%) | |
| | Rarely | xxx (xx%) | xxx (xx%) | |
| | Never | xxx (xx%) | xxx (xx%) | |
| I alter the dose | n | XXX | XXX | |
| | Always | xxx (xx%) | xxx (xx%) | |
| | Often | xxx (xx%) | xxx (xx%) | |
| | Sometimes | xxx (xx%) | xxx (xx%) | |
| | Rarely | xxx (xx%) | xxx (xx%) | |
| | Never | xxx (xx%) | xxx (xx%) | |

Note: MARS-A: Medication Adherence Report Scale for Asthma.

2017N339371\_00 HZA116492


Note: Due to an issue identified with the French translation of the MARS-A, a reminder was sent to centres in France instructing that the questionnaire refers to the patient's preventer inhaler (i.e. their maintenance therapy prior to entering the study, and study medication while on-study).
[1] MARS-A 10-Score is based on the mean score across all ten questions.

Example : EFF\_T10S
Protocol : HZA116492
Population : Intent-to-Treat


Table 2.xx

Summary of Use of Medication Adherence Report Scale for Asthma (MARS-A) During the Study by Status of Patient in Relation to the Reminder Sent to French Centres

Status: Patients in France who had completed all MARS-A assessments prior to the reminder being implemented Visit: Randomisation (Day 0)

| MARS-A Questions | | Usual ICS/LABA<br>(N=xxx) | FF/VI<br>(N=xxx) |
|---|---|---|---|
| | | , | 7 |
| I stop taking it for a while | n | XXX | XXX |
| | Always | xxx (xx%) | xxx (xx%) |
| | Often | xxx (xx%) | xxx (xx%) |
| | Sometimes | xxx (xx%) | xxx (xx%) |
| | Rarely | xxx (xx%) | xxx (xx%) |
| | Never | xxx (xx%) | xxx (xx%) |
| Reserve if treatment doesn't work | n | XXX | XXX |
| | Always | xxx (xx%) | xxx (xx%) |
| | Often | xxx (xx%) | xxx (xx%) |
| | Sometimes | xxx (xx%) | xxx (xx%) |
| | Rarely | xxx (xx%) | xxx (xx%) |
| | Never | xxx (xx%) | xxx (xx%) |
| Before doing something | n | XXX | XXX |
| | Always | xxx (xx%) | xxx (xx%) |
| | Often | xxx (xx%) | xxx (xx%) |
| | Sometimes | xxx (xx%) | xxx (xx%) |
| | Rarely | xxx (xx%) | xxx (xx%) |
| | Never | xxx (xx%) | xxx (xx%) |
| | | . , | . , |

Note: MARS-A: Medication Adherence Report Scale for Asthma.

2017N339371\_00 HZA116492


Note: Due to an issue identified with the French translation of the MARS-A, a reminder was sent to centres in France instructing that the questionnaire refers to the patient's preventer inhaler (i.e. their maintenance therapy prior to entering the study, and study medication while on-study).
[1] MARS-A 10-Score is based on the mean score across all ten questions.

Example : EFF\_T10S
Protocol : HZA116492
Population : Intent-to-Treat


Table 2.xx

Summary of Use of Medication Adherence Report Scale for Asthma (MARS-A) During the Study by Status of Patient in Relation to the Reminder Sent to French Centres

Status: Patients in France, all MARS-A assessments completed pre-reminder

Visit: Randomisation (Day 0)

| MARS-A Questions | | Usual ICS/LABA<br>(N=xxx) | FF/VI<br>(N=xxx) |
|---|---|---|---|
| | | , , | |
| I take less than instructed | n | XXX | XXX |
| | Always | xxx (xx%) | xxx (xx%) |
| | Often | xxx (xx%) | xxx (xx%) |
| | Sometimes | xxx (xx%) | xxx (xx%) |
| | Rarely | xxx (xx%) | xxx (xx%) |
| | Never | xxx (xx%) | xxx (xx%) |
| MARS-A 10-Score [1] | n | XX | XX |
| | Mean | XX.X | XX.X |
| | SD | X.XX | X.XX |
| | Median | XX.X | XX.X |
| | Min. | XX | XX |
| | Max. | XX | XX |

Note: MARS-A: Medication Adherence Report Scale for Asthma.

Note: Due to an issue identified with the French translation of the MARS-A, a reminder was sent to centres in France instructing that the questionnaire refers to the patient's preventer inhaler (i.e. their maintenance therapy prior to entering the study, and study medication while on-study).

[1] MARS-A 10-Score is based on the mean score across all ten questions.

Programming note: Repeat on subsequent pages for Visit = Week 12, Week 24 and Early Withdrawal, and for Status = "Patients in France, some MARS-A assessments completed pre-reminder", "Patients in France, all MARS-A assessments completed post-reminder", "Patients in Germany"

Example : EFF\_T11
Protocol : HZA116492
Population : Intent-to-Treat


Table 2.xx Summary of Severe On-Treatment Asthma Exacerbations

| | Usual ICS/LABA<br>(N=xxx) | FF/VI<br>(N=xxx) |
|---|---|---|
| No. of subjects with one or more severe asthma exacerbation | xx (xx%) | xx (xx%) |
| Total no. of severe asthma exacerbations | xx | XX |
| Number of severe asthma exacerbations per subject 0 1 > 1 | xx (xx%)<br>xx (xx%)<br>xx (xx%) | xx (xx%)<br>xx (xx%)<br>xx (xx%) |
| Duration of severe asthma exacerbation (days) [1] | | |
| n<br>Mean<br>SD<br>Median<br>Min.<br>Max. | XX<br>XX.X<br>X.XX<br>XX.X<br>XX | XX<br>XX.X<br>X.XX<br>XX.X<br>XX |

<sup>[1]</sup> Summary only includes exacerbations for which a date of resolution or death is provided.

Example : EFF\_T11
Protocol : HZA116492
Population : Intent-to-Treat


Table 2.xx Summary of Severe On-Treatment Asthma Exacerbations

| | Usual ICS/LABA<br>(N=xxx) | FF/VI<br>(N=xxx) |
|---|---|---|
| Outcome | | |
| Resolved | xx (xx%) | xx (xx%) |
| Fatal | xx (xx%) | xx (xx%) |
| Not resolved | xx (xx%) | xx (xx%) |
| No. of exacerbations: | | |
| Requiring use of systemic/oral corticosteroids | xx (xx%) | xx (xx%) |
| Leading to hospitalisation | xx (xx%) | xx (xx%) |
| Requiring emergency room visit | xx (xx%) | xx (xx%) |
| No. of exacerbations requiring intubation | xx (xx%) | xx (xx%) |
| No. of exacerbations leading to withdrawal from study | xx (xx%) | xx (xx%) |

<sup>[1]</sup> Summary only includes exacerbations for which a date of resolution or death is provided.

Example : EFF\_T11S
Protocol : HZA116492
Population : Intent-to-Treat


Table 2.xx Summary of Severe On-Treatment Asthma Exacerbations by Season

Season: Spring

| | Usual ICS/LABA<br>(N=xxx) | FF/VI<br>(N=xxx) |
|---|---|---|
| No. of subjects with one or more severe asthma exacerbation | xx (xx%) | xx (xx%) |
| Total no. of severe asthma exacerbations | xx | XX |
| Number of severe asthma exacerbations per subject 0 1 > 1 | xx (xx%)<br>xx (xx%)<br>xx (xx%) | xx (xx%)<br>xx (xx%)<br>xx (xx%) |
| Duration of severe asthma exacerbation (days) [1] | | |
| n | XX | XX |
| Mean | XX.X | XX.X |
| SD | X.XX | X.XX |
| Median | XX.X | XX.X |
| Min. | XX | XX |
| Max. | XX | XX |

Note: Spring = March, April and May; Summer = June, July and August; Autumn = September, October and November; Winter = December, January and February. [1] Summary only includes exacerbations for which a date of resolution or death is provided.

Example : EFF\_T11
Protocol : HZA116492
Population : Intent-to-Treat


Table 2.xx Summary of Severe On-Treatment Asthma Exacerbations by Season

Season: Spring

| | Usual ICS/LABA<br>(N=xxx) | FF/VI<br>(N=xxx) |
|---|---|---|
| Outcome | | |
| Resolved | xx (xx%) | xx (xx%) |
| Fatal | xx (xx%) | xx (xx%) |
| Not resolved | xx (xx%) | xx (xx%) |
| No. of exacerbations: | | |
| Requiring use of systemic/oral corticosteroids | xx (xx%) | xx (xx%) |
| Leading to hospitalisation | xx (xx%) | xx (xx%) |
| Requiring emergency room visit | xx (xx%) | xx (xx%) |
| No. of exacerbations requiring intubation | xx (xx%) | xx (xx%) |
| No. of exacerbations leading to withdrawal from study | xx (xx%) | xx (xx%) |

Note: Spring = March, April and May; Summer = June, July and August; Autumn = September, October and November; Winter = December, January and February. [1] Summary only includes exacerbations for which a date of resolution or death is provided.

Programming note: repeat on subsequent pages for Season = Summer, Autumn, Winter.

Example : EFF\_T12
Protocol : HZA116492
Population : Intent-to-Treat


Table 2.xx
Summary of the Statistical Analysis of Severe On-Treatment Asthma Exacerbations

| | Usual ICS/LABA<br>(N=xxx) | FF/VI<br>(N=xxx) |
|---|---|---|
| | · | · |
| n | XXX | XXX |
| LS Mean Annual Rate | X.XX | X.XX |
| FF/VI vs. Usual ICS/LABA<br>Ratio | | X.XX |
| 95% CI | | (x.xx, x.xx) |
| p-value | | X.XXX |
| Percent Reduction | | X.XX |
| 95% CI | | (x.xx, x.xx) |

Note: The analysis method was Generalised Linear Model assuming an underlying negative binomial distribution with a log-link function and logarithm of time on treatment as an offset variable and adjusted for randomised treatment, number of severe asthma exacerbations in the previous year prior to randomisation, gender, age and country.

Example : EFF\_T13
Protocol : HZA116492
Population : Intent-to-Treat


Table 2.xx
Summary of the Statistical Analysis of Time to First Severe On-Treatment Asthma Exacerbation

| | Usual ICS/LABA<br>(N=xxx) | FF/VI<br>(N=xxx) |
|---|---|---|
| Number of subjects with event<br>Number of subjects censored | xx (xx%)<br>xx (xx%) | xx (xx%)<br>xx (xx%) |
| Probability of having event (%) [1] 95% CI | xx.x<br>(xx.x, xx.x) | xx.x<br>(xx.x, xx.x) |
| FF/VI vs. Usual ICS/LABA<br>Hazard Ratio [2]<br>95% CI<br>p-value | | X.XX<br>(XX.X, XX.X)<br>X.XXX |

Note: At Day 168 all subjects who have not experienced a severe asthma exacerbation are considered censored, regardless of whether their on-treatment phase continues beyond Day 168.

<sup>[1]</sup> Kaplan-Meier estimates.

<sup>[2]</sup> Overall hazard ratios, CIs and p-values are from a Cox proportional hazards model with randomised treatment, gender, age and country as covariates. A hazard ratio <1 indicates a lower risk with FF/VI compared with Usual ICS/LABA.


Example : EFF\_T14 Protocol : HZA116492

: Intent-to-Treat

Table 2.xx

Summary of Percentage of Subjects Who Have an Increase from Baseline of >=0.5 in AQLQ(S) Total Score and Domain Scores

Domain: Total Score

Population

| Visit | Response | Usual ICS/LABA<br>(N=xxx) | FF/VI<br>(N=xxx) |
|---|---|---|---|
| Week 24 | n<br>Responder [1]<br>Non-Responder | xxx<br>xxx (xx%)<br>xxx (xx%) | xxx<br>xxx (xx%)<br>xxx (xx%) |
| Early Withdrawal | n<br>Responder [1]<br>Non-Responder | xxx<br>xxx (xx%)<br>xxx (xx%) | xxx<br>xxx (xx%)<br>xxx (xx%) |

<sup>[1]</sup> Responder is defined as an increase from baseline of >= 0.5.

Programming note: repeat on subsequent pages for Domain = Environmental Stimuli, Symptoms, Activity Limitations, Emotional Function.

Example : EFF\_T15
Protocol : HZA116492
Population : Intent-to-Treat


Table 2.xx Summary of EQ-5D-5L Descriptive System Dimensions

Dimension: Mobility

| | Usual ICS/LABA | FF/VI |
|---|---|---|
| | (N=XXX) | (N=xxx) |
| n | XXX | XXX |
| I am not anxious or depressed | xxx (xx%) | xxx (xx%) |
| I am slightly anxious or depressed | xxx (xx%) | xxx (xx%) |
| I am moderately anxious or depressed | xxx (xx%) | xxx (xx%) |
| I am severely anxious or depressed | xxx (xx%) | xxx (xx%) |
| I am extremely anxious or depressed | xxx (xx%) | xxx (xx%) |
| Missing | xxx (xx%) | xxx (xx%) |
| n | XXX | XXX |
| I am not anxious or depressed | xxx (xx%) | xxx (xx%) |
| I am slightly anxious or depressed | xxx (xx%) | xxx (xx%) |
| I am moderately anxious or depressed | xxx (xx%) | xxx (xx%) |
| I am severely anxious or depressed | xxx (xx%) | xxx (xx%) |
| I am extremely anxious or depressed | xxx (xx%) | xxx (xx%) |
| Missing | xxx (xx%) | xxx (xx%) |
| | I am not anxious or depressed I am slightly anxious or depressed I am moderately anxious or depressed I am severely anxious or depressed I am extremely anxious or depressed Missing n I am not anxious or depressed I am slightly anxious or depressed I am moderately anxious or depressed I am severely anxious or depressed I am extremely anxious or depressed I am extremely anxious or depressed | n xxx I am not anxious or depressed xxx (xx%) I am slightly anxious or depressed xxx (xx%) I am moderately anxious or depressed xxx (xx%) I am severely anxious or depressed xxx (xx%) I am extremely anxious or depressed xxx (xx%) Missing xxx (xx%) Xxx (xx%) Xxx (xx%) I am not anxious or depressed xxx (xx%) I am slightly anxious or depressed xxx (xx%) I am moderately anxious or depressed xxx (xx%) I am severely anxious or depressed xxx (xx%) I am extremely anxious or depressed xxx |

Programming note: repeat on subsequent pages for Visit = Early Withdrawal and for Dimension = Self-Care, Usual Activities, Pain/Discomfort, Anxiety/Depression.

# 12.16.4. Efficacy Figure Shells

Example : EFF\_F1 Protocol : HZA116492

Population : Intent-to-Treat


Figure 2.xx Summary of ACT Total Score

Programming note: present "ACT Total Score" on y-axis and "Visit" on x-axis (Randomisation (Day 0), Week 6, Week 12, Week 18, Week 24). Present mean ACT Total Score ± SD separately for treatment group (FF/VI, Usual ICS/LABA) at each visit, connecting the means with a solid line. Distinguish the treatment groups by different line types and colours.

## Repeat for:

Summary of Change from Baseline in ACT Total Score Per Protocol Population (PP Population)

Summary of Change from Baseline in ACT Total Score by Country (ITT Population)

Country: France
Country: Germany

Example : EFF\_F2
Protocol : HZA116492
Population : Intent-to-Treat


Figure 2.xx
Summary of Primary and Sensitivity Analyses for Change from Baseline in ACT Total Score at Week 12 (Visit 4)



Programming note: present "Treatment difference" on the x-axis, and reverse axis so treatment difference increases from left to right. Replace "Ratio (95% CI)" with "Treatment Difference (95% CI)". Present lines for the following: Primary analysis (ITT), Primary analysis (PP), ANCOVA with LOCF (ITT), Multiple Imputation (Missing at Random) (ITT), Multiple Imputation (Copy Differences from Reference) (ITT), Hodges-Lehmann (ITT), ANCOVA with WOCF (ITT).

## Repeat for:

Summary of Key Secondary and Sensitivity Analyses for Change from Baseline in ACT Total Score at Week 24 (Visit 6)

Example : EFF\_F3
Protocol : HZA116492
Population : Intent-to-Treat


Figure 2.xx
Summary of Interaction Tests for Change from Baseline in ACT Total Score at Week 12 (Visit 4)



Programming note: present "LS Mean Change" on the x-axis, and reverse axis so it increases from left to right. Replace "Ratio (95% CI)" with "LS Mean Change (95% CI)". Present the following subgroups: Country (France, Germany); Number of Severe Asthma Exacerbations in the Previous Year Prior to Randomisation (0, >= 1); Smoking Status at Baseline (Current smoker, Former smoker, Never smoked); Age Group ( $\leq 50$  Years Old, > 50 Years Old); Gender (Male, Female).

2017N339371\_00 HZA116492

Example : EFF\_F4

Protocol : HZA116492 

Population : Intent-to-Treat

Figure 2.xx

Histogram of Percentage of Subjects Who Have Either an ACT Total Score of >= 20 or >= 3 Point Increase from Baseline in ACT Total Score

Programming note: present "Percent of Subjects (%)" on y-axis and "Visit" on x-axis (Week 6, Week 12, Week 18, Week 24, Early Withdrawal). For each visit, present 3 vertical bars distinguished by fill pattern (similar to non-standard EFF\_F6). Each bar represents: "ACT Total Score" >= 20 or >= 3 Point Increase from Baseline in ACT Total Score", "ACT Total Score" and ">= 3 Point Increase from Baseline in ACT Total Score" respectively and should be labelled as such on the legend.

Example : EFF\_F5
Protocol : HZA116492
Population : Intent-to-Treat


Figure 2.xx
Box Plot of Compliance with Study Medication



Programming Note: label y-axis title as "Compliance (%)", maximum of y-axis may be > 100%.

Example : EFF\_F6
Protocol : HZA116492

Population : Intent-to-Treat


Figure 2.xx Histogram of the Questions and Answers of the MARS-A Questionnaire

Randomised Treatment: Usual ICS/LABA Visit: Randomisation (Day 0)



Note: MARS-A = Medication Adherence Report Scale for Asthma.

Programming note: repeat on subsequent pages for Visit = Day 0 and repeated for Week 12, Week 24, and Early Withdrawal; and for Randomised Treatment = FF/VI.

## Repeat for:

Histogram of the Questions and Answers of the MARS-A Questionnaire by Status of Patient in Relation to the Reminder Sent to French Centres (ITT Population)

Status: Patients in France, all MARS-A assessments completed pre-reminder

Status: Patients in France, some MARS-A assessments completed pre-reminder, some post-reminder

Status: Patients in France, all MARS-A assessments completed post-reminder

Status: Patients in Germany

Add the following footnote: "Note: Due to an issue identified with the French translation of the MARS-A, a reminder was sent to centres in France instructing that the questionnaire refers to the patient's preventer inhaler (i.e. their maintenance therapy prior to entering the study, and study medication while on-study)."

Example : EFF\_F7
Protocol : HZA116492

Population

: Intent-to-Treat


Figure 2.xx
Histogram of the Distribution of MARS-A Scores During the Study

Visit: Randomisation (Day 0)



Note: MARS-A = Medication Adherence Report Scale for Asthma.

Note: MARS-A 10-Score is based on the mean score across all ten questions.

Programming note: repeat on subsequent pages for Visit = Week 52 and Early Withdrawal.

## Repeat for:

Histogram of the Distribution of MARS-A Scores During the Study by Status of Patient in Relation to the Reminder Sent to French Centres (ITT Population)

Status: Patients in France, all MARS-A assessments completed pre-reminder

Status: Patients in France, some MARS-A assessments completed pre-reminder, some post-reminder

Status: Patients in France, all MARS-A assessments completed post-reminder

Status: Patients in Germany

Add the following footnote: "Note: Due to an issue identified with the French translation of the MARS-A, a reminder was sent to centres in France instructing that the questionnaire refers to the patient's preventer inhaler (i.e. their maintenance therapy prior to entering the study, and study medication while on-study)."

Example : EFF\_F8
Protocol : HZA116492

: Intent-to-Treat

Population


Figure 2.xx
Box Plot of Severe On-Treatment Asthma Exacerbation Rates Adjusted for Exposure to Treatment



Example : EFF\_F9
Protocol : HZA116492
Population : Intent-to-Treat


Figure 2.xx
Kaplan-Meier Plot of Time to First Severe On-Treatment Asthma Exacerbation



Programming note: display increments of 6 weeks on the x-axis, up to the maximum exposure (e.g. 0, 6, 12, 18, 24).

# 12.16.5. Safety Table Shells

Example : SAFE\_T1
Protocol : HZA116492
Population : Safety


Table 3.xx
On-Treatment Serious Adverse Events and Adverse Drug Reactions Overview

| | Usual ICS/LABA<br>(N=xxx) | FF/VI<br>(N=xxx) |
|---|---|---|
| Any on-treatment ADRs Any on-treatment non serious ADRs | xxx (xx%)<br>xxx (xx%) | xxx (xx%)<br>xxx (xx%) |
| Any on-treatment serious ADRs Any post-treatment serious ADRs | xxx (xx%)<br>xxx (xx%)<br>xxx (xx%) | xxx (xx%)<br>xxx (xx%)<br>xxx (xx%) |
| Any on-treatment SAEs Any post-treatment SAEs | xxx (xx%)<br>xxx (xx%) | xxx (xx%)<br>xxx (xx%) |
| Any SAEs or ADRs leading to permanent discontinuation of study drug or withdrawal from study [1] | xxx (xx%) | xxx (xx%) |
| Any on-treatment fatal serious ADRs | xxx (xx%) | xxx (xx%) |
| Any on-treatment fatal SAEs<br>Any post-treatment fatal SAEs | xxx (xx%)<br>xxx (xx%) | xxx (xx%)<br>xxx (xx%) |

<sup>[1]</sup> Includes both on-treatment and post-treatment SAEs and ADRs.

Programming note: Based on IDSL standard template AE13.

Example : SAFE\_T2
Protocol : HZA116492
Population : Safety


Table 3.xx Summary of On-Treatment Non-Serious Adverse Drug Reactions of Special Interest

| Special Interest Group/ | | |
|--------------------------|----------------|-----------|
| Subgroup | Usual ICS/LABA | FF/VI |
| Preferred Term | (N=xxx) | (N=xxx) |
| Adrenal suppression | | |
| Any event | xxx (xx%) | xxx (xx%) |
| Blood cortisol decreased | xxx (xx%) | xxx (xx%) |
| Cardiovascular effects | | |
| Any event | xxx (xx%) | xxx (xx%) |
| Cardiac Arrhytmia [1] | xxx (xx%) | xxx (xx%) |
| Any event | xxx (xx%) | xxx (xx%) |
| Palpitations | xxx (xx%) | xxx (xx%) |
| Extrasystoles | xxx (xx%) | xxx (xx%) |
| Cardiac Ischaemia [1] | xxx (xx%) | xxx (xx%) |
| Any event | xxx (xx%) | xxx (xx%) |
| Angina pectoris | xxx (xx%) | xxx (xx%) |
| Chest pain | xxx (xx%) | xxx (xx%) |
| Effects on potassium | | |
| Any event | xxx (xx%) | xxx (xx%) |
| XXXXXXX | xxx (xx%) | xxx (xx%) |
| XXXXXXX | xxx (xx%) | xxx (xx%) |
| | . , | • • |

<sup>[1]</sup> This special interest group/subgroup was defined using Special MedDRA Queries.

Programming note: Based on IDSL standard template AE1.

# Repeat for:

Summary of On-Treatment Serious Adverse Drug Reactions of Special Interest (ITT Population)
Summary of On-Treatment Adverse Drug Reactions of Special Interest (ITT Population)
Summary of On-Treatment Serious Adverse Events of Special Interest (ITT Population)
Summary of On-Treatment Fatal Serious Adverse Events of Special Interest (ITT Population)
Summary of On-Treatment Non-Fatal Serious Adverse Events of Special Interest (ITT Population)

Example : SAFE\_T3
Protocol : HZA116492
Population : Safety


Table 3.xx
Top Ten Most Commonly Reported On-Treatment Adverse Drug Reactions Per Treatment Group

| Preferred Term | Usual ICS/LABA<br>(N=xxx) | FF/VI<br>(N=xxx) |
|----------------|---------------------------|------------------|
| XXXXXXX | xxx (xx%) | xxx (xx%) |

Programming note: Present the ten most frequent preferred terms in Usual ICS/LABA, and the ten most frequent in FF/VI (do not use percentages to determine "most frequent").
Page 1

## 12.16.6. Safety Figure Shells

Example : SAFE\_F1 Protocol : HZA116492

of 1

Population : Intent-to-Treat/Safety

Figure 2.xx
Summary of Benefit:Risk for FF/VI vs. Usual ICS/LABA



- \* = Number of subjects with event
- (a) Difference in LS mean change from baseline from an MMRM
- (b) Difference in LS mean change from baseline from an ANCOVA model
- (c) Adjusted odds ratio obtained from a logistic regression model
- (d) Risk difference

Programming note: present the following endpoints:

- Benefits:
- First panel, x-axis decreasing from left to right:
  - Difference in LS mean change from baseline and 95% CI for: change from baseline in ACT total score at Week 12 (Visit 4) and at Week 24 (Visit 6) (labeled (a))
  - Difference in LS mean change from baseline and 95% CI for change from baseline in trough (pre-dose) FEV1 at Week 12 (Visit 4) (labeled (b))
- Second panel, x-axis increasing from left to right:
  - Adjusted odds ratio and 95% CI for: percentage of subjects with correct use of inhaler device at Week 12 (Visit 4) and at Week 24 (Visit 6) (labeled (c))
- Risks:
- Third panel, x-axis increasing from left to right:
  - Risk difference and 95% CI of the following SAEs of special interest:
     asthma/bronchospasm, cardiovascular effects, decreased bone mineral density and
     associated fractures, hypersensitivity, local steroid effects, lower respiratory tract infection
     (LRTI) excluding pneumonia, pneumonia, adrenal suppression, ocular effects, effects on
     glucose, effects on potassium, tremor (labeled (d))

## 12.16.7. Non-ICH Listing Shells

Example : POP\_L1 Protocol : HZA116492

Population : All Subjects Enrolled


Listing x

Subjects Screened but Not in the Intent-to-Treat Population

...

2017N339371\_00 HZA116492

Example : POP\_L2
Protocol : HZA116492
Population : Intent-to-Treat


# Listing x Reasons for Important Protocol Deviations

| Randomised | Site Id./<br>Unique | | Excluded | | |
|---|---|---|---|---|---|
| Treatment | Subject Id. | Important Protocol Deviation | from PP? | Date of Deviation | Study Day of Deviation |
| FF/VI | XXXXX | XXXXXXXXXXX | No | DDMMMYYYY | XX |
| | XXXXX | XXXXXXXXXXX | No | DDMMMYYYY | XX |
| Usual ICS/LABA | xxxxx | XXXXXXXXXXX | No | DDMMMYYYY | XX |
| | XXXXX | XXXXXXXXXXX | Yes | DDMMMYYYY | XX |
| | XXXXX | XXXXXXXXXXX | No | DDMMMYYYY | XX |
| | XXXXX | XXXXXXXXXXX | No | DDMMMYYYY | XX |

....

Example Protocol

: POP\_L3 : HZA116492

XXXXXX

XXXXXXXXXXXX

XX


Protocol : HZAT16492
Population : Intent-to-Treat

Listing x Asthma History

XX

XX

Number of asthma exacerbations in the last 12 months that: Site Id./ Did not require oral/systemic Required oral/systemic corticosteroids (not involving Unique corticosteroids (not involving hospitalisation) hospitalisation) Required hospitalisation Treatment Subject Id. Asthma Duration XXXXXX XXXXXX XXXXXXXXXXXX XX XX XX XXXXXX XX XX XXXXXXXXXXX XX XXXXXX XX XX XX XXXXXXXXXXX

Example : POP\_L4
Protocol : HZA116492
Population : Intent-to-Treat


Listing x Smoking History

| Treatment | Site Id./<br>Unique<br>Subject Id. | Smoking<br>Status | Years Smoked/<br>Cigarettes per day | Smoking<br>Pack Years |
|---|---|---|---|---|
| XXXXXX | Xxxxxx/ | Current | xx/ | XX |
| | XXXXX | | XX | |
| | Xxxxxx/<br>xxxxxx | Former | xx/<br>xx | XX |
| | Xxxxxx/<br>xxxxxx | Never | | |

2017N339371\_00 HZA116492

: POP\_L5 Example Protocol : HZA116492

: Intent-to-Treat


Listing x
Exposure to Study Medication

Treatment: Usual ICS/LABA

Population

| Site Id./<br>Unique<br>Subject Id. | Treatment Start Date/<br>Treatment End date | Start date of dose/<br>End date of dose/<br>Duration of dose (days) | Drug | Dose/ Dose<br>Units/ Dose<br>Frequency | Inhalers<br>Dispensed/<br>Inhalers Returns | Dose counter start/<br>Dose counter stop | Compliance (%) During the study |
|---|---|---|---|---|---|---|---|
| XXXX | DDMMMYYY/ | | | | | | XX.XX |
| | DDMMMYYY | DDMMMYYYY/<br>DDMMMYYYY/ | XXXXXXX | XX/ XX/XXXX | X/X | XXX/XX | |
| | | xx<br>DDMMMYYYY/<br>DDMMMYYYY<br>xx | XXXXXXX | XX/ XX/XXXX | X/X | XXX/XX | |
| XXXX | DDMMMYYY | AA. | | | | | XX.XX |
| | | DDMMMYYYY/<br>DDMMMYYYY/<br>xx | XXXXXXX | XX/ XX/XXXX | X/X | XXX/XX | |

Programming note: Repeat on subsequent pages for Treatment = FF/VI, and use GSK drug synonym as drug name.

Example : EFF\_L1 Protocol : HZA116492


Population : Intent-to-Treat

Listing x ACT Scores

Treatment: Usual ICS/LABA

| Site Id./<br>Unique<br>Subject Id. | Visit/<br>Study Date/<br>Study Day | Impact at<br>home or work<br>[1] | Frequency of shortness of breath [1] | Frequency of sleep trouble [1] | Frequency of rescue medication [1] | Asthma control rating [1] | ACT Total<br>Score [2] /<br>Change from<br>Baseline |
|---|---|---|---|---|---|---|---|
| xxxxxx/<br>xxxxx | Randomisation<br>(Day 0)/<br>DDMMMYYYY/<br>xx | х | Х | X | X | х | xx |
| | Week 6/<br>DDMMMYYYY/<br>xx | X | X | X | X | X | xx /<br>-x |
| | Week 12/<br>DDMMMYYYY/<br>xx | Х | Х | X | Х | Х | xx /<br>x |

<sup>[1]</sup> Responses range between 1 (worst response) and 5 (best response).[2] ACT Total Score ranges between 5 (worst asthma control state) and 25 (best asthma control state).

Example Protocol : EFF\_L2 : HZA116492

Population

: Intent-to-Treat


Listing x Inhaler Device Use

Treatment: Usual ICS/LABA

| 0, 11, 1, 1 | | Critical | Critical errors | | Non-critical errors | |
|---|---|---|---|---|---|---|
| Site Id./<br>Unique<br>Subject Id. | Visit/<br>Study Date/<br>Study Day | Inhaler | Any? | If yes, errors: | Any? | If yes, errors: |
| xxxxxx/<br>xxxxx | Randomisation (Day 0)/<br>DDMMMYYYY/ | Turbuhaler | No | | No | |
| | xx<br>Week 12/<br>DDMMMYYYY/ | Turbuhaler | No | | Yes | Did not hold breath |
| | xx<br>Week 24/<br>DDMMMYYYY/<br>xx | Turbuhaler | Yes | Exhaled directly into mouthpiece | No | |
| xxxxxx/<br>xxxxx | Randomisation (Day 0)/<br>DDMMMYYYY/<br>xx | Diskus | Yes | Did not hold device upright during dose preparation Shook the device after dose preparation | Yes | No exhalation before an inhalation |
| | Week 12/<br>DDMMMYYYY/<br>xx | Diskus | Yes | Shook the device after dose preparation | No | |

2017N339371\_00 HZA116492

Example : EFF\_L3

Protocol : HZA116492 Population : Intent-to-Treat Page 1 of n

Trough (Pre-dose) Percent

Listing x Lung Function Tests

Treatment: Usual ICS/LABA

| | | | Trough (Pr | re-dose) FEV1 (L) | | | cted FEV1 (%) | _ | |
|---|---|---|---|---|---|---|---|---|---|
| Site Id./<br>Unique<br>Subject Id. | Visit | Study Date/<br>Time | Study<br>Day | Absolute | Change from<br>Baseline | Predicted<br>normal FEV1 (L) | Absolute | Change from<br>Baseline | Bronchodilator taken in last 4 hours? |
| xxxxxx/<br>xxxxx | Randomisation (Day 0) | DDMMMYYYY/<br>HH:MM | XX | X.XXX | | X.XXX | XX.X | | No |
| | Week 6 | DDMMMYYYY/<br>HH:MM | XX | X.XXX | X.XXX | x.xxx | XX.X | XX.X | No |
| xxxxxx/<br>xxxxx | Randomisation (Day 0) | DDMMMYYYY/<br>HH:MM | XX | X.XXX | x.xxx | X.XXX | XX.X | XX.X | No |

Example : EFF\_L4 Protocol : HZA116492


Population : Intent-to-Treat

Listing x

Medication Adherence Report Scale for Asthma (MARS-A) Scores

Treatment: Usual ICS/LABA

| Site Id./<br>Unique<br>Subject Id. | Status [1] | Visit/<br>Study Date/<br>Study Day | Assessor Code | MARS-A Questions | Score [2] |
|---|---|---|---|---|---|
| xxxxxx/<br>xxxxx | During | Randomisation<br>(Day 0)/<br>DDMMMYYYY/<br>xx | Subject/Other | I only use it when I need it | Х |
| | | | | Only use it when I feel breathless | Χ |
| | | | | I decide to miss out a dose | Χ |
| | | | | I try to avoid using it | Χ |
| | | | | I forget to take it | X |
| | | | | I alter the dose | Χ |
| | | | | I stop taking it for a while | Χ |
| | | | | Reserve if treatment doesn't work | Χ |
| | | | | Before doing something | Χ |
| | | | | I take less than instructed | Χ |
| | | | | MARS-A 10-Score [3] | X.XX |
| | | Week 12/<br>DDMMMYYYY/<br>xx | Subject/Other | I only use it when I need it | x |
| | | | | Only use it when I feel breathlessetc | Χ |

<sup>[1]</sup> Due to an issue identified with the French translation of the MARS-A, a reminder was sent to centres in France instructing that the questionnaire refers to the patient's preventer inhaler (i.e. their maintenance therapy prior to entering the study, and study medication while on-study. Status = Prior (patient in France who had

completed all MARS-A assessments prior to the reminder), During (patient in France who had completed at least one MARS-A assessment prior to the reminder but also completed at least one MARS-A assessment after the reminder), After (patient in France who had not completed any MARS-A assessments prior to the reminder), Germany (patient in Germany).

[2] Question scores range between 1 (always) and 5 (never).

[3] MARS-A 10-Score is based on the mean score across all ten questions.

Example : EFF\_L5
Protocol : HZA116492


Population : Intent-to-Treat

Listing x
Severe Asthma Exacerbations

Treatment: Usual ICS/LABA

| Site Id./<br>Unique<br>Subject Id.<br>Xxxxxx/<br>xxxxxx | Date of Onset/ Study day/ Date of Resolution/ Study day DDMMMYYYY/ xx/ DDMMMYYYY/ xx | Resolution/<br>Withdrawn from Study?<br>Resolved/<br>N | Required use of systemic/oral corticosteroids? | Led to hospitalisation? | Required<br>emergency<br>room visit?<br>N | Required<br>intubation?<br>N |
|---|---|---|---|---|---|---|
| | DDMMMYYYY/<br>xx/<br>DDMMMYYYY/<br>xx | Resolved/<br>N | N | N | Y | N |
| | DDMMMYYYY/ xx/ DDMMMYYYY/ xx | Fatal/<br>Y | Y | Υ | N | Υ |

Example : EFF\_L6 Protocol

Population

: HZA116492

: Intent-to-Treat


Listing x AQLQ(S) Scores

Treatment: Usual ICS/LABA

| Site Id./<br>Unique<br>Subject Id. | Visit/<br>Study Date/<br>Study Day | Symptoms [1] | Activity Limitations [1] | Emotional<br>Function [1] | Environmental<br>Stimuli [1] | AQLQ(S) Total<br>Score [1] /<br>Change from<br>Baseline |
|---|---|---|---|---|---|---|
| xxxxxx/<br>xxxxx | Randomisation<br>(Day 0)/<br>DDMMMYYYY/<br>xx | X.X | X.X | X.X | X.X | X.X |
| | Week 24/<br>DDMMMYYYY/<br>xx | X.X | X.X | X.X | X.X | x.x /<br>x.x |

[1] Scores range between 1 (lower quality of life) and 7 (higher quality of life) for AQLQ(S) total and domains.

## 2017N339371\_00 HZA116492


Example : EFF\_L7
Protocol : HZA116492
Population : Intent-to-Treat


Listing x

EQ-5D-5L Descriptive System Dimension Scores

Treatment: Usual ICS/LABA

| Site Id./<br>Unique<br>Subject Id. | Visit/<br>Study Date/<br>Study Day | Assessor Code | Subscale/<br>Item | Level of Problem | Score [1] |
|---|---|---|---|---|---|
| xxxxxx/<br>xxxxx | Randomisation<br>(Day 0)<br>DDMMMYYYY/<br>xx | Subject/Other | EQ-5D-5L Utility<br>Score | | XX.XX |
| | | | Mobility Self-Care Usual Activities Pain/Discomfort Anxiety/Depression | 1<br>1<br>1<br>1 | |
| | | | EQ-5D-5L VAS | | XX.XX |
| | Week 12<br>DDMMMYYYY/<br>xx | Subject/Other | EQ-5D-5L Utility<br>Score | | xx.xx |
| | | | Mobilityetc | 1 | |

<sup>[1]</sup> Scores range between 0 (worst imaginable health state) and 1 (best imaginable health state) for EQ-5D-5L Utility Score and range between 0 (worst imaginable health state) and 100 (best imaginable health state) for EQ-5D-5L Visual Analogue Scale (VAS).

Example Protocol : EFF\_L8 : HZA116492 Population : Intent-to-Treat


Listing x PASAP-Q Scores

Treatment: Usual ICS/LABA

Visit/

| Site Id./ | Study Date/ | 5 | | |
|---|---|---|---|---|
| Unique | Study Day | Domain /<br>Question | Response | Coore [1] |
| Subject Id. | Dandamiastian | | | Score [1] |
| xxxxxx/<br>xxxxx | Randomisation<br>(Day 0)<br>DDMMMYYYY/ | Performance | | XX.X |
| | XX | | | |
| | | Overall feeling of inhaling | Χ | |
| | | Inhaled dose goes to lungs | Χ | |
| | | Medication left | Χ | |
| | | Works reliably | Χ | |
| | | Ease of inhaling a dose | Χ | |
| | | Using the inhaler | Χ | |
| | | Speed medicine comes out | Χ | |
| | | Convenience | | XX.X |
| | | Instructions for use | Χ | |
| | | Size of inhaler | Χ | |
| | | Durability of inhaler | Χ | |
| | | Ease of cleaning inhaler | Χ | |
| | | Ease of holding during use | Χ | |
| | | Convenience of carrying | Х | |
| | | Total Score | | XX.X |
| | | Overall Satisfaction | | X |
| | | Willingness to Continue Using Inhaler | | XX.X |

[1] Performance, Convenience, Total Score, and Willingness to Continue Using Inhaler are expressed on a scale of 0 to 100. Overall Satisfaction is expressed on a scale of 1 to 7.

Example Protocol : SAFE\_L1 : HZA116492


Population : Intent

: Intent-to-Treat

# Listing x AE Terms of Special Interest

| Special Interest Group | Subgroup | Preferred Term |
|------------------------|--------------------|-----------------------------|
| XXXXX XXXXX XXXXXX | Xxxxxxx | XXXXXXX |
| | | XXXXXXX XXXXXXX |
| | | XXXX |
| | | XXXXXXX XXX |
| XXXXXXX XXXXXXXXXX | xxxxxxxxxxxxxx [1] | xxxxxx xxxxxx |
| | | XXXXXXX XXXX XXXXX XXXXX |
| | | XXXX |
| XXXXXXXXXX | xxxxxxx [1] | xxxxxxx |
| | | XXXX XXXXXX XXXXXXX |
| XXXXXX XXXXXXX | | XXXXXXXX |
| | | XXXXX XXXXXX XXXXXXX XXXXXX |

<sup>[1]</sup> This special interest group/subgroup was defined using Special MedDRA Queries. Note: All of the pre-specified preferred terms that were assigned to special interest terms are shown, regardless of whether they actually occurred in the study.

Programming Note: The AE special interest dataset and the AE SMQ dataset will be set together in order to report this table and all the subgroups that come from the AE SMQ dataset will be flagged with a [1].

Example Protocol : SAFE\_L2 : HZA116492

Population : Intent-to-Treat Page 1 of n

Listing x
Inhaler Device Malfunctions

| Treatment | Site Id./<br>Unique Subject Id. | Inhaler Device | Comment / Reason for Malfunction |
|---|---|---|---|
| Usual ICS/LABA | xxxxxx/<br>xxxxx | Turbuhaler | XXXXXXXXXX |
| Usual ICS/LABA | xxxxxx/<br>xxxxx | Diskus | XXXXXXXXXX |
| FF/VI | xxxxxx/<br>xxxxx | Ellipta | Powder fell out prior to use<br>Other: XXXXXXXX |

#### The GlaxoSmithKline group of companies

HZA116492

| Division | : Worldwide Development |
|------------------|-------------------------------------|
| Information Type | : Reporting and Analysis Plan (RAP) |

| Title | : | Reporting and Analysis Plan for A 6-month, open label, randomised, efficacy study to evaluate fluticasone furoate (FF, GW685698)/vilanterol (VI, GW642444) Inhalation Powder delivered once daily via the Dry Powder Inhaler Ellipta Compared with usual ICS/LABA maintenance therapy delivered by Dry Powder Inhaler in subjects with Persistent Asthma |
|---|---|---|
| Compound Number | : | GW685698+GW642444 |
| Effective Date | : | 05-DEC-2016 |

#### **Description:**

The purpose of this document is to describe the final planned analyses and output to be included in the Clinical Study Report for Protocol HZA116492.

This RAP is intended to describe the planned efficacy and safety analyses required for the study.

This RAP will be provided to the study team members to convey the content of the final Statistical Analysis Complete (SAC) deliverable.

#### **Author's Name and Functional Area:**

| PPD | | 05-DEC-2016 |
|----------------------|--------------------------|-------------|
| Principal Statistici | an (Clinical Statistics) | 03-DEC-2010 |

#### Approved by:

| PPD | | 05-DEC-2016 |
|----------------|--------------------------------------------|-------------|
| Director, Stat | istics & Programming (Clinical Statistics) | 03-DEC-2010 |

Copyright 2016 the GlaxoSmithKline group of companies. All rights reserved. Unauthorised copying or use of this information is prohibited.

HZA116492

## **TABLE OF CONTENTS**

| | | | PAGE |
|---|---|---|---|
| 1. | SUMM<br>1.1.<br>1.2.<br>1.3.<br>1.4. | ARY OF KEY PROTOCOL INFORMATION Changes to the Protocol Defined Statistical Analysis Plan Study Objectives and Endpoints Statistical Hypotheses Sample Size Assumptions | 8<br>11<br>15 |
| 2. | PLANN<br>2.1.<br>2.2.<br>2.3. | NED ANALYSES Interim Analyses Data Look Final Analyses | 17<br>17 |
| 3. | ANALY<br>3.1. | /SIS POPULATIONSProtocol Deviations | |
| 4. | | IDERATIONS FOR DATA ANALYSES AND DATA HANDLING ENTIONS | 20 |
| 5. | STUDY<br>5.1. | Y POPULATION ANALYSES<br>Overview of Planned Analyses | |
| 6. | PRIMA<br>6.1. | ARY STATISTICAL ANALYSES Efficacy Analyses | 22<br>22 |
| 7. | SECOI<br>7.1.<br>7.2. | NDARY STATISTICAL ANALYSES Efficacy Analyses 7.1.1. Overview of Planned Efficacy Analyses 7.1.2. Planned Efficacy Statistical Analyses Safety Analyses 7.2.1. Overview of Planned Analyses 7.2.2. Benefit:Risk analyses | 26<br>26<br>27<br>29 |
| 8. | OTHER<br>8.1. | R STATISTICAL ANALYSES Other Analyses | 32<br>32 |
| 9. | REFER | RENCES | 37 |
| 10. | APPEN<br>10.1. | Appendix 1: Protocol Deviation Management and Definitions for PP Population | 39 |
| | 10.2.<br>10.3. | 10.1.2. Exclusions from PP Population | 41<br>41 |
| | 10.4. | Appendix 4: Treatment States and Phases | |

HZA116492


| | 10.4.1. | | Phases | |
|---|---|---|---|---|
| | 10.4.2. | | States | |
| | | | Treatment States for Concomitant Medications | |
| | | | Treatment States for Efficacy Measurements | |
| | | | Treatment States for Exacerbation Data | |
| 10.5 | A a ali. | | Treatment States for AE Data | |
| 10.5. | | Study Tro | splay Standards & Handling Conventions | 40 |
| | 10.5.1.<br>10.5.2. | | tment & Sub-group Display Descriptorsefinition & Derivations | |
| | 10.5.2. | | Baseline Definitions | |
| | | | Derivations and Handling of Missing Baseline | 40 |
| | | 10.5.2.2. | Data | 46 |
| | 10.5.3. | Reporting | Process & Standards | |
| 10.6. | | | and Transformed Data | |
| | 10.6.1. | | | |
| | 10.6.2. | | ulation | |
| | 10.6.3. | | | |
| | 10.6.4. | | | |
| 10.7. | Appendix | ι 7: Prematι | ure Withdrawals & Handling of Missing Data | 57 |
| | 10.7.1. | Premature | Withdrawals | 57 |
| | 10.7.2. | | f Missing Data | |
| | | | Handling of Missing or Partial Dates | 57 |
| | | 10.7.2.2. | Handling of Missing Data for Statistical | |
| | | | Analysis | |
| 10.8. | | | of Potential Clinical Importance | |
| 40.0 | 10.8.1. | | | |
| 10.9. | | | nter Studies | |
| 10 10 | 10.9.1. | | or Handling Centres | |
| 10.10. | | | nation of Covariates, Subgroups & Other Strata<br>on of Strata and Covariates | |
| | | | on of subgroups | |
| | | | on of seasonal effect | |
| 10 11 | | | e Comparisons & Multiplicity | |
| 10.11. | | | f Multiple Comparisons & Multiplicity | |
| 10.12. | | | Checking and Diagnostics for Statistical | |
| | | | | 64 |
| | 10.12.1. | Statistical A | Analysis Assumptions | 64 |
| 10.13. | | | g Strategy | |
| | | | viations & Trade Marks | |
| | 10.14.1. | Abbreviation | ons | 68 |
| | | | S | |
| 10.15. | Appendix | c 15: List of | Data Displays | 70 |
| | | | ay Numbering | |
| | | | nple Shell Referencing | |
| | | | e [Priority] | |
| | | | ulation Tables | |
| | | | ulation Figures | |
| | | | ables | |
| | | | guresles | |
| | | | iles | |
| | | ICH Listing | | 102 |

| | | HZA116492 |
|----------|---------------------------------------------|-----------|
| 10.15.11 | .Non-ICH Listings | 103 |
| | ( 16: Example Mock Shells for Data Displays | |
| 10.16.1. | Study Population Table Shells | 105 |
| 10.16.2. | Study Population Figure Shells | 121 |
| 10.16.3. | Efficacy Table Shells | 122 |
| | Efficacy Figure Shells | |
| 10.16.5. | Safety Table Shells | 181 |
| 10.16.6. | Safety Figure Shells | 185 |
| 10.16.7. | Non-ICH Listing Shells | 187 |

HZA116492

## **REPORTING & ANALYSIS PLAN SYNPOSIS**

| Overview | Key Elements of the RAP |
|---|---|
| Purpose | This RAP details all planned analyses and output required for the final Clinical Study Report of study HZA116492. |
| Protocol | This RAP is based on the protocol amendment 02 (Dated: 28-APR-2016) of study HZA116492 (GSK Document No.: 2014N190259_02). |
| Primary<br>Objective | To compare the efficacy of fluticasone furoate (FF)/vilanterol(VI) 92 mcg/22 mcg or FF 184 mcg/22 mcg with usual fixed combinations inhaled corticosteroid / long-acting beta agonist (ICS/LABA) for asthma maintenance therapy at Week 12 (Visit 4). |
| Primary<br>Endpoint | Change from baseline in the Asthma Control Test (ACT) total score at Week 12 (Visit 4). |
| Study<br>Design | This is a Phase IIIb multi-center randomised open label, parallel group study performed in subjects in primary and in respiratory specialist care / research sites who have a diagnosis of asthma and a regular treatment for asthma. Subjects with unsatisfactorily controlled asthma (defined as an ACT < 20) and intended to be treated by usual ICS/LABA maintenance therapy to seek a better control of their asthma will be randomised to receive either FF/VI (FF/VI 92 mcg/22 mcg or FF/VI 184 mcg/22 mcg) once daily or another usual ICS/LABA combination therapy in inhalation powder twice daily (fluticasone propionate[FP]/salmeterol [S] or budesonide[BUD]/formoterol [F]) decided by the physician. Physicians will be allowed during the treatment period to adapt prescription to different doses if necessary as well as to adapt doses of any comparative treatment according to products label. |
| Planned | No interim analysis is planned for this study. |
| Analyses | All decisions regarding final analysis for the reporting effort, as defined in this RAP document, will be made prior to Database Freeze (DBF) (unblinding) of the study data. |
| | All planned analyses will be carried out once DBF has taken place. Once this has been achieved, unblinding will occur and the analyses will be performed. |
| | The open-label study design and the method of recording study medication data in the datasets means that extra steps must be taken to ensure that Statistics and Programming (S&P) remain blinded to study investigator prescribing of study medication until the formal unblinding takes place at DBF. See Section 10.13 for more details. |

HZA116492

| Overview | Key Elements of the RAP |
|---|---|
| Analysis<br>Populations | All Subjects Enrolled (ASE) population: All subjects screened (provided consent) and for whom a record exists on the study database. Note, this population is not identified in the protocol, but is needed for displays that include subjects screened but not in the intent-to-treat (ITT) population (e.g. tabulation of reasons for withdrawal before randomisation). |
| | Intent-to-treat (ITT) population: All randomized subjects having received at least one dose of the prescription of study medication (either FF/VI or usual ICS/LABA asthma maintenance therapy). The ITT population will be used to analyze the primary efficacy endpoint analysis, the secondary efficacy endpoint and other efficacy endpoints. Subjects will be assigned to the treatment group as randomized for the ITT population. |
| | Per protocol (PP) population: all ITT subjects without any protocol deviations specifically defined in this RAP. Protocol deviations will be reviewed and will be classified as important or not important during data review meetings that will be held before DBF. Deviations classified as important will be further defined according to whether they require the patient to be excluded from the PP population. Deviations that exclude a patient from the PP population are defined in this RAP (see Section 10.1.2). Subjects will be assigned to the treatment group as treated for the PP population. |
| | Safety population: All enrolled subjects having received at least one dose of the prescription of study medication (either FF/VI or usual ICS/LABA asthma maintenance therapy) and considered as-treated. The Safety population will be the basis for safety analyses. Subjects will be assigned to the treatment group as treated for the Safety population. |
| Hypothesis | The primary analysis is designed to determine whether the fixed combination FF/VI is non-inferior to any other ICS/LABA combinations in inhalation powder assuming a non-inferiority margin of 1.5. Non-inferiority will be claimed if the 95% two-sided confidence interval (CI) on the difference in mean primary efficacy endpoints (FF/VI versus ICS/LABA comparator) precludes the non-inferiority margin of -1.5. |
| | If (and only if) non-inferiority is significantly achieved at Week 12 (Visit 4) with regard to the primary endpoint, then non-inferiority of the fixed combination FF/VI to any other ICS/LABA combinations will be tested at Week 24 (Visit 6) considering the same non-inferiority margin of 1.5. Non-inferiority will be claimed if the 95% two-sided CI on the difference in mean primary efficacy endpoints (FF/VI versus ICS/LABA comparator) at Week 24 (Visit 6) precludes the non-inferiority margin of -1.5. This step-down testing procedure strongly controls the overall type I error of the non-inferiority endpoints at the 0.05 two-sided level. |
| Primary<br>Analyses | The primary endpoint will be analysed using a mixed model repeated measures (MMRM) approach. The model will include factors and covariates as follows: randomised treatment, scheduled visit time point (Week 6 and Week 12), baseline ACT total score, randomised treatment-by-visit interaction, baseline ACT total score-by-visit interaction, gender, age, country and patient will be fitted as a random factor. The Restricted Maximum Likelihood (REML) estimation approach will be used, and the default covariance structure will be unstructured. Consistent with MMRM model fitting, no explicit imputation of missing assessments for a given time point will be performed. The adjusted means for each treatment and the estimated treatment differences for the treatment comparisons will be presented together with the 95% CIs for the differences (FF/VI versus ICS/LABA comparator) and p-values at Week 12 (Visit 4). |
| | If non-inferiority is statistically achieved at Week 12 (Visit 4), then superiority of FF/VI to any other comparator will be tested at the usual 0.05 two-sided nominal level of significance. |

HZA116492

| Overview | Key Elements of the RAP |
|---|---|
| | The same models and analyses mentioned above will be used to assess the superiority hypothesis. |
| Secondary<br>Analyses | Key secondary analysis |
| Analyses | The key secondary endpoint assessed at Week 24 (Visit 6) will also be analyzed using a MMRM approach where data up to and including Week 24 (Visit 6) will be used in the model. The model will include factors and covariates as follows: randomised treatment, scheduled visit time point (Week 6, Week 12, Week 18 and Week 24), baseline ACT total score, randomised treatment-by-visit interaction, baseline ACT total score-by-visit interaction, gender, age, country and patient will be fitted as a random factor. The REML estimation approach will be used, and the default covariance structure will be unstructured. Consistent with MMRM model fitting, no explicit imputation of missing assessments for a given time point will be performed. The adjusted means for each treatment and the estimated treatment difference for the treatment comparison will be presented together with the 95% CI for the difference (FF/VI versus ICS/LABA comparator) and p-value at Week 24 (Visit 6). If non-inferiority is statistically achieved at Week 24 (Visit 6), then superiority of FF/VI versus any other comparator will be tested at the usual 0.05 two-sided nominal level of significance. The same models and analyses mentioned above will be used to assess the superiority hypothesis. |
| | Other secondary analyses |
| | The other key secondary endpoint will be the correct use of the inhaler device assessed at randomisation (Visit 2), at Week 12 (Visit 4) and at Week 24 (Visit 6). The device will be considered as correctly used if the patient didn't make any critical or non-critical errors at the corresponding visits (randomisation [Visit 2], Week 12 [Visit 4] and Week 24 [Visit 6]). Percentages of subjects correctly using the device will be calculated within each group. A corresponding 95% CI of the difference in percentages will also be provided. |
| | An exploratory analysis of the categorised data will be performed using logistic regression models with covariates as follows: randomised treatment, correct use of inhaler device at baseline, randomised treatment-by-visit interaction, gender, age and country. The estimated treatment differences will be displayed as odds ratios together with 95% CIs and p-values. |

HZA116492

## 1. SUMMARY OF KEY PROTOCOL INFORMATION

## 1.1. Changes to the Protocol Defined Statistical Analysis Plan

Any changes from the originally planned statistical analysis specified in the protocol are outlined in Table 1.

Table 1 Changes to Protocol Defined Analysis Plan

| Protocol | Reporting & Analysis Plan | |
|---|---|---|
| Statistical Analysis Plan | Statistical Analysis Plan | Rationale for Changes |
| • N/A | The open-label study design and the method of recording study medication data in the datasets means that extra steps must be taken to ensure that S&P remain blinded to study investigator prescribing of study medication until the formal unblinding takes place at DBF. See Section 10.13 for more details. | To preserve the integrity of<br>the analyses, S&P will<br>remain blinded prior to<br>formal unblinding at DBF.<br>All planned analyses will be<br>carried out after this point. |
| • N/A | All Subjects Enrolled (ASE) Population: All subjects screened (provided consent) and for whom a record exists on the study database. Note, this population is not identified in the protocol, but is needed for displays that include subjects screened but not in the ITT Population (e.g. tabulation of reasons for withdrawal before randomisation). | Population needed for<br>displays that include<br>subjects screened but not in<br>the ITT population. |
| <ul> <li>Continuous variables will be summarized using descriptive statistics (number of observed and missing data, mean, standard deviation (SD), median, Q1, Q3, minimum, and maximum).</li> <li>Categorical variables will be summarized as numbers of observed and missing data, counts and percentage for each category (reported to the number of non-missing values). For binary variables, 95% confidence</li> </ul> | See Appendix 16: Example Mock Shells for Data Displays for example mock shells for data displays | Continuous and categorical variables will be summarized in line with GSK Integrated Data Standards Library (IDSL) data standards |

HZA116492

| Protocol | | Reporting & Analysis Plan | | | |
|---|---|---|---|---|---|
| Statistical Analysis Plan | | Sta | Statistical Analysis Plan | | Rationale for Changes |
| | intervals for proportions will be estimated based on the Clopper-Pearson method. | | | | |
| • | If treatment is withdrawn, then the missing ACT score at the nearest visit after treatment withdrawal will be replaced by the ACT score assessed at withdrawal time. If no ACT score is assess at withdrawal time, then the ACT missing score at the nearest visit after treatment withdrawal will not be replaced. | • | Consistent with MMRM model fitting, no explicit imputation of missing assessments for a given time point will be performed. | • | The protocol inconsistently describes whether or not missing scores will be imputed. Consistent with MMRM models and the MAR assumption they are based upon, no missing data will be imputed for the primary efficacy analysis. Sensitivity analyses for the primary endpoint are proposed in Section 6.1.2 and will consider imputation of missing data. |
| • | The primary endpoint will be analysed using a mixed model repeated measures (MMRM) approach. The model will include factors and covariates as follows: treatment, scheduled visit time point (Week 6 and Week 12), baseline ACT, treatment by visit interaction, baseline ACT by visit interaction, gender, age and patient will be fitted as a random factor. | • | The primary endpoint will be analysed using a MMRM approach. The model will include factors and covariates as follows: randomised treatment, scheduled visit time point (Week 6 and Week 12), baseline ACT total score, randomised treatment-by-visit interaction, baseline ACT total score-by-visit interaction, gender, age, country and patient will be fitted as a random factor. | • | Clarified that randomised treatment and baseline ACT total score will be included. Additionally country will be included in the model due to the addition of Germany, and separate randomisation schedules for France and Germany achieving stratification by country Same changes for secondary and other analyses |
| • | Sensitivity analyses (for the primary endpoint) | • | Text changed and clarified | • | The text from the protocol regarding sensitivity analyses has been updated and clarified where necessary. Description of the multiple imputation (MI) process has been brought in line with GSK standard text. |
| • | Usual ICS/LABA maintenance therapy | • | Usual ICS/LABA | • | The comparator arm is described as "Usual ICS/LABA" for consistency with reporting of the HZA115150 study (GSK Document No.: 2011N129785_02). |
| • | EQ-5D | • | EQ-5D-5L | • | Clarity as to which version |

HZA116492

| Protocol | Reporting & Analysis Plan | |
|---|---|---|
| Statistical Analysis Plan | Statistical Analysis Plan | Rationale for Changes |
| | | of the EuroQol questionnaire is being used |
| <ul> <li>Binary response defined as an ACT score ≥ 20 at a given visit OR a 3 point increase from baseline in ACT change.</li> <li>The responder analyses will be conducted using a logistic regression model at a given Visit or Phone Call adjusting for treatment and stratification factors (baseline ACT score categorized into two classes, baseline asthma therapy, and potentially season at randomization). Treatment by stratification factors interaction effects will be further investigated in additional logistic models adjusting for these specific effects.</li> </ul> | This endpoint will be analysed using a logistic regression model adjusting for randomised treatment, gender, country, baseline ACT total score, baseline ACT total score squared and age | <ul> <li>Clarified that randomised treatment will be included.</li> <li>Country will be included in the model due to the addition of Germany, and separate randomisation schedules for France and Germany achieving stratification by country</li> <li>Due to this being a composite endpoint, a quadratic relationship is expected between baseline score and probability of response. Baseline ACT total score and baseline ACT total score squared will be included (instead of "baseline ACT score categorised into two classes") to account for this</li> <li>All patients are on the same baseline asthma therapy class (ICS), therefore this will not be included; this is only considered as sensitivity analysis for the primary efficacy endpoint</li> </ul> |
| • N/A | ≥ 3 point increase from baseline in ACT total score at Week 12 (Visit 4) and Week 24 (Visit 6) Time to first severe asthma exacerbation | These endpoints have been added for consistency with the HZA115150 study (GSK Document No.: 2011N129785_02). |

HZA116492

## 1.2. Study Objectives and Endpoints

| Ob | ectives | Endpoints |
|---|---|---|
| | mary Objective | Primary Endpoint |
| • | To compare the efficacy of FF/VI 92 mcg/ 22 mcg or FF 184 mcg/22 mcg with usual fixed combinations ICS/LABA for asthma maintenance therapy at Week 12 (Visit 4). | Change from baseline in the ACT total score at Week 12 (Visit 4). |
| Sec | condary Objectives | Secondary Endpoints |
| • | To assess effect of FF/VI on asthma control compared with usual ICS/LABA fixed combination at Week 24 (Visit 6). | Change from baseline in ACT score at Week 24 (Visit 6). |
| • | To assess Ellipta™ inhaler correct use compared with other dry powder inhaler (DPI) (Diskus™ and Turbuhaler) at Week 12 (Visit 4) and at Week 24 (Visit 6) independently of the use at Week 12 (Visit 4). | <ul> <li>Percentage of subjects with correct use of device<br/>(defined as not making any critical error or non-<br/>critical error) at Week 12 (Visit 4) and at Week 24<br/>(Visit 6) independently of the use at Week 12 (Visit<br/>4).</li> </ul> |
| Oth | ner Objectives | Other Endpoints |
| • | To assess effect of FF/VI on trough (predose) forced expiratory volume in 1 second (FEV1) compared with usual ICS/LABA fixed combination at Week 12 (Visit 4) | Change from baseline in trough (pre-dose) FEV1 at Week 12 (Visit 4). |
| • | To assess the effect of FF/VI on response to treatment at Week 12 (Visit 4) and Week 24 (Visit 6) | <ul> <li>ACT score ≥ 20 or ≥ 3 point increase from baseline in ACT at Week 12 (Visit 4) and Week 24 (Visit 6). Note: A 3 point increase in ACT total score was suggested as the Minimal Clinically Important Difference (MCID) in the literature (Schatz, 2009).</li> <li>ACT score ≥ 20 at Week 12 (Visit 4) and Week 24 (Visit 6).</li> <li>≥ 3 Point Increase from Baseline in ACT Total Score at Week 12 (Visit 4) and Week 24 (Visit 6).</li> <li>Change from baseline in individual question scores for ACT at Weeks 12, 24</li> </ul> |
| • | To assess the compliance with study medication and self-reported adherence to study medication at Week 12 (Visit 4) and Week 24 (Visit 6) | <ul> <li>Compliance with study medication from randomisation (Day 0) to Week 12 (Visit 4), from Week 12 (Visit 4) to Week 24 (Visit 6) and from randomisation (Day 0) to Week 24 (Visit 6).</li> <li>Score of the Medication Adherence Report Scale for Asthma (MARS-A) questionnaire at randomisation (Day 0), Week 12 (Visit 4) and Week 24 (Visit 6).</li> </ul> |
| • | To assess the effect of FF/VI on severe asthma exacerbation over the study period | Number of subject with at least 1 severe asthma<br>exacerbation*, number of severe asthma<br>exacerbation and annual severe exacerbation rate<br>over the study period. |

HZA116492

| Objectives | Endpoints |
|---|---|
| | Time to first severe asthma exacerbation |
| To assess the effect of FF/VI on Health<br>Related Quality of Life at Week 24 (Visit 6) | <ul> <li>Change from baseline in total score and domain scores of standardised Asthma Quality of Life Questionnaire (AQLQ[S]) at Week 24 (Visit 6).</li> <li>An increase from baseline of ≥ 0.5 in AQLQ(s) total score at Week 24 (Visit 6).</li> <li>An increase from baseline of ≥ 0.5 in AQLQ(s) environmental stimuli domain score at Week 24 (Visit 6).</li> <li>Percentage of subjects who have an increase from baseline of ≥ 0.5 in AQLQ(S) individual domain scores at Week 24 (Visit 6).</li> <li>Change from baseline in total score and domain scores of AQLQ(S) at Week 24 (Visit 6).</li> <li>Health status using the EuroQol Questionnaire (EQ-5D-5L) at Week 24 (Visit 6).</li> </ul> |
| To assess Patient Satisfaction and<br>Preference assessment with different<br>inhalers at Week 12 (Visit 4) | Score of Patient Satisfaction and Preference Questionnaire (PASAP-Q) at Week 12 (Visit 4). |
| To evaluate the Safety of FF/VI compared with usual ICS/LABA (FP/S and BUD/F). | Serious Adverse Events (SAE) and non-serious Adverse Drug Reactions (ADR): Frequency and type of SAEs, Frequency and type of non-serious ADRs related to treatment. |

<sup>\*</sup> A severe asthma exacerbation will be defined as deterioration of asthma requiring the use of systemic corticosteroids<sup>2</sup> (tablets, suspension, or injection) for at least 3 days or an inpatient hospitalisation, or emergency department visit due to asthma that required systemic corticosteroids <sup>1,2,3</sup>.

#### Notes defining endpoints:

- 1. Contacts with a doctor or hospitalisation are defined as exacerbation-related contacts if these contacts were a direct result of an acute worsening of asthma symptoms.
- 2. A prescription of systemic corticosteroid is defined as exacerbation-related if the reason the drug was given, in whole or in part, was to treat an acute worsening of asthma symptoms.
- 3. Exacerbation-related hospitalisation includes hospitalisation that is prolonged as a result of an asthma exacerbation.

HZA116492



- A phone call is provided at Week 6 and Week 18 in order to check whether the subject has
  experienced any AEs and then the Investigator calling the patient must determine whether the
  event is related to study medication (either arm) and whether the event is serious. At these
  telephone calls subjects will also be asked to complete the ACT questionnaire and to send it back
  to the Investigator.
- Week 12 (Visit 4) should be scheduled at the same time of day as the randomisation visit (Visit 2).

## Design Features

- This is a Phase IIIb multi-center randomised open label, parallel group study performed in subjects in primary and respiratory specialist care / research sites who have a diagnosis of asthma and a regular treatment for asthma.
- Subjects with unsatisfactorily controlled asthma (defined as ACT total score < 20) and
  intended to be treated by usual ICS/LABA maintenance therapy to seek a better
  control of their asthma will be randomised to receive either FF/VI once daily or another
  usual ICS/LABA combination therapy in inhalation powder twice daily (FP/S or BUD/F)</li>

HZA116492

| Overview of St | udy Design and Key Features | | |
|---|---|---|---|
| | decided by the physician. | | |
| Treatment<br>Assignment | Subjects will be assigned to study schedule. | y treatment in accord | dance with the randomisation |
| | Subjects will be randomised in a 1:1 ratio to one of the 2 following treatment groups: | | |
| | FF/VI (as per dose guidance below) | | |
| | Initiate on usual inhaled dry powder ICS/LABA fixed combination for asthma maintenance therapy (i.e. Seretide Diskus™ or Symbicort Turbuhaler) according to usual physician's prescription. | | |
| | Dose Guidance: | | |
| | For subjects randomised to FF/VI, Investigator can make dosing decision based on the guidance below: | | |
| | FF/VI 92 mcg/22mcg dose once a day is approximately equivalent to FP/S medium dose (250 mcg/50mcg) and BUD/F medium dose (200 mcg/6 mcg) twice a day. See Table 2 for further guidance for doses conversion for other corticosteroids. | | |
| | FF/VI 184 mcg/22 mcg dose once a day is approximately equivalent to FP/S high dose (500 mcg/50 mcg) and to BUD/F high dose (400 mcg/12 mcg) twice a day. See Table 2 for guidance for dose conversion for other corticosteroids. | | |
| | Starting doses are: 92 mcg/22 mcg once daily for FF/VI; 250 mcg/50 mcg twice daily for FP/S and 200 mcg/6 mcg twice daily for BUD/F. | | |
| | Table 2 ICS/LABA Daily Dose (SmPC Seretide Diskus™; Symbicort Turbuhaler) | | |
| | Formulation | Inhaler Devices | Doses Available (mcg)<br>ICS/LABA and<br>Inhalations/day |
| | Fluticasone propionate/salmeterol | DPI (Diskus) | 1 inhalation x 2 |
| | | | Medium-dose 250/50 |
| | | | High-dose 500/50 |
| | Budesonide/formoterol | DPI (Turbuhaler) | 1-2 inhalations x 2 |
| | | | Medium-dose 200/6 |
| | | | High-dose 400/12 |
| Information extracted from Global Initiative for Asthma (GINA, 2012). For patients with moderate to severe hepatic impairment, the 92/22 micro | | | A, 2012). |
| | FF/VI should be used and patients should be monitored for systemic corticosteroid-related | | |

HZA116492

| Overview of Study Design and Key Features | |
|---|---|
| | adverse reactions. |
| | Planned Dose Adjustments |
| | Subjects randomised to the usual ICS/LABA asthma maintenance therapy arm can have their treatment adjusted as would be normal clinical practice at the Investigator's discretion. This will not require the subject to be withdrawn from the study. These subjects should not receive FF/VI, if the medication is marketed during the study period. |
| | Subjects randomized to the FF/VI arm and for whom it is considered appropriate/ necessary to adjust treatment, can have their regimen changed as required as per normal clinical practice at any point in the study and the subject could remain in the study. Subjects on FF/VI arm can also change between the two FF/VI doses as appropriate and at the Investigator's discretion. |
| Interim<br>Analysis | No interim analysis is planned for this study. |

From this point onwards in the RAP, usual ICS/LABA maintenance therapy will be referred to as usual ICS/LABA.

### 1.3. Statistical Hypotheses

The primary endpoint is defined as the change from baseline in the ACT total score assessed at Week 12 (Visit 4). The primary analysis will assess the non-inferiority of fixed combination FF/VI to usual ICS/LABA in inhalation powder assuming a non-inferiority margin of 1.5. Non-inferiority will be claimed if the 95% two-sided confidence interval on the difference in mean primary efficacy endpoints (FF/VI versus usual ICS/LABA) precludes the non-inferiority margin of -1.5.

If (and only if) non-inferiority is significantly achieved at Week 12 (Visit 4) with regard to the primary endpoint, then non-inferiority of the fixed combination FF/VI to usual ICS/LABA will be tested at Week 24 (Visit 6) considering the same non-inferiority margin of 1.5. Non-inferiority will be claimed if the 95% two-sided confidence interval on the difference in mean primary efficacy endpoints (FF/VI versus usual ICS/LABA) at Week 24 (Visit 6) precludes the non-inferiority margin of -1.5.

Of note, as the two tests for non-inferiority are sequentially performed, the closure principle holds and there is no need to adjust the two-sided nominal level of significance (i.e. 0.05) for each test.

### 1.4. Sample Size Assumptions

Results based on the HZA106829 study have shown that the estimated SD of the change in ACT score was 3.7. Unpublished data have shown that the standard deviation of change of ACT ranged from 3.8 to 4.8. Therefore, a somewhat conservative choice of SD of 4.5 point is retained.

Based on the literature (Schatz, 2009), the Minimally Important Difference (MID) of the ACT could be considered as 3 points. Half this MID (i.e. 1.5) could therefore be used to define the non-inferiority margin.

HZA116492

Assuming a 4.5 point standard deviation for the change in ACT total score at Week 12 (Visit 4), a 1.5 point non-inferiority margin, and a two-sided nominal significance level of 0.05, the sample size needed per group to achieve at least a 90% power is 191 (i.e. a total of 382 subjects). Assuming a 10% dropout rate, around 422 subjects must be randomized either to FF/VI or to usual ICS/LABA in 1:1 ratio to achieve at least a 90% power.

HZA116492

### 2. PLANNED ANALYSES

## 2.1. Interim Analyses

Not applicable.

#### 2.2. Data Look

At a date agreed by the study team and the contract research organisation (CRO) (selected to execute the statistical analyses specified in this RAP), a data look will be performed using blinded treatment codes on a subset of the data. The aim of the data look is solely to ensure that all of the required tables, figures and listings are being produced and formatted correctly, such that the output produced on unblinded data at the end of the study is correct and complete. This data look will be performed when sufficient data are available, but early enough to leave time for changes to be made to the planned outputs and methods prior to database release (DBR). Any changes will be documented before DBR.

## 2.3. Final Analyses

All planned analyses will be performed after the completion of the following sequential steps:

- 1. All subjects have completed the study as defined in the protocol
- 2. All required database cleaning activities have been completed and final DBR has been declared by Data Management.
- 3. All protocol deviations (PDs) have been confirmed
- 4. All criteria for unblinding the randomisation codes have been met.
- 5. Randomisation codes have been distributed according to RandAll NG procedures.
- 6. DBF has been declared by Data Management.
HZA116492

# 3. ANALYSIS POPULATIONS

| Population | Definition / Criteria | Analyses Evaluated |
|---|---|---|
| All Subjects<br>Enrolled (ASE) | Comprise of all subjects screened (provided consent) and for whom a record exists on the study database. | Subject disposition tables |
| | Note, this population is not identified in the protocol, but is needed for displays that include subjects screened but not in the ITT Population (e.g. tabulation of reasons for withdrawal before randomisation) | |
| Intent-To-Treat<br>(ITT) | Comprise of all randomized subjects having<br>received at least one dose of the prescription of<br>study medication (either FF/VI or usual ICS/LABA) | Study Population Efficacy |
| | Subjects will be assigned to the treatment group as randomized for the ITT population | |
| Per Protocol (PP) | Comprise of all ITT subjects without any major violations of study procedures. | This population will be used for summaries |
| | Major protocol violations will be identified prior to database lock. | and analyses of the<br>primary efficacy<br>secondary efficacy |
| | Protocol deviations will be reviewed and classified as minor or major during a data review meeting that will be held before database lock. | endpoints. |
| | Exclusion of subjects from the PP population are defined in Section 3.1 (Protocol Deviations) and Appendix 1: Protocol Deviation Management and Definitions for PP Population | |
| | Subjects will be assigned to the treatment group as treated for the PP population | |
| Safety | <ul> <li>Comprise of all enrolled subjects having received at least one dose of study medication (either FF/VI or usual ICS/LABA) and considered as-treated.</li> <li>Subjects will be assigned to the treatment group as treated for the Safety population</li> </ul> | Safety |

# NOTES:

 Please refer to Appendix 15: List of Data Displays which details the population to be used for each displays being generated.

HZA116492

# 3.1. Protocol Deviations

All PDs (any deviation from the protocol) are tracked and monitored during the study. Important PDs are those deviations that may compromise subject rights, safety, or well-being, and/or data integrity, and/or study end-points, and are defined in the protocol deviation management plan (PDMP). Apart from any incorrect treatment deviations, all full and partial protocol deviations will be agreed upon prior the unblinding and the freezing of the database. All deviations from the inclusion/exclusion criteria, and important PDs will be summarised. A listing of treatment misallocations will be produced.

HZA116492

# 4. CONSIDERATIONS FOR DATA ANALYSES AND DATA HANDLING CONVENTIONS

Table 3 provides an overview of appendices within the RAP for outlining general considerations for data analyses and data handling conventions.

# Table 3 Overview of Appendices

| Section | Component |
|---|---|
| 10.1 | Appendix 1: Protocol Deviation Management and Definitions for PP Population |
| 10.2 | Appendix 2: Time & Events |
| 10.3 | Appendix 3: Assessment Windows |
| 10.4 | Appendix 4: Treatment States and Phases |
| 10.5 | Appendix 5: Data Display Standards & Handling Conventions |
| 10.6 | Appendix 6: Derived and Transformed Data |
| 10.7 | Appendix 7: Premature Withdrawals & Handling of Missing Data |
| 10.8 | Appendix 8: Values of Potential Clinical Importance |
| 10.9 | Appendix 9: Multicenter Studies |
| 10.10 | Appendix 10: Examination of Covariates, Subgroups & Other Strata |
| 10.11 | Appendix 11: Multiple Comparisons & Multiplicity |
| 10.12 | Appendix 12: Model Checking and Diagnostics for Statistical Analyses |
| 10.13 | Appendix 13: Blinding Strategy |
| 10.14 | Appendix 14: Abbreviations & Trade Marks |
| 10.15 | Appendix 15: List of Data Displays |
| 10.16 | Appendix 16: Example Mock Shells for Data Displays |

HZA116492

# 5. STUDY POPULATION ANALYSES

# 5.1. Overview of Planned Analyses

The study population analyses will be based on the ITT population, unless otherwise specified.

Table 4 provides an overview of the planned study population analyses, with full details of data displays being presented in Appendix 15: List of Data Displays.

Table 4 Overview of Planned Study Population Analyses

| Display Type | Data Displays Generated | | |
|---|---|---|---|
| | Table | Figure | Listing |
| Subject Disposition | | | |
| Subject Populations | <b>Y</b> [1] | | Υ |
| Inclusion/exclusion Criteria Failures for Subjects Not | <b>Y</b> [1] | | |
| Starting Treatment | I, i, i | | |
| End of Study Record | <b>Y</b> [2] | | Υ |
| Attendance at Each Clinic Visit and Phone Call Visit | Υ | | |
| Number of Subjects by Country and Centre | <b>Y</b> [2,3] | | |
| Randomised and Actual Treatments | | | Υ |
| Protocol Deviations | | | |
| Deviations from the Inclusion/Exclusion Criteria | Υ | | Υ |
| Important Protocol Deviations | Υ | | Υ |
| Important Protocol Deviations Resulting in Exclusion from | Υ | | Υ |
| the PP Population | Ī | | ľ |
| Treatment Misallocations | | | Υ |
| Demographic and Baseline Characteristics | | | |
| Demographic Characteristics | Y <sup>[2,4]</sup> | | Υ |
| Race and Racial Combinations | Υ | | Υ |
| Race and Racial Combinations Details | Υ | | |
| Current and Past Medical Conditions | Y | | |
| Asthma Duration at Baseline | <b>Y</b> [2] | | Υ |
| Asthma Exacerbation History at Baseline | <b>Y</b> [2] | | Υ |
| Lung Function at Baseline | Y | | |
| Smoking History at Baseline | <b>Y</b> [2] | | Υ |
| Concomitant Medications | | | |
| Pre-Treatment Concomitant Medications | Y | | Υ |
| On-Treatment Concomitant Medications | Y | | Y |
| On-Treatment Asthma Concomitant Medications | Y | | |
| Relationship between Ingredient and Verbatim Text | | | Υ |
| Exposure and Medication Modifications | | | |
| Study Medication Dosage Modification | Y | | |
| Extent of Exposure to Study Medication (Regardless of | Υ | Υ | Y |
| Modification to Study Medication Dosage) | ſ | Ť | Ť |
| Extent of Exposure to Study Medication (up to First | Υ | | |
| Modification of Study Medication Dosage) | ī | | |
| Extent of Exposure to Study Medication by Medication and | Υ | | |
| Dosage | | | |
| Number of Subjects by Subgroup | Υ | | |

H7A116492

#### NOTES:

- Y = Yes display generated.
- [1]: Display will be based on ASE population
- [2]: Display will be repeated for the PP population
- [3]: Display will be repeated for the ASE population
- [4]: Display will be repeated for the Safety population

# 6. PRIMARY STATISTICAL ANALYSES

# 6.1. Efficacy Analyses

# 6.1.1. Overview of Planned Efficacy Analyses

The primary efficacy analyses will be based on the ITT population and repeated for the PP population, unless otherwise specified.

Table 5 provides an overview of the planned efficacy analyses, with full details of data displays being presented in: List of Data Displays.

Table 5 Overview of Planned Efficacy Analyses

| Endpoint | Data displays generated | | | | | | |
|---|---|---|---|---|---|---|---|
| - | Stats Analysis | | | Summary | | Individual | |
| | T | F | L | T | F | F | L |
| ACT Total Score | | | | | | | |
| Change from Baseline | Y[1,2,3,4,5,6, | | | Y[1,2,3,4,5,7] | <b>Y</b> [1] | | Y[8] |
| in the ACT Total Score<br>at Week 12 (Visit 4) | 7] | | | | | | |

#### NOTES:

- T = Table, F = Figure, L = Listing, Y = Yes display generated.
- Stats Analysis = Represents TFL related to any formal statistical analyses (i.e. modelling) conducted.
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.
- Display will be repeated for the following subgroups (ITT only) (see Section 10.10 for more details):
  - [1]: Country
  - [2]: Number of severe asthma exacerbations in the previous year prior to randomisation
  - [3]: Smoking status at baseline
  - [4]: Age group
  - [5]: Gender
- [6]: Sensitivity analyses will be produced for the following approaches:
  - Last observation carried forward (LOCF) (ITT only)
  - MI analyses utilizing covariates (ITT only)
  - Semi-parametric Hodges-Lehmann (HL) approach (ITT only)
  - Worst observation carried forward (WOCF) for treatment withdrawals (ITT only)
  - · Adjusting for seasonal effect
- [7]: Display will be repeated for:
  - FF/VI versus the subset of Usual ICS/LABA subjects prescribed FP/S at randomisation (only if ≥25% of Usual ICS/LABA patients are prescribed FP/S at randomisation)
  - FF/VI versus the subset of Usual ICS/LABA subjects prescribed BUD/F at randomisation (only if ≥25% of Usual ICS/LABA patients are prescribed BUD/F at randomisation)
- [8]: Display will be produced for the ITT population only.

HZA116492

# 6.1.2. Planned Efficacy Statistical Analyses

## **Primary Statistical Analyses**

#### Endpoint(s)

Change from Baseline in the ACT Total Score at Week 12 (Visit 4)

#### **Model Specification**

- The primary endpoint will be performed on both the ITT and the PP populations, and analysed using an MMRM model utilizing the REML estimation approach and a default covariance structure of unstructured
- Terms fitted in the model will include:

Response : Change from Baseline in ACT Total Score

Fixed Categorical : Randomised treatment, visit (Week 6 and Week 12), gender, country

Fixed Continuous : Baseline ACT total score, age

Interaction terms : Randomised treatment-by-visit, baseline ACT total score-by-visit

Random effect : Subject

# SAS Code to Perform Analysis

```
proc mixed data=input data;
```

class trtcd gender country visit subjid;

model ACT = trtcd gender country age baseline

visit visit\*baseline visit\*trtcd / ddfm=kr;

repeated visit / subject=subjid type=un;

random intercept / subject=subjid;

Ismeans visit\*trtcd / cl diff e om=OMdset at (baseline age)=(&blm. &agem.);

run;

where OMdset is a dataset with a row for every visit-subject combination that contains all of the covariates and blm and agem are macro variables containing the means for baseline and age for the subjects used in the analysis. These are used to derive the adjusted means using coefficients which are based on the subjects used in the analysis.

#### **Model Checking & Diagnostics**

Refer to Appendix 12: Model Checking and Diagnostics for Statistical Analyses.

#### **Model Results Presentation**

- For Week 12 (Visit 4), the adjusted (least squares [LS]) mean change from baseline for each treatment and the estimated treatment difference for FF/VI versus Usual ICS/LABA (i.e. the difference in LS mean change from baseline) will be presented together with the associated 95% CI and p-value.
- Summary statistics will be produced for absolute value of and change from baseline in ACT total score
  at each post-baseline visit (Week 6 [Visit 3], Week 12 [Visit 4], Week 18 [Visit 5] and Week 24 [Visit 6]).
- A listing of ACT total and change from baseline scores will be provided.
- Mean ACT total score ± SD will be plotted by visit.

#### **Subgroup Analyses**

- For the analyses by country (France, Germany) and gender (male, female), the model will additionally
  include the randomised treatment-by-subgroup and randomised treatment-by-subgroup-by-visit
  interactions as a covariate.
- For the analyses by number of severe asthma exacerbations in the previous year prior to randomisation (0, >1) and smoking status at baseline (non-smoker, former smoker, current smoker), the model will additionally include the subgroup, randomised treatment-by-subgroup interaction and randomised treatment-by-subgroup-by-visit interaction as covariates.
- For the analysis by age group (<50 years, ≥50 years), the continuous covariate age will be replaced by age group, randomised treatment-by-age group interaction and randomised treatment-by-age group-byvisit interaction.

HZA116492

#### **Sensitivity and Supportive Statistical Analyses**

# **Justification for Sensitivity Analyses Handling Missing Data**

• While subjects missing Week 12 (Visit 4) data but having earlier data will be included in the MMRM primary analysis, the interpretability of the results from the primary model will depend on the missing data satisfying the Missing at Random (MAR) assumption. To support the validity of the conclusions drawn from this analysis, several sensitivity analyses will be performed to explore the dropout pattern and its possible impact on treatment comparisons. These sensitivity analyses will be performed on the ITT population only as subjects with missing ACT total score at Week 12 (Visit 4) are excluded from the PP population.

#### **Last Observation Carried Forward**

• Missing values at Week 12 (Visit 4) will be replaced by the last available post-randomization value (either the Week 6 (Visit 2) ACT score or the ACT score at treatment withdrawal time, if applicable), i.e. based on the LOCF method. The change from baseline in ACT at Week 12 (Visit 4) will be analyzed using an analysis of covariance (ANCOVA) model adjusting for randomised treatment, baseline ACT score, gender, country and age. For Week 12 (Visit 4), the LS mean change from baseline for each treatment and estimated LS mean change from baseline difference for FF/VI versus Usual ICS/LABA will be presented together with the associated 95% CI and p-value.

## **Multiple Imputation**

- Sensitivity analyses will be performed using MI methods based on pattern mixture models. First, a
  repeated measures Normal model will be fitted to the data using a Bayesian approach, with noninformative priors for the mean and variance-covariance matrix to provide a joint posterior for the
  parameters in this model. The repeated measures Normal model will include separate mean profiles for
  each treatment group and the same covariates as those in the primary efficacy analysis.
- Independent samples will then be drawn from the posterior distributions for the mean and variance-covariance matrix to provide inputs into an imputation model. For each subject with missing data, these sampled values of the parameters for mean vectors and the variance-covariance matrices specify a joint distribution for their observed and unobserved outcome data.
- The post-withdrawal part of each pattern-specific distribution will be modelled using the approach discussed below. This imputation model will have the same covariates as those in the primary efficacy analysis.
- Based on this imputation model, a single set of data will be sampled for the missing data based on the
  distribution for the subject's missing data conditional upon their observed data. Each imputed data set
  will then be analysed using simple ANCOVA at Week 12 (Visit 4) and the resulting treatment
  differences and their standard errors combined using Rubin's rules.
- The post-withdrawal part of each pattern-specific distribution will be modelled using these two approaches:
  - MAR Approach. The means and variance-covariances following withdrawal are chosen to reflect the subject's own treatment group. This approach will provide similar results to using a mixed effects model where the unstructured covariance matrix is estimated separately for each arm, and all covariates are crossed with treatment. As such it is not truly a sensitivity analysis as we expect to get very similar results. Like the MMRM this answers an on-treatment question.
  - Copy Differences from Reference Approach. This approach addresses a potential pattern of informative missingness, in which subjects withdrawn from the test groups would have followed the same trend over time (difference in mean value between time-points) as those in the reference group, had they continued in the study. Therefore, this approach may be considered conservative because it will assume that following withdrawal from a test treatment arm, imputation for their missingness will be derived from observed reference data. The intention is to represent an ITT-like approach.
- For each method, the LS mean change from baseline at Week 12 (Visit 4) for each treatment and

HZA116492

## Sensitivity and Supportive Statistical Analyses

estimated LS mean change from baseline difference for FF/VI versus Usual ICS/LABA will be presented together with the associated 95% CI and p-value.

# Hodges-Lehmann Approach

A sensitivity analysis based on the semi parametric HL approach will be proposed to assess the
robustness of the MMRM Model-based non-inferiority results. The HL difference between groups at
Week 12 (Visit 4) and corresponding 95% CI will be provided.

#### **Worst Observation Carried Forward**

• When treatment withdrawal occurs, an alternative method for imputing the missing value at the nearest visit after withdrawal time will be proposed: the primary endpoint missing value will be estimated by the worst ACT score observed between baseline visit and withdrawal time, inclusive – i.e. using the WOCF method. An ANCOVA model adjusting for randomised treatment, baseline ACT score, gender, country and age will be used to analyse this imputed data, with the LS mean change from baseline for each treatment presented at Week 12 (Visit 4) together with the estimated LS mean change from baseline difference and associated 95% CI and p-value

#### **Summary of Sensitivity Statistical Analyses**

 A plot will be produced displaying the treatment differences and 95% CIs for the primary analysis and each of the sensitivity analyses described above.

#### Seasonal effect

A sensitivity analysis adjusting for seasonal effect will be performed by repeating the primary efficacy
analysis with the addition of season at randomisation, randomised treatment-by-season at
randomisation interaction and randomised treatment-by-season at randomisation-by-visit interaction.
 See Section 10.10.3 for the definition of season at randomisation. The LS mean change from baseline
at Week 12 (Visit 4) for each treatment and estimated LS mean change from baseline difference will be
displayed for each season at randomisation together with the associated 95% CI and p-value, and the
interaction p-value.

HZA116492

# 7. SECONDARY STATISTICAL ANALYSES

# 7.1. Efficacy Analyses

# 7.1.1. Overview of Planned Efficacy Analyses

The secondary efficacy analyses will be based on the ITT population, unless specified otherwise.

Table 6 provides an overview of the planned efficacy analyses, with further details of data displays being presented in Appendix 15: List of Data Displays.

Table 6 Overview of Planned Efficacy Analyses

| Endpoint | Data displays generated | | | | | | |
|---|---|---|---|---|---|---|---|
| | St | ats Analysi | | Summary | | Individual | |
| | T | F | L | T | F | F | L |
| ACT Total Score | | | | | | | |
| Change from Baseline | Y[1,2,3,4] | Υ | | Y[1,2,4,5,6,7, | Y[1,2] | | |
| in the ACT Total Score | | | | 8] | | | |
| at Week 24 (Visit 4) | | | | | | | |
| Correct Use of Device | | | | | | | |
| Percentage of Subjects | <b>Y</b> [1] | | | <b>Y</b> [1] | | | Υ |
| with Correct Use of | | | | | | | |
| Inhaler Device at Week | | | | | | | |
| 12 (Visit 4) and at | | | | | | | |
| Week 24 (Visit 6) | | | | | | | |
| Independently of the | | | | | | | |
| Use at Week 12 (Visit | | | | | | | |
| 4) | | | | | | | |

#### NOTES:

- T = Table, F = Figure, L = Listing, Y = Yes display generated.
- Stats Analysis = Represents TFL related to any formal statistical analyses (i.e. modelling) conducted.
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.
- [1]: Display will be repeated for the PP population
- [2]: Display will be repeated by Country (ITT only)
- [3]: Sensitivity analyses will be produced for the following approaches:
  - LOCF (ITT only)
  - MI analyses utilizing covariates (ITT only)
  - Semi-parametric HL approach (ITT only)
  - WOCF for treatment withdrawals (ITT only)
  - Adjusting for seasonal effect
- [4]: Display will be repeated for:
  - FF/VI versus the subset of Usual ICS/LABA subjects prescribed FP/S at randomisation (only if ≥25% of Usual ICS/LABA patients are prescribed FP/S at randomisation)
  - FF/VI versus the subset of Usual ICS/LABA subjects prescribed BUD/F at randomisation (only if ≥25% of Usual ICS/LABA patients are prescribed BUD/F at randomisation)
- Display will be repeated for the following subgroups (ITT only) (see Section 10.10 for more details):
  - [5]: Number of severe asthma exacerbations in the previous year prior to randomisation
  - [6]: Smoking status at baseline
  - [7]: Age group
  - [8]: Gender

HZA116492

# 7.1.2. Planned Efficacy Statistical Analyses

## **Secondary Statistical Analyses**

## Endpoint(s)

• Change from Baseline in the ACT Total Score at Week 24 (Visit 6)

#### **Model Specification**

- This endpoint will be performed on both the ITT and the PP populations, and analysed using an MMRM model utilizing the REML estimation approach and a default variance-covariance structure of unstructured
- Terms fitted in the model will include:

Response : Change from Baseline in ACT Total Score

Fixed Categorical : Randomised treatment, visit (Week 6, Week 12, Week 18 and Week 24),

gender, country

Fixed Continuous : Baseline ACT total score, age

Interaction terms : Randomised treatment-by-visit, baseline ACT total score-by-visit

Random effect : Subject

# **Model Checking & Diagnostics**

Refer to Appendix 12: Model Checking and Diagnostics for Statistical Analyses.

#### **Model Results Presentation**

- For Week 24 (Visit 6), the LS mean change from baseline for each treatment and the estimated difference in LS mean change from baseline for FF/VI versus Usual ICS/LABA will be presented together with the associated 95% CI and p-value.
- Summary statistics, a listing and plots of mean ACT total score  $\pm$  SD will be produced as part of the primary efficacy endpoint analysis (see Section 6.1.2).

#### **Subgroup Analysis**

 For the analysis by country (France, Germany), the model will additionally include the randomised treatment-by-country and randomised treatment-by-country-by-visit interactions as a covariate.

#### **Sensitivity and Supportive Statistical Analyses**

 The same sensitivity analyses as those described for the primary endpoint will be performed for the key secondary endpoint of change from baseline in the ACT total score at Week 24 (Visit 6).

# **Secondary Statistical Analyses**

## Endpoint(s)

Percentage of subjects with correct use of inhaler device at Week 12 (Visit 4) and at Week 24 (Visit 6) independently of the use at Week 12 (Visit 4)

#### **Model Specification**

- These endpoints will be analysed for both the ITT and the PP populations using logistic regression models
- Terms fitted in the model will include:

Response : Endpoint

Fixed Categorical : Randomised treatment, correct use of inhaler device at baseline, gender,

country

Fixed Continuous : Age

# SAS Code to Perform Analysis

proc logistic data=input data plots=(all);

class trtcd country baseline gender / ref=first param=ref;

model corr\_use (event="Y") = trtcd baseline age gender country;

contrast "Trt\_effect" trtcd 1 / estimate=exp;

run;

HZA116492

# **Secondary Statistical Analyses**

# **Model Checking & Diagnostics**

• Refer to Appendix 12: Model Checking and Diagnostics for Statistical Analyses.

# Model Results Presentation

- The number and percentage of subjects with correct use within each randomised treatment group will be presented by visit, together with the adjusted odds ratio comparing FF/VI with Usual ICS/LABA, associated p-value and 95% CI.
- A summary and listing of correct use / errors of inhaler use will be produced.

HZA116492

# 7.2. Safety Analyses

# 7.2.1. Overview of Planned Analyses

The safety analyses will be based on the Safety population.

Table 7 provides an overview of the planned analyses, with further details of data displays being presented in Appendix 15: List of Data Displays.

Table 7 Overview of Planned Safety Analyses

| Endpoint | | D | Data displays generated | | | |
|---|---|---|---|---|---|---|
| | Stats A | Stats Analysis | | mary | Indiv | idual |
| | Т | F | Τ | F | F | L |
| Adverse Events | | | | | | |
| SAEs and ADRs Overview | | | Υ | | | |
| Non-Serious ADRs | | | Υ | | | Υ |
| Serious ADRs | | | Υ | | | |
| All ADRs | | | Υ | | | |
| SAEs | | | Υ | | | Υ |
| SAEs and ADRs Leading to Permanent | | | Υ | | | Υ |
| Discontinuation of Study Medication or | | | | | | |
| Withdrawal from Study | | | | | | |
| SAEs Leading to Permanent | | | Υ | | | |
| Discontinuation of Study Medication or | | | | | | |
| Withdrawal from Study | | | | | | |
| ADRs Leading to Permanent | | | Υ | | | |
| Discontinuation of Study Medication or | | | | | | |
| Withdrawal from Study | | | | | | |
| Non-Serious ADRs Leading to | | | | | | Υ |
| Permanent Discontinuation of Study | | | | | | |
| Medication or Withdrawal from Study | | | | | | |
| Most Frequent Non-Serious ADRs, | | | Υ | | | |
| Reported by ≥1% or More of Subjects in | | | | | | |
| Any Treatment Group | | | | | | |
| Non-Serious ADRs of Special Interest | | | Υ | | | |
| Serious ADRs of Special Interest | | | Υ | | | |
| All ADRs of Special Interest | | | Υ | | | |
| SAEs of Special Interest | | | Υ | | | |
| Fatal SAEs | | | Υ | | | Υ |
| Fatal Serious ADRs | | | Υ | | | |
| Fatal SAEs of Special Interest | | | Υ | | | |
| Non-Fatal SAEs | | | Υ | | | Υ |
| Non-Fatal SAEs of Special Interest | | | Υ | | | |
| AE terms of Special Interest | | | | | | Υ |
| Top Ten Most Commonly Reported On- | | | Υ | | | |
| treatment ADRs per Treatment Group | | | | | | |
| Vital Signs | | | | | | |
| Vital Signs | | | Υ | | | Υ |

HZA116492

| Endpoint | Data displays generated | | | | | |
|---|---|---|---|---|---|---|
| | Stats A | nalysis | Sum | mary | Individual | |
| | T | F | T | F | F | L |
| Inhaler Device Malfunctions | | | | | | |
| Inhaler Device Malfunctions | | | | | | Υ |
| Liver chemistry | | | | | | |
| Liver event | | | | | | Υ |
| Liver biopsy | | | | | | Υ |
| Liver imaging | | | | | | Υ |
| Other | | | | | | |
| Pregnancy | | | | | | Y |

#### NOTES:

- T = Table, F = Figure, L = Listing, Y = Yes display generated.
- Stats Analysis = Represents TFL related to any formal statistical analyses (i.e. modelling) conducted.
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.

# 7.2.2. Benefit:Risk analyses

Benefit:Risk analyses will be based on the ITT population for Benefit, and Safety population for Risk.

Table 8 provides an overview of the planned analyses, with further details of data displays being presented in Appendix 15: List of Data Displays.

Table 8 Overview of Planned Benefit:Risk Analyses

| Endpoint | Data displays generated | | | | |
|---|---|---|---|---|---|
| | Stats Analysis | | Summary | | Individual |
| | T | F | Т | F | L |
| Summary of Benefit:Risk | | Υ | | | |

#### NOTES:

- T = Table, F = Figure, L = Listing, Y = Yes display generated.
- Stats Analysis = Represents TFL related to any formal statistical analyses (i.e. modelling) conducted.
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.

# **Benefit Risk Statistical Safety Analyses**

## Endpoint(s)

 Summary of Benefit:Risk: various endpoints analyses in the context of safety and effectiveness analyses

#### **Model Specification**

- Estimates and their 95% CIs obtained from selected safety and effectiveness analyses will be
  presented for the ITT population on a multiple panel forest plot which will display effectiveness and
  safety data.
- For certain endpoints, the x-axis may be reversed to ensure benefit/risk to either FF/VI or Usual ICS/LABA is shown accurately.
- Due to endpoints being presented using different scales, the forest plot will be split into additional
  panels to allow better visibility of the results.

HZA116492

## **Benefit Risk Statistical Safety Analyses**

# **Model Checking & Diagnostics**

Model checking and diagnostics are described in each endpoint analysis section.

# **Model Results Presentation**

- The top panel ("Benefits") of the forest plot will display:
  - difference in LS mean change from baseline from the MMRM analysis of the primary efficacy endpoint, defined as the change from baseline in ACT total score at Week 12 (Visit 4), as described in Section 6.1.2
  - difference in LS mean change from baseline from the MMRM analysis of the change from baseline in ACT total score at Week 24 (Visit 6), as described in Section 7.1.2
  - adjusted odds ratio from the logistic regression analysis of percentage of subjects with correct use of inhaler device at Week 12 (Visit 4), as described in Section 7.1.2
  - adjusted odds ratio from the logistic regression analysis of percentage of subjects with correct use of inhaler device at Week 24 (Visit 6) independently of the use at Week 12 (Visit 4), as described in Section 7.1.2
- The bottom panel ("Risks") of the forest plot will display the risk difference for FF/VI vs. usual ICS/LABA
  of the incidence of the following SAEs of special interest:
  - Asthma/bronchospasm, cardiovascular effects, decreased bone mineral density and associated fractures, hypersensitivity, local steroid effects, lower respiratory tract infection (LRTI) excluding pneumonia, pneumonia, adrenal suppression, ocular effects, effects on glucose, effects on potassium, tremor

HZA116492

# 8. OTHER STATISTICAL ANALYSES

# 8.1. Other Analyses

# 8.1.1. Overview of Planned Other Analyses

The other statistical analyses will be based on the ITT population, unless otherwise specified.

Table 9 provides an overview of the planned other analyses, with full details of data displays being presented in Appendix 15: List of Data Displays.

Table 9 Overview of Planned Other Analyses

| Endpoint | Absolute | | | | | | |
|---|---|---|---|---|---|---|---|
| | Stats Analysis | | | Sum | mary | | ridual |
| | T | F | L | T | F | F | L |
| Trough (Pre-dose) FEV | | | | | | | |
| Change from Baseline<br>in Trough (Pre-dose)<br>FEV1 at Week 12<br>(Visit 4) | Y | | | Y | | | Y |
| ACT | | | | | | | |
| ACT Total Score ≥ 20<br>or ≥ 3 Point Increase<br>from Baseline in ACT<br>Total Score at Week<br>12 (Visit 4) and Week<br>24 (Visit 6) | Y | | | Y | Y | | |
| ACT Total Score ≥ 20<br>at Week 12 (Visit 4)<br>and Week 24 (Visit 6) | | | | Y | Y | | |
| ≥ 3 Point Increase<br>from Baseline in ACT<br>Total Score at Week<br>12 (Visit 4) and Week<br>24 (Visit 6) | | | | Y | Y | | |
| Change from Baseline<br>in Individual ACT<br>Questions at Week 12<br>(Visit 4) and Week 24<br>(Visit 6) | | | | Y | | | |
| Compliance with Study | / Medication | | | | | | |
| Compliance with Study Medication from Randomisation (Day 0) to Week 12 (Visit 4), from Week 12 (Visit 4) to Week 24 (Visit 6) and from Randomisation (Day 0) to Week 24 (Visit 6) | | | | <b>Y</b> [1] | Y | | Y |

HZA116492

| Endpoint | Absolute | | | | | | |
|---|---|---|---|---|---|---|---|
| | S | tats Analysis | | | mary | Indiv | idual |
| | T | F | L | T | F | F | |
| MARS-A Score at | | | _ | Y[2] | Y[2] | | Y |
| Randomisation (Day | | | | • | | | |
| 0), Week 12 (Visit 4) | | | | | | | |
| and Week 24 (Visit 6). | | | | | | | |
| Severe asthma exacerb | nations | l. | | | | | |
| Number of Subjects | ations | I | | <b>Y</b> [3] | | I | Y |
| With at Least 1 Severe | | | | 1 | | | ' |
| Asthma Exacerbation | | | | | | | |
| and Number of Severe | | | | | | | |
| Asthma Exacerbations | | | | | | | |
| Annual Severe Asthma | Υ | Y | | | | | |
| | ĭ | Ť | | | | | |
| Exacerbation Rate | | | | | | | |
| over the Study Period | | | | | | - | |
| Time to First Severe | Υ | Y | | | | | |
| Asthma Exacerbation | | | | | | | |
| Asthma Quality of Life | Questionna | ire (AQLQ[S | []) | | ı . | 1 | |
| Change from Baseline | | | | Υ | | | Υ |
| in Total Score and | | | | | | | |
| Domain Scores of | | | | | | | |
| AQLQ(S) at Week 24 | | | | | | | |
| (Visit 6) | | | | | | | |
| An Increase from | Υ | | | Υ | | | |
| Baseline of ≥ 0.5 in | | | | | | | |
| AQLQ(s) Total Score | | | | | | | |
| at Week 24 (Visit 6) | | | | | | | |
| An Increase from | Υ | | | Υ | | | |
| Baseline of ≥ 0.5 in | | | | | | | |
| AQLQ(s) | | | | | | | |
| Environmental Stimuli | | | | | | | |
| Domain Score at Week | | | | | | | |
| 24 (Visit 6) | | | | | | | |
| An Increase from | | | | Υ | | | |
| Baseline of ≥ 0.5 in | | | | | | | |
| AQLQ(S) Individual | | | | | | | |
| Domain Scores | | | | | | | |
| (Symptoms, Activity | | | | | | | |
| limitations and | | | | | | | |
| Emotional Function) at | | | | | | | |
| Week 24 (Visit 6) | | | | | | | |
| EQ-5D-5L | | | | | | | |
| EQ-5D-5L Descriptive | Υ | | | Υ | | | Υ |
| System Dimensions at | | | | | | | |
| Week 24 (Visit 6) | | | | | | | |
| EQ-5D-5L Utility Score | Υ | | | Υ | | | Υ |
| at Week 24 (Visit 6) | | | | | | | |
| EQ-5D-5L Visual | Υ | | | Υ | | | Υ |
| Analogue Scale (VAS) | • | | | | | | |
| Score at Week 24 | | | | | | | |
| (Visit 6) | | | | | | | |
| ( viole o) | | I | | I | I | ı | L |

HZA116492

| Endpoint | Absolute | | | | | | |
|-------------------|----------------|---|---|---------|---|------------|---|
| | Stats Analysis | | | Summary | | Individual | |
| | T | F | L | T | F | F | L |
| PASAP-Q | | | | | | | |
| PASAP-Q Scores at | | | | Υ | | | Υ |
| Week 12 (Visit 4) | | | | | | | |

#### NOTES:

- T = Table, F = Figure, L = Listing, Y = Yes display generated.
- Stats Analysis = Represents TFL related to any formal statistical analyses (i.e. modelling) conducted.
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.
- [1]: Display will be repeated for the PP population
- [2]: A reminder was sent to centres in France instructing that the MARS-A questionnaire refers to the patient's
  preventer inhaler (i.e. their maintenance therapy prior to entering the study, and study medication while on-study).
   See Section 10.6.3 for further details. Display will be repeated split by:
  - Patients in France who had completed all MARS-A assessments prior to the reminder being implemented
  - Patients in France who had completed at least one MARS-A assessment prior to the reminder being
    implemented but also completed at least one MARS-A assessment after the reminder being implemented
  - Patients in France who had not completed any MARS-A assessments prior to the reminder being implemented
  - Patients in Germany
- [3]: Display will be repeated by season.

# 8.1.2. Planned Other Statistical Analyses

| Other Statistical Analyses |
|----------------------------|

# Endpoint(s)

- Change from baseline in trough (pre-dose) FEV1 at Week 12 (Visit 4)
- Change from baseline in EQ-5D-5L Utility Score at Week 24 (Visit 6)
- Change from baseline in EQ-5D-5L VAS Score at Week 24 (Visit 6)

#### **Model Specification**

- These endpoints will be analysed for the ITT population using ANCOVA models
- Terms fitted in the model will include:

Response : Endpoint

Fixed Categorical : Randomised treatment, gender, country

Fixed Continuous FEV1 endpoint: Baseline trough (pre-dose) FEV1 and age

EQ-5D-5L Utility Score endpoint: Baseline EQ-5D-5L Utility Score

and age

EQ-5D-5L VAS Score endpoint: Baseline EQ-5D-5L VAS Score

and age

#### **Model Checking & Diagnostics**

Refer to Appendix 12: Model Checking and Diagnostics for Statistical Analyses.

# SAS Code to Perform Analysis

proc mixed data=input\_data;

class trtcd gender country;

model FEV1 = trtcd gender country age baseline / ddfm=kr;

Ismeans trtcd / cl diff e;

run;

#### **Model Results Presentation**

 The LS mean change from baseline for each treatment and the difference in estimated LS mean change from baseline for FF/VI versus Usual ICS/LABA will be presented together with the associated 95% CI and p-value.

HZA116492

#### **Other Statistical Analyses**

- Summary statistics.
- Listings will be provided.

## **Other Statistical Analyses**

#### Endpoint(s)

- Percentage of subjects who had either an ACT total score ≥ 20 or ≥ 3 point increase from baseline in ACT total score at Week 12 (Visit 4) and Week 24 (Visit 6)
- Percentage of subjects who have an increase from baseline of ≥ 0.5 in AQLQ(S) total score at Week 24 (Visit 6)
- Percentage of subjects who have an increase from baseline of ≥ 0.5 in AQLQ(S) environmental stimuli domain score at Week 24 (Visit 6)
- Percentage of subjects with 'no problems' in each dimension of the EQ-5D-5L questionnaire at Week 24 (Visit 6)

#### **Model Specification**

• These endpoints will be analysed for the ITT population using logistic regression models

Terms fitted in the model will include:

Response : Endpoint

Fixed Categorical : Randomised treatment, gender, country

Fixed Continuous ACT endpoints: Baseline ACT total score, baseline ACT total

score squared and age

AQLQ(S) endpoints: Baseline AQLQ(S) score and age

EQ-5D-5L endpoints: Baseline EQ-5D-5L dimension score and

age

# **Model Checking & Diagnostics**

• Refer to Appendix 12: Model Checking and Diagnostics for Statistical Analyses.

#### **Model Results Presentation**

- The number and percentage of subjects with a response within each randomised treatment group will be presented by visit, together with the adjusted odds ratio comparing FF/VI with Usual ICS/LABA, associated 95% CIs and p-values.
- The number and percentage of subjects with ACT total score ≥20 or ≥3 point increase from baseline in ACT total score will be summarized by visit to include the tabulations of frequencies together and separately.
- The number and percentage of subjects with an increase from baseline of ≥ 0.5 in AQLQ(S) total and
  individual domain scores at Week 24 (Visit 6) will be summarized.
- The responses to each EQ-5D-5L dimension will be descriptively summarised

#### **Other Statistical Analyses**

#### Endpoint(s)

Annual severe asthma exacerbation rate over the study period

## **Model Specification**

- This endpoint will be analysed for the ITT population using a generalised linear model (GLM), assuming the Negative Binomial distribution
- Terms fitted in the model will include:

Response : Annual severe asthma exacerbation rate over the study period Fixed Categorical : Randomised treatment, gender, country, number of severe

: Randomised treatment, gender, country, number of severe asthma exacerbations in the previous year prior to randomisation

(0, ≥1)

Fixed Continuous : Age

HZA116492

#### Other Statistical Analyses

Offset variable : Logarithm of time on treatment

#### **Model Checking & Diagnostics**

Refer to Appendix 12: Model Checking and Diagnostics for Statistical Analyses.

#### SAS Code to Perform Analysis

proc genmod data=input data;

class trtcd gender country;

model no exac = trtcd exacbl gender country age / dist=negbin link=log offset=log\_tm type3; Ismeans trtcd /cl diff=control("0") om exp;

run;

#### **Model Results Presentation**

- The LS mean number / annual rate, adjusted treatment ratio and associated 95% CI and p-value will be
- Percentage reduction in mean number / annual rate and associated 95% CI will also be presented.
- The severe asthma exacerbation data will be summarized to include the tabulations of exacerbation frequencies, exacerbation duration (days) and the outcome, the prescription of oral corticosteroids and/or antibiotics to treat exacerbations, hospitalisations and emergency department visits due to an exacerbation, intubations due to an exacerbation and withdrawal of IP or withdrawal from the study as a result of an exacerbation.
- A listing of severe exacerbations will be provided.
- Box plots will be provided for the severe annual exacerbation rates.

## **Other Statistical Analyses**

#### Endpoint(s)

Time to first severe asthma exacerbation

#### **Model Specification**

- The cumulative distribution of this endpoint will be illustrated for the ITT population using Kaplan-Meier estimates and evaluated using the Wald Chi-Square test based on a Cox proportional hazards model.
- The analyses and summaries will include on-treatment exacerbations, from start date of exposure to min(stop date of exposure + 1 day, date of study discontinuation).
- The exact method for handling ties in times will be used.
- Terms fitted in the model will include:

Response : Time to first severe asthma exacerbation Fixed Categorical : Randomised treatment, gender, country **Fixed Continuous** 

: Age

#### **Model Checking & Diagnostics**

Refer to Appendix 12: Model Checking and Diagnostics for Statistical Analyses.

#### **Model Results Presentation**

- The hazard ratio for FF/VI versus Usual ICS/LABA with associated 95% CI and p-value will be presented.
- Cumulative incidence curves of time to first severe asthma exacerbation will be presented.
- Summary statistics will also be presented.

HZA116492

# 9. REFERENCES

Devlin N., Shah K., Feng Y., Mulhern B., Van Hou, B. Valuing Health-Related Quality of Life: An EQ-5D-5L Value Set for England. Office of Health Economics. January 2016.

Efron, B. The Efficiency of Cox's Likelihood Function for Censored Data. J Am Stat Assoc. 1977;72:557–565.

EuroQol. EQ-5D-3L User Guide. EuroQol, Europe: 2013. Version 5.

Firth D. Bias Reduction of Maximum Likelihood Estimates. Biometrika. 1993;80:27–38.

GINA 2012, http://www.ginasthma.org/local/uploads/files/GINA Report March13.pdf

GlaxoSmithKline Document Number 2011N129785\_02 Study ID HZA115150. A 12-month, open label, randomised, effectiveness study to evaluate fluticasone furoate (FF, GW685698)/vilanterol (VI, GW642444) Inhalation Powder delivered once daily via a Novel Dry Powder Inhaler compared with usual maintenance therapy in subjects with Asthma. Report Date 11-Mar-2014.

GlaxoSmithKline Document number 2014N190259\_02. Study HZA116492: A 6-month, open label, randomised, efficacy study to evaluate fluticasone furoate (FF, GW685698)/vilanterol (VI, GW642444) Inhalation Powder delivered once daily via the Dry Powder Inhaler Ellipta<sup>TM</sup> compared with usual ICS/LABA maintenance therapy delivered by Dry Powder Inhaler in subjects with Persistent Asthma.

Juniper E.F., Guyatt G.H, Ferrie P.J., Griffith L.E. Measuring quality of life in asthma. Am Rev Respir Dis. 1993;147:832–838.

Kozma C.M., Slaton T.L., Monz B.U., Hodder R., Reese P.R. Development and Validation of a Patient Satisfaction and Preference Questionnaire for Inhalation Devices (PASAPQ). Treat Respir Med. 2005; 4 (1): 41-52.

Schatz M., Kosinski M., Yarlas A.S., Hanlon J., Watson M.E., Jhingran P. The minimally important difference of the Asthma Control Test. J Allergy Clin Immunol. 2009;124(4):719–23.

HZA116492

# 10. APPENDICES

| Section | Appendix |
|---|---|
| RAP Section 3 : Analysis Populations | |
| Section 10.1 | Appendix 1: Protocol Deviation Management and Definitions for PP Population |
| RAP Section 4: | General Considerations for Data Analyses & Data Handling Conventions |
| Section 10.2 | Appendix 2: Time & Events |
| Section 10.3 | Appendix 3: Assessment Windows |
| Section 10.4 | Appendix 4: Treatment States and Phases |
| Section 10.5 | Appendix 5: Data Display Standards & Handling Conventions |
| Section 10.6 | Appendix 6: Derived and Transformed Data |
| Section 10.7 | Appendix 7: Premature Withdrawals & Handling of Missing Data |
| Section 10.8 | Appendix 8: Values of Potential Clinical Importance |
| Section 10.9 | Appendix 9: Multicenter Studies |
| Section 10.10 | Appendix 10: Examination of Covariates, Subgroups & Other Strata |
| Section 10.11 | Appendix 11: Multiple Comparisons & Multiplicity |
| Section 10.12 | Appendix 12: Model Checking and Diagnostics for Statistical Analyses |
| Other RAP Appe | ndices |
| Section 10.13 | Appendix 13: Blinding Strategy |
| Section 10.14 | Appendix 14: Abbreviations & Trade Marks |
| Section 10.15 | Appendix 15: List of Data Displays |
| Section 10.16 | Appendix 16: Example Mock Shells for Data Displays |

HZA116492

# 10.1. Appendix 1: Protocol Deviation Management and Definitions for PP Population

#### 10.1.1. Protocol Deviations

All PDs (any deviation from the protocol) are tracked and monitored during the study. Important PDs are those deviations that may compromise subject rights, safety, or well-being, and/or data integrity, and/or study end-points, and are defined in the PDMP. Apart from any incorrect treatment deviations, all full and partial protocol deviations will be agreed upon prior the unblinding and the freezing of the database. All deviations from the inclusion/exclusion criteria, and important PDs will be summarised. A listing of treatment misallocations will be produced.

# 10.1.2. Exclusions from PP Population

**Important** PDs that will result in exclusion from the PP population are specified in Table 10, and will be summarised in a data display.

Table 10 PDs resulting in exclusion from the PP population

| <b>Deviation Category</b> | Deviation Subcategory |
|---|---|
| Informed consent | Signed informed consent/assent not available on site |
| | Wrong informed consent/assent version signed <sup>[1]</sup> |
| | Informed consent/assent not signed and/or dated by |
| | subject (parent/Legally Acceptable representative, if applicable) |
| | Informed consent/assent not signed and/or dated by appropriate site staff. [1] |
| | Informed consent/assent not signed prior to any study procedure <sup>[1]</sup> |
| | Other informed consent/assent deviations <sup>[1]</sup> |
| Eligibility criteria not met – | Informed consent |
| inclusion criteria | Gender and Age <sup>[2]</sup> |
| | Type of subject |
| | Current Asthma Therapy |
| | Inability of subject to complete questionnaires |
| Eligibility criteria not met – | History of Life-threatening asthma |
| exclusion criteria | Subjects having a severe and unstable asthma |
| | COPD Respiratory Disease |
| | Other diseases/abnormalities <sup>[1]</sup> |
| | Subjects with a history of adverse reaction to any |
| | intranasal, inhaled, or systemic corticosteroid and LABA |
| | therapy and to components of the inhalation powder <sup>[1]</sup> |
| | Investigational Medications used within 30 days or five |
| | half-lives of prior study <sup>[1]</sup> |
| | Chronic user of systemic corticosteroids |
| | Subjects treated by the monoclonal antibody omalizumab |
| | (Xolair) or mepolizumab (Nucala <sup>TM</sup> ) |
| | Subjects involved in other clinical trials <sup>[1]</sup> |
| Not withdrawn after developing | Not withdrawn from study <sup>[1]</sup> |

HZA116492

| <b>Deviation Category</b> | Deviation Subcategory |
|---|---|
| withdrawal criteria | Not discontinued from study treatment <sup>[1]</sup> |
| | Other deviation of not being withdrawn after developing |
| | withdrawal criteria <sup>[1]</sup> |
| Excluded medication, vaccine | • Medication, excluded by the protocol, was administered <sup>[3]</sup> |
| or device | Other excluded medication, vaccine or device deviation <sup>[3]</sup> |
| Visit completion | Missed visit/phone contact <sup>[4]</sup> |
| | Out of window visit/phone contact <sup>[4]</sup> |
| | Other visit window deviation <sup>[4]</sup> |
| Wrong study treatment / | Study treatment not administered per protocol <sup>[1]</sup> |
| administration / dose | Wrong study treatment or assignment administered |
| | Expired study treatment administered <sup>[1]</sup> |
| | Use of study treatment impacted by a temperature |
| | excursion which was not reported or approved or which was disapproved for further use. [1] |
| | Study treatment not available at site for administration <sup>[1]</sup> |
| | Other deviations related to wrong study |
| | treatment/administration/dose <sup>[1]</sup> |
| Study procedures | Non study treatment supply procedures <sup>[1]</sup> |
| | Equipment procedures <sup>[1]</sup> |
| | Other deviations from study procedures <sup>[1]</sup> |

<sup>[1]:</sup> To be reviewed on a case-by-case basis

<sup>[2]:</sup> Patients < 18 years will be excluded from PP population, others will be reviewed on a case-by-case basis

<sup>[3]:</sup> To be judged by the medical monitor

<sup>[4]:</sup> Missed or out of window Visit 4 will lead to exclusion from the PP population, missed or out of window other visits will not

HZA116492

# 10.2. Appendix 2: Time & Events

# 10.2.1. Protocol Defined Time & Events

| Study Visits | Visit 1*<br>Screening | Visit 2*<br>Randomisation | Visit 3<br>Phone<br>call 1 | Visit<br>4** | Visit 5<br>Phone<br>call 2 | Visit 6 | Early<br>Withdrawal |
|---|---|---|---|---|---|---|---|
| Study Week (± specified no. of days) | Day -7 to -<br>1 | Day 0 | Week<br>6 (±3<br>days) | Week<br>12<br>(±7<br>days) | Week<br>18 (±3<br>days) | Week<br>24<br>(±14<br>days) | Early<br>Withdrawal |
| Visit | Х | х | | Х | | Х | х |
| Phone interview | | | X | | X | | |
| Assessments | | | | | | | |
| Informed Consent | x | | | | | | |
| Eligibility criteria | X | X | | | | | |
| Demography | х | | | | | | |
| Smoking status | X | | | | | | |
| Medical/Family history of consented subjects including CV Risk factors and exacerbation history | х | | | | | | |
| PGx (saliva sample)*** | | X | | | | | |
| Physical examination | х | Х | | X | | X | X |
| Safety Assessments | | | | | | | |
| Urine Pregnancy Test¥ | | X | | Х | | X | X |
| Exacerbation<br>Assessment | | X | Х | Х | Х | Х | X |
| Vital signs | Х | Х | | X | | X | X |
| Serious Adverse Event<br>and Adverse Drug<br>Reaction Assessment <sup>1</sup> | | X | x | X | x | X | x |
| Efficacy Assessments | | | | | | | |
| Spirometry Testing (Predose trough FEV1) | | х | | х | | | X **** |
| Subject Questionnaires | | | | | | | |
| Asthma Control Test | X | X | X | X | X | X | х |
| EQ-5D | | X | | | | X | x |
| Asthma Quality of<br>Life Questionnaire | | X | | | | x | x |
| MARS-A questionnaire | | х | | Х | | X | х |
| Patient Satisfaction and Preference (PASAP-Q) | | | | х | | | X |
| Inhaler correct use assessment | | | | | | | |
| Type A/overall errors record | | X | | х | | х | |
| Medication | | | | | | | |

HZA116492

| Study Visits | Visit 1*<br>Screening | Visit 2*<br>Randomisation | Visit 3<br>Phone<br>call 1 | Visit<br>4** | Visit 5<br>Phone<br>call 2 | Visit 6 | Early<br>Withdrawal |
|---|---|---|---|---|---|---|---|
| Study Week (± specified no. of days) | Day -7 to -<br>1 | Day 0 | Week<br>6 (±3<br>days) | Week<br>12<br>(±7<br>days) | Week<br>18 (±3<br>days) | Week<br>24<br>(±14<br>days) | Early<br>Withdrawal |
| Visit | Х | х | | Х | | Х | х |
| Phone interview | | | х | | х | | |
| Assessments | | | | | | | |
| Concomitant Medication Assessment | X | x | | X | | х | х |
| Dispense Study<br>Medication <sup>2</sup> | | х | | x | | | |
| Collect Study<br>Medication <sup>2</sup> | | | | x | | х | х |
| RAMOS/eCRF | | | | | | | |
| RAMOS NG | | X | | X | | | |
| eCRF | x | X | х | X | X | х | x |

SAE and ADR monitoring will occur from Day 1. SAE related to study participation should begin from signing of informed consent form (ICF). An additional safety and ACT check is provided by phone at Week 6 and 18.

<sup>2.</sup> Throughout the study the study medication will be dispensed and collected by the investigator site.

<sup>\*</sup> Visit 1 and Visit 2 can be combined if the subject did not take his usual asthma medication before coming on site. Then this visit will be Day 0 and all baseline characteristics will be collected at this visit. Written Informed Consent must be obtained prior to initiation of study procedures or initiating changes in medications.

<sup>\*\*</sup> Visit 4 (Week 12) should be scheduled at the same time of day as Visit 2 (Randomisation visit).

<sup>\*\*\*</sup>PGx saliva sample collected at Visit 2 (Randomisation) or any scheduled clinic visit thereafter.

<sup>\*\*\*\*</sup> Only if early withdrawal occurs before Week 12.

<sup>¥</sup> Only for childbearing women.

HZA116492

# 10.3. Appendix 3: Assessment Windows

Clinic visits/phone calls are scheduled to take place as specified in the protocol. For the ACT and MARS-A questionnaires, measurements that are not within  $\pm 7$  days of the visit target day for Week 6 (Visit 3) and Week 18 (Visit 5), or  $\pm 14$  days for Week 12 (Visit 4) and Week 24 (Visit 6) will be excluded from the analyses. For EQ-5D-5L and AQLQ(S), measurements that are not within  $\pm 14$  days of the visit target day of Week 24 (Visit 6) will be excluded from the summaries. For PASAP-Q, measurements that are not within  $\pm 14$  days of the visit target day of Week 12 (Visit 4) will be excluded from the summaries.

Table 11 Visit slotting rules for ACT and MARS-A

| Days relative to randomisation * | Target Study Day | Visit Slot |
|--------------------------------------|------------------|-------------------|
| 35 – 49 | 42 | Week 6 (Visit 3) |
| 70 – 98 | 84 | Week 12 (Visit 4) |
| 119 – 133 | 126 | Week 18 (Visit 5) |
| 154 – 182 | 168 | Week 24 (Visit 6) |
| * Date of assessment – Randomisation | date + 1 | • |

Table 12 Visit slotting rules for EQ-5D-5L and AQLQ(S)

| Days relative to randomisation * | Target Study Day | Visit Slot |
|---|---|---|
| 154 – 182 | 168 | Week 24 (Visit 6) |
| * Date of assessment – Randomisation date + 1 | | |

Table 13 Visit slotting rules for PASAP-Q

| Days relative to randomisation * | Target Study Day | Visit Slot |
|---|---|---|
| 70 – 98 | 84 | Week 12 (Visit 4) |
| * Date of assessment – Randomisation da | te + 1 | |

For all other endpoints, individual measurements collected outside of the assessment window for scheduled visits will be included in the ITT and PP analyses without adjustment.

If multiple measurements are collected within the same assessment window, the last valid value prior to randomisation will be used as the baseline value and the value closest to the target day for that window will be used for all post-randomisation visits.

HZA116492

# 10.4. Appendix 4: Treatment States and Phases

# 10.4.1. Treatment Phases

In general, assessments and events will be classified according to the time of occurrence relative to study treatment, unless otherwise specified. Endpoint/measurement specific definitions are defined in Section 10.4.2.

| Treatment Phase | Definition |
|---|---|
| Pre-Treatment | Date < Study Treatment Start Date |
| On-Treatment | Study Treatment Start Date ≤ Date ≤ Study Treatment Stop Date + 1 |
| Post-Treatment | Date > Study Treatment Stop Date + 1 |

#### NOTES:

 If it is not possible to determine the treatment phase of an assessment or event it will be considered as On-Treatment.

#### 10.4.2. Treatment States

Assessments and events will be classified according to time of occurrence relative to the start and/or stop date of the study treatment. The earliest and latest exposure treatment start and stop dates will be used to determine whether an assessment or event was pre-treatment, on-treatment or post-treatment. If it is not possible to tell whether an assessment or event was on-treatment or not it will be considered as on-treatment.

#### 10.4.2.1. Treatment States for Concomitant Medications

| Treatment State | Definition |
|---|---|
| Pre-Treatment | (Start Date of Medication < Study Treatment Start Date) and (End Date of Medication < Study Treatment Start Date) |
| On-Treatment | [(Start Date of Medication < Study Treatment Start Date) and (End Date of Medication ≥ Study Treatment Start Date)] or (Study Treatment Start Date ≤ Start Date of Medication ≤ Study Treatment Stop Date + 1) |
| Post-Treatment | Start Date of Medication > Study Treatment Stop Date +1 |

HZA116492

# 10.4.2.2. Treatment States for Efficacy Measurements

| Treatment State | Definition |
|---|---|
| Pre-Treatment | Date of Measurement ≤ Study Treatment Start Date |
| On-Treatment | Study Treatment Start Date < Date of Measurement ≤ Study Treatment Stop Date + 1 |
| Post-Treatment | Date of Measurement > Study Treatment Stop Date +1 |

#### 10.4.2.3. Treatment States for Exacerbation Data

| Treatment State | Definition |
|---|---|
| Pre-Treatment | Exacerbation Onset Date < Study Treatment Start Date |
| On-Treatment | Study Treatment Start Date ≤ Exacerbation Onset Date ≤ Study Treatment Stop Date + 1 |
| Post-Treatment | Exacerbation Onset Date > Study Treatment Stop Date + 1 |

# NOTES:

- If the study treatment stop date is missing then the exacerbation will be considered to be On-Treatment
- See Section 10.6.3 for details on missing onset and/or resolution dates.

# 10.4.2.4. Treatment States for AE Data

Treatment states for adverse events are described below. Severe asthma exacerbations will be treated in the same way, with the exacerbation start date used in place of the AE start date.

| Treatment State | Definition |
|---|---|
| Pre-Treatment | AE Onset Date < Study Treatment Start Date |
| On-Treatment | Study Treatment Start Date ≤ AE Onset Date ≤ Study Treatment Stop Date + 1 |
| Post-Treatment | AE Onset Date > Study Treatment Stop Date + 1 |
| Onset Time<br>Since 1st Dose<br>(Days) | If Study Treatment Start Date > AE Onset Date = AE Onset Date - Study Treatment Start Date If Study Treatment Start Date ≤ AE Onset Date = AE Onset Date - Study Treatment Start Date +1 Missing otherwise. |
| Duration (Days) | AE Resolution Date – AE Onset Date + 1 |
| Drug-related | If relationship is marked 'YES' or is missing on the AE case report form (CRF) page. |

#### NOTES:

• If the study treatment stop date is missing then the AE will be considered to be On-Treatment.

HZA116492

# 10.5. Appendix 5: Data Display Standards & Handling Conventions

# 10.5.1. Study Treatment & Sub-group Display Descriptors

| Treatment Group Descriptions | | | |
|---|---|---|---|
| RandAll NG | | Data Displays for Reportin | g |
| Code | Description | Description | Order [1] |
| А | Fluticasone furoate /vilanterol inhalation<br>Powder delivered once daily | FF/VI | 2 |
| В | Usual ICS/LABA maintenance therapy delivered by Dry Powder Inhaler | Usual ICS/LABA | 1 |

# NOTES:

#### 10.5.2. Baseline Definition & Derivations

#### 10.5.2.1. Baseline Definitions

For all endpoints the baseline value will be the last assessment prior to randomisation.

# 10.5.2.2. Derivations and Handling of Missing Baseline Data

| Definition | Reporting Details |
|---|---|
| Change from Baseline | = Post-Dose Visit Value – Baseline |
| % Change from Baseline | = 100 x [(Post-Dose Visit Value – Baseline) / Baseline] |
| Maximum Change from Baseline | = Calculate the change from baseline at each given timepoint and determine the maximum change |

#### NOTES:

- Unless otherwise specified, the baseline definitions specified in Section 10.5.2.1 will be used for derivations for endpoints / parameters and indicated on summaries and listings.
- Unless otherwise stated, if baseline data is missing no derivation will be performed and will be set to missing.
- The baseline definition will be footnoted on all change from baseline displays.

#### 10.5.3. Reporting Process & Standards

| Reporting Process | |
|---|---|
| Software | |
| The currently supported versions of SAS software will be used. | |
| Reporting Area | |
| HARP Server | : uk1salx00175 |
| HARP Area | : /arenv/arprod/gw685698_gw642444/hza116492/final |
| QC Spreadsheet | : /arenv/arwork/gw685698_gw642444/hza116492/final/qc |
| Analysis Datasets | |
| Analysis datasets will be created according to CDISC standards. | |

<sup>1.</sup> Order represents treatments being presented in data displays, as appropriate.

HZA116492

# **Reporting Process**

 For creation of ADaM datasets (e.g. ADCM, ADAE) the same version of dictionary datasets will be implemented for conversion from SI to SDTM.

#### Generation of RTF Files

RTF files will be generated for all tables in the final reporting effort.

#### **Reporting Standards**

#### General

- The current GSK IDSL will be applied for reporting, unless otherwise stated:
  - 4.03 to 4.23: General Principles
  - 5.01 to 5.08: Principles Related to Data Listings
  - 6.01 to 6.11: Principles Related to Summary Tables
  - 7.01 to 7.13: Principles Related to Graphics

#### **Formats**

- All data will be reported according to the treatment the subject was randomised to unless otherwise stated
- GSK IDSL Statistical Principles (5.03 & 6.06.3) for decimal places (DPs) will be adopted for reporting of data based on the raw data collected.
- Numeric data will be reported at the precision collected on the electronic case report form (eCRF) or recorded in the raw dataset if from non eCRF sources.
- The reported precision from non eCRF sources will follow the IDSL statistical principles but may be adjusted to a clinically interpretable number of DP's.

#### **Planned and Actual Times**

- Reporting for tables, figures and formal statistical analyses :
  - Planned time relative to dosing will be used in figures, summaries, statistical analyses and calculation of any derived parameters, unless otherwise stated.
  - The impact of any major deviation from the planned assessment times and/or scheduled visit days on the analyses and interpretation of the results will be assessed as appropriate.
- Reporting for Data Listings:
  - Planned and actual time relative to study drug dosing will be shown in listings (Refer to IDSL Statistical Principle 5.05.1).
  - Unscheduled or unplanned readings will be presented within the subject's listings.
  - For visits outside the time-windows, please see Section 10.3.

# **Unscheduled Visits**

- Unscheduled visits will not be included in summary tables or figures.
- All unscheduled visits will be included in listings.

# **Descriptive Summary Statistics**

| Continuous Data | Refer to IDSL Statistical Principle 6.06.1 |
|--------------------|--------------------------------------------|
| Categorical Data | N, n, frequency, % |
| Graphical Displays | |

Refer to IDSL Statistical Principals 7.01 to 7.13.

HZA116492

#### 10.6. **Appendix 6: Derived and Transformed Data**

#### 10.6.1. General

## Multiple Measurements at One Time Point

- If there are multiples values within a time window the last valid value prior to randomisation will be used as the baseline value and the value closest to the target day for that window will be used for all postrandomisation visits. If values are the same distance from the target then the mean will be taken.
- Subjects having both High and Low values for Normal Ranges at any post-baseline visits for safety parameters will be counted in both the High and Low categories of "Any visit post-baseline" row of related summary tables. This will also be applicable to relevant Potential Clinical Importance summary tables.

#### Study Day

- Calculated as the number of days from randomisation date :
  - Ref Date = Missing
- → Study Day = Missing
- Ref Date < Randomisation Date → Study Day = Ref Date Randomisation Date
- Ref Data ≥ Randomisation Date → Study Day = Ref Date (Randomisation Date) + 1

#### **Time Since First Dose**

- Calculated as the number of days from the date of first dose :
  - Ref Date = Missing
- → Time Since First Dose = Missing
- Ref Date < First Dose Date → Time Since First Dose = Ref Date First Dose Date
- Ref Date ≥ First Dose Date → Time Since First Dose = Ref Date (First Dose Date) + 1

#### **Study Treatment Discontinuation**

In this study, subjects who are intentionally and permanently withdrawn from study medication may not continue in the study attending the remaining visits (excluding the Follow-up contact) and completing the scheduled assessments.

#### 10.6.2. **Study Population**

# **Demographics**

## Age

- GSK standard IDSL algorithms will be used for calculating age where birth date will be imputed as
  - Any subject with a missing day will have this imputed as day '15'.
  - Any subject with a missing date and month will have this imputed as '30th June'.
- Birth date will be presented in listings as 'YYYY'.
- Completely missing dates of birth will remain as missing, with no imputation applied. Consequently, the age of the subject will not be calculated and will remain missing.
- Age, in whole years, will be calculated with respect to the date of screening (Visit 1).

# **Body Mass Index**

Calculated as Weight (kg) / [Height (m)]<sup>2</sup>

#### Race

In the demographic summary table race will be summarised as follows: White is defined as those subjects who chose only the White (Arabic/North African Heritage) and/or White

HZA116492

# **Demographics**

(White/Caucasian/European Heritage) categories on the CRF, Black is defined as those subjects who chose only the African American/African Heritage category on the CRF, and Other is defined as those subjects who chose any of the other races on the CRF.

### **Extent of Exposure**

Subjects randomised to FF/VI or to Usual ICS/LABA can have their treatment dosage adjusted at the investigators discretion, and will be recorded in the eCRF. Treatment sequence identifier will be incremented by 1 each time the study medication is modified, and recorded on eCRF.

Extent of exposure will be presented in three different ways:

 The extent of exposure to study medication, regardless of study medication dosage modifications during the study, will be defined as the number of days on study medication and will be calculated for each subject as follows:

Exposure = (study medication stop date - study medication start date) + 1

If medication start date is missing then the randomisation date (i.e. date of Visit 2) of the subject will be used for medication start date. If the medication stop date is missing, the Visit 6 date or early withdrawal visit date will be used instead. If all these dates are missing, then the extent of exposure will be set to missing.

- The extent of exposure to study medication, up to first study medication dosage modification
- The extent of exposure to each dose of study medication, presented separately for FF/VI 92 mcg/22 mcg, FF/VI 184 mcg/22mcg, FP/S 250 mcg/50 mcg, FP/S 500 mcg/50 mcg, BUD/F 200 mcg/6 mcg, BUD/F 400 mcg/12 mcg

#### 10.6.3. Efficacy

#### **Primary Endpoint**

# ACT

The ACT is a validated self-administered questionnaire utilising 5 questions to assess asthma control during the past 4 Weeks on a 5-point categorical scale (1 to 5).

By answering all 5 questions, a subject with asthma can obtain a score that may range between 5 and 25, with higher scores indicating better control. An ACT score of 5 to 19 suggests that the subject's asthma is unlikely to be well controlled. A score of 20 to 25 suggests that the subject's asthma is likely to be well controlled. The MID for ACT is 3 (Schatz, 2009).

The total score is calculated as the sum of the scores from all 5 questions, provided all scores are non-missing; if any individual scores are missing then the overall score will be set to missing.

HZA116492

# **Secondary Endpoint**

#### **Correct Use of Device**

Inhaler use will be assessed at Randomisation (Visit 2), Week 12 (Visit 4) and Week 24 (Visit 6). Correct use of device is defined as making no critical or non-critical errors.

#### **Critical and Non-Critical Errors for Ellipta**

#### Critical errors:

- Failed to open cover
- Shook the device upside down after dose preparation
- Exhaled directly into mouthpiece
- No seal by the lips around the mouthpiece during the inhalation

#### Non-critical errors:

- No exhalation before an inhalation
- Inhalation manoeuvre was not:
  - long
  - steady
  - deep
- Blocked air inlet during inhalation manoeuvre
- Did not hold breath
- Did not close the device (Note: this is an error but one which does not affect the medication that is inhaled)

#### **Critical and Non-Critical Errors for Diskus**

# Critical errors:

- Failed to open cover
- · Lever is not pushed back
- Shook the device after dose preparation
- Exhaled directly into mouthpiece
- No seal by the lips round the mouthpiece during the inhalation

#### Non-critical errors:

- No exhalation before an inhalation
- Inhalation manoeuvre was not:
  - steady
  - deep
- Did not hold breath
- Did not close the device (Note: this is an error but one which does not affect the medication that is inhaled)

# **Critical and Non-Critical Errors for Turbuhaler**

#### Critical errors:

- Failed to remove cap
- Did not hold device upright (±45° OK) during dose preparation
- Base not twisted fully backwards and forwards, no click heard
- Shook the device after dose preparation
- Exhaled directly into mouthpiece
- No seal by the lips round the mouthpiece during the inhalation

HZA116492

# **Primary Endpoint**

Non-critical errors:

- Device tipped downwards after dose preparation
- No exhalation before an inhalation
- Inhalation manoeuvre was not:
  - forceful
  - deep
- Blocked air inlet during inhalation manoeuvre
- Did not hold breath
- Did not close the device (Note: this is an error but one which does not affect the medication that is inhaled)

#### **Other Endpoints**

#### FEV1

FEV1 will be measured to assess lung function at Randomisation (Visit 2) and Week 12 (Visit 4). Visit 4 should be scheduled at the same time of day as Visit 2, FEV1 measurements should be taken pre-dose and subjects should be instructed not to take their asthma medication/study drug prior to coming into the clinic at these visits. Subjects should also withhold from using their rescue medication for at least 4 hours prior to Visit 2 and Visit 4.

All sites will use standardised spirometry equipment provided by GSK. For each observation, at least 3 (with no more than 8) efforts will be obtained. At least two of the spirometry efforts should be acceptable and repeatable. The best FEV1 value will be recorded in the eCRF.

# MARS-A

The MARS-A questionnaire is a 10-item questionnaire. The response to all ten questions will be presented and included in the calculation of the MARS-A 10-score.

The responses to the MARS-A questions will be scored as follows: Always=1, Often=2, Sometimes=3, Rarely=4, Never=5. The MARS-A 10-Score will be calculated for each subject as the sum of scores for each of the ten questions divided by the number of non-missing responses to the ten questions.

If some responses are missing the MARS-A 10-score is calculated as follows for each subject:

- If eight or more of the questions have been answered, the missing responses for that subject will be imputed to the average score
- If less than eight of the questions have been answered, the overall MARS-A 10-score for that subject will be set to missing

The French translation of the MARS-A questionnaire did not go through cognitive debriefing; therefore while the study was ongoing it was determined that there is no word for "preventer" in French. "Preventer inhaler" was translated as "dispositif d'inhalation" (i.e., "inhalation device"). A reminder was sent to centres in France instructing that the MARS-A questionnaire refers to the patient's preventer inhaler (i.e. their maintenance therapy prior to entering the study, and study medication while on-study) as opposed to their reliever inhaler. The German translation went through cognitive debriefing and was correctly translated. The MARS-A data displays will therefore be repeated split by:

 Patients in France who had completed all MARS-A assessments prior to the reminder being implemented

HZA116492

# Other Endpoints

- Patients in France who had completed at least one MARS-A assessment prior to the reminder being implemented but also completed at least one MARS-A assessment after the reminder being implemented
- Patients in France who had not completed any MARS-A assessments prior to the reminder being implemented
- Patients in Germany

The reminder was sent on 17OCT2016, and it was assumed that the centres started implementing the instructions two days after this, i.e. on 19OCT2016.

#### **Severe Asthma Exacerbations**

Missing onset or resolution dates will be handled as follows:

- Single event with missing onset and/or resolution dates:
  - (a) Missing onset date: set onset date = study treatment start date
  - (b) Missing resolution date: set resolution date = study treatment stop date
  - (c) Both missing: imputed per both (a) and (b)
- Multiple events, one event with some missing onset/resolution dates; on the assumption any partial date information does not occur during the other events:
  - (a) Missing onset date: set onset date = max[(resolution date of the nearest previous event) + 1 day, study treatment start date]
  - (b) Missing resolution date: set resolution date = min[(onset date of the nearest subsequent event) -1 day, study treatment stop date]
  - (c) Both missing: determine the largest gap between study treatment start date and first event onset date, between first event resolution date and next event(s) onset dates (if any), between last event resolution date and study treatment stop date. If there is more than one gap which is the largest, then take the first occurrence. Then impute as follows:

onset date = (onset date of largest gap) + 1 day resolution date = (resolution date of largest gap) + 1 day

# Time to First Severe Asthma Exacerbation

The date of a severe asthma exacerbation is defined as the exacerbation onset date. Subjects who complete the study without a severe asthma exacerbation will be censored. Time to first severe asthma exacerbation is measured from the date of randomisation (i.e., study treatment start date) to the onset date of first severe asthma exacerbation, as recorded on eCRF, or study treatment stop date (Visit 6 or early withdrawal visit) for subject who complete the study without any severe asthma exacerbations (censored). Analyses of time to first severe asthma exacerbation will be censored at Day 168.

#### AQLQ(S) Domain and Total Scores

The AQLQ(S) contains 32 items in four domains: activity limitation (11 items), symptoms (12 items), emotional function (5 items) and environmental stimuli (4 items). The following items are included in each of the 4 domains:

- Symptoms: 6, 8, 10, 12, 14, 16, 18, 20, 22, 24, 29, 30
- Activity Limitation: 1, 2, 3, 4, 5, 11, 19, 25, 28, 31, 32
- Emotional Function: 7, 13, 15, 21, 27
- Environmental Stimuli: 9, 17, 23, 26

The response format consists of a seven-point scale where a value of 1 indicates "total impairment" and a value of 7 indicates "no impairment". The total AQLQ(S) score is the mean of all 32 items in the questionnaire and each individual domain score is calculated as the mean of the items within that domain. Hence, the total and domain scores are also each defined on a range from 1 to 7 with higher scores

HZA116492

#### Other Endpoints

indicating a higher quality of life. The MID for AQLQ(S) is 0.5 (Juniper, 1993).

For the total AQLQ(S) score, the score for a subject at any time point will only be calculated if at least 90% of the questions were answered (calculated as the mean of those non-missing questions). If fewer than 90% of the questions were answered then the mean score for that subject at that time point will be considered missing.

For each individual domain of the AQLQ(S) score, the score for a subject at any time point will only be calculated if at least 90% of the questions for that domain were answered (calculated as the mean of those non-missing questions). If fewer than 90% of the questions were answered for that domain then the mean score for that subject and domain at that time point will be considered missing.

# **EQ-5D-5L Utility and VAS Scores**

The EQ-5D-5L is administered at randomisation (Visit 2), Week 24 (Visit 6) and Early Withdrawal. The EQ-5D-5L consists of 2 parts: the EQ-5D-5L descriptive system and the EQ VAS.

The EQ-5D-5L descriptive system comprises the following 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels, where Level 1 (coded as '1') = 'No problems', Level 2 (coded as '2') = 'Slight problems', Level 3 (coded as '3') = 'Moderate problems', Level 4 (coded as '4') = 'Severe problems' and Level 5 (coded as '5') = 'Extreme problems'. Subjects indicate their health state for each dimension by ticking (or placing a cross) in the box of the most appropriate level for that dimension. Ambiguous values (e.g. 2 boxes are ticked for a single dimension) will be considered missing. Missing values will be coded as '9'. The responses (1, 2, 3, 4 or 5) to the five questions will be converted into a single utility score using the developer's instructions (EuroQol, 2013): the responses (1, 2, 3, 4 or 5) to the five questions in the descriptive system can be represented as one of 5<sup>5</sup>=3125 possible health states (11111, 11112, ..., 55555). These will be converted into a single summary index (y) that attaches value to each of the levels in each dimension by applying the formula below, which is based on the EQ-5D-5L value set for England (Devlin, 2016).

```
\begin{array}{l} y = 1 - 0.9675 \times (0.051M_2 + 0.063M_3 + 0.212M_4 + 0.275M_5 + 0.057S_2 + 0.076S_3 \\ &\quad + 0.181S_4 + 0.217S_5 + 0.051U_2 + 0.067U_3 + 0.174U_4 + 0.190U_5 + 0.060P_2 \\ &\quad + 0.075P_3 + 0.276P_4 + 0.341P_5 + 0.079A_2 + 0.104A_3 + 0.296A_4 \\ &\quad + 0.301A_5) \end{array}
```

where variables with subscript n are indicator variables equal to 1 when the corresponding level for the dimension is 'n' and equal to 0 otherwise,  $M_m$  variables represent responses for the mobility domain,  $S_m$  variables represent responses for the self-care domain,  $U_n$  variables represent responses for the usual activities domain,  $P_n$  variables represent responses for the pain / discomfort domain, and  $A_n$  variables represent responses for the anxiety / depression domain.

For example, health state where domains MSUPA = 11223 would be equal to:

$$1 - 0.9675 \times (0.051 + 0.060 + 0.104) \approx 0.7920$$

The EQ VAS records the subject's self-rated health state on a vertical, VAS where 0='worst imaginable health state' and 100='best imaginable health state'. Subjects indicate their own health state by drawing a line from the box on the left of the scale to whichever point on the scale indicates how good or bad their own health state is that day. Ambiguous values (e.g. the line crosses the VAS twice) will be considered missing. Missing values will be coded as '999'.

Only validated EuroQoLs completed in the same language as that completed at Baseline (Visit 2) will be
HZA116492

# **Other Endpoints**

summarised.

#### **PASAP-Q Domain and Total Scores**

The PASAP-Q is a self-administered 16-item questionnaire measuring satisfaction and preference with inhaler devices (Kozma, 2005). Two domains (performance and convenience) are calculated from 13 satisfaction items, measured on a Likert-type scale where a value of 1 indicates "very dissatisfied" and 7 indicates "very satisfied". The performance and convenience domains together form the total score. The other items include an overall satisfaction question (again measured from 1 to 7), a preference question (not applicable and so not asked for this study) and a question on willingness to continue using the device in the future, measured on a scale of 0 (not willing) to 100 (definitely willing).

The performance and convenience domains include the following items:

• Performance: 1, 2, 3, 4, 5, 10, 11

• Convenience: 6, 7, 8, 9, 12, 13

If the patient completes at least half of the items in a domain, values for missing items are imputed using the mean of the completed items in that domain. The domain score is then transformed to a scale from 0 (least) to 100 (most) as follows:

Domain Score = 
$$[Mean(responses for items in domain) - 1] \times \frac{100}{6}$$

If the patient completes less than half of the items in a domain, then the missing items are not imputed and the domain score is set to missing. The total score can be calculated only when both domain scores are computable and substitution for missing items at the domain level has taken place, and is calculated on the same scale as:

Total Score = 
$$[Mean(responses for all 13 items) - 1] \times \frac{100}{6}$$

The overall satisfaction and willingness questions are summarised on their original scales of 1 to 7 and 0 to 100 respectively.

HZA116492

# **Other Endpoints**

#### **Treatment Compliance**

Overall percentage treatment compliance for every subject will be calculated for each type of inhaler (Diskus, Turbuhaler and Ellipta) separately.

Compliance for Diskus, Turbuhaler and Ellipta will be based on the total number of inhalations taken from each type of inhaler and the expected number of inhalations to be taken. The expected number of inhalations will be derived as the expected number of inhalations per day (from each inhaler) multiplied by the number of days on study drug based on the subjects treatment start and stop date for that type of inhaler.

The total number of inhalations taken will be based on the dose counter for each type of inhaler, all of which are re-supplied during the study. If there is no dose counter information at all then the compliance will be missing; however, as long as the information from one dose counter is present, the compliance will be calculated. If a dose counter start count is missing then it will be assumed to be 30 for Ellipta and 60 for both Diskus and Turbuhaler.

In each calculation, all inhalers dispensed will be used, provided the dose counter stop counts are non-missing. The following formula will be used:

$$Compliance = \frac{Total\ number\ of\ inhalations\ taken}{Dose\ frequency\ \times\ (Stop\ date\ -\ Start\ date)} \times 100$$

where Total number of inhalations taken is the sum of (dose counter start count – dose counter stop count) for all inhalers used during the time period, Dose frequency is equal to 1 for Ellipta and 2 for Diskus and Turbuhaler, and Start date and Stop date are the earliest treatment start date and latest treatment stop date respectively recorded for all inhalers used during the time period.

# 10.6.4. Safety

#### **SAEs of Special Interest**

SAE groups of special interest have been defined as SAEs which are included in specified areas of interest for one or more of the treatment groups (FF/VI, FF and/or VI). They are identified by groupings of preferred terms based on the Medical Dictionary for Regulatory Activities (MedDRA) dictionary version used in each reporting effort. Groupings or subgroups may be defined, based on relevant combination of preferred terms, or on Standardised MedDRA queries (SMQs).

SAEs of special interest will be confirmed prior to final data, based on the MedDRA version in use at the time.

| Special Interest SAE Group |
|---------------------------------------------------------|
| Asthma/bronchospasm |
| Cardiovascular effects |
| Decreased bone mineral density and associated fractures |
| Hypersensitivity |
| Local steroid effects |
| LRTI excluding pneumonia |
| Pneumonia |
| Adrenal suppression |
| Ocular effects |
| Effects on glucose |
| Effects on potassium |
| Tremor |

HZA116492

# **Laboratory Parameters**

- If a laboratory value which is expected to have a numeric value for summary purposes, has a non-detectable level reported in the database, where the numeric value is missing, but typically a character value starting with '<x' or '>x' (or indicated as less than x or greater than x in the comment field) is present, the number of significant digits in the observed values will be used to determine how much to add or subtract in order to impute the corresponding numeric value.
  - Example 1: 2 Significant Digits = '< x ' becomes x 0.01</li>
  - Example 2: 1 Significant Digit = '> x' becomes x + 0.1
  - Example 3: 0 Significant Digits = '< x' becomes x 1</li>

HZA116492

# 10.7. Appendix 7: Premature Withdrawals & Handling of Missing Data

# 10.7.1. Premature Withdrawals

| Element | Reporting Detail |
|---|---|
| General | <ul> <li>Subject study completion was defined in the protocol as a subject who has completed all study visits. The end of the study is defined as the last subject's last visit.</li> <li>The definition of subject early withdrawal from the study will be any subject who is randomised and, for any reason, does not complete all study visits.</li> <li>Withdrawn subjects will not be replaced in the study.</li> <li>All available data from subjects who were withdrawn from the study will be listed and all available planned data will be included in summary tables and figures, unless otherwise specified.</li> </ul> |

# 10.7.2. Handling of Missing Data

| Element | Reporting Detail |
|---|---|
| General | Missing data occurs when any requested data is not provided, leading to blank fields on the collection instrument: |
| | These data will be indicated by the use of a "blank" in subject<br>listing displays (if applicable). Unless all data for a specific visit are missing in<br>which case the data is excluded from the table. |
| | <ul> <li>Answers such as "Not applicable" and "Not evaluable" are not<br/>considered to be missing data and should be displayed as such.</li> </ul> |
| Outliers | <ul> <li>Any subjects excluded from the summaries and/or statistical<br/>analyses will be documented along with the reason for exclusion in the clinical study<br/>report.</li> </ul> |
| Exposure start and stop date | If a subject's treatment start date is missing then their Visit 2 date will be assumed to be the exposure start date. If a subject's treatment stop date is missing, this will be taken to be the date of Week 24 (Visit 6) (if the subject completes Visit 6) or the early withdrawal visit date. |

# 10.7.2.1. Handling of Missing or Partial Dates

| Element | Reporting Detail |
|---|---|
| General | Partial dates will be displayed as captured in subject listing displays. |
| SAEs and<br>ADRs | • The eCRF does not allow the possibility of partial dates (i.e., only month and year) to be recorded for SAE and ADR start and end dates; |
| | <ul> <li>Completely missing start or end dates will remain missing, with no imputation applied.</li> <li>Consequently, time to onset and duration of such events will be missing.</li> </ul> |
| Concomitant<br>Medications | Partial dates for any concomitant medications recorded in the CRF will be imputed using the following convention: |
| | <ul> <li>If the partial date is a start date, a '01' will be used for the day and 'Jan' will be<br/>used for the month</li> </ul> |
| | <ul> <li>If the partial date is a stop date, a '28/29/30/31' will be used for the day<br/>(dependent on the month and year) and 'Dec' will be used for the month.</li> </ul> |

HZA116492

| Element | Reporting Detail |
|---------|----------------------------------------------------------|
| | The recorded partial date will be displayed in listings. |

# 10.7.2.2. Handling of Missing Data for Statistical Analysis

In general, missing data will not be imputed except for the sensitivity analyses defined in Section 6.1.2.

HZA116492

# 10.8. Appendix 8: Values of Potential Clinical Importance

# 10.8.1. Vital Signs

| Vital Sign Parameter | Units | Clinical Concern Range | |
|--------------------------------|-------|------------------------|-------|
| (Absolute) | | Lower | Upper |
| Systolic Blood Pressure (SBP) | mmHg | < 85 | > 160 |
| Diastolic Blood Pressure (DBP) | mmHg | < 45 | > 100 |
| Heart Rate (HR) | bpm | < 40 | > 110 |

| Vital Sign Parameter | Units | Clinical Concern Range | | | |
|---|---|---|---|---|---|
| (Change from Baseline) Decrease | | Incre | Increase | | |
| | | Lower | Upper | Lower | Upper |
| SBP | mmHg | ≥ 20 | ≥ 40 | ≥ 20 | ≥ 40 |
| DBP | mmHg | ≥ 10 | ≥ 20 | ≥ 10 | ≥ 20 |
| HR | bpm | ≥ 15 | ≥ 30 | ≥ 15 | ≥ 30 |

HZA116492

# 10.9. Appendix 9: Multicenter Studies

# 10.9.1. Methods for Handling Centres

In this multicentre study conducted in France and Germany, enrolment will be presented by investigative site.

HZA116492

# 10.10. Appendix 10: Examination of Covariates, Subgroups & Other Strata

#### 10.10.1. Examination of Strata and Covariates

The following is a list of covariates that may be used in descriptive summaries and statistical analyses, some of which may also be used for subgroup analyses.

Additional covariates of clinical interest may also be considered.

| Category | Covariates and / or Subgroups |
|---|---|
| Strata | Separate randomisation schedules were utilised for France and Germany respectively thereby stratifying the randomisation by country. Country will be included in all analyses as a covariate. A sensitivity analysis will examine the randomized treatment-by-country interaction for the primary and key secondary endpoints. |
| Covariates | For the primary efficacy analysis, the following baseline variables will be adjusted for: Randomised treatment (FF/VI, Usual ICS/LABA) Baseline ACT total score Age Gender Country Similar covariates will be considered for all other analyses; in each case the relevant baseline score (e.g. baseline AQLQ[S] score for the AQLQ[S] endpoints) will be included instead of baseline ACT total score. |

# 10.10.2. Examination of subgroups

- If the percentage of subjects is small within a particular subgroup, then the subgroup categories may be refined prior to unblinding the trial.
- If the category cannot be refined further, then descriptive rather than statistical comparisons may be performed for the particular subgroup.
- For statistical analyses by subgroup, models will include subgroup and treatment by subgroup interaction as covariates.

| Category | Subgroups |
|------------------------------------|-----------------|
| Country | France |
| | Germany |
| Number of severe asthma | • 0 |
| exacerbations in the previous year | • ≥1 |
| prior to randomisation | |
| Smoking Status at Baseline | Current smokers |

HZA116492

| Category | Subgroups |
|-----------|---------------------|
| | Former smokers |
| | Non-smokers |
| Age Group | • 18 – 50 years old |
| | > 50 years old |
| Gender | Male |
| | Female |

# 10.10.3. Examination of seasonal effect

A sensitivity analysis for the primary efficacy endpoint examining seasonal effect is defined in Section 6.1.2, specifying a season at randomisation covariate defined as follows:

| Season at Randomisation | Calendar Month of Randomisation |
|-------------------------|---------------------------------|
| Spring | March |
| | April |
| | May |
| Summer | June |
| | • July |
| | August |
| Autumn | September |
| | October |
| | November |
| Winter | December |
| | January |
| | February |

Furthermore, the summary of severe asthma exacerbations will be repeated by season using the same definition (according to calendar month) as specified above.

HZA116492

# 10.11. Appendix 11: Multiple Comparisons & Multiplicity

# 10.11.1. Handling of Multiple Comparisons & Multiplicity

Non inferiority of FF/VI to ICS/LABA will be first tested at the 0.05 two-sided nominal level of significance. If non-inferiority is statistically achieved, then superiority of FF/VI to ICS/LABA will be tested at the 0.05 two-sided nominal level of significance.

If and only if non-inferiority is achieved for the primary endpoint at Week 12 (Visit 4), then the key secondary endpoint, i.e. the change from baseline in the total ACT score assessed at Week 24 (Visit 6) will be tested. At Week 24 (Visit 6), non inferiority of FF/VI to ICS/LABA will be first tested at the 0.05 two-sided nominal level of significance. If non-inferiority is achieved, then superiority of FF/VI to ICS/LABA will be tested at the 0.05 two-sided nominal level of significance.

Of note, this step-down testing procedure still strongly controls the overall type I error at the 0.05 two-sided level for the non-inferiority endpoints. The overall type I error is not controlled for the superiority tests at Week 12 (Visit 4) and Week 24 (Visit 6).

HZA116492

# 10.12. Appendix 12: Model Checking and Diagnostics for Statistical Analyses

#### 10.12.1. Statistical Analysis Assumptions

| Endpoint(s) | Change from Baseline in the ACT Total Score at Week 12 (Visit 4) |
|---|---|
| | Change from Baseline in the ACT Total Score at Week 24 (Visit 6) |
| Analysis | MMRM (ANCOVA for LOCF and WOCF sensitivity analyses) |

- Should computational issues be encountered when running the model with an unstructured variancecovariance matrix, other structures including autoregressive 1 and compound symmetry will be considered.
- Distributional assumptions underlying the model will be checked with graphical methods (including
  quantile-quantile (Q-Q) plots of studentized residuals, plots of studentized residuals versus fitted
  values, etc.). To investigate the relationship between baseline ACT total score and the change from
  baseline in ACT total score, baseline ACT total will be categorized according to the distribution quartiles
  and the model will be fitted using this categorized variable in place of continuous baseline ACT total
  score.
- If the distributional assumption of normality fails then the LS means, estimated LS mean treatment
  difference and associated 95% CI from the model will be presented, with the p-value for the difference
  between treatment groups from a model on the rank-transformed values. Should the distributional
  assumption of normality also fail for the ranked model, other methods of analysis will be investigated.

# Percentage of subjects with correct use of inhaler device at Week 12 (Visit 4) and at Week 24 (Visit 6) independently of the use at Week 12 (Visit 4) ACT total score of ≥ 20 or ≥ 3 point increase from baseline in ACT total score at Week 12 (Visit 4) and Week 24 (Visit 6) Increase from baseline of ≥ 0.5 in AQLQ(S) total score at Week 24 (Visit 6) Increase from baseline of ≥ 0.5 in AQLQ(S) environmental stimuli domain score at Week 24 (Visit 6) Proportion of subjects with 'no problems' at Endpoint in the EQ-5D-5L questionnaire Analysis

- If the likelihood maximisation algorithm fails to converge due to complete or quasi-complete separation
  of the data then Firth's penalized likelihood (Firth, 1993) will be implemented by use of the FIRTH
  option on the MODEL statement in PROC LOGISTIC.
- The fit of the logistic regression model will be assessed by examining the ROC curve and other diagnostic plots.

| Endpoint(s) | Change from baseline in trough (pre-dose) FEV1 at Week 12 (Visit 4) |
|---|---|
| | Change from baseline in EQ-5D Utility Score |
| | Change from baseline in EQ-5D VAS Score |
| Analysis | ANCOVA model |

- Distributional assumptions underlying the model will be checked with graphical methods (including quantile-quantile (Q-Q) plots of studentized residuals, plots of studentized residuals versus fitted values, etc.).
- If the distributional assumption of normality fails then the LS means, estimated LS mean treatment difference and associated 95% CI from the ANCOVA model will be presented, with the p-value for the

HZA116492

difference between treatment groups from an ANCOVA model on the rank-transformed values. Should the distributional assumption of normality also fail for the ranked ANCOVA, an exact p-value from a two-sample Wilcoxon Rank Sum test will be presented for the difference between treatment groups.

| Endpoint(s) | Annual severe asthma exacerbation rate over the study period |
|-------------|--------------------------------------------------------------|
| Analysis | GLM assuming the Negative Binomial distribution |

If a GLM assuming the Negative Binomial distribution cannot be fitted due to the lack of repeat events
within a subject, a GLM assuming the Poisson distribution will be used. The underlying assumption for
the Poisson distribution that the mean and variance of the response variable are equal will be
examined. If the variance of the fitted model exceeds the mean (over-dispersion), the dispersion
parameter will be estimated as a ratio of the Pearson Chi-Square to its associated degrees of freedom
(using the PSCALE option in PROC GENMOD).

| Endpoint(s) | • | Time to first severe asthma exacerbation |
|-------------|---|------------------------------------------|
| Analysis | • | Cox proportional hazards model |

- Proportional hazards assumptions will be checked by plotting the log of the negative log of the
  estimated survivor functions against log time, for each treatment group. If hazards are proportional, the
  lines should be approximately parallel.
- If the assumption of proportionality is not met, the use of other models such as models including timedependent covariates will be considered.
- If there are computational issues in implementing the exact method for handling ties, then the Efron method (Efron, 1977) will be used instead.

HZA116492

# 10.13. Appendix 13: Blinding Strategy

#### **Purpose**

- The trial design (open label) and the ways the study medication data are recorded in the
  datasets means that extra steps must be taken to ensure that S&P remain blinded to
  investigational product (IP) data until the formal unblinding takes place at DBF.
   Maintaining the blind prior to DBF is a requirement for the French Ethics Committee.
- S&P also need to be able to have sufficient data to pre-program up to the point of DBF. This needs to done on sufficient 'real' data to ensure the programs can handle all possibilities of data, particularly regarding treatment modifications during the study.
- Datasets containing IP data that need to be considered: EXPOSURE and INVPCOMP
- Other datasets that contain data that could unblind S&P and therefore also need to be considered: DS, DV1, FADTH, INDEVERR, and IPDEVMAL
- Note: assigning subjects to dummy (blinded) randomised treatment group (FF/VI or Other ICS/LABA) prior to DBF will be done in the usual way using standard GSK procedures.
- To ensure unblinding does not occur through other sources, access to INFORM, E-Track, Study Explorer, DMENV (\\uk1salx00175.corpnet2.com\dmenv\dmwork\gw685698\_gw642444\hza116492) and SPECTRE is prohibited for S&P.

# Proposal for the EXPOSURE dataset

Prior to DBF:

Data Management (DM) to provide two datasets to S&P based on the source EXPOSURE dataset

- (1) Dataset EXPOSURE same as the source EXPOSURE dataset but with EXINVPCD (study treatment code) and EXINVP (study treatment) blanked out as '999' and 'CENSORED' respectively. This will allow S&P to use the subjects' real exposure start dates and times and stop dates in order to assign other data items to pre, during and post treatment, derive study day, overall exposure duration etc
- (2) Dataset named DUM\_EXP\_SP, which will be a scrambled sample of the EXPOSURE dataset. Each time S&P are provided a new update of data from DM a different scrambled sample of data will be used.

The method to be used by DM to sample and scramble the data is as follows:

Select a sample of subjects, in the EXPOSURE dataset using a random sampling method
which uses a seed (so that the same ones could be chosen again if it needs to be re-run).
The exact size of this sample will change according to the number of subjects in the
EXPOSURE dataset at that time, ensuring that no more than ≈50% of the total sample
size (N=422) is used at any point and defined per the following table:

| No. of subjects in EXPOSURE dataset | Percentage of subjects used for sampling |
|---|---|
| ≤ 199 | 94% |
| 200 to 299 inclusive | 70% |
| ≥ 300 | 40% |

HZA116492

- Store which subjects have been chosen so it can be checked over time that all subjects get seen by programmers before DBR
- Make a random adjustment to the dates and times in the sample, such that e.g. the first subject has 10 days added to all their dates and 34 minutes added to their start times, the second subject has 17 days subtracted from all their dates and 95 minutes added to their start times this means they do not match with any real dates or times in the EXPOSURE dataset above, but it means the within-subject integrity of dates remains. The range of the date adjustment is set at the range ± 60 days, and the range of the time adjustment is set at the range ± 120 minutes.
- Rename subjid to orig\_subj this enables DM to be able to trace the subject in the event
  of data queries from S&P
- Randomly map this sampled data onto the SUBJIDs in the EXPOSURE dataset, so that
  every true SUBJID in the EXPOSURE dataset has scrambled subject data assigned to it
- Data management keep a copy of this with the orig\_subj number in it
- Data management remove orig subj and pass this data to S&P

#### At DBF:

DM will provide to S&P the one unmodified version of EXPOSURE dataset, with all variables uncensored.

# Proposal for the INVPCOMP, INDEVERR and IPDEVMAL datasets

#### Prior to DBF:

DM to provide a single version of each dataset to S&P based on the source datasets.

(1) Dataset named DUM\_INVP\_SP, DUM\_IERR\_SP and DUM\_IMAL\_SP which will be a scrambled (subjid) sample of the INVPCOMP, INDEVERR and IPDEVMAL datasets respectively. Each time S&P are provided a new update of data from DM a different scrambled sample of data will be used.

These datasets must be produced in conjunction with DUM\_EXP so that the same subjects get selected, the same date adjustment per subject is made and the same merging onto real subject data gets done.

#### At DBF:

DM will provide the single unmodified versions of INVPCOMP, INDEVERR and IPDEVMAL datasets, with all variables uncensored

Other datasets and variables to be censored before being sent to S&P up until DBF

| Dataset | Variables to be censored before being sent to |
|---------|-----------------------------------------------|
| | S&P up until DBF |
| DS | DSRSSP, DSSBRSSP |
| DV1 | DVTERM |
| FADTH | DDORRSTX, DDORRSSP |

#### **Documentation**

Once this blinding strategy has been agreed between S&P and DM, and approved by the study Clinical Investigation Lead (CIL), the Data Quality Lead (DQL) will send an email to S&P stating that the blinding strategy is in place and is being followed.

HZA116492

# 10.14. Appendix 14: Abbreviations & Trade Marks

# 10.14.1. Abbreviations

| Abbreviation | Description |
|--------------|---------------------------------------------------|
| ACT | Asthma Control Test |
| ADR | Adverse Drug Reaction |
| AE | Adverse Event |
| AESI | Adverse Event of Special Interest |
| ANCOVA | Analysis of Covariance |
| AQLQ(S) | Standardised Asthma Quality of Life Questionnaire |
| ASE | All Subjects Enrolled |
| BMI | Body Mass Index |
| BUD | Budesonide |
| CI | Confidence Interval |
| CIL | Clinical Investigational Lead |
| CRF | Case Report Form |
| CRO | Contract Research Organisation |
| DBF | Database Freeze |
| DBP | Diastolic Blood Pressure |
| DBR | Database Release |
| DM | Data Management |
| DP | Decimal Place |
| DPI | Dry Powder Inhaler |
| DQL | Data Quality Lead |
| eCRF | Electronic Case Report Form |
| EQ-5D-5L | EuroQol Questionnaire |
| F | Formoterol |
| FEV1 | Forced Expiratory Volume in 1 Second |
| FF | Fluticasone Furoate |
| FP | Fluticasone Propionate |
| GINA | Global Initiative for Asthma |
| GLM | Generalised Linear Model |
| GSK | GlaxoSmithKline |
| HL | Hodges-Lehmann |
| HR | Heart Rate |
| ICF | Informed Consent Form |
| ICS | Inhaled Corticosteroid |
| IDSL | Integrated Data Standards Library |
| IP | Investigational Product |
| ITT | Intent-to-Treat |
| LABA | Long-acting Beta Agonist |
| LOCF | Last Observation Carried Forward |
| LRTI | Lower Respiratory Tract Infection |
| LS | Least Squares |
| MAR | Missing at Random |
| MARS-A | Medication Adherence Report Scale for Asthma |
| MCID | Minimal Clinically Important Difference |
| MedDRA | Medical Dictionary for Regulatory Activities |

HZA116492

| Abbreviation | Description |
|--------------|---------------------------------------------------|
| MI | Multiple Imputation |
| MID | Minimally Important Difference |
| MMRM | Mixed Model Repeated Measures |
| PASAP-Q | Patient Satisfaction and Preference Questionnaire |
| PD | Protocol Deviation |
| PDMP | Protocol Deviation Management Plan |
| PP | Per Protocol |
| Q-Q | Quantile-Quantile |
| RAP | Reporting and Analysis Plan |
| REML | Restricted Maximum Likelihood |
| S | Salmeterol |
| S&P | Statistics and Programming |
| SAC | Statistical Analysis Complete |
| SAE | Serious Adverse Event |
| SBP | Systolic Blood Pressure |
| SD | Standard Deviation |
| SMQ | Standardised MedDRA Query |
| VAS | Visual Analogue Scale |
| VI | Vilanterol |
| WOCF | Worst Observation Carried Forward |

# 10.14.2. Trademarks

| Trademarks of the GlaxoSmithKline Group of Companies |
|------------------------------------------------------|
| DISKUS |
| ELLIPTA |
| GSK |
| NUCALA |
| SERETIDE |

| Trademarks not owned by the GlaxoSmithKline Group of Companies |
|----------------------------------------------------------------|
| ACT |
| Asthma Quality of Life Questionnaire - |
| AQLQ(S) |
| EQ-5D |
| MARS-A Questionnaire |
| PASAP Questionnaire |
| Symbicort Turbuhaler |
| TURBUHALER |
| XOLAIR |

HZA116492

# 10.15. Appendix 15: List of Data Displays

# 10.15.1. Data Display Numbering

The following numbering will be applied for RAP generated displays:

| Section | Tables | Figures |
|------------------|------------|------------|
| Study Population | 1.1 to 1.n | 1.1 to 1.n |
| Efficacy | 2.1 to 2.n | 2.1 to 2.n |
| Safety | 3.1 to 3.n | 3.1 to 3.n |
| Section | Listings | |
| ICH Listings | 1 t | 0 X |
| Other Listings | y t | 0 Z |

# 10.15.2. Mock Example Shell Referencing

Non IDSL specifications will be referenced as indicated and if required an example mock-up displays provided in Appendix 11: Example Mock Shells for Data Displays

.

| Section | Figure | Table | Listing |
|------------------|---------|---------|---------|
| Study Population | POP_Fn | POP_Tn | POP_Ln |
| Efficacy | EFF_Fn | EFF_Tn | EFF_Ln |
| Safety | SAFE Fn | SAFE Tn | SAFE Ln |

# NOTES:

Non-Standard displays are indicated in the 'IDSL / TST ID / Example Shell' or 'Programming Notes' column as '[Non-Standard] + Reference.'

# 10.15.3. Deliverable [Priority]

| Delivery [Priority] [1] | Description |
|-------------------------|-------------------------------------|
| Data Look [1] | Data Look Outputs (blinded review) |
| SAC [2] | Final Statistical Analysis Complete |

#### NOTES:

1. Indicates priority (i.e. order) in which displays will be generated for the reporting effort.

HZA116492

# 10.15.4. Study Population Tables

| Study F | Study Population: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Subject | Subject Disposition | | | | |
| 1.1. | All Enrolled<br>Subjects | Non-Standard<br>POP_T1 | Summary of Subject Populations | Randomised population line will provide the denominators for the ITT, PP and Safety percentages. | Data Look [1]<br>SAC [2] |
| 1.2. | All Enrolled<br>Subjects | IE2 | Summary of Inclusion/Exclusion Criteria Failures for Subjects Not Starting Treatment | | Data Look [1]<br>SAC [2] |
| 1.3. | ITT | ES1 | Summary of End of Study Record | | Data Look [1]<br>SAC [2] |
| 1.4. | PP | ES1 | Summary of End of Study Record<br>Per Protocol Population | | Data Look [1]<br>SAC [2] |
| 1.5. | ITT | Non-Standard<br>POP_T2 | Summary of Attendance at Each Clinic Visit and Phone Call Visit | | Data Look [1]<br>SAC [2] |
| 1.6. | All Enrolled<br>Subjects | NS3 | Summary of Number of Subjects by Country and Centre | | SAC [2] |
| 1.7. | ITT | NS3 | Summary of Number of Subjects by Country and Centre | | Data Look [1]<br>SAC [2] |
| 1.8. | PP | NS3 | Summary of Number of Subjects by Country and Centre Per Protocol Population | | SAC [2] |
| Protoco | ol Deviations | | | | |
| 1.9. | ITT | IE2 | Summary of Deviations from the Inclusion/Exclusion Criteria | | Data Look [1]<br>SAC [2] |
| 1.10. | ITT | Non-Standard<br>POP_T3 | Summary of Important Protocol Deviations | | Data Look [1]<br>SAC [2] |

| Study F | Study Population: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 1.11. | ITT | Non-Standard<br>POP_T3 | Summary of Important Protocol Deviations Resulting in Exclusion from the PP Population | | Data Look [1]<br>SAC [2] |
| Demog | raphic and Bas | eline Characteris | tics | • | |
| 1.12. | ITT | DM1 | Summary of Demographic Characteristics | | Data Look [1]<br>SAC [2] |
| 1.13. | PP | DM1 | Summary of Demographic Characteristics Per Protocol Population | | SAC [2] |
| 1.14. | Safety | DM1 | Summary of Demographic Characteristics<br>Safety Population | | SAC [2] |
| 1.15. | All Enrolled<br>Subjects | DM11 | Summary of Age Ranges | | Data Look [1]<br>SAC [2] |
| 1.16. | ITT | DM5 | Summary of Race and Racial Combinations | | Data Look [1]<br>SAC [2] |
| 1.17. | ITT | DM6 | Summary of Race and Racial Combinations Details | | Data Look [1]<br>SAC [2] |
| 1.18. | ITT | MH4 | Summary of Current Medical Conditions | | Data Look [1]<br>SAC [2] |
| 1.19. | ITT | MH4 | Summary of Past Medical Conditions | | SAC [2] |
| 1.20. | ITT | Non-Standard<br>POP_T4 | Summary of Asthma Duration at Baseline | | Data Look [1]<br>SAC [2] |
| 1.21. | PP | Non-Standard<br>POP_T4 | Summary of Asthma Duration at Baseline<br>Per Protocol Population | | Data Look [1]<br>SAC [2] |
| 1.22. | ITT | Non-Standard<br>POP_T5 | Summary of Asthma Exacerbation History at Baseline | | Data Look [1]<br>SAC [2] |

| Study F | Study Population: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 1.23. | PP | Non-Standard<br>POP_T5 | Summary of Asthma Exacerbation History at Baseline<br>Per Protocol Population | | Data Look [1]<br>SAC [2] |
| 1.24. | ITT | Non-Standard<br>POP_T6 | Summary of Smoking History at Baseline | | Data Look [1]<br>SAC [2] |
| 1.25. | PP | Non-Standard<br>POP_T6 | Summary of Smoking History at Baseline<br>Per Protocol Population | | SAC [2] |
| Concor | nitant Medicati | ons | | | |
| 1.26. | ITT | CM8 | Summary of Pre-Treatment Concomitant Medications | | SAC [2] |
| 1.27. | ITT | CM8 | Summary of On-Treatment Concomitant Medications | | SAC [2] |
| 1.28. | ITT | CM8 | Summary of On-Treatment Asthma Concomitant Medications | | Data Look [1]<br>SAC [2] |
| Exposi | ire | | | | |
| 1.29. | ITT | Non-Standard<br>POP_T7 | Summary of Study Medication Dosage Modification | | Data Look [1]<br>SAC [2] |
| 1.30. | ITT | Non-Standard<br>POP_T8 | Summary of Extent of Exposure to Study Medication (Regardless of Modification to Study Medication Dosage) | | Data Look [1]<br>SAC [2] |
| 1.31. | ITT | Non-Standard<br>POP_T8 | Summary of Extent of Exposure to Study Medication (up to First Modification to Study Medication Dosage) | | SAC [2] |

| Study Population: Tables | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 1.32. | ITT | Non-Standard<br>POP_T9 | Summary of Extent of Exposure to Study Medication by Medication and Dosage | Repeat on subsequent pages for Medication/Dosage = FF/VI 184 mcg/22 mcg OD, FP/S 250 mcg/50 mcg BID, FP/S 500 mcg/50 mcg BID, BUD/F 200 mcg/6 mcg BID (1 inhalation per dose), BUD/F 200 mcg/6 mcg BID (2 inhalations per dose), BUD/F 400 mcg/12 mcg BID (1 inhalation per dose), BUD/F 400 mcg/12 mcg BID (2 inhalations per dose). | Data Look [1]<br>SAC [2] |
| Number | Number of Subjects by Subgroup | | | | |
| 1.33. | ITT | Non-Standard<br>POP_T10 | Summary of Number of Subjects by Subgroup | | SAC [2] |

HZA116492

# 10.15.5. Study Population Figures

| Study Population: Figures | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Exposure | | | | | |
| 1.1. | ITT | Non-Standard<br>POP_F1 | Plot of Exposure to Study Medication (Regardless of Modification to Study Medication Dosage) | Display increments of 6 weeks on the x-axis, up to the maximum exposure (e.g. 0, 6, 12, 18, 24, 30). | Data Look [1]<br>SAC [2] |

HZA116492

# 10.15.6. Efficacy Tables

| Efficac | Efficacy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Change | from Baseline | in ACT Total Sco | re at Week 12 (Visit 4) | | |
| 2.1. | ITT | Non-Standard<br>EFF_T1 | Summary of Change from Baseline in ACT Total Score | | Data Look [1]<br>SAC [2] |
| 2.2. | PP | Non-Standard<br>EFF_T1 | Summary of Change from Baseline in ACT Total Score<br>Per Protocol Population | | SAC [2] |
| 2.3. | ITT | Non-Standard<br>EFF_T2 | Summary of the Statistical Analysis of Change from Baseline in ACT Total Score at Week 12 (Visit 4) | | Data Look [1]<br>SAC [2] |
| 2.4. | PP | Non-Standard<br>EFF_T2 | Summary of the Statistical Analysis of Change from Baseline in ACT Total Score at Week 12 (Visit 4) Per Protocol Population | | SAC [2] |
| 2.5. | ІТТ | Non-Standard<br>EFF_T2 | Summary of the Statistical Analysis of Change from Baseline in ACT Total Score at Week 12 (Visit 4) (ANCOVA with LOCF) | Footnotes as follows: "Note: The analysis method was an ANCOVA model adjusted for randomised treatment, baseline ACT total score, gender, age and country. Note: Missing values at Week 12 (Visit 4) were replaced by last available post-randomization value based on the last observation carried forward (LOCF) method." | Data Look [1]<br>SAC [2] |

| Efficacy | Efficacy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.6. | ІТТ | Non-Standard<br>EFF_T2 | Summary of the Statistical Analysis of Change from Baseline in ACT Total Score at Week 12 (Visit 4) (Multiple Imputation – Missing at Random Approach) | Footnotes as follows: "Note: Missing values post- randomisation were imputed using multiple imputation methods based on pattern mixture models. Note: Each imputed data set was analysed using an ANCOVA model at Week 12 (Visit 4) adjusted for randomised treatment, baseline ACT total score, gender, age and country and the resulting treatment differences and their standard errors combined using Rubin's rules." | Data Look [1]<br>SAC [2] |
| 2.7. | ІТТ | Non-Standard<br>EFF_T2 | Summary of the Statistical Analysis of Change from Baseline in ACT Total Score at Week 12 (Visit 4) (Multiple Imputation – Copy Differences from Reference Approach) | Footnotes as follows: "Note: Missing values post- randomisation were imputed using multiple imputation methods based on pattern mixture models. Note: Each imputed data set was analysed using an ANCOVA model at Week 12 (Visit 4) adjusted for randomised treatment, baseline ACT total score, gender, age and country and the resulting treatment differences and their standard errors combined using Rubin's rules." | Data Look [1]<br>SAC [2] |

| Efficacy | Efficacy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.8. | ITT | Non-Standard<br>EFF_T2 | Summary of the Statistical Analysis of Change from Baseline in ACT Total Score at Week 12 (Visit 4) (Hodges-Lehmann Approach) | Present the "Difference" and "95% CI" lines of "FF/VI vs. Usual ICS/LABA" section only. Footnotes as follows: "Note: The difference between treatment groups at Week 12 (Visit 4) was calculated using the Hodges-Lehmann approach." | Data Look [1]<br>SAC [2] |
| 2.9. | ITT | Non-Standard<br>EFF_T2 | Summary of the Statistical Analysis of Change from Baseline in ACT Total Score at Week 12 (Visit 4) (ANCOVA with WOCF) | Footnotes as follows: "Note: The analysis method was an ANCOVA model adjusted for randomised treatment, baseline ACT total score, gender, age and country. Note: Missing values at Week 12 (Visit 4) due to treatment withdrawal prior to this time point were replaced by worst post-randomisation value based on the worst observation carried forward (WOCF) method." | Data Look [1]<br>SAC [2] |
| 2.10. | ITT | Non-Standard<br>EFF_T3 | Summary of the Statistical Analysis of Change from Baseline in ACT Total Score at Week 12 (Visit 4), Adjusting for Seasonal Effect | Repeat on subsequent pages for<br>Season at randomisation = Summer,<br>Autumn, Winter. | Data Look [1]<br>SAC [2] |
| 2.11. | PP | Non-Standard<br>EFF_T3 | Summary of the Statistical Analysis of Change from Baseline in ACT Total Score at Week 12 (Visit 4), Adjusting for Seasonal Effect Per Protocol Population | Repeat on subsequent pages for Season at randomisation = Summer, Autumn, Winter. | SAC [2] |
| 2.12. | ITT | Non-Standard<br>EFF_T1 | Summary of Change from Baseline in ACT Total Score, FF/VI Versus the Subset of Usual ICS/LABA Subjects Prescribed FP/S at Randomisation | | Data Look [1]<br>SAC [2] |

| Efficacy | Efficacy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.13. | ITT | Non-Standard<br>EFF_T2 | Summary of the Statistical Analysis of Change from Baseline in ACT Total Score at Week 12 (Visit 4), FF/VI Versus the Subset of Usual ICS/LABA Subjects Prescribed FP/S at Randomisation | Output only to be produced if ≥25% of Usual ICS/LABA patients are prescribed FP/S at randomisation. | Data Look [1]<br>SAC [2] |
| 2.14. | ITT | Non-Standard<br>EFF_T1 | Summary of Change from Baseline in ACT Total Score, FF/VI<br>Versus the Subset of Usual ICS/LABA Subjects Prescribed<br>BUD/F at Randomisation | | SAC [2] |
| 2.15. | ITT | Non-Standard<br>EFF_T2 | Summary of the Statistical Analysis of Change from Baseline in ACT Total Score at Week 12 (Visit 4), FF/VI Versus the Subset of Usual ICS/LABA Subjects Prescribed BUD/F at Randomisation | Output only to be produced if ≥75% of Usual ICS/LABA patients are prescribed BUD/F at randomisation. | SAC [2] |
| 2.16. | ITT | Non-Standard<br>EFF_T1S | Summary of Change from Baseline in ACT Total Score by Country | | Data Look [1]<br>SAC [2] |
| 2.17. | ITT | Non-Standard<br>EFF_T2S | Summary of the Statistical Analysis of Change from Baseline in ACT Total Score at Week 12 (Visit 4) by Country | | Data Look [1]<br>SAC [2] |
| 2.18. | ITT | Non-Standard<br>EFF_T1S | Summary of Change from Baseline in ACT Total Score by<br>Number of Severe Asthma Exacerbations in the Previous Year<br>Prior to Randomisation | | SAC [2] |

| Efficacy | Efficacy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.19. | ІТТ | Non-Standard<br>EFF_T2S | Summary of the Statistical Analysis of Change from Baseline in ACT Total Score at Week 12 (Visit 4) by Number of Severe Asthma Exacerbations in the Previous Year Prior to Randomisation | First footnote as follows: "Note: The analysis method was an MMRM adjusted for randomised treatment, visit (Week 6 and Week 12), baseline ACT total score, baseline ACT total score-by-visit interaction, gender, age, country, number of severe asthma exacerbations in the previous year prior to randomisation, two- and three- way interactions between randomised treatment, visit and number of severe asthma exacerbations in the previous year prior to randomisation, and patient fitted as a random factor." | SAC [2] |
| 2.20. | ITT | Non-Standard<br>EFF_T1S | Summary of Change from Baseline in ACT Total Score by Smoking Status at Baseline | | SAC [2] |
| 2.21. | ITT | Non-Standard<br>EFF_T2S | Summary of the Statistical Analysis of Change from Baseline in ACT Total Score at Week 12 (Visit 4) by Smoking Status at Baseline | First footnote as follows: "Note: The analysis method was an MMRM adjusted for randomised treatment, visit (Week 6 and Week 12), baseline ACT total score, baseline ACT total score-by-visit interaction, gender, age, country, smoking status at baseline, two- and three- way interactions between randomised treatment, visit and smoking status at baseline, and patient fitted as a random factor." | SAC [2] |
| 2.22. | ITT | Non-Standard<br>EFF_T1S | Summary of Change from Baseline in ACT Total Score by Age Group | | SAC [2] |

| Efficacy | Efficacy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.23. | ІТТ | Non-Standard<br>EFF_T2S | Summary of the Statistical Analysis of Change from Baseline in ACT Total Score at Week 12 (Visit 4) by Age Group | First footnote as follows: "Note: The analysis method was an MMRM adjusted for randomised treatment, visit (Week 6 and Week 12), baseline ACT total score, baseline ACT total score-by-visit interaction, gender, country, age group, two- and three- way interactions between randomised treatment, visit and age group, and patient fitted as a random factor." | SAC [2] |
| 2.24. | ITT | Non-Standard<br>EFF_T1S | Summary of Change from Baseline in ACT Total Score by Gender | | SAC [2] |
| 2.25. | ITT | Non-Standard<br>EFF_T2S | Summary of the Statistical Analysis of Change from Baseline in ACT Total Score at Week 12 (Visit 4) by Gender | First footnote as follows: "Note: The analysis method was an MMRM adjusted for randomised treatment, visit (Week 6 and Week 12), baseline ACT total score, baseline ACT total score-by-visit interaction, gender, age, country, two- and three- way interactions between randomised treatment, visit and gender, and patient fitted as a random factor." | SAC [2] |

| Efficac | Efficacy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Change | from Baseline | in ACT Total Sco | re at Week 24 (Visit 6) | | |
| 2.26. | ІТТ | Non-Standard<br>EFF_T2 | Summary of the Statistical Analysis of Change from Baseline in ACT Total Score at Week 24 (Visit 6) | First footnote as follows: "Note: The analysis method was an MMRM adjusted for randomised treatment, visit (Week 6, Week 12, Week 18 and Week 24), baseline ACT total score, randomised treatment-by-visit interaction, baseline ACT total score-by-visit interaction, gender, age, country and patient fitted as a random factor." | Data Look [1]<br>SAC [2] |
| 2.27. | PP | Non-Standard<br>EFF_T2 | Summary of the Statistical Analysis of Change from Baseline in ACT Total Score at Week 24 (Visit 6) Per Protocol Population | First footnote as follows: "Note: The analysis method was an MMRM adjusted for randomised treatment, visit (Week 6, Week 12, Week 18 and Week 24), baseline ACT total score, randomised treatment-by-visit interaction, baseline ACT total score-by-visit interaction, gender, age, country and patient fitted as a random factor." | SAC [2] |
| 2.28. | ІТТ | Non-Standard<br>EFF_T2 | Summary of the Statistical Analysis of Change from Baseline in ACT Total Score at Week 24 (Visit 6) (ANCOVA with LOCF) | Footnotes as follows: "Note: The analysis method was an ANCOVA model adjusted for randomised treatment, baseline ACT total score, gender, age and country. Note: Missing values at Week 24 (Visit 6) were replaced by last available post-randomization value based on the last observation carried forward (LOCF) method." | SAC [2] |

| Efficacy | Efficacy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.29. | ΙΤΤ | Non-Standard<br>EFF_T2 | Summary of the Statistical Analysis of Change from Baseline in ACT Total Score at Week 24 (Visit 6) (Multiple Imputation – Missing at Random Approach) | Footnotes as follows: "Note: Missing values post- randomisation were imputed using multiple imputation methods based on pattern mixture models. Note: Each imputed data set was analysed using an ANCOVA model at Week 24 (Visit 6) adjusted for randomised treatment, baseline ACT total score, gender, age and country and the resulting treatment differences and their standard errors combined using Rubin's rules." | SAC [2] |
| 2.30. | ΙΠ | Non-Standard<br>EFF_T2 | Summary of the Statistical Analysis of Change from Baseline in ACT Total Score at Week 24 (Visit 6) (Multiple Imputation – Copy Differences from Reference Approach) | Footnotes as follows: "Note: Missing values post- randomisation were imputed using multiple imputation methods based on pattern mixture models. Note: Each imputed data set was analysed using an ANCOVA model at Week 24 (Visit 6) adjusted for randomised treatment, baseline ACT total score, gender, age and country and the resulting treatment differences and their standard errors combined using Rubin's rules." | SAC [2] |

| Efficacy | Efficacy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.31. | ITT | Non-Standard<br>EFF_T2 | Summary of the Statistical Analysis of Change from Baseline in ACT Total Score at Week 24 (Visit 6) (Hodges-Lehmann Approach) | Present the "Difference" and "95% CI" lines of "FF/VI vs. Usual ICS/LABA" section only. Footnotes as follows: "Note: The difference between treatment groups at Week 24 (Visit 6) was calculated using the Hodges-Lehmann approach." | SAC [2] |
| 2.32. | ІТТ | Non-Standard<br>EFF_T2 | Summary of the Statistical Analysis of Change from Baseline in ACT Total Score at Week 24 (Visit 6) (ANCOVA with WOCF) | Footnotes as follows: "Note: The analysis method was an ANCOVA model adjusted for randomised treatment, baseline ACT total score, gender, age and country. Note: Missing values at Week 24 (Visit 6) due to treatment withdrawal prior to this time point were replaced by worst post-randomisation value based on the worst observation carried forward (WOCF) method." | SAC [2] |
| 2.33. | ITT | Non-Standard<br>EFF_T3 | Summary of the Statistical Analysis of Change from Baseline in ACT Total Score at Week 24 (Visit 6), Adjusting for Seasonal Effect | First footnote as follows: "Note: The analysis method was an MMRM adjusted for randomised treatment, visit (Week 6, Week 12, Week 18 and Week 24), baseline ACT total score, baseline ACT total score, baseline ACT total score-by-visit interaction, gender, age, country, season at randomisation, two-and three- way interactions between randomised treatment, visit and season at randomisation, and patient fitted as a random factor." | SAC [2] |

| Efficacy | Efficacy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.34. | PP | Non-Standard<br>EFF_T3 | Summary of the Statistical Analysis of Change from Baseline in ACT Total Score at Week 24 (Visit 6), Adjusting for Seasonal Effect Per Protocol Population | First footnote as follows: "Note: The analysis method was an MMRM adjusted for randomised treatment, visit (Week 6, Week 12, Week 18 and Week 24), baseline ACT total score, baseline ACT total score, baseline ACT total score-by-visit interaction, gender, age, country, season at randomisation, two-and three- way interactions between randomised treatment, visit and season at randomisation, and patient fitted as a random factor." | SAC [2] |
| 2.35. | ITT | Non-Standard<br>EFF_T2 | Summary of the Statistical Analysis of Change from Baseline in ACT Total Score at Week 24 (Visit 6), FF/VI Versus the Subset of Usual ICS/LABA Subjects Prescribed FP/S at Randomisation | Output only to be produced if ≥25% of Usual ICS/LABA patients are prescribed FP/S at randomisation. First footnote as follows: "Note: The analysis method was an MMRM adjusted for randomised treatment, visit (Week 6, Week 12, Week 18 and Week 24), baseline ACT total score, randomised treatment-by-visit interaction, baseline ACT total score-by-visit interaction, gender, age, country and patient fitted as a random factor." | SAC [2] |

| Efficacy | Efficacy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.36. | ITT | Non-Standard<br>EFF_T2 | Summary of the Statistical Analysis of Change from Baseline in ACT Total Score at Week 12 (Visit 4), FF/VI Versus the Subset of Usual ICS/LABA Subjects Prescribed BUD/F at Randomisation | Output only to be produced if ≥25% of Usual ICS/LABA patients are prescribed BUD/F at randomisation. First footnote as follows: "Note: The analysis method was an MMRM adjusted for randomised treatment, visit (Week 6, Week 12, Week 18 and Week 24), baseline ACT total score, randomised treatment-by-visit interaction, baseline ACT total score-by-visit interaction, gender, age, country and patient fitted as a random factor." | SAC [2] |
| 2.37. | ІТТ | Non-Standard<br>EFF_T2S | Summary of the Statistical Analysis of Change from Baseline in ACT Total Score at Week 24 (Visit 6) by Country | First footnote as follows: "Note: The analysis method was an MMRM adjusted for randomised treatment, visit (Week 6, Week 12, Week 18 and Week 24), baseline ACT total score, baseline ACT total score, by-visit interaction, gender, age, country, two- and three- way interactions between randomised treatment, visit and country, and patient fitted as a random factor." | SAC [2] |
| Correct | Correct Use of Inhaler Device | | | | |
| 2.38. | ITT | Non-Standard<br>EFF_T4 | Summary of Inhaler Device Use Errors | Repeat on subsequent pages for Visit = Week 12 and Week 24. "Number of patients using" line will provide the denominators for each section's percentages. | Data Look [1]<br>SAC [2] |

| Efficacy | Efficacy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.39. | PP | Non-Standard<br>EFF_T4 | Summary of Inhaler Device Use Errors<br>Per Protocol Population | Repeat on subsequent pages for Visit = Week 12 and Week 24. "Number of patients using" line will provide the denominators for each section's percentages. | SAC [2] |
| 2.40. | ITT | Non-Standard<br>EFF_T5 | Summary of Correct Use of Inhaler Device | | Data Look [1]<br>SAC [2] |
| 2.41. | PP | Non-Standard<br>EFF_T5 | Summary of Correct Use of Inhaler Device<br>Per Protocol Population | | SAC [2] |
| 2.42. | ITT | Non-Standard<br>EFF_T6 | Summary of the Statistical Analysis of Correct Use of Inhaler<br>Device at Week 12 (Visit 4) and at Week 24 (Visit 6)<br>Independently of the Use at Week 12 (Visit 4) | | Data Look [1]<br>SAC [2] |
| 2.43. | PP | Non-Standard<br>EFF_T6 | Summary of the Statistical Analysis of Correct Use of Inhaler<br>Device at Week 12 (Visit 4) and at Week 24 (Visit 6)<br>Independently of the Use at Week 12 (Visit 4)<br>Per Protocol Population | | SAC [2] |
| Lung F | unction Tests | | | | |
| 2.44. | ITT | Non-Standard<br>EFF_T1 | Summary of Change from Baseline in Lung Function Tests | Present an additional column to the left of "Visit", labelled "Test" with values "Trough (Pre-dose) FEV1" and "Trough (Pre-dose) Percent Predicted FEV1" to allow presentation of results by Test. Present the following visits: Day 0, Week 12, Change from Baseline at Week 12, Early Withdrawal and Change from Baseline at Early Withdrawal. | Data Look [1]<br>SAC [2] |

| Efficacy | Efficacy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.45. | ITT | Non-Standard<br>EFF_T2 | Summary of the Statistical Analysis of Change from Baseline in Trough (Pre-dose) FEV1 at Week 12 (Visit 4) | Footnote as follows: "Note: The analysis method was an ANCOVA model adjusted for randomised treatment, baseline trough (pre-dose) FEV1, gender, age and country." | Data Look [1]<br>SAC [2] |
| Subject | s Who Have Ei | ther an ACT Total | Score >= 20 or >= 3 Point Increase from Baseline in ACT Total | Score | |
| 2.46. | ITT | Non-Standard<br>EFF_T7 | Summary of Percentage of Subjects Who Have Either an ACT Total Score >= 20 or >= 3 Point Increase from Baseline in ACT Total Score | Repeat for Visit = Week 18, Week 24, Early Withdrawal. | Data Look [1]<br>SAC [2] |
| 2.47. | ІТТ | Non-Standard<br>EFF_T6 | Summary of the Statistical Analysis of Percentage of Subjects Who Have Either an ACT Total Score >= 20 or >= 3 Point Increase from Baseline in ACT Total Score at Week 12 (Visit 4) and Week 24 (Visit 6) | Replace "With correct use [1]" with "Responder [1]" and "Without correct use" with "Non-Responder". Footnotes as follows: "[1] Responder is defined as an ACT total score >= 20 or >= 3 point increase from baseline in ACT total score at that visit. Note: The analysis method was logistic regression adjusted for randomised treatment, baseline ACT total score, baseline ACT total score squared, gender, age and country." | SAC [2] |

| Efficac | Efficacy: Tables | | | | | | |
|---|---|---|---|---|---|--|--|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] | | |
| Individ | ual ACT Questi | on Scores | | | | | |
| 2.48. | ITT | Non-Standard<br>EFF_T8 | Summary of Individual ACT Question Scores | Repeat on subsequent pages for Question = 2. Shortness of breath, 3. Asthma symptoms woken up at night or earlier than usual, 4. Used rescue inhaler or nubuliser medication, 5. Asthma control. | Data Look [1]<br>SAC [2] | | |
| Compli | ance with Stud | y Medication | | | | | |
| 2.49. | ITT | Non-Standard<br>EFF_T9 | Summary of Compliance with Study Medication | | Data Look [1]<br>SAC [2] | | |
| 2.50. | PP | Non-Standard<br>EFF_T9 | Summary of Compliance with Study Medication Per Protocol Population | | SAC [2] | | |
| MARS- | A | | | | | | |
| 2.51. | ITT | Non-Standard<br>EFF_T10 | Summary of Use of Medication Adherence Report Scale for Asthma (MARS-A) During the Study | Repeat on subsequent pages for Visit = Week 12, Week 24 and Early Withdrawal. | Data Look [1]<br>SAC [2] | | |
| 2.52. | ITT | Non-Standard<br>EFF_T10S | Summary of Use of Medication Adherence Report Scale for Asthma (MARS-A) During the Study by Status of Patient in Relation to the Reminder Sent to French Centres | Repeat on subsequent pages for Visit = Week 12, Week 24 and Early Withdrawal, and for Status = Patients in France who had completed at least one MARS-A assessment prior to the reminder being implemented but also completed at least one MARS-A assessment after the reminder being implemented, Patients in France who had not completed any MARS-A assessments prior to the reminder being implemented, Patients in Germany. | Data Look [1]<br>SAC [2] | | |
| Efficacy | Efficacy: Tables | | | | | | | |
|---|---|---|---|---|---|--|--|--|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] | | | |
| Severe | On-Treatment | Asthma Exacerba | tions | | | | | |
| 2.53. | ITT | Non-Standard<br>EFF_T11 | Summary of Severe On-Treatment Asthma Exacerbations | | Data Look [1]<br>SAC [2] | | | |
| 2.54. | ITT | Non-Standard<br>EFF_T11S | Summary of Severe On-Treatment Asthma Exacerbations by Season | Repeat on subsequent pages for Season = Summer, Autumn, Winter. | Data Look [1]<br>SAC [2] | | | |
| 2.55. | ITT | Non-Standard<br>EFF_T12 | Summary of the Statistical Analysis of Severe On-Treatment Asthma Exacerbations | | Data Look [1]<br>SAC [2] | | | |
| 2.56. | ITT | Non-Standard<br>EFF_T13 | Summary of the Statistical Analysis of Time to First Severe On-<br>Treatment Asthma Exacerbation | | Data Look [1]<br>SAC [2] | | | |
| AQLQ( | 5) | | | | | | | |
| 2.57. | ІТТ | Non-Standard<br>EFF_T1 | Summary of Change from Baseline in AQLQ(S) Total Score and Domain Scores | Present an additional column to the left of "Visit", labelled "Domain" with values "Total Score", "Environmental Stimuli", "Symptoms", "Activity Limitations" and "Emotional Function" to allow presentation of results by Domain. Present the following visits: Day 0, Week 24, Change from Baseline at Week 24, Early Withdrawal and Change from Baseline at Early Withdrawal. | SAC [2] | | | |
| 2.58. | ITT | Non-Standard<br>EFF_T14 | Summary of Percentage of Subjects Who Have an Increase from Baseline of >=0.5 in AQLQ(S) Total Score and Domain Scores | Repeat on subsequent pages for<br>Domain = Environmental Stimuli,<br>Symptoms, Activity Limitations and<br>Emotional Function. | Data Look [1]<br>SAC [2] | | | |

| Efficacy | Efficacy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.59. | ІТТ | Non-Standard<br>EFF_T6 | Summary of the Statistical Analysis of Percentage of Subjects Who Have an Increase from Baseline of >=0.5 in AQLQ(S) Total Score and Environmental Stimuli Domain Score at Week 24 (Visit 6) | Replace "With correct use [1]" with "Responder [1]" and "Without correct use" with "Non-Responder". Do not display the "Visit" column. Footnotes as follows: "[1] Responder is defined as an increase from baseline of >= 0.5. Note: The analysis method was logistic regression adjusted for randomised treatment, baseline score, gender, age and country." | SAC [2] |
| EQ-5D- | 5L | | | | |
| 2.60. | ITT | Non-Standard<br>EFF_T15 | Summary of EQ-5D-5L Descriptive System Dimensions | Repeat on subsequent pages for Visit =<br>Early Withdrawal and for Dimension =<br>Mobility, Pain/Discomfort, Self-care,<br>Usual activities. | Data Look [1]<br>SAC [2] |
| 2.61. | ІТТ | Non-Standard<br>EFF_T6 | Summary of the Statistical Analysis of Proportion of Responders<br>According to EQ-5D-5L Descriptive System Dimensions at Week<br>24 (Visit 6) | Replace "With correct use [1]" with "Responder [1]" and "Without correct use" with "Non-Responder". Do not display the "Visit" column. Footnotes as follows: "[1] Responder is defined as a score of 1 ('no problems'). Note: The analysis method was logistic regression adjusted for randomised treatment, baseline EQ-5D-5L domain score, gender, age and country." | SAC [2] |

| Efficacy | Efficacy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.62. | ITT | Non-Standard<br>EFF_T1 | Summary of EQ-5D-5L Utility Score | Present the following visits: Day 0,<br>Week 24, Change from Baseline at<br>Week 24, Early Withdrawal and<br>Change from Baseline at Early<br>Withdrawal. | Data Look [1]<br>SAC [2] |
| 2.63. | ITT | Non-Standard<br>EFF_T2 | Summary of the Statistical Analysis of Change from Baseline in EQ-5D-5L Utility Score at Week 24 (Visit 6) | Footnote as follows: "Note: The analysis method was an ANCOVA model adjusted for randomised treatment, baseline EQ-5D-5L utility score, gender, age and country." | SAC [2] |
| 2.64. | ITT | Non-Standard<br>EFF_T1 | Summary of EQ-5D-5L Visual Analogue Scale (VAS) Score | Present the following visits: Day 0,<br>Week 24, Change from Baseline at<br>Week 24, Early Withdrawal and<br>Change from Baseline at Early<br>Withdrawal. | SAC [2] |
| 2.65. | ITT | Non-Standard<br>EFF_T2 | Summary of the Statistical Analysis of Change from Baseline in EQ-5D-5L Visual Analogue Scale (VAS) Score at Week 24 (Visit 6) | Footnote as follows: "Note: The analysis method was an ANCOVA model adjusted for randomised treatment, baseline EQ-5D-5L VAS score, gender, age and country." | SAC [2] |

| Efficacy | Efficacy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| PASAP | -Q | | | | |
| 2.66. | ІТТ | Non-Standard<br>EFF_T1 | Summary of PASAP-Q Scores | Present an additional column to the left of "Visit", labelled "Score" with values "Performance", "Convenience", "Overall Satisfaction", "Total Score" and "Willingness to Continue Using Inhaler" to allow presentation of results by Domain. Present the following visits: Week 12 and Early Withdrawal. Add the following footnotes: "Note: Performance, Convenience, Total Score, and Willingness to Continue Using Inhaler are expressed on a scale of 0 to 100. Note: Overall Satisfaction is expressed on a scale of 1 to 7." | SAC [2] |

HZA116492

# 10.15.7. Efficacy Figures

| Efficacy | Efficacy: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Change | from Baseline | in ACT Total Sco | re at Week 12 (Visit 4) | | |
| 2.1. | Ш | Non-Standard<br>EFF_F1 | Summary of Change from Baseline in ACT Total Score | Present "ACT Total Score" on y-axis and "Visit" on x-axis (Day 0, Week 6, Week 12, Week 18, Week 24). Present mean ACT Total Score ± SD separately for treatment group (FF/VI, Usual ICS/LABA) at each visit, connecting the means with a solid line. Distinguish the treatment groups by different line types. | Data Look [1]<br>SAC [2] |
| 2.2. | PP | Non-Standard<br>EFF_F1 | Summary of Change from Baseline in ACT Total Score<br>Per Protocol Population | Present "ACT Total Score" on y-axis and "Visit" on x-axis (Day 0, Week 6, Week 12, Week 18, Week 24). Present mean ACT Total Score ± SD separately for treatment group (FF/VI, Usual ICS/LABA) at each visit, connecting the means with a solid line. Distinguish the treatment groups by different line types. | SAC [2] |
| 2.3. | ITT | Non-Standard<br>EFF_F1 | Summary of Change from Baseline in ACT Total Score by Country | Present "ACT Total Score" on y-axis and "Visit" on x-axis (Day 0, Week 6, Week 12, Week 18, Week 24). Present mean ACT Total Score ± SD separately for treatment group (FF/VI, Usual ICS/LABA) at each visit, connecting the means with a solid line. Distinguish the treatment groups by different line types. | SAC [2] |

| Efficacy | Efficacy: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.4. | ITT/PP | Non-Standard<br>EFF_F2 | Summary of Primary and Sensitivity Analyses for Change from Baseline in ACT Total Score at Week 12 (Visit 4) | Present "Treatment difference" on the x-axis, and reverse axis so treatment difference increases from left to right. Replace "Ratio (95% CI)" with "Treatment Difference (95% CI)". Present lines for the following: Primary analysis (ITT), Primary analysis (PP), ANCOVA with LOCF (ITT), Multiple Imputation (Missing at Random) (ITT), Multiple Imputation (Copy Differences from Reference) (ITT), Hodges-Lehmann (ITT), ANCOVA with WOCF (ITT). | Data Look [1]<br>SAC [2] |
| 2.5. | ІТТ | Non-Standard<br>EFF_F3 | Summary of Interaction Tests for Change from Baseline in ACT Total Score at Week 12 (Visit 4) | Present "LS Mean Change" on the x-axis, and reverse axis so it increases from left to right. Replace "Ratio (95% CI)" with "LS Mean Change (95% CI)". Present the following subgroups: Country (France, Germany); Number of Severe Asthma Exacerbations in the Previous Year Prior to Randomisation (0, >= 1); Smoking Status at Baseline (Current Smokers, Former Smokers, Never Smoked); Age Group (18 – 50 Years Old, > 50 Years Old); Gender (Male, Female). | Data Look [1]<br>SAC [2] |

| Efficacy | Efficacy: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Change | from Baseline | in ACT Total Sco | ore at Week 24 (Visit 6) | | |
| 2.6. | ITT/PP | Non-Standard<br>EFF_F2 | Summary of Key Secondary and Sensitivity Analyses for Change from Baseline in ACT Total Score at Week 24 (Visit 6) | Present "Treatment difference" on the x-axis, and reverse axis so treatment difference increases from left to right. Replace "Ratio (95% CI)" with "Treatment Difference (95% CI)". Present lines for the following: Primary analysis (ITT), Primary analysis (PP), ANCOVA with LOCF (ITT), Multiple Imputation (Missing at Random) (ITT), Multiple Imputation (Copy Differences from Reference) (ITT), Hodges-Lehmann (ITT), ANCOVA with WOCF (ITT). | SAC [2] |
| Subject | ts Who Have Ei | ther an ACT Total | Score >= 20 or >= 3 Point Increase from Baseline in ACT Total | Score | |
| 2.7. | ITT | Non-Standard<br>EFF_F4 | Summary of Percentage of Subjects Who Have Either an ACT Total Score >= 20 or >= 3 Point Increase from Baseline in ACT Total Score | Present "Percent of Subjects (%)" on y-axis and "Visit" on x-axis (Week 6, Week 12, Week 18, Week 24, Early Withdrawal). For each visit, present 3 vertical bars distinguished by fill pattern (similar to non-standard EFF_F6). Each bar represents: "ACT Total Score >= 20 or >= 3 Point Increase from Baseline in ACT Total Score", "ACT Total Score >= 20" and ">= 3 Point Increase from Baseline in ACT Total Score" respectively and should be labelled as such on the legend. | Data Look [1]<br>SAC [2] |

| Efficacy | Efficacy: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Compli | ance with Stud | y Medication | | | |
| 2.8. | ITT | Non-Standard<br>EFF_F5 | Box Plot of Compliance with Study Medication | Label y-axis title as "Compliance (%)", maximum of y-axis may be > 100%. | Data Look [1]<br>SAC [2] |
| MARS- | A | | | | |
| 2.9. | ITT | Non-Standard<br>EFF_F6 | Histogram of the Questions and Answers of the MARS-A Questionnaire | Repeat on subsequent pages for Visit = Week 24, Week 52 and Early Withdrawal; and for Randomised Treatment = FF/VI. | Data Look [1]<br>SAC [2] |
| 2.10. | ITT | Non-Standard<br>EFF_F6 | Histogram of the Questions and Answers of the MARS-A Questionnaire by Status of Patient in Relation to the Reminder Sent to French Centres | Present bylines and footnotes per<br>"Repeat for" programming note on<br>shell. | SAC [2] |
| 2.11. | ITT | Non-Standard<br>EFF_F7 | Histogram of the Distribution of MARS-A Scores During the Study | Repeat on subsequent pages for Visit = Week 52 and Early Withdrawal. | Data Look [1]<br>SAC [2] |
| 2.12. | ITT | Non-Standard<br>EFF_F7 | Histogram of the Distribution of MARS-A Scores During the Study by Status of Patient in Relation to the Reminder Sent to French Centres | Present bylines and footnotes per<br>"Repeat for" programming note on<br>shell. | SAC [2] |
| Severe | On-Treatment | Asthma Exacerba | tions | | |
| 2.13. | ITT | Non-Standard<br>EFF_F8 | Box Plot of Severe On-Treatment Asthma Exacerbation Rates<br>Adjusted for Exposure to Treatment | | Data Look [1]<br>SAC [2] |
| 2.14. | ITT | Non-Standard<br>EFF_F9 | Kaplan-Meier Plot of Time to First Severe On-Treatment Asthma Exacerbation | Display increments of 6 weeks on the x-axis, up to the maximum exposure (e.g. 0, 6, 12, 18, 24, 30). | Data Look [1]<br>SAC [2] |

HZA116492

# 10.15.8. Safety Tables

| Safety | Safety : Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| SAEs and ADRs | | | | | |
| 3.1. | Safety | Non-Standard<br>SAFE_T1 | On-Treatment Serious Adverse Events and Adverse Drug Reactions Overview | Based on IDSL standard template AE13. | Data Look [1]<br>SAC [2] |
| 3.2. | Safety | AE1 | Summary of On-Treatment Non-Serious Adverse Drug Reactions | | SAC [2] |
| 3.3. | Safety | AE1 | Summary of On-Treatment Serious Adverse Drug Reactions | | SAC [2] |
| 3.4. | Safety | AE1 | Summary of On-Treatment Adverse Drug Reactions | | Data Look [1]<br>SAC [2] |
| 3.5. | Safety | AE1 | Summary of On-Treatment Serious Adverse Events | | Data Look [1]<br>SAC [2] |
| 3.6. | Safety | AE1 | Summary of On-Treatment or Post-Treatment Serious Adverse<br>Events and Adverse Drug Reactions Leading to Permanent<br>Discontinuation of Study Drug or Withdrawal from the Study | | SAC [2] |
| 3.7. | Safety | AE1 | Summary of On-Treatment or Post-Treatment Serious Adverse<br>Events Leading to Permanent Discontinuation of Study Drug or<br>Withdrawal from the Study | | SAC [2] |
| 3.8. | Safety | AE1 | Summary of On-Treatment or Post-Treatment Adverse Drug<br>Reactions Leading to Permanent Discontinuation of Study Drug<br>or Withdrawal from the Study | | SAC [2] |
| 3.9. | Safety | AE1 | Summary of Most Frequent On-Treatment Non-Serious Adverse Drug Reactions, Reported by 1% or More of Subjects in Any Treatment Group | | SAC [2] |

| Safety | Safety : Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| SAEs a | nd ADRs of Sp | ecial Interest | | | |
| 3.10. | Safety | Non-Standard<br>SAFE_T2 | Summary of On-Treatment Non-Serious Adverse Drug<br>Reactions of Special Interest | Based on IDSL standard template AE1. | Data Look [1]<br>SAC [2] |
| 3.11. | Safety | Non-Standard<br>SAFE_T2 | Summary of On-Treatment Serious Adverse Drug Reactions of Special Interest | Based on IDSL standard template AE1. | SAC [2] |
| 3.12. | Safety | Non-Standard<br>SAFE_T2 | Summary of On-Treatment Adverse Drug Reactions of Special Interest | Based on IDSL standard template AE1. | SAC [2] |
| 3.13. | Safety | Non-Standard<br>SAFE_T2 | Summary of On-Treatment Serious Adverse Events of Special Interest | Based on IDSL standard template AE1. | SAC [2] |
| Fatal S | AEs and ADRs | | | | |
| 3.14. | Safety | AE1 | Summary of On-Treatment Fatal Serious Adverse Events | | SAC [2] |
| 3.15. | Safety | AE1 | Summary of On-Treatment Fatal Serious Adverse Drug Reactions | | SAC [2] |
| 3.16. | Safety | Non-Standard<br>SAFE_T2 | Summary of On-Treatment Fatal Serious Adverse Events of Special Interest | Based on IDSL standard template AE1. | SAC [2] |
| Non-Fa | tal SAEs and A | DRs | | | |
| 3.17. | Safety | AE1 | Summary of On-Treatment Non-Fatal Serious Adverse Events | | SAC [2] |
| 3.18. | Safety | Non-Standard<br>SAFE_T2 | Summary of On-Treatment Non-Fatal Serious Adverse Events of Special Interest | Based on IDSL standard template AE1. | SAC [2] |
| Top Te | n Most Commo | nly Reported ADF | Rs . | | |
| 3.19. | Safety | Non-Standard<br>SAFE_T3 | Top Ten Most Commonly Reported On-Treatment Adverse Drug<br>Reactions Per Treatment Group | Present the ten most frequent preferred terms in Usual ICS/LABA, and the ten most frequent in FF/VI (do not use percentages to determine "most frequent") | Data Look [1]<br>SAC [2] |

| Safety : | Safety: Tables | | | |
|---|---|---|---|---|
| No. | No. Population IDSL / TST ID / Example Shell Title Programming Notes Delive [Prior | | | |
| Vital Sig | gns | | | |
| 3.20. | Safety | VS1 | Summary of Vital Signs | SAC [2] |
| 3.21. | Safety | VS2 | Summary of Vital Sign Data Outside Clinical Concern Range | SAC [2] |

HZA116492

# 10.15.9. Safety Figures

| Safety : | Safety : Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Benefit | :Risk | | | | |
| 3.1. | ITT/Safety | Non-Standard<br>SAFE_F1 | Summary of Benefit:Risk for FF/VI vs. Usual ICS/LABA | | Data Look [1]<br>SAC [2] |

HZA116492

# 10.15.10. ICH Listings

| ICH:L | istings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Study I | Population | | | | |
| 1. | ITT | ES2 | Reasons for Study Withdrawal | | SAC [2] |
| 2. | ITT | TA1 | Randomised and Actual Treatments | For subjects with multiple 'actual' treatments, present in the order the treatments were received. | SAC [2] |
| 3. | ITT | IE3 | Subjects with Inclusion, Exclusion or Randomisation Criteria Deviations | | SAC [2] |
| 4. | ITT | DM2 | Demographic Characteristics | | SAC [2] |
| 5. | ITT | DM9 | Race | | SAC [2] |
| Advers | se Events | | | | |
| 6. | Safety | AE7 | Subject Numbers for Individual Serious Adverse Events and Non-Serious Adverse Drug Reactions | | SAC [2] |
| 7. | Safety | AE8 | All Serious Adverse Events and Non-Serious Adverse Drug Reactions | | SAC [2] |
| 8. | Safety | AE8 | Fatal Serious Adverse Events | | SAC [2] |
| 9. | Safety | AE8 | Serious Adverse Events Leading to Permanent Discontinuation of Study Drug or Withdrawal from the Study | | SAC [2] |
| 10. | Safety | AE8 | Non-Serious Adverse Drug Reactions Leading to Permanent Discontinuation of Study Drug or Withdrawal from the Study | | SAC [2] |
| 11. | Safety | AE7 | Subject Numbers for Individual Serious Adverse Events and Non-Serious Adverse Drug Reactions | | SAC [2] |

HZA116492

# 10.15.11. Non-ICH Listings

| Non-IC | H : Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Study F | opulation | | | • | |
| 12. | ASE | Non-Standard POP_L1 | Subjects Screened but Not in the Intent-to-Treat Population | | SAC [2] |
| 13. | ITT | Non-Standard<br>POP_L2 | Reasons for Important Protocol Deviations | | SAC [2] |
| 14. | ITT | MH3 | Medical Conditions | | SAC [2] |
| 15. | ITT | Non-Standard<br>POP_L3 | Asthma History | | SAC [2] |
| 16. | ITT | Non-Standard<br>POP_L4 | Smoking History | | SAC [2] |
| 17. | ITT | CM3 | Concomitant Medications | Only include medications included in pre-treatment and on-treatment summary tables. | SAC [2] |
| 18. | ITT | CM6 | Relationship between Ingredient and Verbatim Text | | SAC [2] |
| 19. | ITT | Non-Standard<br>POP_L5 | Exposure to Study Medication | Repeat on subsequent pages for<br>Treatment = FF/VI, and use GSK drug<br>synonym as drug name. | SAC [2] |
| Efficac | у | | | | |
| 20. | ITT | Non-Standard<br>EFF_L1 | ACT Scores | Repeat on subsequent pages for Treatment = FF/VI. | SAC [2] |
| 21. | ITT | Non-Standard<br>EFF_L2 | Inhaler Device Use | Repeat on subsequent pages for<br>Treatment = FF/VI. | SAC [2] |
| 22. | ITT | Non-Standard<br>EFF_L3 | Lung Function Tests | Repeat on subsequent pages for Treatment = FF/VI. | SAC [2] |

| Non-IC | H : Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 23. | ITT | Non-Standard<br>EFF_L4 | Medication Adherence Report Scale for Asthma (MARS-A)<br>Scores | Repeat on subsequent pages for<br>Treatment = FF/VI. | SAC [2] |
| 24. | ITT | Non-Standard<br>EFF_L5 | Severe Asthma Exacerbations | Repeat on subsequent pages for<br>Treatment = FF/VI. | SAC [2] |
| 25. | ITT | Non-Standard<br>EFF_L6 | AQLQ(S) Scores | Repeat on subsequent pages for<br>Treatment = FF/VI. | SAC [2] |
| 26. | ITT | Non-Standard<br>EFF_L7 | EQ-5D-5L Descriptive System Dimension Scores | Repeat on subsequent pages for<br>Treatment = FF/VI. | SAC [2] |
| 27. | ITT | Non-Standard<br>EFF_L8 | PASAP-Q Scores | Repeat on subsequent pages for<br>Treatment = FF/VI. | SAC [2] |
| Safety | | | | | |
| 28. | Safety | Non-Standard<br>SAFE_L1 | AE Terms of Special Interest | The AE special interest dataset and the AE SMQ dataset will be set together in order to report this table and all the subgroups that come from the AE SMQ dataset will be flagged with a [1]. | SAC [2] |
| 29. | Safety | VS4 | Vital Signs | | SAC [2] |
| 30. | Safety | Non-Standard<br>SAFE_L2 | Inhaler Device Malfunctions | | SAC [2] |
| Liver C | hemistry | | | | |
| 31. | Safety | LIVER5 | Liver Event Results and Time of Event Relative to Treatment | | SAC [2] |
| 32. | Safety | LIVER6 | Liver Event Information for RUCAM Score | | SAC [2] |
| 33. | Safety | LIVER7 | Liver Biopsy Details | | SAC [2] |
| 34. | Safety | LIVER8 | Liver Imaging Details | | SAC [2] |

HZA116492

# 10.16. Appendix 16: Example Mock Shells for Data Displays

# 10.16.1. Study Population Table Shells

Example : POP\_T1 Protocol : HZA116492

Population : All Subjects Enrolled


Table 1.xx Summary of Subject Populations

| Population | Usual ICS/LABA | FF/VI | Total |
|-----------------------------|----------------|-----------|-----------|
| All Subjects Enrolled (ASE) | | | XXX |
| Randomised | XXX | XXX | XXX |
| Intent-to-Treat (ITT) | xxx (xx%) | xxx (xx%) | xxx (xx%) |
| Per Protocol (PP) | xxx (xx%) | xxx (xx%) | xxx (xx%) |
| Safety | xxx (xx%) | xxx (xx%) | xxx (xx%) |

ASE: All subjects screened and for whom a record exists on the study database.

ITT: All randomised subjects having received at least one dose of the prescription of study medication (FF/VI or Usual ICS/LABA).

PP: All ITT subjects who without any protocol deviations excluding them from this population.

Safety. All randomised subjects having received at least one dose of the prescription of study medication (FF/VI or Usual ICS/LABA).

Note: The randomised summary is not a defined population and consists of all subjects who were randomised and given a randomisation number.

Programming Note: randomised population line will provide the denominators for the ITT, PP and Safety percentages.

HZA116492

Example Protocol : POP\_T2 : HZA116492


Population : Intent-to-Treat

Table 1.xx Summary of Attendance at Each Clinic Visit

| | Usual ICS/LABA<br>(N=xxx) | FF/VI<br>(N=xxx) | Total<br>(N=xxx) |
|---|---|---|---|
| Visit 1: Screening | xxx (xx%) | xxx (xx%) | xxx (xx%) |
| Visit 1: Goldening Visit 2: Randomisation (Day 0) | xxx (xx%) | xxx (xx%) | xxx (xx%) |
| Visit 3: Week 6 | xxx (xx%) | xxx (xx%) | xxx (xx%) |
| Visit 4: Week 12 | xxx (xx%) | xxx (xx%) | xxx (xx%) |
| Visit 5: Week 18 | xxx (xx%) | xxx (xx%) | xxx (xx%) |
| Visit 6: Week 24 | xxx (xx%) | xxx (xx%) | xxx (xx%) |
| Early Withdrawal | xxx (xx%) | xxx (xx%) | xxx (xx%) |

Note: Weeks 6 and 18 are telephone contacts.

HZA116492

Example : POP\_T3 Protocol : HZA116492


Population : Intent-to-Treat

Table 1.xx Summary of Important Protocol Deviations

| | Usual ICS/LABA<br>(N=xxx) | FF/VI<br>(N=xxx) | Total<br>(N=xxx) |
|---|---|---|---|
| Any Important Protocol Deviation | xxx (xx%) | xxx (xx%) | xxx (xx%) |
| Reason 1 | xxx (xx%) | xxx (xx%) | xxx (xx%) |
| Reason 2 | xxx (xx%) | xxx (xx%) | xxx (xx%) |
| Reason 3 | xxx (xx%) | xxx (xx%) | xxx (xx%) |
| | xxx (xx%) | xxx (xx%) | xxx (xx%) |

Note: A subject may have more than one protocol deviation. Note: Includes any important deviation from the protocol.

# Repeat for:

Summary of Important Protocol Deviations Resulting in Exclusion from the PP Population (ITT Population)

HZA116492

Example Protocol : POP\_T4 : HZA116492


Population : Intent-to-Treat

Table 1.xx Summary of Asthma Duration at Baseline

| | Usual ICS/LABA<br>(N=xxx) | FF/VI<br>(N=xxx) | Total<br>(N=xxx) |
|---|---|---|---|
| | (14-7///) | (14-7/7/) | (14-222) |
| Duration of Asthma | | | |
| < 6 months | xxx (xx%) | xxx (xx%) | xxx (xx%) |
| >= 6 months to < 1 year | xxx (xx%) | xxx (xx%) | xxx (xx%) |
| >= 1 year to < 5 years | xxx (xx%) | xxx (xx%) | xxx (xx%) |
| >= 5 years to < 10 years | xxx (xx%) | xxx (xx%) | xxx (xx%) |
| >= 10 years | xxx (xx%) | xxx (xx%) | xxx (xx%) |
| Duration of Asthma (years): | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | X.XX | X.XX | X.XX |
| Median | XX.X | XX.X | XX.X |
| Min. | XX | XX | XX |
| Max. | XX | XX | Xx |

Repeat for: Summary of Asthma Duration at Baseline (PP Population)

HZA116492

Example : POP\_T5 Protocol : HZA116492


Protocol : HZA116492
Population : Intent-to-Treat

Table 1.xx Summary of Asthma Exacerbation History at Baseline

| | Usual ICS/LABA<br>(N=xxx) | FF/VI<br>(N=xxx) | Total<br>(N=xxx) |
|---|---|---|---|
| Did not require oral/systemic corticosteroids (not involving | | | |
| hospitalisation) | | | |
| n | XX | XX | XX |
| 0 | xx (xx%) | xx (xx%) | xx (xx%) |
| 1 | xx (xx%) | xx (xx%) | xx (xx%) |
| >1 | xx (xx%) | xx (xx%) | xx (xx%) |
| Required oral/systemic corticosteroids (not involving hospitalisation) | | | |
| n | XX | XX | XX |
| 0 | xx (xx%) | xx (xx%) | xx (xx%) |
| 1 | xx (xx%) | xx (xx%) | xx (xx%) |
| >1 | xx (xx%) | xx (xx%) | xx (xx%) |
| Required hospitalisation | | | |
| n | XX | XX | XX |
| 0 | xx (xx%) | xx (xx%) | xx (xx%) |
| 1 | xx (xx%) | xx (xx%) | xx (xx%) |
| >1 | xx (xx%) | xx (xx%) | xx (xx%) |

Note: Number of severe asthma exacerbations reported in the 12 months prior to Day 0.

HZA116492

Example : POP\_T5 Protocol : HZA116492


Protocol : HZA116492
Population : Intent-to-Treat

# Table 1.xx Summary of Asthma Exacerbation History at Baseline

| | Usual ICS/LABA<br>(N=xxx) | FF/VI<br>(N=xxx) | Total<br>(N=xxx) |
|---|---|---|---|
| Total number of exacerbations during the 12 months prior to randomisation | | | |
| n | XX | XX | XX |
| 0 | xx (xx%) | xx (xx%) | xx (xx%) |
| 1 | xx (xx%) | xx (xx%) | xx (xx%) |
| >1 | xx (xx%) | xx (xx%) | xx (xx%) |
| Number of exacerbations during the 12 months prior to randomisation | l | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | X.XX | X.XX | X.XX |
| Median | XX.X | XX.X | XX.X |
| Min. | XX | XX | XX |
| Max. | XX | XX | XX |

Note: Number of severe asthma exacerbations reported in the 12 months prior to Visit 2 (Day 0).

# Repeat for:

Summary of Asthma Exacerbation History at Baseline (PP Population)

HZA116492

Example : POP\_T6
Protocol : HZA116492
Population : Intent-to-Treat


# Table 1.xx Summary of Smoking History at Baseline

| | | Usual ICS/LABA<br>(N=xxx) | FF/VI<br>(N=xxx) | Total<br>(N=xxx) |
|---|---|---|---|---|
| History of Smoking Use | Current Smokers<br>Former Smokers<br>Never Smoked | xxx (xx%)<br>xxx (xx%)<br>xxx (xx%) | xxx (xx%)<br>xxx (xx%)<br>xxx (xx%) | xxx (xx%)<br>xxx (xx%)<br>xxx (xx%) |
| For Current and Former Smokers: | | | | |
| Years Smoked | n | XX | XX | XX |
| | Mean | XX.X | XX.X | XX.X |
| | SD | X.XX | X.XX | X.XX |
| | Median | XX.X | XX.X | XX.X |
| | Min. | XX | XX | XX |
| | Max. | XX | XX | XX |
| Cigarettes/Day | n | XX | XX | XX |
| , | Mean | XX.X | XX.X | XX.X |
| | SD | X.XX | X.XX | X.XX |
| | Median | XX.X | XX.X | XX.X |
| | Min. | XX | XX | XX |
| | Max. | XX | XX | XX |

<sup>[1]</sup> Smoking Pack Years = (Number of cigarettes smoked per day/20) x number of years smoked.

HZA116492

Example : POP\_T6
Protocol : HZA116492
Population : Intent-to-Treat


# Table 1.xx Summary of Smoking History at Baseline

| | | Usual ICS/LABA<br>(N=xxx) | FF/VI<br>(N=xxx) | Total<br>(N=xxx) |
|---|---|---|---|---|
| Smoking Pack Years[1] | | | | |
| Overall | n | XX | W | XX |
| Overall | n<br>Maan | | XX | |
| | Mean | XX.X | XX.X | XX.X |
| | SD | X.XX | X.XX | X.XX |
| | Median | XX.X | XX.X | XX.X |
| | Min. | XX | XX | XX |
| | Max. | XX | XX | XX |
| Current Smokers | n | XX | XX | XX |
| | Mean | XX.X | XX.X | XX.X |
| | SD | X.XX | X.XX | X.XX |
| | Median | XX.X | XX.X | XX.X |
| | Min. | XX | XX | XX |
| | Max. | XX | XX | XX |
| Former Smokers | n | XX | XX | XX |
| | Mean | XX.X | XX.X | XX.X |
| | SD | X.XX | X.XX | X.XX |
| | Median | XX.X | XX.X | XX.X |
| | Min. | XX | XX | XX |
| | Max. | | | |
| | IVIAX. | XX | XX | XX |

<sup>[1]</sup> Smoking Pack Years = (Number of cigarettes smoked per day/20) x number of years smoked. *Repeat for:* 

HZA116492

Summary of Smoking History at Baseline (PP Population)

HZA116492

Example : POP\_T7 Protocol : HZA116492


Population : Intent-to-Treat

# Table 1.xx Summary of Study Medication Dosage Modification

| Dosage Modification / Prescription | Usual ICS/LABA | FF/VI | Total |
|---|---|---|---|
| Treatment Path | (N=xxx) | (N=xxx) | (N=xxx) |
| Did Not Modify Dose During the Study<br>Modified Dose at Least Once During the Study | xxx (xx%)<br>xxx (xx%) | xxx (xx%)<br>xxx (xx%) | xxx (xx%)<br>xxx (xx%) |
| Randomised to FF/VI<br>FF/VI 92 mcg/22 mcg OD<br>FF/VI 92 mcg/22 mcg OD -> FF/VI 184 mcg/22 mcg OD | | xxx<br>xxx (xx%)<br>xxx (xx%) | xxx<br>xxx (xx%)<br>xxx (xx%) |
| Randomised to Usual ICS/LABA and Prescribed FP/S FP/S 250 mcg/50 mcg BID FP/S 250 mcg/50 mcg BID -> FP/S 500 mcg/50 mcg BID | xxx<br>xxx (xx%)<br>xxx (xx%) | | xxx<br>xxx (xx%)<br>xxx (xx%) |
| Randomised to Usual ICS/LABA and Prescribed BUD/F BUD/F 200 mcg/6 mcg BID (1 inh) BUD/F 200 mcg/6 mcg BID (1 inh) -> BUD/F 200 mcg/6 mcg BID (2 inh) BUD/F 200 mcg/6 mcg BID (1 inh) -> BUD/F 400 mcg/12 mcg BID (1 inh) BUD/F 200 mcg/6 mcg BID (2 inh) BUD/F 200 mcg/6 mcg BID (2 inh) -> BUD/F 400 mcg/12 mcg BID (1 inh) BUD/F 200 mcg/6 mcg BID (2 inh) -> BUD/F 400 mcg/12 mcg BID (2 inh) | xxx<br>xxx (xx%)<br>xxx (xx%)<br>xxx (xx%)<br>xxx (xx%)<br>xxx (xx%)<br>xxx (xx%) | xxx (xx%)<br>xxx (xx%)<br>xxx (xx%)<br>xxx (xx%)<br>xxx (xx%)<br>xxx (xx%) | xxx<br>xxx (xx%)<br>xxx (xx%)<br>xxx (xx%)<br>xxx (xx%)<br>xxx (xx%)<br>xxx (xx%) |

Note: 1 inh = 1 inhalation per dose, 2 inh = 2 inhalations per dose.

Note: Subjects randomised to FF/VI initiated treatment on 92 mcg/22 mcg OD and could increase to 184 mcg/22 mcg OD.

Note: Subjects randomised to Usual ICS/LABA and prescribed FP/S initiated treatment on 250 mcg/50 mcg BID and could increase to 500 mcg/50 mcg BID.

HZA116492

Note: Subjects randomised to Usual ICS/LABA and prescribed BUD/F could: initiate treatment on 200 mcg/6 mcg BID (1 inh) and increase to 200 mcg/6 mcg BID (2 inh) or 400 mcg/12 mcg BID (1 inh); or initiate on 200 mcg/6 mcg BID (2 inh) and modify to 400 mcg/12 mcg BID (1 inh) or increase to 400 mcg/12 mcg BID (2 inh).

HZA116492

Example : POP\_T8
Protocol : HZA116492


Protocol : HZA116492
Population : Intent-to-Treat

Table 1.xx
Summary of Extent of Exposure to Study Medication (Regardless of Modification to Study Medication Dosage)

| Overall | | Usual ICS/LABA<br>(N=xxx) | FF/VI<br>(N=xxx) |
|---|---|---|---|
| Exposure (days) [1] | n<br>Mean<br>SD<br>Median<br>Min.<br>Max. | XX<br>XX.X<br>X.XX<br>XX.X<br>XX | XX<br>XX.X<br>X.XX<br>XX.X<br>XX |
| Total Years Exposed (yrs) | | XX | xx |
| Range of Exposure (days) | <= 6 weeks<br><= 12 weeks<br><= 18 weeks<br><= 24 weeks<br>> 24 weeks | xxx (xx%)<br>xxx (xx%)<br>xxx (xx%)<br>xxx (xx%)<br>xxx (xx%) | xxx (xx%)<br>xxx (xx%)<br>xxx (xx%)<br>xxx (xx%)<br>xxx (xx%) |
| Subjects Exposed for six months (24 weeks ± 2 weeks) | | xxx (xx%) | xxx (xx%) |

<sup>[1]</sup> Exposure to study medication = treatment stop date – treatment start date + 1, regardless of dosage modification.

HZA116492

# Repeat for:

Summary of Summary of Extent of Exposure to Study Medication (up to First Modification to Study Medication Dosage) (ITT Population)
Footnote: "[1] Exposure to study medication = treatment stop date - treatment start date + 1."

HZA116492

Example : POP\_T9
Protocol : HZA116492
Population : Intent-to-Treat


Table 1.xx
Summary of Extent of Exposure to Study Medication by Medication and Dosage

| Medication/Dosage | Overall | | Usual ICS/LABA<br>(N=xxx) | FF/VI<br>(N=xxx) |
|---|---|---|---|---|
| FF/VI 92 mcg/22 mcg OD | Exposure (days) [1] | n<br>Mean<br>SD<br>Median<br>Min.<br>Max. | XX<br>XX.X<br>X.XX<br>XX.X<br>XX | XX<br>XX.X<br>X.XX<br>XX.X<br>XX |
| | Total Years Exposed (yrs) | | XX | xx |
| | Range of Exposure (days) | <= 6 weeks<br><= 12 weeks<br><= 18 weeks<br><= 24 weeks<br>> 24 weeks | xxx (xx%)<br>xxx (xx%)<br>xxx (xx%)<br>xxx (xx%)<br>xxx (xx%) | xxx (xx%)<br>xxx (xx%)<br>xxx (xx%)<br>xxx (xx%)<br>xxx (xx%) |
| | Subjects Exposed for six months (24 weeks ± 2 weeks) | | xxx (xx%) | xxx (xx%) |

<sup>[1]</sup> Exposure to study medication = treatment stop date – treatment start date + 1.

Programming note: repeat on subsequent pages for Medication/Dosage = FF/VI 184 mcg/22 mcg OD, FP/S 250 mcg/50 mcg BID, FP/S 500 mcg/50 mcg BID, BUD/F 200 mcg/6 mcg BID (1 inhalation per dose), BUD/F 200 mcg/6 mcg BID (2 inhalations per dose), BUD/F 400 mcg/12 mcg BID (1 inhalations per dose), BUD/F 400 mcg/12 mcg BID (2 inhalations per dose).

HZA116492

Example : POP\_T10
Protocol : HZA116492
Population : Intent-to-Treat


# Table 1.xx Summary of Number of Subjects by Subgroup

| | Usual ICS/LABA<br>(N=xxx) | FF/VI<br>(N=xxx) | Total<br>(N=xxx) |
|---|---|---|---|
| Country | | | |
| n | XXX | XXX | XXX |
| France | xxx (xx%) | xxx (xx%) | xxx (xx%) |
| Germany | xxx (xx%) | xxx (xx%) | xxx (xx%) |
| Number of Severe Asthma Exacerbations in the Previous Year Prior to Randomisation | | | |
| n | XXX | XXX | XXX |
| 0 | xxx (xx%) | xxx (xx%) | xxx (xx%) |
| >= 1 | xxx (xx%) | xxx (xx%) | xxx (xx%) |
| Smoking Status at Baseline | | | |
| n | XXX | XXX | XXX |
| Current smokers | xxx (xx%) | xxx (xx%) | xxx (xx%) |
| Former smokers | xxx (xx%) | xxx (xx%) | xxx (xx%) |
| Never smoked | xxx (xx%) | xxx (xx%) | xxx (xx%) |
| Age Group | | | |
| n | XXX | XXX | XXX |
| 18 – 50 years old | xxx (xx%) | xxx (xx%) | xxx (xx%) |
| > 50 years old | xxx (xx%) | xxx (xx%) | xxx (xx%) |

Note: Spring = March, April and May; Summer = June, July and August; Autumn = September, October and November; Winter = December, January and February.

HZA116492

Example : POP\_T10 Protocol : HZA116492

Population

: HZA116492  : Intent-to-Treat

Table 1.xx Summary of Number of Subjects by Subgroup

| | Usual ICS/LABA<br>(N=xxx) | FF/VI<br>(N=xxx) | Total<br>(N=xxx) |
|---|---|---|---|
| Gender | | | |
| n | XXX | XXX | XXX |
| Male | xxx (xx%) | xxx (xx%) | xxx (xx%) |
| Female | xxx (xx%) | xxx (xx%) | xxx (xx%) |
| Season at randomisation | | | |
| n | XXX | XXX | XXX |
| Spring | xxx (xx%) | xxx (xx%) | xxx (xx%) |
| Summer | xxx (xx%) | xxx (xx%) | xxx (xx%) |
| Autumn | xxx (xx%) | xxx (xx%) | xxx (xx%) |
| Winter | xxx (xx%) | xxx (xx%) | xxx (xx%) |

Note: Spring = March, April and May; Summer = June, July and August; Autumn = September, October and November; Winter = December, January and February.

HZA116492


# 10.16.2. Study Population Figure Shells

Example : POP\_F1
Protocol : HZA116492
Population : Intent-to-Treat

Figure 1.xx
Plot of Exposure to Study Medication (Regardless of Modification to Study Medication Dosage)



Programming note: display increments of 6 weeks on the x-axis, up to the maximum exposure (e.g. 0, 6, 12, 18, 24, 30).

HZA116492

# 10.16.3. Efficacy Table Shells

Example : EFF\_T1
Protocol : HZA116492
Population : Intent-to-Treat


Table 2.xx Summary of Change from Baseline in ACT Total Score

| Visit | | Usual ICS/LABA<br>(N=xxx) | FF/VI<br>(N=xxx) |
|---|---|---|---|
| Day 0 | n | XX | XX |
| | Mean | XX.X | XX.X |
| | SD | X.XX | X.XX |
| | Median | XX.X | XX.X |
| | Min. | XX | XX |
| | Max. | XX | XX |
| Week 6 | n | XX | XX |
| | Mean | XX.X | XX.X |
| | SD | X.XX | X.XX |
| | Median | XX.X | XX.X |
| | Min. | XX | XX |
| | Max. | XX | XX |
| Change from Baseline at Week 6 | n | XX | XX |
| | Mean | XX.X | XX.X |
| | SD | X.XX | X.XX |
| | Median | XX.X | XX.X |

HZA116492

Min. xx xx XX Max. xx xx

Programming note: repeat for Week 12, Change from Baseline at Week 18, Week 18, Change from Baseline at Week 24, Change from Baseline at Week 24, Change from Baseline at Early Withdrawal.

#### Repeat for:

Summary of Change from Baseline in ACT Total Score Per Protocol Population (PP Population)

Summary of Change from Baseline in Lung Function Tests (ITT Population)

Programming note: Present an additional column to the left of "Visit", labelled "Test" with values "Trough (Pre-dose) FEV1" and "Trough (Pre-dose) Percent Predicted FEV1" to allow presentation of results by Test. Present the following visits: Day 0, Week 12, Change from Baseline at Week 12, Early Withdrawal and Change from Baseline at Early Withdrawal.

Summary of Change from Baseline in AQLQ(S) Total Score and Domain Scores (ITT Population)

Programming note: Present an additional column to the left of "Visit", labelled "Domain" with values "Total Score", "Environmental Stimuli", "Symptoms", "Activity Limitations" and "Emotional Function" to allow presentation of results by Domain. Present the following visits: Day 0, Week 24, Change from Baseline at Week 24, Early Withdrawal and Change from Baseline at Early Withdrawal.

Summary of PASAP-Q Scores (ITT Population)

Programming note: Present an additional column to the left of "Visit", labelled "Score" with values "Performance", "Convenience", "Overall Satisfaction", "Total Score" and "Willingness to Continue Using Inhaler" to allow presentation of results by Domain. Present the following visits: Week 12 and Early Withdrawal.

Add the following footnotes:

"Note: Performance, Convenience, Total Score, and Willingness to Continue Using Inhaler are expressed on a scale of 0 to 100.

Note: Overall Satisfaction is expressed on a scale of 1 to 7."

Summary of EQ-5D-5L Utility Score (ITT Population)

Summary of EQ-5D-5L Visual Analogue Scale (VAS) Score (ITT Population)

Programming note: Present the following visits: Day 0, Week 24, Change from Baseline at Week 24, Early Withdrawal, Change from Baseline at Early Withdrawal.

HZA116492

Example Protocol : EFF\_T1S : HZA116492


Population : Intent-to-Treat

# Table 2.xx Summary of Change from Baseline in ACT Total Score by Country

Country: France

| Visit | | Usual ICS/LABA<br>(N=xxx) | FF/VI<br>(N=xxx) |
|---|---|---|---|
| Day 0 | n | XX | xx |
| , - | Mean | XX.X | XX.X |
| | SD | X.XX | X.XX |
| | Median | XX.X | XX.X |
| | Min. | XX | XX |
| | Max. | XX | XX |
| Week 6 | n | XX | XX |
| | Mean | XX.X | XX.X |
| | SD | X.XX | X.XX |
| | Median | XX.X | XX.X |
| | Min. | XX | XX |
| | Max. | XX | XX |
| Change from Baseline at Week 6 | n | XX | XX |
| | Mean | XX.X | XX.X |
| | SD | X.XX | X.XX |
| | Median | XX.X | XX.X |
| | Min. | XX | XX |
| | Max. | XX | XX |

HZA116492

Example : EFF\_T1S Protocol : HZA116492

Population : Intent-to-Treat


Table 2.xx Summary of Change from Baseline in ACT Total Score by Country

Country: Germany

| Visit | | Usual ICS/LABA<br>(N=xxx) | FF/VI<br>(N=xxx) |
|---|---|---|---|
| D 0 | | | |
| Day 0 | n | XX | XX |
| | Mean | XX.X | XX.X |
| | SD | X.XX | X.XX |
| | Median | XX.X | XX.X |
| | Min. | XX | XX |
| | Max. | XX | XX |
| Week 6 | n | XX | XX |
| | Mean | XX.X | XX.X |
| | SD | X.XX | X.XX |
| | Median | XX.X | XX.X |
| | Min. | XX | XX |
| | Max. | XX | XX |
| Change from Baseline at Week 6 | n | XX | XX |
| | Mean | XX.X | XX.X |
| | SD | X.XX | X.XX |
| | Median | XX.X | XX.X |
| | Min. | XX | XX |
| | Max. | XX | XX |
HZA116492

## Repeat for:

Summary of Change from Baseline in ACT Total Score by Number of Severe Asthma Exacerbations in the Previous Year Prior to Randomisation (ITT Population)
Number of Severe Asthma Exacerbations in the Previous Year Prior to Randomisation: 0

Number of Severe Asthma Exacerbations in the Previous Year Prior to Randomisation: >= 1

Summary of Change from Baseline in ACT Total Score by Smoking Status at Baseline (ITT Population)

Smoking Status at Baseline: Current Smokers Smoking Status at Baseline: Former Smokers Smoking Status at Baseline: Never Smoked

Summary of Change from Baseline in ACT Total Score by Age Group (ITT Population)

Age Group: 18 – 50 Years Old Age Group: > 50 Years Old

Summary of Change from Baseline in ACT Total Score by Gender (ITT Population)

Gender: Male Gender: Female

HZA116492

Example : EFF\_T2 Protocol : HZA116492

ZA116492 

Population : Intent-to-Treat

Table 2.xx

Summary of the Statistical Analysis of Change from Baseline in ACT Total Score at Week 12 (Visit 4)

| | Usual ICS/LABA<br>(N=xxx) | FF/VI<br>(N=xxx) |
|---|---|---|
| n<br>LS Mean Change (SE) | xx<br>xx.xx (x.xxx) | xx<br>xx.xx (x.xxx) |
| FF/VI vs. Usual ICS/LABA | | |
| Difference | | XX.X |
| 95% CI | | (xx.x, xx.x) |
| p-value | | X.XXX |

Note: The analysis method was an MMRM adjusted for randomised treatment, visit (Week 6 and Week 12), baseline ACT total score, randomised treatment-by-visit interaction, baseline ACT total score-by-visit interaction, gender, age, country and patient fitted as a random factor.

Note: The Restricted Maximum Likelihood (REML) estimation approach was used with a default covariance structure of unstructured.

Programming note: Should computational issues be encountered when using an unstructured covariance structure, other structures including AR1 and CS should be considered and the second footnote updated as appropriate. Should the distributional assumption of normality fail then the p-value from a model on the rank-transformed values should be presented and the following footnote added: "Note: the p-value presented was obtained from an MMRM on the rank-transformed values of change from baseline in ACT total score at Week 12 (Visit 4) with the same specification as the untransformed model."

HZA116492

#### Repeat for:

Summary of the Statistical Analysis of Change from Baseline in ACT Total Score at Week 12 (Visit 4) Per Protocol Population (PP Population)

Summary of the Statistical Analysis of Change from Baseline in ACT Total Score at Week 12 (Visit 4) (ANCOVA with LOCF) (ITT Population)

Programming note: Should the distributional assumption of normality fail then the p-value from a model on the rank-transformed values should be presented and the following footnote added: "Note: the p-value presented was obtained from an ANCOVA on the rank-transformed values of change from baseline in ACT total score at Week 12 (Visit 4) with the same specification as the untransformed model."

Footnotes as follows:

"Note: The analysis method was an ANCOVA model adjusted for randomised treatment, baseline ACT total score, gender, age and country.

Note: Missing values at Week 12 (Visit 4) were replaced by last available post-randomisation value based on the last observation carried forward (LOCF) method."

Summary of the Statistical Analysis of Change from Baseline in ACT Total Score at Week 12 (Visit 4) (Multiple Imputation – Missing at Random Approach) (ITT Population)

Summary of the Statistical Analysis of Change from Baseline in ACT Total Score at Week 12 (Visit 4) (Multiple Imputation – Copy Differences from Reference Approach) (ITT Population)

Programming note: Present the "FF/VI vs. Usual ICS/LABA" section only. Footnotes as follows:

"Note: Missing values post-randomisation were imputed using multiple imputation methods based on pattern mixture models.

Note: Each imputed data set was analysed using an ANCOVA model at Week 12 (Visit 4) adjusted for randomised treatment, baseline ACT total score, gender, age and country and the resulting treatment differences and their standard errors combined using Rubin's rules."

Summary of the Statistical Analysis of Change from Baseline in ACT Total Score at Week 12 (Visit 4) (Hodges-Lehmann Approach) (ITT Population)

Programming note: Present the "Difference" and "95% CI" lines of "FF/VI vs. Usual ICS/LABA" section only. Footnotes as follows:

"Note: The difference between treatment groups at Week 12 (Visit 4) was calculated using the Hodges-Lehmann approach."

Summary of the Statistical Analysis of Change from Baseline in ACT Total Score at Week 12 (Visit 4) (ANCOVA with WOCF) (ITT Population)

Programming note: Should the distributional assumption of normality fail then the p-value from a model on the rank-transformed values should be presented and the following footnote added: "Note: the p-value presented was obtained from an ANCOVA on the rank-transformed values of change from baseline in ACT total score at Week 12 (Visit 4) with the same specification as the untransformed model."

Footnotes as follows:

"Note: The analysis method was an ANCOVA model adjusted for randomised treatment, baseline ACT total score, gender, age and country.

Note: Missing values at Week 12 (Visit 4) due to treatment withdrawal prior to this time point were replaced by worst post-randomisation value based on the worst observation carried forward (WOCF) method."

HZA116492

Summary of the Statistical Analysis of Change from Baseline in ACT Total Score at Week 12 (Visit 4), FF/VI Versus the Subset of Usual ICS/LABA Subjects Prescribed FP/S at Randomisation (ITT Population)

Summary of the Statistical Analysis of Change from Baseline in ACT Total Score at Week 12 (Visit 4), FF/VI Versus the Subset of Usual ICS/LABA Subjects Prescribed BUD/F at Randomisation (ITT Population)

Summary of the Statistical Analysis of Change from Baseline in ACT Total Score at Week 24 (Visit 6) (ITT Population)

Summary of the Statistical Analysis of Change from Baseline in ACT Total Score at Week 24 (Visit 6) Per Protocol Population (PP Population)

Programming note: first footnote as follows:

"Note: The analysis method was an MMRM adjusted for randomised treatment, visit (Week 6, Week 12, Week 18 and Week 24), baseline ACT total score, randomised treatment-by-visit interaction, baseline ACT total score-by-visit interaction, gender, age, country and patient fitted as a random factor."

Summary of the Statistical Analysis of Change from Baseline in ACT Total Score at Week 24 (Visit 6) (ANCOVA with LOCF) (ITT Population)

Programming note: Should the distributional assumption of normality fail then the p-value from a model on the rank-transformed values should be presented and the following footnote added: "Note: the p-value presented was obtained from an ANCOVA on the rank-transformed values of change from baseline in ACT total score at Week 24 (Visit 6) with the same specification as the untransformed model."

Footnotes as follows:

"Note: The analysis method was an ANCOVA model adjusted for randomised treatment, baseline ACT total score, gender, age and country.

Note: Missing values at Week 24 (Visit 6) were replaced by last available post-randomisation value based on the last observation carried forward (LOCF) method."

Summary of the Statistical Analysis of Change from Baseline in ACT Total Score at Week 24 (Visit 6) (Multiple Imputation – Missing at Random Approach) (ITT Population)

Summary of the Statistical Analysis of Change from Baseline in ACT Total Score at Week 24 (Visit 6) (Multiple Imputation – Copy Differences from Reference Approach) (ITT Population)

Programming note: Present the "FF/VI vs. Usual ICS/LABA" section only. Footnotes as follows:

"Note: Missing values post-randomisation were imputed using multiple imputation methods based on pattern mixture models.

Note: Each imputed data set was analysed using an ANCOVA model at Week 24 (Visit 6) adjusted for randomised treatment, baseline ACT total score, gender, age and country and the resulting treatment differences and their standard errors combined using Rubin's rules."

Summary of the Statistical Analysis of Change from Baseline in ACT Total Score at Week 24 (Visit 6) (Hodges-Lehmann Approach) (ITT Population)

Present the "Difference" and "95% CI" lines of "FF/VI vs. Usual ICS/LABA" section only. Footnotes as follows:

"Note: The difference between treatment groups at Week 24 (Visit 6) was calculated using the Hodges-Lehmann approach."

Summary of the Statistical Analysis of Change from Baseline in ACT Total Score at Week 24 (Visit 6) (ANCOVA with WOCF) (ITT Population)

HZA116492

Programming note: Should the distributional assumption of normality fail then the p-value from a model on the rank-transformed values should be presented and the following footnote added: "Note: the p-value presented was obtained from an ANCOVA on the rank-transformed values of change from baseline in ACT total score at Week 24 (Visit 6) with the same specification as the untransformed model."

Footnotes as follows:

"Note: The analysis method was an ANCOVA model adjusted for randomised treatment, baseline ACT total score, gender, age and country.

Note: Missing values at Week 24 (Visit 6) due to treatment withdrawal prior to this time point were replaced by worst post-randomisation value based on the worst observation carried forward (WOCF) method."

Summary of the Statistical Analysis of Change from Baseline in ACT Total Score at Week 24 (Visit 6), FF/VI Versus the Subset of Usual ICS/LABA Subjects Prescribed FP/S at Randomisation (ITT Population)

Programming note: Output only to be produced if ≥25% of Usual ICS/LABA patients are prescribed FP/S at randomisation. First footnote as follows:

"Note: The analysis method was an MMRM adjusted for randomised treatment, visit (Week 6, Week 12, Week 18 and Week 24), baseline ACT total score, randomised treatment-by-visit interaction, baseline ACT total score-by-visit interaction, gender, age, country and patient fitted as a random factor."

Summary of the Statistical Analysis of Change from Baseline in ACT Total Score at Week 24 (Visit 6), FF/VI Versus the Subset of Usual ICS/LABA Subjects Prescribed BUD/F at Randomisation (ITT Population)

Programming note: Output only to be produced if ≥25% of Usual ICS/LABA patients are prescribed BUD/F at randomisation. First footnote as follows:

"Note: The analysis method was an MMRM adjusted for randomised treatment, visit (Week 6, Week 12, Week 18 and Week 24), baseline ACT total score, randomised treatment-by-visit interaction, baseline ACT total score-by-visit interaction, gender, age, country and patient fitted as a random factor."

Summary of the Statistical Analysis of Change from Baseline in Trough (Pre-dose) FEV1 at Week 12 (Visit 4) (ITT Population)

Programming note: Should the distributional assumption of normality fail then the p-value from a model on the rank-transformed values should be presented and the following footnote added: "Note: the p-value presented was obtained from an ANCOVA on the rank-transformed values of change from baseline in trough (pre-dose) FEV1 at Week 12 (Visit 4) with the same specification as the untransformed model." Footnote as follows:

"Note: The analysis method was an ANCOVA model adjusted for randomised treatment, baseline trough (pre-dose) FEV1, gender, age and country."

Summary of the Statistical Analysis of Change from Baseline in EQ-5D-5L Utility Score at Week 24 (Visit 6) (ITT Population)

Programming note: Should the distributional assumption of normality fail then the p-value from a model on the rank-transformed values should be presented and the following footnote added: "Note: the p-value presented was obtained from an ANCOVA on the rank-transformed values of change from baseline in EQ-5D-5L utility score at Week 24 (Visit 6) with the same specification as the untransformed model."

Footnote as follows:

"Note: The analysis method was an ANCOVA model adjusted for randomised treatment, baseline EQ-5D-5L utility score, gender, age and country."

HZA116492

Summary of the Statistical Analysis of Change from Baseline in EQ-5D-5L Visual Analogue Scale (VAS) Score at Week 24 (Visit 6) (ITT Population)
Programming note: Should the distributional assumption of normality fail then the p-value from a model on the rank-transformed values should be presented and the following footnote added: "Note: the p-value presented was obtained from an ANCOVA on the rank-transformed values of change from baseline in EQ-5D-5L VAS score at Week 24 (Visit 6) with the same specification as the untransformed model."
Footnote as follows:

"Note: The analysis method was an ANCOVA model adjusted for randomised treatment, baseline EQ-5D-5L VAS score, gender, age and country."

HZA116492

Example : EFF\_T2S Protocol : HZA11649

: HZA116492 

Population : Intent-to-Treat

Table 2.xx

Summary of the Statistical Analysis of Change from Baseline in ACT Total Score at Week 12 (Visit 4) by Country

# Country: France

| | Usual ICS/LABA<br>(N=xxx) | FF/VI<br>(N=xxx) |
|--------------------------|---------------------------|------------------|
| n | XX | XX |
| LS Mean Change (SE) | xx.xx (x.xxx) | xx.xx (x.xxx) |
| FF/VI vs. Usual ICS/LABA | | |
| Difference | | XX.X |
| 95% CI | | (xx.x, xx.x) |

Note: The analysis method was an MMRM adjusted for randomised treatment, visit (Week 6 and Week 12), baseline ACT total score, baseline ACT total score-by-visit interaction, gender, age, country, two- and three- way interactions between randomised treatment, visit and country, and patient fitted as a random factor.

Note: The Restricted Maximum Likelihood (REML) estimation approach was used with a default covariance structure of unstructured.

HZA116492

Example : EFF\_T2S Protocol : HZA11649

: HZA116492 

Population : Intent-to-Treat

Table 2.xx

Summary of the Statistical Analysis of Change from Baseline in ACT Total Score at Week 12 (Visit 4) by Country

# Country: Germany

| | Usual ICS/LABA<br>(N=xxx) | FF/VI<br>(N=xxx) |
|--------------------------|---------------------------|------------------|
| n | XX | XX |
| LS Mean Change (SE) | xx.xx (x.xxx) | xx.xx (x.xxx) |
| FF/VI vs. Usual ICS/LABA | | |
| Difference | | XX.X |
| 95% CI | | (xx.x, xx.x) |

Note: The analysis method was an MMRM adjusted for randomised treatment, visit (Week 6 and Week 12), baseline ACT total score, randomised treatment-by-visit interaction, baseline ACT total score-by-visit interaction, gender, age, country, randomised treatment-by-country interaction and patient fitted as a random factor. Note: The Restricted Maximum Likelihood (REML) estimation approach was used with a default covariance structure of unstructured.

Programming note: Should computational issues be encountered when using an unstructured covariance structure, other structures including AR1 and CS should be considered and the second footnote updated as appropriate.

HZA116492

#### Repeat for:

Summary of the Statistical Analysis of Change from Baseline in ACT Total Score at Week 12 (Visit 4) by Number of Severe Asthma Exacerbations in the Previous Year Prior to Randomisation (ITT Population)

Number of Severe Asthma Exacerbations in the Previous Year Prior to Randomisation: 0

Number of Severe Asthma Exacerbations in the Previous Year Prior to Randomisation: >= 1

Programming note: first footnote as follows:

"Note: The analysis method was an MMRM adjusted for randomised treatment, visit (Week 6 and Week 12), baseline ACT total score, baseline ACT total score-by-visit interaction, gender, age, country, number of severe asthma exacerbations in the previous year prior to randomisation, two- and three- way interactions between randomised treatment, visit and number of severe asthma exacerbations in the previous year prior to randomisation, and patient fitted as a random factor."

Summary of the Statistical Analysis of Change from Baseline in ACT Total Score at Week 12 (Visit 4) by Smoking Status at Baseline (ITT Population) Programming note: first footnote as follows:

"Note: The analysis method was an MMRM adjusted for randomised treatment, visit (Week 6 and Week 12), baseline ACT total score, baseline ACT total score-by-visit interaction, gender, age, country, smoking status at baseline, two- and three- way interactions between randomised treatment, visit and smoking status at baseline, and patient fitted as a random factor."

Summary of the Statistical Analysis of Change from Baseline in ACT Total Score at Week 12 (Visit 4) by Age Group (ITT Population) Programming note: first footnote as follows:

"Note: The analysis method was an MMRM adjusted for randomised treatment, visit (Week 6 and Week 12), baseline ACT total score, baseline ACT total score, baseline ACT total score, baseline ACT total score by-visit interaction, gender, country, age group, two- and three- way interactions between randomised treatment, visit and age group, and patient fitted as a random factor."

Summary of the Statistical Analysis of Change from Baseline in ACT Total Score at Week 12 (Visit 4) by Gender (ITT Population) Programming note: first footnote as follows:

"Note: The analysis method was an MMRM adjusted for randomised treatment, visit (Week 6 and Week 12), baseline ACT total score, baseline ACT total score-by-visit interaction, gender, age, country, two- and three- way interactions between randomised treatment, visit and gender, and patient fitted as a random factor."

Summary of the Statistical Analysis of Change from Baseline in ACT Total Score at Week 24 (Visit 6) by Country (ITT Population) Programming note: first footnote as follows:

"Note: The analysis method was an MMRM adjusted for randomised treatment, visit (Week 6, Week 12, Week 18 and Week 24), baseline ACT total score, baseline ACT total score-by-visit interaction, gender, age, country, two- and three- way interactions between randomised treatment, visit and country, and patient fitted as a random factor."

HZA116492

Example : EFF\_T3 Protocol : HZA116492


Population : Intent-to-Treat

Table 2.xx

Summary of the Statistical Analysis of Change from Baseline in ACT Total Score at Week 12 (Visit 4), Adjusting for Seasonal Effect

| | Usual ICS/LABA<br>(N=xxx) | FF/VI<br>(N=xxx) |
|---|---|---|
| Randomised treatment-by-season at randomisation interaction p-value | | X.XXX |
| Season at randomisation: Spring<br>n<br>LS Mean Change (SE) | xx<br>xx.xx (x.xxx) | xx<br>xx.xx (x.xxx) |
| FF/VI vs. Usual ICS/LABA<br>Difference<br>95% CI | | xx.x<br>(xx.x, xx.x) |

Note: The analysis method was an MMRM adjusted for randomised treatment, visit (Week 6 and Week 12), baseline ACT total score, baseline ACT total score-by-visit interaction, gender, age, country, season at randomisation, two- and three- way interactions between randomised treatment, visit and season at randomisation, and patient fitted as a random factor.

Note: The Restricted Maximum Likelihood (REML) estimation approach was used with a default covariance structure of unstructured.

Note: Spring = March, April and May; Summer = June, July and August; Autumn = September, October and November; Winter = December, January and February.

Programming note: repeat on subsequent pages for Season at randomisation = Summer, Autumn, Winter. Should computational issues be encountered when using an unstructured covariance structure, other structures including AR1 and CS should be considered and the second footnote updated as appropriate.

HZA116492

#### Repeat for:

Summary of the Statistical Analysis of Change from Baseline in ACT Total Score at Week 12 (Visit 4), Adjusting for Seasonal Effect Per Protocol Population (PP Population)

Summary of the Statistical Analysis of Change from Baseline in ACT Total Score at Week 24 (Visit 6), Adjusting for Seasonal Effect (ITT Population)
Summary of the Statistical Analysis of Change from Baseline in ACT Total Score at Week 24 (Visit 6), Adjusting for Seasonal Effect Per Protocol Population (PP Population)

First footnote as follows:

"Note: The analysis method was an MMRM adjusted for randomised treatment, visit (Week 6, Week 12, Week 18 and Week 24), baseline ACT total score, baseline ACT total score-by-visit interaction, gender, age, country, season at randomisation, two- and three- way interactions between randomised treatment, visit and season at randomisation, and patient fitted as a random factor."

HZA116492

Example : EFF\_T4
Protocol : HZA116492
Population : Intent-to-Treat


Table 2.xx Summary of Inhaler Device Use Errors

| Visit | | Usual ICS/LABA<br>(N=xxx) | FF/VI<br>(N=xxx) |
|---|---|---|---|
| VIOIC | | (IT AXX) | (IV AAA) |
| Day 0 | Number of patients using Ellipta | | XXX |
| | Number of patients with correct use [1] | | xxx (xx%) |
| | Number of patients without correct use | | xxx (xx%) |
| | Number of patients with at least one critical error<br>Type of critical error: | | xxx (xx%) |
| | Failed to open cover | | xxx (xx%) |
| | Shook the device upside down after dose preparation Exhaled directly into mouthpiece | | xxx (xx%)<br>xxx (xx%) |
| | No seal by the lips around the mouthpiece during the inhalation | | xxx (xx%) |
| | Number of patients with at least one non-critical error Type of non-critical error: | | xxx (xx%) |
| | No exhalation before an inhalation | | xxx (xx%) |
| | Inhalation manoeuvre was not: long, steady and deep | | xxx (xx%) |
| | Blocked air inlet during inhalation manoeuvre | | xxx (xx%) |
| | Did not hold breath | | xxx (xx%) |
| | Did not close the device | | xxx (xx%) |

<sup>[1]</sup> Correct use is defined as not making any critical or non-critical errors at that visit.

HZA116492

Example : EFF\_T4
Protocol : HZA116492
Population : Intent-to-Treat


# Table 2.xx Summary of Inhaler Device Use Errors

| Visit | | Usual ICS/LABA<br>(N=xxx) | FF/VI<br>(N=xxx) |
|---|---|---|---|
| Day 0 | Number of patients using Diskus | xxx | |
| | Number of patients with correct use [1] | xxx (xx%) | |
| | Number of patients without correct use | xxx (xx%) | |
| | Number of patients with at least one critical error Type of critical error: | xxx (xx%) | |
| | Failed to open cover | xxx (xx%) | |
| | Lever is not pushed back | xxx (xx%) | |
| | Shook the device after dose preparation | xxx (xx%) | |
| | Exhaled directly into mouthpiece | xxx (xx%) | |
| | No seal by the lips around the mouthpiece during the inhalation | xxx (xx%) | |
| | Number of patients with at least one non-critical error Type of non-critical error: | xxx (xx%) | |
| | No exhalation before an inhalation | xxx (xx%) | |
| | Inhalation manoeuvre was not: steady and deep | xxx (xx%) | |
| | Did not hold breath | xxx (xx%) | |
| | Did not close the device | xxx (xx%) | |

<sup>[1]</sup> Correct use is defined as not making any critical or non-critical errors at that visit.

HZA116492

Example : EFF\_T4
Protocol : HZA116492
Population : Intent-to-Treat


# Table 2.xx Summary of Inhaler Device Use Errors

| Visit | | Usual ICS/LABA<br>(N=xxx) | FF/VI<br>(N=xxx) |
|---|---|---|---|
| Day 0 | Number of patients using Turbuhaler | xxx | |
| | Number of patients with correct use [1]<br>Number of patients without correct use | xxx (xx%)<br>xxx (xx%) | |
| | Number of patients with at least one critical error Type of critical error: Failed to remove cap Did not hold device upright during dose preparation Base not twisted fully backwards and forwards, no click heard Shook the device after dose preparation Exhaled directly into mouthpiece No seal by the lips around the mouthpiece during the inhalation Number of patients with at least one non-critical error Type of non-critical error: Device tipped downwards after dose preparation No exhalation before an inhalation Inhalation manoeuvre was not: forceful and deep | xxx (xx%) | |
| | Blocked air inlet during inhalation manoeuvre Did not hold breath Did not close the device | xxx (xx%)<br>xxx (xx%)<br>xxx (xx%) | |

HZA116492

[1] Correct use is defined as not making any critical or non-critical errors at that visit.

Programming note: repeat on subsequent pages for Visit = Week 12 and Week 24. "Number of patients using..." line will provide the denominators for each section's percentages.

# Repeat for:

Summary of Inhaler Device Use Errors Per Protocol Population (PP Population)

HZA116492

Example : EFF\_T5
Protocol : HZA116492

: Intent-to-Treat

Population


Table 2.xx Summary of Correct Use of Inhaler Device

| Visit | | Usual ICS/LABA<br>(N=xxx) | FF/VI<br>(N=xxx) |
|---|---|---|---|
| Day 0 | n | XXX | xxx |
| , - | Number of patients with correct use [1] | xxx (xx%) | xxx (xx%) |
| | Number of patients without correct use | xxx (xx%) | xxx (xx%) |
| | Number of patients with at least one critical error | xxx (xx%) | xxx (xx%) |
| | Number of patients with at least one non-critical error | xxx (xx%) | xxx (xx%) |
| Week 12 | n | XXX | XXX |
| | Number of patients with correct use [1] | xxx (xx%) | xxx (xx%) |
| | Number of patients without correct use | xxx (xx%) | xxx (xx%) |
| | Number of patients with at least one critical error | xxx (xx%) | xxx (xx%) |
| | Number of patients with at least one non-critical error | xxx (xx%) | xxx (xx%) |
| Week 24 | n | XXX | XXX |
| | Number of patients with correct use [1] | xxx (xx%) | xxx (xx%) |
| | Number of patients without correct use | xxx (xx%) | xxx (xx%) |
| | Number of patients with at least one critical error | xxx (xx%) | xxx (xx%) |
| | Number of patients with at least one non-critical error | xxx (xx%) | xxx (xx%) |

[1] Correct use is defined as not making any critical or non-critical errors at that visit.

# Repeat for:

Summary of Correct Use of Inhaler Device Per Protocol Population (PP Population)

HZA116492


Example

: EFF\_T6 : HZA116492 Protocol Population : Intent-to-Treat

# Table 2.xx

Summary of the Statistical Analysis of Correct Use of Inhaler Device at Week 12 (Visit 4) and at Week 24 (Visit 6) Independently of the Use at Week 12 (Visit 4)

| Visit | | Usual ICS/LABA<br>(N=xxx) | FF/VI<br>(N=xxx) |
|---|---|---|---|
| Violt | | (IV-XXX) | (14-222) |
| Week 12 | n | XXX | XXX |
| | With correct use [1] | xxx (xx%) | xxx (xx%) |
| | Without correct use | xxx (xx%) | xxx (xx%) |
| | FF/VI vs. Usual ICS/LABA | | |
| | Adjusted Odds Ratio | | X.XX |
| | 95% CI | | (x.xx, x.xx) |
| | p-value | | X.XXX |
| Week 24 | n | XXX | XXX |
| | With correct use [1] | xxx (xx%) | xxx (xx%) |
| | Without correct use | xxx (xx%) | xxx (xx%) |
| | FF/VI vs. Usual ICS/LABA | | |
| | Adjusted Odds Ratio | | X.XX |
| | 95% CI | | (x.xx, x.xx) |
| | p-value | | X.XXX |

<sup>[1]</sup> Correct use is defined as not making any critical or non-critical errors at that visit.

HZA116492

Note: The analysis method was logistic regression adjusted for randomised treatment, correct use of inhaler device at baseline, gender, age and country.

Programming note: If the likelihood maximisation algorithm fails to converge due to complete or quasi-complete separation of the data then implement Firth's penalized likelihood and add the following footnote: "Note: Firth's penalized likelihood was implemented due to [complete / quasi-complete] separation of data.", deleting "complete" or "quasi-complete" as appropriate.

#### Repeat for:

Summary of the Statistical Analysis of Correct Use of Inhaler Device at Week 12 (Visit 4) and at Week 24 (Visit 6) Independently of the Use at Week 12 (Visit 4) Per Protocol Population (PP Population)

Summary of the Statistical Analysis of Percentage of Subjects Who Have Either an ACT Total Score >= 20 or >= 3 Point Increase from Baseline in ACT Total Score at Week 12 (Visit 4) and Week 24 (Visit 6) (ITT Population)

Programming note: Replace "With correct use [1]" with "Responder [1]" and "Without correct use" with "Non-Responder".

Footnotes as follows:

"[1] Responder is defined as an ACT total score >= 20 or >= 3 point increase from baseline in ACT total score at that visit.

Note: The analysis method was logistic regression adjusted for randomised treatment, baseline ACT total score, baseline ACT total score squared, gender, age and country."

Summary of the Statistical Analysis of Percentage of Subjects Who Have an Increase from Baseline of >=0.5 in AQLQ(S) Total Score and Environmental Stimuli Domain Score at Week 24 (Visit 6) (ITT Population)

Domain: Total Score

Domain: Environmental Stimuli

Programming note: Replace "With correct use [1]" with "Responder [1]" and "Without correct use" with "Non-Responder". Do not display the "Visit" column.

Footnotes as follows:

"[1] Responder is defined as an increase from baseline of >= 0.5.

Note: The analysis method was logistic regression adjusted for randomised treatment, baseline score, gender, age and country."

Summary of the Statistical Analysis of Proportion of Responders According to EQ-5D-5L Descriptive System Dimensions at Week 24 (Visit 6) (ITT Population)

Dimension: Anxiety/Depression

Dimension: Mobility

Dimension: Pain/Discomfort

Dimension: Self-care

HZA116492

Dimension: Usual activities

Programming note: Replace "With correct use [1]" with "Responder [1]" and "Without correct use" with "Non-Responder". Do not display the "Visit" column. Footnotes as follows:

"[1] Responder is defined as a score of 1 ('no problems').

Note: The analysis method was logistic regression adjusted for randomised treatment, baseline EQ-5D-5L domain score, gender, age and country."

HZA116492

Example

: EFF\_T7 : HZA116492 Protocol Population : Intent-to-Treat


Table 2.xx

Summary of Percentage of Subjects Who Have Either an ACT Total Score of >= 20 or >= 3 Point Increase from Baseline in ACT Total Score

| Visit | | Usual ICS/LABA<br>(N=xxx) | FF/VI<br>(N=xxx) |
|---|---|---|---|
| Week 6 | n ACT Total Score >= 20 or >= 3 Point Increase from Baseline ACT Total Score >= 20 >= 3 Point Increase from Baseline | xxx<br>xxx (xx%)<br>xxx (xx%)<br>xxx (xx%) | xxx<br>xxx (xx%)<br>xxx (xx%)<br>xxx (xx%) |
| Week 12 | n ACT Total Score >= 20 or >= 3 Point Increase from Baseline ACT Total Score >= 20 >= 3 Point Increase from Baseline | xxx<br>xxx (xx%)<br>xxx (xx%)<br>xxx (xx%) | xxx<br>xxx (xx%)<br>xxx (xx%)<br>xxx (xx%) |

Programming note: repeat for Visit = Week 18, Week 24, Early Withdrawal.

HZA116492

Example : EFF\_T8
Protocol : HZA116492
Population : Intent-to-Treat


Table 2.xx Summary of Individual ACT Question Scores

Question: 1. Getting as much done at work, school or home

| Visit | Response | Usual ICS/LABA<br>(N=xxx) | FF/VI<br>(N=xxx) |
|---|---|---|---|
| Day 0 | n | XXX | XXX |
| , | 1. All of the time | xxx (xx%) | xxx (xx%) |
| | 2. Most of the time | xxx (xx%) | xxx (xx%) |
| | 3. Some of the time | xxx (xx%) | xxx (xx%) |
| | <ol><li>A little of the time</li></ol> | xxx (xx%) | xxx (xx%) |
| | 5. None of the time. | xxx (xx%) | xxx (xx%) |
| Week 6 | n | XXX | XXX |
| | 1. All of the time | xxx (xx%) | xxx (xx%) |
| | 2. Most of the time | xxx (xx%) | xxx (xx%) |
| | 3. Some of the time | xxx (xx%) | xxx (xx%) |
| | <ol><li>A little of the time</li></ol> | xxx (xx%) | xxx (xx%) |
| | 5. None of the time. | xxx (xx%) | xxx (xx%) |
| Week 12 | n | XXX | XXX |
| | 1. All of the time | xxx (xx%) | xxx (xx%) |
| | 2. Most of the time | xxx (xx%) | xxx (xx%) |
| | <ol><li>Some of the time</li></ol> | xxx (xx%) | xxx (xx%) |
| | <ol><li>A little of the time</li></ol> | xxx (xx%) | xxx (xx%) |
| | <ol><li>None of the time.</li></ol> | xxx (xx%) | xxx (xx%) |

HZA116492

Example : EFF\_T8
Protocol : HZA116492

Population : Intent-to-Treat


# Table 2.xx Summary of Individual ACT Question Scores

Question: 1. Getting as much done at work, school or home

| Visit | Response | Usual ICS/LABA<br>(N=xxx) | FF/VI<br>(N=xxx) |
|---|---|---|---|
| Week 18 | n | XXX | XXX |
| | 1. All of the time | xxx (xx%) | xxx (xx%) |
| | 2. Most of the time | xxx (xx%) | xxx (xx%) |
| | 3. Some of the time | xxx (xx%) | xxx (xx%) |
| | 4. A little of the time | xxx (xx%) | xxx (xx%) |
| | 5. None of the time. | xxx (xx%) | xxx (xx%) |
| Week 24 | n | XXX | xxx |
| | 1. All of the time | xxx (xx%) | xxx (xx%) |
| | 2. Most of the time | xxx (xx%) | xxx (xx%) |
| | 3. Some of the time | xxx (xx%) | xxx (xx%) |
| | <ol><li>A little of the time</li></ol> | xxx (xx%) | xxx (xx%) |
| | 5. None of the time. | xxx (xx%) | xxx (xx%) |
| Early Withdrawal | n | XXX | XXX |
| • | 1. All of the time | xxx (xx%) | xxx (xx%) |
| | 2. Most of the time | xxx (xx%) | xxx (xx%) |
| | <ol><li>Some of the time</li></ol> | xxx (xx%) | xxx (xx%) |
| | <ol><li>A little of the time</li></ol> | xxx (xx%) | xxx (xx%) |
| | <ol><li>None of the time.</li></ol> | xxx (xx%) | xxx (xx%) |

HZA116492

Programming note: repeat on subsequent pages for Question = 2. Shortness of breath, 3. Asthma symptoms woken up at night or earlier than usual, 4. Used rescue inhaler or nubuliser medication, 5. Asthma control.

HZA116492

Example : EFF\_T9
Protocol : HZA116492

Population : Intent-to-Treat


# Table 2.xx Summary of Compliance with Study Medication

| Time period | Compliance (%) | Usual ICS/LABA<br>(N=xxx) | FF/VI<br>(N=xxx) |
|---|---|---|---|
| Day 0 to Week 24 | n | XXX | XXX |
| Day o to Wook 21 | < 80% | xxx (xx%) | xxx (xx%) |
| | 80% to 120% inclusive | xxx (xx%) | xxx (xx%) |
| | > 120% | xxx (xx%) | xxx (xx%) |
| | n | XX | XX |
| | Mean | XX.X | XX.X |
| | SD | X.XX | X.XX |
| | Median | XX.X | XX.X |
| | Min. | XX | XX |
| | Max. | XX | XX |

Note: Compliance =  $\{[Total no. of inhalations taken]/[Dose frequency x (Stop date - Start date)]\} x 100.$ 

Note: Total number of inhalations taken is the sum of (dose counter start count – dose counter stop count) for all inhalers used during the time period, Dose frequency is equal to 1 for Ellipta, 2 for Diskus and 2 or 4 for Turbuhaler, and Start date and Stop date are the earliest treatment start date and latest treatment stop date respectively recorded for all inhalers used during the time period.

Programming note: repeat on subsequent pages for Time period = Day 0 to Week 12, Week 12 to Week 24.

#### Repeat for:

Summary of Compliance with Study Medication Per Protocol Population (PP Population)

HZA116492

: EFF\_T10 : HZA116492 Example Protocol

Population : Intent-to-Treat 

Table 2.xx

Summary of Use of Medication Adherence Report Scale for Asthma (MARS-A) During the Study

Visit: Day 0

| MARS-A Questions | | Usual ICS/LABA<br>(N=xxx) | FF/VI<br>(N=xxx) |
|---|---|---|---|
| I only use it when I need it | n | XXX | XXX |
| Tonly use it when theed it | Always | xxx (xx%) | xxx (xx%) |
| | Often | xxx (xx%) | xxx (xx%) |
| | Sometimes | xxx (xx%) | xxx (xx%) |
| | Rarely | xxx (xx%) | xxx (xx%) |
| | Never | xxx (xx%) | xxx (xx%) |
| | Nevel | XXX (XX70) | XXX (XX 70) |
| Only use it when I feel breathless | n | XXX | XXX |
| | Always | xxx (xx%) | xxx (xx%) |
| | Often | xxx (xx%) | xxx (xx%) |
| | Sometimes | xxx (xx%) | xxx (xx%) |
| | Rarely | xxx (xx%) | xxx (xx%) |
| | Never | xxx (xx%) | xxx (xx%) |
| I decide to miss out a dose | n | XXX | XXX |
| | Always | xxx (xx%) | xxx (xx%) |
| | Often | xxx (xx%) | xxx (xx%) |
| | Sometimes | xxx (xx%) | xxx (xx%) |
| | Rarely | xxx (xx%) | xxx (xx%) |
| | Never | xxx (xx%) | xxx (xx%) |

Note: MARS-A: Medication Adherence Report Scale for Asthma.
[1]: MARS-A 10-Score is based on the mean score across all ten questions.

HZA116492

: EFF\_T10 : HZA116492 Example

Protocol Population : Intent-to-Treat 

Table 2.xx Summary of Use of Medication Adherence Report Scale for Asthma (MARS-A) During the Study

Visit: Day 0

| MARS-A Questions | | Usual ICS/LABA<br>(N=xxx) | FF/VI<br>(N=xxx) |
|---|---|---|---|
| I try to avoid using it | n | XXX | XXX |
| 3, | Always | xxx (xx%) | xxx (xx%) |
| | Often | xxx (xx%) | xxx (xx%) |
| | Sometimes | xxx (xx%) | xxx (xx%) |
| | Rarely | xxx (xx%) | xxx (xx%) |
| | Never | xxx (xx%) | xxx (xx%) |
| I forget to take it | n | XXX | XXX |
| • | Always | xxx (xx%) | xxx (xx%) |
| | Often | xxx (xx%) | xxx (xx%) |
| | Sometimes | xxx (xx%) | xxx (xx%) |
| | Rarely | xxx (xx%) | xxx (xx%) |
| | Never | xxx (xx%) | xxx (xx%) |
| I alter the dose | n | XXX | XXX |
| | Always | xxx (xx%) | xxx (xx%) |
| | Often | xxx (xx%) | xxx (xx%) |
| | Sometimes | xxx (xx%) | xxx (xx%) |
| | Rarely | xxx (xx%) | xxx (xx%) |
| | Never | xxx (xx%) | xxx (xx%) |

Note: MARS-A: Medication Adherence Report Scale for Asthma.
[1]: MARS-A 10-Score is based on the mean score across all ten questions.

HZA116492

: EFF\_T10 : HZA116492 Example Protocol

Population : Intent-to-Treat 

Table 2.xx

Summary of Use of Medication Adherence Report Scale for Asthma (MARS-A) During the Study

Visit: Day 0

| MARS-A Questions | | Usual ICS/LABA<br>(N=xxx) | FF/VI<br>(N=xxx) |
|---|---|---|---|
| I stop taking it for a while | n | XXX | XXX |
| | Always | xxx (xx%) | xxx (xx%) |
| | Often | xxx (xx%) | xxx (xx%) |
| | Sometimes | xxx (xx%) | xxx (xx%) |
| | Rarely | xxx (xx%) | xxx (xx%) |
| | Never | xxx (xx%) | xxx (xx%) |
| Reserve if treatment doesn't work | n | XXX | XXX |
| | Always | xxx (xx%) | xxx (xx%) |
| | Often | xxx (xx%) | xxx (xx%) |
| | Sometimes | xxx (xx%) | xxx (xx%) |
| | Rarely | xxx (xx%) | xxx (xx%) |
| | Never | xxx (xx%) | xxx (xx%) |
| Before doing something | n | XXX | XXX |
| 5 | Always | xxx (xx%) | xxx (xx%) |
| | Often | xxx (xx%) | xxx (xx%) |
| | Sometimes | xxx (xx%) | xxx (xx%) |
| | Rarely | xxx (xx%) | xxx (xx%) |
| | Never | xxx (xx%) | xxx (xx%) |

Note: MARS-A: Medication Adherence Report Scale for Asthma.
[1]: MARS-A 10-Score is based on the mean score across all ten questions.

HZA116492

Example : EFF\_T10

Protocol : HZA116492 Population : Intent-to-Treat 

Table 2.xx

Summary of Use of Medication Adherence Report Scale for Asthma (MARS-A) During the Study

Visit: Day 0

| MARS-A Questions | | Usual ICS/LABA<br>(N=xxx) | FF/VI<br>(N=xxx) |
|---|---|---|---|
| With the 71 Queeneries | | (11 700) | (14 7000) |
| I take less than instructed | n | XXX | XXX |
| | Always | xxx (xx%) | xxx (xx%) |
| | Often | xxx (xx%) | xxx (xx%) |
| | Sometimes | xxx (xx%) | xxx (xx%) |
| | Rarely | xxx (xx%) | xxx (xx%) |
| | Never | xxx (xx%) | xxx (xx%) |
| MARS-A 10-Score [1] | n | XX | XX |
| • • | Mean | XX.X | XX.X |
| | SD | X.XX | X.XX |
| | Median | XX.X | XX.X |
| | Min. | XX | XX |
| | Max. | XX | XX |

Note: MARS-A: Medication Adherence Report Scale for Asthma.

[1]: MARS-A 10-Score is based on the mean score across all ten questions.

Programming note: Repeat on subsequent pages for Visit = Week 12, Week 24 and Early Withdrawal.

HZA116492

Example : EFF\_T10S

Protocol : HZA116492 

Population : Intent-to-Treat

Table 2.xx

Summary of Use of Medication Adherence Report Scale for Asthma (MARS-A) During the Study by Status of Patient in Relation to the Reminder Sent to French Centres

Status: Patients in France who had completed all MARS-A assessments prior to the reminder being implemented Visit: Day 0

| MARS-A Questions | | Usual ICS/LABA<br>(N=xxx) | FF/VI<br>(N=xxx) |
|---|---|---|---|
| I only use it when I need it | n | xxx | xxx |
| | Always | xxx (xx%) | xxx (xx%) |
| | Often | xxx (xx%) | xxx (xx%) |
| | Sometimes | xxx (xx%) | xxx (xx%) |
| | Rarely | xxx (xx%) | xxx (xx%) |
| | Never | xxx (xx%) | xxx (xx%) |
| Only use it when I feel breathless | n | xxx | xxx |
| | Always | xxx (xx%) | xxx (xx%) |
| | Often | xxx (xx%) | xxx (xx%) |
| | Sometimes | xxx (xx%) | xxx (xx%) |
| | Rarely | xxx (xx%) | xxx (xx%) |
| | Never | xxx (xx%) | xxx (xx%) |
| I decide to miss out a dose | n | xxx | xxx |
| | Always | xxx (xx%) | xxx (xx%) |
| | Often | xxx (xx%) | xxx (xx%) |
| | Sometimes | xxx (xx%) | xxx (xx%) |
| | Rarely | xxx (xx%) | xxx (xx%) |
| | Never | xxx (xx%) | xxx (xx%) |

Note: MARS-A: Medication Adherence Report Scale for Asthma.

HZA116492

Note: Due to an issue identified with the French translation of the MARS-A, a reminder was sent to centres in France instructing that the questionnaire refers to the patient's preventer inhaler (i.e. their maintenance therapy prior to entering the study, and study medication while on-study).
[1]: MARS-A 10-Score is based on the mean score across all ten questions.

HZA116492

Example : EFF\_T10S Protocol : HZA116492

otocol : HZA116492 

Population : Intent-to-Treat

Table 2.xx

Summary of Use of Medication Adherence Report Scale for Asthma (MARS-A) During the Study by Status of Patient in Relation to the Reminder Sent to French Centres

Status: Patients in France who had completed all MARS-A assessments prior to the reminder being implemented Visit: Day 0

| MARS-A Questions | | Usual ICS/LABA<br>(N=xxx) | FF/VI<br>(N=xxx) |
|---|---|---|---|
| I try to avoid using it | n | XXX | XXX |
| | Always | xxx (xx%) | xxx (xx%) |
| | Often | xxx (xx%) | xxx (xx%) |
| | Sometimes | xxx (xx%) | xxx (xx%) |
| | Rarely | xxx (xx%) | xxx (xx%) |
| | Never | xxx (xx%) | xxx (xx%) |
| I forget to take it | n | XXX | XXX |
| - | Always | xxx (xx%) | xxx (xx%) |
| | Often | xxx (xx%) | xxx (xx%) |
| | Sometimes | xxx (xx%) | xxx (xx%) |
| | Rarely | xxx (xx%) | xxx (xx%) |
| | Never | xxx (xx%) | xxx (xx%) |
| I alter the dose | n | XXX | XXX |
| | Always | xxx (xx%) | xxx (xx%) |
| | Often | xxx (xx%) | xxx (xx%) |
| | Sometimes | xxx (xx%) | xxx (xx%) |
| | Rarely | xxx (xx%) | xxx (xx%) |
| | Never | xxx (xx%) | xxx (xx%) |

Note: MARS-A: Medication Adherence Report Scale for Asthma.

HZA116492

Note: Due to an issue identified with the French translation of the MARS-A, a reminder was sent to centres in France instructing that the questionnaire refers to the patient's preventer inhaler (i.e. their maintenance therapy prior to entering the study, and study medication while on-study).
[1]: MARS-A 10-Score is based on the mean score across all ten questions.

HZA116492


Example : EFF\_T10S Protocol : HZA116492

Population : Intent-to-Treat

Table 2.xx

Summary of Use of Medication Adherence Report Scale for Asthma (MARS-A) During the Study by Status of Patient in Relation to the Reminder Sent to French Centres

Status: Patients in France who had completed all MARS-A assessments prior to the reminder being implemented Visit: Day 0

| MARS-A Questions | | Usual ICS/LABA<br>(N=xxx) | FF/VI<br>(N=xxx) |
|---|---|---|---|
| I stop taking it for a while | n | xxx | xxx |
| | Always | xxx (xx%) | xxx (xx%) |
| | Often | xxx (xx%) | xxx (xx%) |
| | Sometimes | xxx (xx%) | xxx (xx%) |
| | Rarely | xxx (xx%) | xxx (xx%) |
| | Never | xxx (xx%) | xxx (xx%) |
| Reserve if treatment doesn't work | n | xxx | xxx |
| | Always | xxx (xx%) | xxx (xx%) |
| | Often | xxx (xx%) | xxx (xx%) |
| | Sometimes | xxx (xx%) | xxx (xx%) |
| | Rarely | xxx (xx%) | xxx (xx%) |
| | Never | xxx (xx%) | xxx (xx%) |
| Before doing something | n | xxx | xxx |
| | Always | xxx (xx%) | xxx (xx%) |
| | Often | xxx (xx%) | xxx (xx%) |
| | Sometimes | xxx (xx%) | xxx (xx%) |
| | Rarely | xxx (xx%) | xxx (xx%) |
| | Never | xxx (xx%) | xxx (xx%) |

Note: MARS-A: Medication Adherence Report Scale for Asthma.

HZA116492

Note: Due to an issue identified with the French translation of the MARS-A, a reminder was sent to centres in France instructing that the questionnaire refers to the patient's preventer inhaler (i.e. their maintenance therapy prior to entering the study, and study medication while on-study).
[1]: MARS-A 10-Score is based on the mean score across all ten questions.

HZA116492


Example : EFF\_T10S Protocol : HZA116492

Population : Intent-to-Treat

Table 2.xx

Summary of Use of Medication Adherence Report Scale for Asthma (MARS-A) During the Study by Status of Patient in Relation to the Reminder Sent to French Centres

Status: Patients in France who had completed all MARS-A assessments prior to the reminder being implemented Visit: Day 0

| MARS-A Questions | | Usual ICS/LABA<br>(N=xxx) | FF/VI<br>(N=xxx) |
|---|---|---|---|
| I take less than instructed | n<br>Always<br>Often<br>Sometimes<br>Rarely<br>Never | xxx<br>xxx (xx%)<br>xxx (xx%)<br>xxx (xx%)<br>xxx (xx%)<br>xxx (xx%) | xxx<br>xxx (xx%)<br>xxx (xx%)<br>xxx (xx%)<br>xxx (xx%)<br>xxx (xx%) |
| MARS-A 10-Score [1] | n<br>Mean<br>SD<br>Median<br>Min.<br>Max. | XX<br>XX.X<br>X.XX<br>XX.X<br>XX | XX<br>XX.X<br>X.XX<br>XX.X<br>XX |

Note: MARS-A: Medication Adherence Report Scale for Asthma.

Note: Due to an issue identified with the French translation of the MARS-A, a reminder was sent to centres in France instructing that the questionnaire refers to the patient's preventer inhaler (i.e. their maintenance therapy prior to entering the study, and study medication while on-study).

[1]: MARS-A 10-Score is based on the mean score across all ten questions.

HZA116492

Programming note: Repeat on subsequent pages for Visit = Week 12, Week 24 and Early Withdrawal, and for Status = Patients in France who had completed at least one MARS-A assessment prior to the reminder being implemented but also completed at least one MARS-A assessment after the reminder being implemented, Patients in France who had not completed any MARS-A assessments prior to the reminder being implemented, Patients in Germany.
HZA116492

Example : EFF\_T11
Protocol : HZA116492
Population : Intent-to-Treat


# Table 2.xx Summary of Severe On-Treatment Asthma Exacerbations

| | Usual ICS/LABA<br>(N=xxx) | FF/VI<br>(N=xxx) |
|---|---|---|
| No. of subjects with one or more severe asthma exacerbation | xx (xx%) | xx (xx%) |
| Total no. of severe asthma exacerbations | xx | XX |
| Number of severe asthma exacerbations per subject 0 1 > 1 | xx (xx%)<br>xx (xx%)<br>xx (xx%) | xx (xx%)<br>xx (xx%)<br>xx (xx%) |
| Duration of severe asthma exacerbation (days) [1] | | |
| n | XX | XX |
| Mean | XX.X | XX.X |
| SD | X.XX | X.XX |
| Median | XX.X | XX.X |
| Min. | XX | XX |
| Max. | XX | XX |

<sup>[1]</sup> Summary only includes exacerbations for which a date of resolution or death is provided.

HZA116492

Example : EFF\_T11
Protocol : HZA116492
Population : Intent-to-Treat


# Table 2.xx Summary of Severe On-Treatment Asthma Exacerbations

| | Usual ICS/LABA<br>(N=xxx) | FF/VI<br>(N=xxx) |
|---|---|---|
| Outcome | | |
| Resolved | xx (xx%) | xx (xx%) |
| Fatal | xx (xx%) | xx (xx%) |
| Not resolved | xx (xx%) | xx (xx%) |
| Total no. of severe asthma exacerbations | XX | XX |
| No. of exacerbations: | | |
| Requiring use of systemic/oral corticosteroids | xx (xx%) | xx (xx%) |
| Leading to hospitalisation | xx (xx%) | xx (xx%) |
| Requiring emergency room visit | xx (xx%) | xx (xx%) |
| No. of exacerbations requiring intubation | xx (xx%) | xx (xx%) |
| No. of exacerbations leading to withdrawal from study | xx (xx%) | xx (xx%) |

<sup>[1]</sup> Summary only includes exacerbations for which a date of resolution or death is provided.

HZA116492

Example : EFF\_T11S Protocol : HZA116492

HZA116492 

Population : Intent-to-Treat

# Table 2.xx Summary of Severe On-Treatment Asthma Exacerbations by Season

Season: Spring

| | Usual ICS/LABA<br>(N=xxx) | FF/VI<br>(N=xxx) |
|---|---|---|
| No. of subjects with one or more severe asthma exacerbation | xx (xx%) | xx (xx%) |
| Total no. of severe asthma exacerbations | XX | XX |
| Number of severe asthma exacerbations per subject 0 1 > 1 | xx (xx%)<br>xx (xx%)<br>xx (xx%) | xx (xx%)<br>xx (xx%)<br>xx (xx%) |
| Duration of severe asthma exacerbation (days) [1] | | |
| n | XX | XX |
| Mean | XX.X | XX.X |
| SD | X.XX | X.XX |
| Median | XX.X | XX.X |
| Min. | XX | XX |
| Max. | XX | XX |

Note: Spring = March, April and May; Summer = June, July and August; Autumn = September, October and November; Winter = December, January and February. [1] Summary only includes exacerbations for which a date of resolution or death is provided.

HZA116492

Example : EFF\_T11 Protocol : HZA116492

: HZA116492 

Population : Intent-to-Treat

# Table 2.xx Summary of Severe On-Treatment Asthma Exacerbations by Season

Season: Spring

| | Usual ICS/LABA<br>(N=xxx) | FF/VI<br>(N=xxx) |
|---|---|---|
| Outcome | | |
| Resolved | xx (xx%) | xx (xx%) |
| Fatal | xx (xx%) | xx (xx%) |
| Not resolved | xx (xx%) | xx (xx%) |
| Total no. of severe asthma exacerbations | xx | XX |
| No. of exacerbations: | | |
| Requiring use of systemic/oral corticosteroids | xx (xx%) | xx (xx%) |
| Leading to hospitalisation | xx (xx%) | xx (xx%) |
| Requiring emergency room visit | xx (xx%) | xx (xx%) |
| No. of exacerbations requiring intubation | xx (xx%) | xx (xx%) |
| No. of exacerbations leading to withdrawal from study | xx (xx%) | xx (xx%) |

Note: Spring = March, April and May; Summer = June, July and August; Autumn = September, October and November; Winter = December, January and February. [1] Summary only includes exacerbations for which a date of resolution or death is provided.

Programming note: repeat on subsequent pages for Season = Summer, Autumn, Winter.

HZA116492

Example : EFF\_T12
Protocol : HZA116492
Population : Intent-to-Treat


Table 2.xx Summary of the Statistical Analysis of Severe On-Treatment Asthma Exacerbations

| | Usual ICS/LABA<br>(N=xxx) | FF/VI<br>(N=xxx) |
|---|---|---|
| n | XXX | XXX |
| LS Mean Annual Rate | X.XX | X.XX |
| FF/VI vs. Usual ICS/LABA<br>Ratio | | X.XX |
| 95% CI | | (x.xx, x.xx) |
| p-value | | X.XXX |
| Percent Reduction<br>95% CI | | x.xx<br>(x.xx, x.xx) |

Note: The analysis method was Generalised Linear Model assuming an underlying negative binomial distribution with a log-link function and logarithm of time on treatment as an offset variable and adjusted for randomised treatment, number of severe asthma exacerbations in the previous year prior to randomisation, gender, age and country.

HZA116492

Example : EFF\_T13
Protocol : HZA116492
Population : Intent-to-Treat


Table 2.xx
Summary of the Statistical Analysis of Time to First Severe On-Treatment Asthma Exacerbation

| | Usual ICS/LABA<br>(N=xxx) | FF/VI<br>(N=xxx) |
|---|---|---|
| Number of subjects with event<br>Number of subjects censored | xx (xx%)<br>xx (xx%) | xx (xx%)<br>xx (xx%) |
| Probability of having event (%) [1] 95% CI | xx.x<br>(xx.x, xx.x) | xx.x<br>(xx.x, xx.x) |
| FF/VI vs. Usual ICS/LABA<br>Hazard Ratio [2]<br>95% CI<br>p-value | | X.XX<br>(XX.X, XX.X)<br>X.XXX |

<sup>[1]</sup> Kaplan-Meier estimates.

Note: At Day 168 all subjects who have not experienced a severe asthma exacerbation are considered censored, regardless of whether their on-treatment phase continues beyond Day 168.

<sup>[2]</sup> Overall hazard ratios, CIs and p-values are from a Cox proportional hazards model with randomised treatment, gender, age and country as covariates. A hazard ratio <1 indicates a lower risk with FF/VI compared with Usual ICS/LABA.

HZA116492

Example : EFF\_T14

Protocol : HZA116492 Page 1 of 5

Population : Intent-to-Treat

Table 2.xx

Summary of Percentage of Subjects Who Have an Increase from Baseline of >=0.5 in AQLQ(S) Total Score and Domain Scores

Domain: Total Score

| Visit | Response | Usual ICS/LABA<br>(N=xxx) | FF/VI<br>(N=xxx) |
|---|---|---|---|
| Week 24 | n | xxx | xxx |
| | Responder [1] | xxx (xx%) | xxx (xx%) |
| | Non-Responder | xxx (xx%) | xxx (xx%) |
| Early Withdrawal | n | xxx | xxx |
| | Responder [1] | xxx (xx%) | xxx (xx%) |
| | Non-Responder | xxx (xx%) | xxx (xx%) |

[1] Responder is defined as an increase from baseline of >= 0.5.

Programming note: repeat on subsequent pages for Domain = Environmental Stimuli, Symptoms, Activity Limitations and Emotional Function.

HZA116492

Example : EFF\_T15 Protocol : HZA116492


Protocol : HZA116492
Population : Intent-to-Treat

Table 2.xx Summary of EQ-5D-5L Descriptive System Dimensions

Dimension: Anxiety/Depression

| Visit | | Usual ICS/LABA<br>(N=xxx) | FF/VI<br>(N=xxx) |
|---|---|---|---|
| Day 0 | n | XXX | XXX |
| | I am not anxious or depressed | xxx (xx%) | xxx (xx%) |
| | I am slightly anxious or depressed | xxx (xx%) | xxx (xx%) |
| | I am moderately anxious or depressed | xxx (xx%) | xxx (xx%) |
| | I am severely anxious or depressed | xxx (xx%) | xxx (xx%) |
| | I am extremely anxious or depressed | xxx (xx%) | xxx (xx%) |
| | Missing | xxx (xx%) | xxx (xx%) |
| Week 24 | n | XXX | XXX |
| | I am not anxious or depressed | xxx (xx%) | xxx (xx%) |
| | I am slightly anxious or depressed | xxx (xx%) | xxx (xx%) |
| | I am moderately anxious or depressed | xxx (xx%) | xxx (xx%) |
| | I am severely anxious or depressed | xxx (xx%) | xxx (xx%) |
| | I am extremely anxious or depressed | xxx (xx%) | xxx (xx%) |
| | Missing | xxx (xx%) | xxx (xx%) |

Programming note: repeat on subsequent pages for Visit = Early Withdrawal and for Dimension = Mobility, Pain/Discomfort, Self-care, Usual activities.

HZA116492

# 10.16.4. Efficacy Figure Shells

Example : EFF\_F1

Protocol : HZA116492 

Population : Intent-to-Treat

Figure 2.xx Summary of ACT Total Score

Programming note: present "ACT Total Score" on y-axis and "Visit" on x-axis (Day 0, Week 6, Week 12, Week 18, Week 24). Present mean ACT Total Score ± SD separately for treatment group (FF/VI, Usual ICS/LABA) at each visit, connecting the means with a solid line. Distinguish the treatment groups by different line types and colours.

# Repeat for:

Summary of Change from Baseline in ACT Total Score Per Protocol Population (PP Population)

Summary of Change from Baseline in ACT Total Score by Country (ITT Population)

Country: France Country: Germany

HZA116492

Example : EFF\_F2
Protocol : HZA116492
Population : Intent-to-Treat


Figure 2.xx
Summary of Primary and Sensitivity Analyses for Change from Baseline in ACT Total Score at Week 12 (Visit 4)



Programming note: present "Treatment difference" on the x-axis, and reverse axis so treatment difference increases from left to right. Replace "Ratio (95% CI)" with "Treatment Difference (95% CI)". Present lines for the following: Primary analysis (ITT), Primary analysis (PP), ANCOVA with LOCF (ITT), Multiple Imputation (Missing at Random) (ITT), Multiple Imputation (Copy Differences from Reference) (ITT), Hodges-Lehmann (ITT), ANCOVA with WOCF (ITT).

HZA116492

#### Repeat for:

Summary of Key Secondary and Sensitivity Analyses for Change from Baseline in ACT Total Score at Week 24 (Visit 6)

Example : EFF\_F3
Protocol : HZA116492
Population : Intent-to-Treat


Figure 2.xx
Summary of Interaction Tests for Change from Baseline in ACT Total Score at Week 12 (Visit 4)



Programming note: present "LS Mean Change" on the x-axis, and reverse axis so it increases from left to right. Replace "Ratio (95% CI)" with "LS Mean Change (95% CI)". Present the following subgroups: Country (France, Germany); Number of Severe Asthma Exacerbations in the Previous Year Prior to Randomisation (0, >= 1); Smoking Status at Baseline (Current Smokers, Former Smokers, Never Smoked); Age Group (18 – 50 Years Old, > 50 Years Old); Gender (Male, Female).

HZA116492

Example : EFF\_F4
Protocol : HZA116492


Population : Intent-to-Treat

Figure 2.xx

Histogram of Percentage of Subjects Who Have Either an ACT Total Score of >= 20 or >= 3 Point Increase from Baseline in ACT Total Score

Programming note: present "Percent of Subjects (%)" on y-axis and "Visit" on x-axis (Week 6, Week 12, Week 18, Week 24, Early Withdrawal). For each visit, present 3 vertical bars distinguished by fill pattern (similar to non-standard EFF\_F6). Each bar represents: "ACT Total Score >= 20 or >= 3 Point Increase from Baseline in ACT Total Score", "ACT Total Score >= 20" and ">= 3 Point Increase from Baseline in ACT Total Score" respectively and should be labelled as such on the legend.

HZA116492

Example : EFF\_F5
Protocol : HZA116492
Population : Intent-to-Treat


Figure 2.xx
Box Plot of Compliance with Study Medication



Programming Note: label y-axis title as "Compliance (%)", maximum of y-axis may be > 100%.

HZA116492

Example : EFF\_F6

Protocol : HZA116492 Population : Intent-to-Treat 

Figure 2.xx Histogram of the Questions and Answers of the MARS-A Questionnaire

Randomised Treatment: Usual ICS/LABA Visit: Day 0



Note: MARS-A = Medication Adherence Report Scale for Asthma.

Programming note: repeat on subsequent pages for Visit = Week 24, Week 52 and Early Withdrawal; and for Randomised Treatment = FF/VI.

HZA116492

#### Repeat for:

Histogram of the Questions and Answers of the MARS-A Questionnaire by Status of Patient in Relation to the Reminder Sent to French Centres (ITT Population)

Status: Patients in France who had completed all MARS-A assessments prior to the reminder being implemented

Status: Patients in France who had completed at least one MARS-A assessment prior to the reminder being implemented but also completed at least one MARS-A assessment after the reminder being implemented

Status: Patients in France who had not completed any MARS-A assessments prior to the reminder being implemented

Status: Patients in Germany

Add the following footnote: "Note: Due to an issue identified with the French translation of the MARS-A, a reminder was sent to centres in France instructing that the questionnaire refers to the patient's preventer inhaler (i.e. their maintenance therapy prior to entering the study, and study medication while on-study)."

HZA116492

Example : EFF\_F7
Protocol : HZA1164

: HZA116492 Page 1 of 4

Population : Intent-to-Treat

Figure 2.xx Histogram of the Distribution of MARS-A Scores During the Study



Note: MARS-A = Medication Adherence Report Scale for Asthma.

Note: MARS-A 10-Score is based on the mean score across all ten questions.

Programming note: repeat on subsequent pages for Visit = Week 52 and Early Withdrawal.

HZA116492

#### Repeat for:

Histogram of the Distribution of MARS-A Scores During the Study by Status of Patient in Relation to the Reminder Sent to French Centres (ITT Population)

Status: Patients in France who had completed all MARS-A assessments prior to the reminder being implemented

Status: Patients in France who had completed at least one MARS-A assessment prior to the reminder being implemented but also completed at least one MARS-A assessment after the reminder being implemented

Status: Patients in France who had not completed any MARS-A assessments prior to the reminder being implemented

Status: Patients in Germany

Add the following footnote: "Note: Due to an issue identified with the French translation of the MARS-A, a reminder was sent to centres in France instructing that the questionnaire refers to the patient's preventer inhaler (i.e. their maintenance therapy prior to entering the study, and study medication while on-study)."

HZA116492

Example : EFF\_F8
Protocol : HZA116492
Population : Intent-to-Treat


Figure 2.xx
Box Plot of Severe On-Treatment Asthma Exacerbation Rates Adjusted for Exposure to Treatment



HZA116492

Example : EFF\_F9
Protocol : HZA116492
Population : Intent-to-Treat


Figure 2.xx
Kaplan-Meier Plot of Time to First Severe On-Treatment Asthma Exacerbation



Programming note: display increments of 6 weeks on the x-axis, up to the maximum exposure (e.g. 0, 6, 12, 18, 24, 30).

HZA116492

# 10.16.5. Safety Table Shells

Example : SAFE\_T1
Protocol : HZA116492
Population : Safety


# Table 3.xx On-Treatment Serious Adverse Events and Adverse Drug Reactions Overview

| | Usual ICS/LABA<br>(N=xxx) | FF/VI<br>(N=xxx) |
|---|---|---|
| Any on-treatment ADRs Any on-treatment non serious ADRs Any on-treatment serious ADRs Any post-treatment serious ADRs | xxx (xx%)<br>xxx (xx%)<br>xxx (xx%)<br>xxx (xx%) | xxx (xx%)<br>xxx (xx%)<br>xxx (xx%)<br>xxx (xx%) |
| Any on-treatment SAEs Any post-treatment SAEs | xxx (xx%)<br>xxx (xx%) | xxx (xx%)<br>xxx (xx%) |
| Any SAEs or ADRs leading to permanent discontinuation of study drug or withdrawal from study [1] | xxx (xx%) | xxx (xx%) |
| Any on-treatment fatal serious ADRs | xxx (xx%) | xxx (xx%) |
| Any on-treatment fatal SAEs<br>Any post-treatment fatal SAEs | xxx (xx%)<br>xxx (xx%) | xxx (xx%)<br>xxx (xx%) |

[1] Includes both on-treatment and post-treatment SAEs and ADRs.

Programming note: Based on IDSL standard template AE13.

HZA116492

Example : SAFE\_T2
Protocol : HZA116492
Population : Safety


Table 3.xx
Summary of On-Treatment Non-Serious Adverse Drug Reactions of Special Interest

| Special Interest Group/ | | |
|--------------------------|----------------|-----------|
| Subgroup | Usual ICS/LABA | FF/VI |
| Preferred Term | (N=xxx) | (N=xxx) |
| Adrenal suppression | | |
| Any event | xxx (xx%) | xxx (xx%) |
| Blood cortisol decreased | xxx (xx%) | xxx (xx%) |
| Cardiovascular effects | | |
| Any event | xxx (xx%) | xxx (xx%) |
| Cardiac Arrhytmia [1] | xxx (xx%) | xxx (xx%) |
| Any event | xxx (xx%) | xxx (xx%) |
| Palpitations | xxx (xx%) | xxx (xx%) |
| Extrasystoles | xxx (xx%) | xxx (xx%) |
| Cardiac Ischaemia [1] | xxx (xx%) | xxx (xx%) |
| Any event | xxx (xx%) | xxx (xx%) |
| Angina pectoris | xxx (xx%) | xxx (xx%) |
| Chest pain | xxx (xx%) | xxx (xx%) |
| Effects on potassium | | |
| Any event | xxx (xx%) | xxx (xx%) |
| XXXXXXX | xxx (xx%) | xxx (xx%) |
| XXXXXXX | xxx (xx%) | xxx (xx%) |
| | () | ( , , , , |

[1]: This subgroup was defined using Special MedDRA queries.

Programming note: Based on IDSL standard template AE1.

HZA116492

# Repeat for:

Summary of On-Treatment Serious Adverse Drug Reactions of Special Interest (ITT Population)
Summary of On-Treatment Adverse Drug Reactions of Special Interest (ITT Population)
Summary of On-Treatment Serious Adverse Events of Special Interest (ITT Population)
Summary of On-Treatment Fatal Serious Adverse Events of Special Interest (ITT Population)
Summary of On-Treatment Non-Fatal Serious Adverse Events of Special Interest (ITT Population)

HZA116492

Example : SAFE\_T3
Protocol : HZA116492

Population : Safety


Table 3.xx
Top Ten Most Commonly Reported On-Treatment Adverse Drug Reactions Per Treatment Group

| Preferred Term | Usual ICS/LABA<br>(N=xxx) | FF/VI<br>(N=xxx) |
|----------------|---------------------------|------------------|
| XXXXXXX | xxx (xx%) | xxx (xx%) |

Programming note: Present the ten most frequent preferred terms in Usual ICS/LABA, and the ten most frequent in FF/VI (do not use percentages to determine "most frequent").

HZA116492

# 10.16.6. Safety Figure Shells

Example : SAFE\_F1 Protocol : HZA116492

Page 1

of 1

Population : Intent-to-Treat/Safety

Figure 2.xx Summary of Benefit:Risk for FF/VI vs. Usual ICS/LABA



<sup>\* =</sup> Number of subjects with event

- (a) Difference in LS mean change from baseline from an MMRM
- (b) Difference in LS mean change from baseline from an ANCOVA model
- (c) Adjusted odds ratio obtained from a logistic regression model
- (d) Risk difference

HZA116492

Programming note: present the following endpoints:

- Benefits:
- First panel, x-axis decreasing from left to right:
  - o Difference in LS mean change from baseline and 95% CI for: change from baseline in ACT total score at Week 12 (Visit 4) and at Week 24 (Visit 6) (labeled (a))
  - Difference in LS mean change from baseline and 95% CI for change from baseline in trough (pre-dose) FEV1 at Week 12 (Visit 4) (labeled (b))
- Second panel, x-axis increasing from left to right:
  - Adjusted odds ratio and 95% CI for: percentage of subjects with correct use of inhaler device at Week 12 (Visit 4) and at Week 24 (Visit 6) (labeled (c))
- Risks:
- Third panel, x-axis increasing from left to right:
  - Risk difference and 95% CI of the following SAEs of special interest: asthma/bronchospasm, cardiovascular effects, decreased bone mineral density and associated fractures, hypersensitivity, local steroid effects, lower respiratory tract infection (LRTI) excluding pneumonia, pneumonia, adrenal suppression, ocular effects, effects on glucose, effects on potassium, tremor (labeled (d))

HZA116492

# 10.16.7. Non-ICH Listing Shells

Example Protocol Population

: POP\_L1 : HZA116492 : All Subjects Enrolled Page 1 of n

Listing x
Subjects Screened but Not in the Intent-to-Treat Population

Randomised

| Treatment | lnv. | Subj. | Disposition Status | Reason for Screen Failure/Withdrawal |
|---|---|---|---|---|
| Screen Failure | XXXXXX | XXXXXX | Screen Failure | Xxxxxxxxxxx |
| FF/VI | XXXXXX | XXXXXX | Early Withdrawal | Xxxxxxxxxxx |

HZA116492

Example : POP\_L2 Protocol : HZA116492


Protocol : HZA116492
Population : Intent-to-Treat

# Listing x Reasons for Important Protocol Deviations

| Randomised | | | | Excluded | | |
|---|---|---|---|---|---|---|
| Treatment | lnv. | Subj. | Important Protocol Deviation | from PP? | Date of Deviation | Study Day of Deviation |
| FF/VI | XXXXX | XXXXX | XXXXXXXXXXX | No | DDMMMYYYY | XX |
| | XXXXX | XXXXX | XXXXXXXXXXX | No | DDMMMYYYY | XX |
| Usual ICS/LABA | xxxxx | xxxxx | XXXXXXXXXX | No | DDMMMYYYY | XX |
| | XXXXX | XXXXX | XXXXXXXXXXX | Yes | DDMMMYYYY | XX |
| | XXXXX | XXXXX | XXXXXXXXXXX | No | DDMMMYYYY | XX |
| | XXXXX | XXXXX | XXXXXXXXXXX | No | DDMMMYYYY | XX |

....

# 2017N339371\_00


HZA116492

Example Protocol Population : POP\_L3 : HZA116492

: Intent-to-Treat


Listing x Asthma History

| | | | | Number of asthma exacerbation | lumber of asthma exacerbations in the last 12 months that: | |
|---|---|---|---|---|---|---|
| | | | | Did not require oral/systemic corticosteroids (not involving | Required oral/systemic corticosteroids (not involving | |
| Treatment | lnv. | Subj. | Asthma Duration | hospitalisation) | hospitalisation) | Required hospitalisation |
| XXXXXX | XXXXXX | XXXXXX | XXXXXXXXXXX | XX | XX | XX |
| | XXXXXX | XXXXXX | XXXXXXXXXXXX | XX | XX | XX |
| | XXXXXX | XXXXXX | XXXXXXXXXXX | XX | XX | XX |
| | XXXXXX | XXXXXX | XXXXXXXXXXX | XX | XX | XX |

# 2017N339371\_00


HZA116492

Example : POP\_L4
Protocol : HZA116492
Population : Intent-to-Treat


Listing x Smoking History

| Treatment | Inv./<br>Subj.<br>Xxxxxx/<br>xxxxxx | Smoking<br>Status<br>Current | Years Smoked/<br>Cigarettes per day<br>xx/<br>xx | Smoking<br>Pack Years<br>xx |
|---|---|---|---|---|
| | Xxxxxx/<br>xxxxxx | Former | xx/<br>xx | XX |
| | Xxxxxx/<br>xxxxxx | Never | | |

HZA116492

Example Protocol : POP\_L5 : HZA116492

: Intent-to-Treat Population


Listing x
Exposure to Study Medication

Treatment: Usual ICS/LABA

| Inv./<br>Subj. | Treatment Start Date/<br>Treatment End date | Start date of dose/<br>End date of dose/<br>Duration of dose (days) | Drug | Dose/ Dose<br>Units/ Dose<br>Frequency | Inhalers<br>Dispensed/<br>Inhalers Returns | Dose counter start/<br>Dose counter stop | Compliance (%) During the study |
|---|---|---|---|---|---|---|---|
| XXXX | DDMMMYYY/ | | | | | | XX.XX |
| | DDMMMYYY | DDMMMYYYY/<br>DDMMMYYYY/ | XXXXXXX | XX/ XX/XXXX | X/X | XXX/XX | |
| | | XX<br>DDMMMYYYY/<br>DDMMMYYYY | XXXXXXX | XX/ XX/XXXX | X/X | XXX/XX | |
| XXXX | DDMMMYYY | XX | | | | | XX.XX |
| | | DDMMMYYYY/<br>DDMMMYYYY/<br>xx | XXXXXXX | XX/ XX/XXXX | X/X | XXX/XX | |

Programming note: Repeat on subsequent pages for Treatment = FF/VI, and use GSK drug synonym as drug name.

HZA116492

Example : EFF\_L1 Protocol

: HZA116492 Page 1 of n

Population : Intent-to-Treat

Listing x ACT Scores

Treatment: Usual ICS/LABA

| Inv./<br>Subj. | Visit/<br>Study Date/<br>Study Day | Impact at<br>home or work<br>[1] | Frequency of shortness of breath [1] | Frequency of sleep trouble [1] | Frequency of rescue medication [1] | Asthma control rating [1] | ACT Total<br>Score [2] /<br>Change from<br>Baseline |
|---|---|---|---|---|---|---|---|
| xxxxxx/<br>xxxxx | Day 0/<br>DDMMMYYYY/ | X | X | Х | X | X | XX |
| | xx<br>Week 6/<br>DDMMMYYYY/<br>xx | x | х | Х | х | х | xx /<br>-x |
| | Week 12/<br>DDMMMYYYY/<br>xx | X | Х | Х | Х | X | xx /<br>x |

<sup>[1]</sup> Responses range between 1 (worst response) and 5 (best response).
[2] ACT Total Score ranges between 5 (worst asthma control state) and 25 (best asthma control state).

HZA116492

Example : EFF\_L2
Protocol : HZA116492
Population : Intent-to-Treat


Listing x Inhaler Device Use

Treatment: Usual ICS/LABA

| | Visit/ | | Critical e | Critical errors | | Non-critical errors |
|---|---|---|---|---|---|---|
| Inv./<br>Subj. | Study Date/<br>Study Day | Inhaler | Any? | If yes, errors: | Any? | If yes, errors: |
| xxxxxx/<br>xxxxx | Day 0/<br>DDMMMYYYY/ | Turbuhaler | No | | No | |
| | xx<br>Week 12/<br>DDMMMYYYY/ | Turbuhaler | No | | Yes | Did not hold breath |
| | xx<br>Week 24/<br>DDMMMYYYY/<br>xx | Turbuhaler | Yes | Exhaled directly into mouthpiece | No | |
| xxxxxx/<br>xxxxx | Day 0/<br>DDMMMYYYY/<br>xx | Diskus | Yes | Did not hold device upright during dose preparation Shook the device after dose preparation | Yes | No exhalation before an inhalation |
| | Week 12/<br>DDMMMYYYY/<br>xx | Diskus | Yes | Shook the device after dose preparation | No | |

HZA116492

Example : EFF\_L3

Protocol : HZA116492


Trough (pre-dose) percent

Population : Intent-to-Treat

Listing x Lung Function Tests

Treatment: Usual ICS/LABA

predicted normal FEV1 (%) Trough (pre-dose) FEV1 (L) Bronchodilator Predicted Inv./ Study Date/ Study Change from Change from taken in last 4 Baseline normal FEV1 (L) Absolute Subj. Absolute Visit Time Day Baseline hours? DDMMMYYYY/ Day 0 No xxxxxx/ XX X.XXX X.XXX XX.X HH:MM XXXXX Week 6 DDMMMYYYY/ No XX X.XXX X.XXX X.XXX XX.X XX.X HH:MM xxxxxx/ Day 0 DDMMMYYYY/ No X.XXX X.XXX X.XXX XX.X XX.X HH:MM XXXXX

HZA116492

Example : EFF\_L4
Protocol : HZA11649

: HZA116492 Page 1 of n

Population : Intent-to-Treat

Listing x

Medication Adherence Report Scale for Asthma (MARS-A) Scores

Treatment: Usual ICS/LABA

| Inv./ | | Visit/<br>Study Date/ | | | |
|---|---|---|---|---|---|
| Subj. | Status [1] | Study Day | Assessor Code | MARS-A Questions | Score [2] |
| xxxxxx/<br>xxxxx | During | Day 0/<br>DDMMMYYYY/ | Subject/Other | I only use it when I need it | Х |
| | | XX | | Only was it when I feel has all less | |
| | | | | Only use it when I feel breathless | Х |
| | | | | I decide to miss out a dose | Χ |
| | | | | I try to avoid using it | X |
| | | | | I forget to take it | X |
| | | | | I alter the dose | Χ |
| | | | | I stop taking it for a while | Χ |
| | | | | Reserve if treatment doesn't work | Χ |
| | | | | Before doing something | Χ |
| | | | | I take less than instructed | Χ |
| | | | | MARS-A 10-Score [3] | X.XX |
| | | Week 12/<br>DDMMMYYYY/<br>xx | Subject/Other | I only use it when I need it | х |
| | | ٨٨ | | Only use it when I feel breathlessetc | х |

<sup>[1]</sup> Due to an issue identified with the French translation of the MARS-A, a reminder was sent to centres in France instructing that the questionnaire refers to the patient's preventer inhaler (i.e. their maintenance therapy prior to entering the study, and study medication while on-study. Status = Prior (patient in France who had completed all MARS-A assessments prior to the reminder), During (patient in France who had completed at least one MARS-A assessment prior to the reminder but

HZA116492

also completed at least one MARS-A assessment after the reminder), After (patient in France who had not completed any MARS-A assessments prior to the reminder), Germany (patient in Germany).

- [2] Question scores range between 1 (always) and 5 (never).
  [3] MARS-A 10-Score is based on the mean score across all ten questions.

HZA116492

Example Protocol

: EFF\_L5 : HZA116492 Population : Intent-to-Treat


Listing x
Severe Asthma Exacerbations

Treatment: Usual ICS/LABA

| Inv./<br>Subj. | Date of Onset/<br>Study day/<br>Date of Resolution/<br>Study day | Resolution/<br>Withdrawn from Study? | Required use of systemic/oral corticosteroids? | Led to hospitalisation? | Required emergency room visit? | Required intubation? |
|---|---|---|---|---|---|---|
| Xxxxxx/<br>xxxxx | DDMMMYYYY/<br>xx/<br>DDMMMYYYY/<br>xx | Resolved/<br>N | Y | N | N | N |
| | DDMMMYYYY/<br>xx/<br>DDMMMYYYY/<br>xx | Resolved/<br>N | N | N | Υ | N |
| | DDMMMYYYY/<br>xx/<br>DDMMMYYYY/<br>xx | Fatal/<br>Y | Υ | Υ | N | Υ |

HZA116492

Example

: EFF\_L6 : HZA116492 Protocol


Population : Intent-to-Treat

Listing x AQLQ(S) Scores

Treatment: Usual ICS/LABA

| Inv./<br>Subj. | Visit/<br>Study Date/<br>Study Day | Symptoms [1] | Activity Limitations | Emotional<br>Function [1] | Environmental<br>Stimuli [1] | AQLQ(S) Total<br>Score [1] /<br>Change from<br>Baseline |
|---|---|---|---|---|---|---|
| xxxxxx/ | Day 0/ | X.X | X.X | X.X | X.X | X.X |
| XXXXX | DDMMMYYYY/ | | | | | |
| | XX | | | | | 1 |
| | Week 24/ | X.X | X.X | X.X | X.X | x.x / |
| | DDMMMYYYY/ | | | | | X.X |
| | XX | | | | | |

[1] Scores range between 1 (lower quality of life) and 7 (higher quality of life) for AQLQ(S) total and domains.

HZA116492

Example : EFF\_L7
Protocol : HZA116492


Population : Intent-to-Treat

Listing x

EQ-5D-5L Descriptive System Dimension Scores

Treatment: Usual ICS/LABA

| | Visit/ | | | | |
|---|---|---|---|---|---|
| Inv./ | Study Date/ | | Subscale/ | | |
| Subj. | Study Day | Assessor Code | Item | Level of Problem | Score [1] |
| xxxxxx/ | Day 0 | Subject/Other | EQ-5D-5L Utility | | XX.XX |
| XXXXX | DDMMMYYYY/ | | Score | | |
| | XX | | | | |
| | | | Mobility | 1 | |
| | | | Self-Care | 1 | |
| | | | Usual Activities | 1 | |
| | | | Pain/Discomfort | 1 | |
| | | | Anxiety/Depression | 1 | |
| | | | EQ-5D-5L VAS | | XX.XX |
| | Week 12 | Subject/Other | EQ-5D-5L Utility | | XX.XX |
| | DDMMMYYYY/ | | Score | | |
| | XX | | | | |
| | | | Mobilityetc | 1 | |

<sup>[1]</sup> Scores range between 0 (worst imaginable health state) and 1 (best imaginable health state) for EQ-5D-5L Utility Score and range between 0 (worst imaginable health state) and 100 (best imaginable health state) for EQ-5D-5L Visual Analogue Scale (VAS).

HZA116492

Example : EFF\_L8
Protocol : HZA116492
Population : Intent-to-Treat


Listing x PASAP-Q Scores

Treatment: Usual ICS/LABA

| | Visit/ | | | |
|---|---|---|---|---|
| Inv./ | Study Date/ | Domain / | | |
| Subj. | Study Day | Question | Response | Score [1] |
| xxxxxx/ | Day 0 | Performance | | XX.X |
| XXXXX | DDMMMYYYY/ | | | |
| | XX | | | |
| | | Overall feeling of inhaling | X | |
| | | Inhaled dose goes to lungs | X | |
| | | Medication left | X | |
| | | Works reliably | X | |
| | | Ease of inhaling a dose | X | |
| | | Using the inhaler | X | |
| | | Speed medicine comes out | X | |
| | | Convenience | | XX.X |
| | | Instructions for use | X | |
| | | Size of inhaler | X | |
| | | Durability of inhaler | X | |
| | | Ease of cleaning inhaler | X | |
| | | Ease of holding during use | X | |
| | | Convenience of carrying | X | |
| | | Total Score | | XX.X |

Willingness to Continue Using Inhaler xx.x

[1] Performance, Convenience, Total Score, and Willingness to Continue Using Inhaler are expressed on a scale of 0 to 100. Overall Satisfaction is expressed on a scale of 1 to 7.

Overall Satisfaction

Χ

HZA116492

HZA116492

Example : SAFE\_L1 Protocol : HZA116492

Population

: Intent-to-Treat


Listing x
AE Terms of Special Interest

| Special Interest Term | Subgroup | Preferred Term |
|-----------------------|--------------------|-----------------------------|
| XXXXX XXXXX XXXXXX | Xxxxxxx | XXXXXXX |
| | | XXXXXXX XXXXXXX |
| | | XXXX |
| | | XXXXXXX XXX |
| XXXXXXX XXXXXXXXX | xxxxxxxxxxxxxx [1] | XXXXXXX XXXXXX |
| | | XXXXXXX XXXX XXXXX XXXXX |
| | | XXXX |
| XXXXXXXXXX | xxxxxxx [1] | XXXXXXX |
| | | XXXX XXXXXX XXXXXXX |
| XXXXXX XXXXXXX | | xxxxxxxx |
| | | XXXXX XXXXXX XXXXXXX XXXXXX |

<sup>[1]:</sup> This special interest term was defined using Special MedDRA Queries.

Note: All of the pre-specified preferred terms that were assigned to special interest terms are shown, regardless of whether they actually occurred in the study.

Programming Note: The AE special interest dataset and the AE SMQ dataset will be set together in order to report this table and all the subgroups that come from the AE SMQ dataset will be flagged with a [1].

# 2017N339371\_00


HZA116492

Example Protocol Population : SAFE\_L2 : HZA116492

: Intent-to-Treat


Listing x
Inhaler Device Malfunctions

| Treatment | Inv./<br>Subj. | Inhaler Device | Comment / Reason for Malfunction |
|---|---|---|---|
| Usual ICS/LABA | xxxxxx/<br>xxxxx | Turbuhaler | XXXXXXXXX |
| Usual ICS/LABA | xxxxxx/<br>xxxxx | Diskus | XXXXXXXXX |
| FF/VI | xxxxxx/<br>xxxxx | Ellipta | Powder fell out prior to use<br>Other: XXXXXXXX |